An Open-label, Baseline-controlled, Multicenter, Phase 3 Dosetitration Study Followed by a Fixed-dose Observation Period to Evaluate Efficacy, Safety and Pharmacokinetics of Mirabegron in Children and Adolescents From 3 to Less Than 18 Years of Age with Neurogenic Detrusor Overactivity (NDO) on Clean Intermittent Catheterization (CIC)

Open-label Phase 3 Study with Mirabegron in Children From 3 to Less Than 18 Years of Age with Neurogenic Detrusor Overactivity (Crocodile Study)

ISN/Protocol 178-CL-206A

ClinicalTrials.gov Identifier: NCT02751931

**Date of SAP v3: 21 May 2019** 

Sponsor: Astellas Pharma Europe B.V. (APEB)

Sylviusweg 62 2333 BE Leiden, the Netherlands

### STATISTICAL ANALYSIS PLAN

Final Version 3.0, dated 21-May-2019

An Open-label, Baseline-controlled, Multicenter, Phase 3 Dose-titration Study Followed by a Fixed-dose Observation Period to Evaluate Efficacy, Safety and Pharmacokinetics of Mirabegron in Children and Adolescents From 3 to Less Than 18 Years of Age with Neurogenic Detrusor Overactivity (NDO) on Clean Intermittent Catheterization (CIC)

Open-label Phase 3 Study with Mirabegron in Children From 3 to Less Than 18 Years of Age with Neurogenic Detrusor Overactivity (Crocodile Study)

ISN: 178-CL-206A

EudraCT number: 2015-002876-25

IND number: IND 69,416

Astellas Pharma Europe B.V. (APEB)/ Sylviusweg 62 2333 BE Leiden, the Netherlands

.-----

This confidential document is the property of the sponsor. No unpublished information contained in this document may be disclosed without prior written approval of the sponsor.

## **Table of Contents**

| TA | TABLE OF CONTENTS ······ 2 | | |
|---|---|---|---|
| LI | LIST OF TABLES·······6 | | |
| LI | LIST OF ABBREVIATIONS AND KEY TERMS ······ 7 | | |
| 1 | INTRODUCTION······11 | | |
| 2 | | FLO | OW CHART AND VISIT SCHEDULE ······12 |
| 3 | | STU | JDY OBJECTIVE(S) AND DESIGN······15 |
| | 3.1 | L | Study Objective(s) ·····15 |
| | | 3.1.1 | Primary Objectives · · · · · 15 |
| | | 3.1.2 | Secondary Objectives · · · · · · 15 |
| | 3.2 | 2 | Study Design |
| | 3.3 | | Assignment and Allocation · · · · · 17 |
| 4 | | SAI | MPLE SIZE······18 |
| 5 | | AN. | ALYSIS SETS ·····19 |
| | 5.1 | 1 | All Screened Set |
| | 5.2 | 2 | All Allocated Set · · · · · 19 |
| | 5.3 | 3 | Full Analysis Set (FAS) ·····19 |
| | <b>5.</b> 4 | 1 | Per Protocol Set (PPS) 19 |
| | | 5.4.1 | Reasons for Exclusion From PPS · · · · · 20 |
| | 5.5 | 5 | Safety Analysis Set (SAF) ·····21 |
| | 5.6 | 6 | Pharmacokinetics Analysis Set (PKAS)······21 |
| | 5.7 | 7 | Pharmacodynamic Analysis Set (PDAS)······22 |
| 6 | | AN. | ALYSIS VARIABLES ······23 |
| | 6.1 | l | Efficacy Endpoints · · · · 23 |
| | | 6.1.1 | Primary Efficacy Endpoint · · · · · 30 |
| | | 6.1.2 | Primary Estimand ······30 |
| | | 6.1.3 | Secondary Efficacy Endpoints · · · · 31 |
| | | 6.1.4 | Exploratory Efficacy Endpoints |
| | 6.2 | 2 | Safety Endpoints 37 |
| | | 6.2.1 | Vital signs ······40 |
| | | 6.2.2 | Adverse Events · · · · 43 |
| | | 6.2.3 | Clinical Laboratory Variables45 |

| 6. | | 6.2.4 | Physical Examinations | 17 |
|---|---|---|---|---|
| | | 6.2.5 | 12-lead Electrocardiogram (ECG)····· | 18 |
| | | 6.2.6 | Estimated Glomerular Filtration Rate and Upper Urinary Tract Ultrasound ·····4 | 18 |
| | | 6.2.7 | Height, Weight and BMI · | -49 |
| | 6.3 | 3 | Pharmacokinetic Variables | 19 |
| | <b>6.</b> 4 | l | Pharmacodynamic Variables 5 | 50 |
| | 6.5 | 5 | Other Variables | 50 |
| | | 6.5.1 | Baseline Characteristics5 | 50 |
| | | 6.5.2 | Previous and Concomitant Medications and Therapies5 | 50 |
| | | 6.5.3 | Exposure to Study Drug5 | 51 |
| | | 6.5.4 | Compliance to Study Drug5 | 52 |
| 7 | | STA | ATISTICAL METHODOLOGY ······5 | 56 |
| | 7.1 | | General Considerations5 | 56 |
| | 7.2 | 2 | Study Population | 56 |
| | | 7.2.1 | Disposition of Subjects5 | 56 |
| | | 7.2.2 | Protocol Deviations5 | 57 |
| | | 7.2.3 | Demographic and Other Baseline Characteristics5 | 57 |
| | | 7.2.4 | Previous and Concomitant Medications · · · · 5 | 58 |
| | 7.3 | } | Study Drugs · · · · 5 | 59 |
| | | 7.3.1 | Dosing ·····5 | 59 |
| | | 7.3.2 | Exposure ···································· | 50 |
| | | 7.3.3 | Treatment Compliance 6 | |
| | <b>7.</b> 4 | | Analysis of Efficacy ··································· | 51 |
| | | 7.4.1 | Analysis of Primary Endpoint ···································· | 51 |
| | | 7.4.2 | Analysis of Secondary Endpoints · | |
| | | 7.4.3 | Analysis of Exploratory Endpoints · | 55 |
| | | 7.4.4 | Analysis of Other Variables · | |
| | | 7.4.5 | Sensitivity Analysis · | |
| | 7.5 | 5 | Analysis of Safety 6 | 56 |
| | _ | 7.5.1 | Adverse Events · | |
| | | 7.5.2 | Clinical Laboratory Evaluation · | |
| | | 7.5.3 | Vital Signs····· | |
| | | 7.5.4 | Height and Weight ····· | 13 |
| | | 7.5.5 | Electrocardiograms (ECGs) · | 74 |

| | 7.5.6 | Pregnancies 75 |
|---|---|---|
| _ | 7.5.7 | 11 2 |
| 7 | .6 | Analysis of PK······75 |
| | 7.6.1 | Estimation of Pharmacokinetic Parameters ······75 |
| | 7.6.2 | Statistical Analysis · |
| 7 | .7 | Analysis of PD······76 |
| 7 | .8 | Subgroups of Interest ······76 |
| 7 | .9 | Other Analyses ······77 |
| 7 | .10 | Interim Analysis (and Early Discontinuation of the Clinical Study) ······77 |
| 7 | .11 | Handling of Missing Data, Outliers, Visit Windows, and Other Information · · · · · · · 77 |
| | 7.11.1 | 1 Missing Data · |
| | 7.11.2 | 2 Outliers ·····80 |
| | 7.11.3 | 3 Visit Windows ·····80 |
| 8 | DO | CUMENT REVISION HISTORY ······82 |
| 9 | RE | FERENCES88 |
| 10 | APl | PENDICES90 |
| 10.1 Appendix 1: Inclusion and Exclusion Criteria | | Appendix 1: Inclusion and Exclusion Criteria · · · · · 90 |
| 10.2 Appendix 2: List of Excluded Concomitant Medication | | Appendix 2: List of Excluded Concomitant Medications93 |
| 1 | 0.3 | Appendix 3: AEs of Interest not covered by Standard MedDRA SMQs V16.0 ······94 |
| 1 | 0.4 | Appendix 4: Questionnaires 95 |
| | Appe | endix 4.1 Pediatric Incontinence Questionnaire · · · · · 95 |
| | Appe | endix 4.2 Patient Global Impression of Severity Scale ·····96 |
| | | endix 4.3 Acceptability Questionnaire for Tablets ······97 |
| | Appe | endix 4.4 Acceptability Questionnaire for Oral Suspension ······98 |
| | Appe | endix 4.5 Clinical Global Impression of Change Scale · · · · · 100 |
| 1 | 0.5 | Appendix 5 Centiles of heart rate for normal children from birth to 18 years of |
| | | age [Fleming et al, 2011] |
| 1 | 0.6 | Appendix 6 CDC Data Table of Stature-for-age Chart for Males · · · · · 102 |
| 1 | 0.7 | Appendix 7 CDC Data Table of Stature-for-age Chart for Females |
| 1 | 0.8 | Appendix 8 CDC Data Table of Weight-for-age Chart for Males |
| 1 | 0.9 | Appendix 9 CDC Data Table of Weight-for-age Chart for Females · · · · · 122 |
| 1 | 0.10 | Blood Pressure Levels for Males by Age and Height Percentile · · · · · 128 |
| _ | Appe | ndix 10.1 Fourth (4th) Report ······ 128 |

| | Appendix 10.2 | 2017 Clinical Practice Guidelines 129 |
|---|---|---|
| 10. | 11 Blood Pr | essure Levels for Females by Age and Height Percentile |
| | Appendix 11.1 | Fourth (4th) Report · · · · 130 |
| | Appendix 11.2 | 2017 Clinical Practice Guidelines 131 |
| 10. | 12 Appendi | x 12: Calculation of Z-Scores for Height, Weight and BMI for Age and |
| | Sex Nor | ms · · · · · 132 |
| 10. | 13 Appendi | x 13: ECG Abnormality Codes · · · · 154 |
| 10. | 14 Appendi | x 14: Key Contributors and Approvers · · · · · 159 |

# **List of Tables**

| Table 1 | Schedule of Assessments 13 |
|---|---|
| Table 2 | Efficacy Endpoints |
| Table 3 | Summary of Efficacy Endpoints · · · · · 28 |
| Table 4 | Safety Endpoints · · · · 38 |
| Table 5 | Summary of Safety Endpoints |
| Table 6 | Coefficients for Conversion of Blood Pressure to Percentiles |
| Table 7 | Percentiles for Resting Pulse Rate in Relation to Age and Gender43 |
| Table 8 | Standardized MedDRA Queries, Version 16.0 |
| Table 9 | Laboratory Assessments 46 |
| Table 10 | Number of Kits to be Dispensed at each Visit54 |
| Table 11 | Weight based Doses for Suspension54 |
| Table 12 | Definitions of Blood Pressure Categories and Stages70 |
| Table 13 | Percentiles for Pulse Rate in Relation to Age71 |
| Table 14 | Systolic and Diastolic Home Blood Pressure Values · · · · · · 72 |
| Table 15 | Time Windows for Summary of Plasma Concentration Data76 |
| Table 16 | Visit Windows for Efficacy and Safety Parameters 80 |

### ISN/Protocol 178-CL-206A

### LIST OF ABBREVIATIONS AND KEY TERMS

### **List of Abbreviations**

| Abbreviation | Description |
|---|---|
| APEB | Astellas Pharma Europe B.V. |
| APGD | Astellas Pharma Global Development |
| ASCM | Analysis Set Classification Meeting |
| AE | adverse event |
| ALP | alkaline phosphatase |
| ALT | alanine aminotransferase |
| ANCOVA | analysis of covariance |
| AST | aspartate aminotransferase |
| $AUC_{24}$ | Area under the plasma concentration-time curve from time zero to 24 h |
| CIC | clean intermittent catheterization |
| CGI-C | Clinician Global Impression of Change |
| CL/F | apparent total clearance of the drug from plasma after oral administration |
| $C_{max}$ | maximum (peak) plasma drug concentration |
| CRO | contract research organization |
| CSR | clinical study report |
| $C_{trough}$ | trough plasma concentration (measured concentration at the end of a dosing |
| liough | interval at steady state) |
| CYP | cytochrome P450 |
| DRM | Data Review Meeting |
| DSMB | Data and Safety Monitoring Board |
| EBC | Expected Bladder Capacity |
| ECG Electrocardiogram | |
| eCRF electronic case report form | |
| e-diary | electronic diary |
| eGFR | estimated glomerular filtration rate |
| EOS | end of study |
| EOT | end of treatment |
| FAS | full analysis set |
| FSI | First Subject In |
| HLT | High Level Term |
| IB | Investigator's Brochure |
| ICF | informed consent form |
| ICH | International Conference on Harmonisation |
| IEC | Independent Ethics Committee |
| IRB | Institutional Review Board |
| ISN | international study number |
| IUD | intrauterine device |
| IUS | intrauterine system |
| LOCF last observation carried forward | |
| LQTS long QT syndrome | |
| MCC | maximum cystometric capacity |
| M&S | Modeling & Simulation |
| · · · | |
| NDO neurogenic detrusor overactivity OAB overactive bladder | |
| PCR Potentially Clinically Relevant | |
| | · |
| PED | pediatric equivalent dose |

| Abbreviation | Description |
|---|---|
| PDAS | Pharmacodynamic Data Set |
| PGI-S | Patient Global Impression of Severity Scale |
| P-gp | P-glycoprotein |
| PIN-Q | Pediatric Incontinence Questionnaire |
| PK | Pharmacokinetic(s) |
| PKAS | Pharmacokinetics Analysis Set |
| PKDAP | Pharmacokinetic Data Analysis Plan |
| PKMS | Pharmacokinetics, Modeling, and Simulation |
| PPS | per protocol set |
| PR | Pulse Rate |
| QTcB | QT interval corrected by Bazett's formula |
| QTcF | QT interval corrected by Fridericia's formula |
| SAE | serious adverse event |
| SAF | safety analysis set |
| SAP | statistical analysis plan |
| SBPM | self blood pressure measurement |
| TEAE | treatment-emergent adverse event |
| TBL | total bilirubin |
| TLF | tables, listings and figures |
| t <sub>max</sub> | time to reach maximum (peak) plasma concentration following drug |
| | administration |
| ULN | upper limit of normal |
| UTI | urinary tract infection |
| V <sub>z</sub> /F | apparent volume of distribution after nonintravenous administration |

# **List of Key Terms**

| Terms | Definition of terms |
|---|---|
| Baseline | Observed values/findings which are considered to be the starting point for comparison. |
| Discontinuation | The act of concluding participation in a trial by an enrolled subject, prior to completion of all protocol required elements. |
| | Note: subject discontinuation does not necessarily imply exclusion of subject data from analysis that was collected prior to discontinuation. |
| Enroll | To register or enter into a clinical trial, i.e., signing the informed consent form (ICF). Once a subject has been enrolled, the clinical trial protocol applies to the subject. |
| Investigational period | Period of time where major interests of protocol objectives are observed, and where the study drug is given to a subject. This period continues until the last assessment after completing the last dose of the study drug. |
| Pediatric equivalent dose (PEDx) | Weight-range based doses predicted to achieve plasma concentrations equivalent to steady state exposures expected with "x" mg mirabegron administered once daily in adults. |
| Postinvestigational period | Period of time after the last assessment of the protocol. Follow-up observations for sustained adverse events and/or survival are done in this period. |
| Screening | A process of active consideration of potential subjects for a trial. |
| Screening period | Period of time before entering the investigational period, usually from the time the subject signed informed consent until just before the first dose of the study drug is given to a subject. |
| Screening failure | Screened subject who did not fulfill protocol inclusion and/or exclusion criteria, or decided not to participate anymore (withdrew consent) prior to first dose of study drug. |
| Source data | All information in original records or certified copies of original records of clinical findings, observations, or other activities in a clinical trial necessary for the reconstruction and evaluation of the trial. Source data are contained in source documents (original records, certified copies). |
| Source documents | Original documents, data, and records including source data. |
| Steady state | When the amount of drug intake is equilibrium with the rate of drug elimination. |
| | Note: for mirabegron steady state is considered to be reached after 10 days of daily dosing. |
| Study period | Period of time from the first site initiation date to the last site completing the study. |
| Subject | An individual in the population of interest who participates in a clinical trial as recipient of the investigational product. |
| Treatment emergent adverse event | An adverse event observed after starting administration of the study drug. |

# Sponsor: Astellas Pharma Global Development, Inc. ${\rm ISN/Protocol~178\text{-}CL\text{-}206A}$

| Terms | Definition of terms |
|---|---|
| Trough sample | Pharmacokinetic sample taken just prior to the next dose of study medication. |

### 1 INTRODUCTION

This Statistical Analysis Plan (SAP) contains a more technical and detailed elaboration of the principal features of the analysis described in the protocol 178-CL-206A (version 2.0, dated 02 November 2016), the current EU PIP (EMEA-000597-PIP-03-M03, EMA Decision 17 March 2017, ref. P/0056/2017) and US Written Request (NDA 202611, dated 18 March 2016), and includes detailed procedures for executing the statistical analysis of the primary and secondary endpoints and safety data.

The SAP will be finalized and signed prior to First Subject In (FSI). If needed, revisions to the approved SAP may be made prior to the database hard lock. Revisions will be version controlled.

This statistical analysis is coordinated by the responsible biostatistician of Astellas Pharma Global Development, Inc. (APGD). Any changes from the analyses planned in the SAP will be justified in the Clinical Study Report (CSR).

Prior to database hard lock, a final review of data and Tables Listings and Figures (TLFs) meeting will be held to allow a review of the clinical trial data and to verify the data that will be used for analysis set classification. If required, consequences for the statistical analysis will be discussed and documented. A meeting to determine analysis set classifications may also be held prior to database hard lock.

Pharmacokinetic (PK) analyses will be described in a separate data analysis plan (PKDAP) which will be finalized prior to the analysis commencement and will be reported separately.

A SAP for the Data and Safety Monitoring Board (DSMB) will also be provided separately and finalized prior to FSI. If needed, revisions to the approved DSMB SAP may be made prior to the database hard lock. Revisions will be version controlled.

### 2 FLOW CHART AND VISIT SCHEDULE

### **Flow Chart**

| | Study Period<br>(56 weeks) | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| 1 | Pretreatment Period<br>(4 weeks) | l | | Effica | Long-term Safety Period ‡<br>(28 weeks) | | | | |
| Visit 1 | Visit 2/TC 1 | Visit 3 | Visit 4/TC 2<br>Week 2 | Visit 5<br>Week 4 | Visit 6/TC 3<br>Week 8 | Visit 7<br>Week 12 | Visit 8<br>Week 24 | Visit 9/TC 4<br>Week 36 | Visit 10/EOS<br>Week 52 |
| Screening | Group A & B §:<br>Review of 2-day<br>e-diary<br>Group B:<br>Start washout on<br>day -15 | Baseline | 1 <sup>st</sup> up-titration<br>possibility | 2 <sup>nd</sup> up-titration<br>possibility | 3 <sup>rd</sup> up-titration<br>possibility | Fixed dose | Fixed dose | Fixed dose | End of Study |

TC: telephone contact; EOS: end of study

<sup>†</sup> The efficacy treatment period begins with the first dose, the day after baseline measurements on visit 3/baseline.

<sup>‡</sup> The long-term safety period begins immediately after visit 8/week 24.

<sup>§</sup> Group A: Subjects who are currently not receiving any prohibited medication including any oral drug treatment to manage their NDO, or when botulinum toxin is no longer considered effective. Group B: Subjects who currently are receiving oral drug treatment to manage their NDO or receive any other prohibited medication.

Table 1 Schedule of Assessments

| | Visit 1 | Visit 2 /TC 1 | Visit 3 | Visit 4<br>/TC 2 <sup>†</sup> | Visit 5 | Visit 6<br>/TC 3 † | Visit 7 | Visit 8 | Visit 9<br>/TC 4 <sup>†</sup> | Visit 10<br>/EOS <sup>‡</sup> |
|---|---|---|---|---|---|---|---|---|---|---|
| Assessments | Screening | Start of<br>Washout ††† | Baseline | Week 2 | Week 4 | Week 8 | Week 12 | Week 24 | Week 36 | Week 52 |
| | Day -28 to<br>Day -15 | Day -15 to<br>Day -8 | Day -1 | Day 14<br>(+3 days) | Day 28<br>(+3 days) | Day 56<br>(±7 days) | Day 84<br>(±7 days) | Day 168<br>(±7 days) | Day 252<br>(±14 days) | Day 364<br>(±14 days) |
| Signing informed consent form | X | | | | | | | | | |
| Inclusion/Exclusion criteria | X | | X | | | | | | | |
| Demographics | X | | | | | | | | | |
| Height & weight | X | | X | | | | | X | | X |
| Medical history (including NDO) | X | | | | | | | | | |
| Current NDO medications | X | X | | | | | | | | |
| Vital signs (triplicate) and body temperature (ear) § | Х | | x | | x | | x | х | | x |
| Physical examination | X | | | | | | | | | X |
| 12-lead ECG (triplicate) ¶ | X | | X | | X | | X | X | | X |
| Hematology/Biochemistry/eGFR | X | | (X) <sup>††</sup> | | | | X | | | X |
| Urinalysis | X | | X | | X | | X | X | | X |
| Pregnancy test <sup>‡‡</sup> | X | | X | | X | | X | X | | X |
| Pharmacokinetics §§ | | | | | (X) | (X) | (X) | (X) | (X) | (X) |
| Upper urinary tract ultrasound | | | X | | | | | | | X |
| Urodynamic assessments ¶ | | | X | | X | | | X | | |
| Dose-titration assessment | | | | X | X | X | | | | |
| Dispense study drug ††† | | | X | | X | | X | X | (X) | |
| Bladder diary and collection of catheterized volume <sup>‡‡‡</sup> | | X | X | X | X | Х | X | Х | X | Х |
| SBPM (triplicate) §§§ | | X | X | X | X | X | X | X | X | X |
| PIN-Q, PGI-S | | | X | | | | | X | | X |
| CGI-C | | | | | | | | X | | X |
| Acceptability questionnaires | | | | | X | | | X | | X |
| Adverse events and previous and | | | | | | | | | | |
| concomitant medication | | • | | | | | | | | _ |

ECG: Electrocardiogram; EOS: end of study; CGI-C: Clinician Global Impression of Change scale; NDO: neurogenic detrusor overactivity; PGI-S: Patient Global Impression of Severity Scale; PIN-Q: Pediatric Incontinence Questionnaire; SBPM: self blood pressure measurement; TC: telephone contact.

See Footnotes on next page

# **Sponsor: Astellas Pharma Global Development, Inc.** ISN/Protocol 178-CL-206A

- † For the visits where a TC is indicated there is no need for the subject to visit the clinic, provided that the e-diary data is reviewed by the investigator prior to the TC and discussed and confirmed with the subject or the subject's parent(s)/caregiver(s) during the TC.
- Subjects who withdraw early from the study after having received study drug should complete the EOS visit. If the final dose is reached before the last possibility for up-titration at 8 weeks, the fixed-dose treatment period will be extended to keep the entire treatment period 364 days as a minimum. The maximum is 378 days in order to allow for visit windows.
- Triplicate vital signs with an interval of approximately 2 minutes in the sitting position (when possible, otherwise supine, but always in the same position). Preferably the right arm should be used. Subject should have been calm and without distress for at least 5 minutes. Clinic measurements will be used to assess eligibility. Single measurements for body temperature must be performed with an ear thermometer.
- Triplicate 12-lead ECG with an interval of about 30 seconds to 5 minutes in the supine position (when possible, but always in the same position). Subject should have been calm and without distress for at least 5 minutes.
- †† Additional hematology/biochemistry taken at baseline only if an AE related to hematology/biochemistry parameters occurred between visit 1/screening and visit 3/baseline. The first group of subjects (minimum of 5, maximum of 10) who reach study visit 5/week 4 will have an additional blood draw for a DSMB-mandated interim safety check at this visit. For sampling, preferably the left arm should be used. Blood sampling should occur after vital signs and ECG measurements.
- ‡‡ Pregnancy test in female subjects of childbearing potential in serum (if blood is drawn) or urine (at other visits).
- A total of 4 pharmacokinetic samples will be collected, divided over 2 sampling days. Sampling day 1: 1 trough sample; Sampling day 2: 1 trough and 2 post-dose samples between 2 h and 5 h post-dose, with at least 1 hour in between the samples. These 2 sampling days do not have to be in a specific order and can be selected from the given options. To allow for an early assessment of the dose-response relationship by the DSMB, it is preferred the pharmacokinetic sampling takes place as early in the study as possible. Dosing on a sampling day with post-dose samples must occur within 1 hour after completion of breakfast [Protocol Section 5.3.4]. On days where a pharmacokinetic visit is planned in the clinic, breakfast and dosing should occur in the clinic. Blood sampling should occur after vital signs and ECG measurements.
- Mandatory at visit 3/baseline, visit 5/week 4 and visit 8/week 24. When the urodynamic trace is believed not to be in accordance with the subject's clinical condition, it is allowed to repeat the urodynamic assessment once. Additional urodynamic assessments at other visits may be performed if deemed necessary by the Investigator
- ††† Daily study drug administration will begin on Day 1 (the day after visit 3/baseline). Due to shelf-life limitations, an additional dispensing visit is foreseen at visit 9/week 36 for subjects receiving mirabegron oral suspension. This dispensing visit does not need to be accompanied by the subject.
- After a successful screening visit, all subjects start with the completion of a 2-day weekend e-diary visit to get acquainted with the e-diary and the assessments. Completion of this diary should start in the weekend prior to visit 2. Completion of subsequent bladder diaries should start approximately 7 days prior to the indicated visit (or TC). If successful completion of the 2-day weekend e-diary is confirmed at visit 2, subjects from group A start with collection of the 7-day baseline e-diary, followed by the baseline visit. Subjects in group B start with a 14-day washout. In the second week of the washout period, collection of their 7-day baseline e-diary starts, followed by the baseline visit.
- Triplicate SBPM will be performed in the morning and evening during the 2-day weekend e-diary collection period and on 2 consecutive days at around 1 and 2 weeks after start of dosing with PED25 (day 1) and after up-titration to PED50, if not already covered by the scheduled SBPM. Measurements to be taken with an interval of approximately 2 minutes in the sitting position (when possible, otherwise supine, but always in the same position). Preferably the right arm should be used. Morning measurements should be taken after waking-up, before breakfast and before study drug intake, evening measurements prior to bedtime. Subject should have been calm and without distress for at least 5 minutes.

## 3 STUDY OBJECTIVE(S) AND DESIGN

# 3.1 Study Objective(s)

### 3.1.1 Primary Objectives

• To evaluate the efficacy of mirabegron after multiple-dose administration in the pediatric population.

### 3.1.2 Secondary Objectives

- To evaluate the safety and tolerability of mirabegron after multiple-dose administration in the pediatric population.
- To evaluate the pharmacokinetics of mirabegron after multiple-dose administration in the pediatric population.

## 3.2 Study Design

This is a phase 3, open-label, baseline-controlled, multicenter study in male and female children and adolescents aged 3 to less than 18 years of age with NDO on CIC. Approximately 50 enrolling study centers in Europe, Latin America, Africa, Middle East, and Asia-Pacific are planned. At least 44 evaluable subjects (estimate of 63 enrolled), with at least 10 subjects from each age group (children aged 3 to less than 12 years of age; adolescents aged 12 to less than 18 years of age) are planned.

The study consists of 3 periods:

- Pretreatment period: for a maximum of 28 days before baseline, including screening (visit 1), washout (if applicable) (visit 2) and baseline (visit 3)
- Efficacy treatment period: beginning the day after baseline and continuing to visit 8/week 24
- Long-term safety period: beginning after visit 8/week 24 and continuing to visit 10/week 52 (end of study [EOS]), or to the end of treatment (EOT).

### Pretreatment Period: From screening (visit 1) to baseline (visit 3)

After informed consent and visit 1/screening, subjects are grouped according to their current NDO therapy and/or other medication:

- Group A: Subjects who are currently not receiving any prohibited medication including any oral drug treatment to manage their NDO, or when botulinum toxin is no longer considered effective.
- Group B: Subjects who currently are receiving oral drug treatment to manage their NDO or receive any other prohibited medication.

After the screening visit, a 2-day weekend e-diary has to be completed by the subjects to get acquainted with the e-diary and the home assessments:

• Group A: Following successful completion of the first 2-day weekend e-diary, confirmed at visit 2, the subjects will start to complete the 7-day baseline e-diary followed by visit 3/baseline.

• Group B: Following successful completion of the first 2-day weekend e-diary, confirmed at visit 2, the subjects will start their 2-week washout period. In the second week of their washout period, they will complete the 7-day baseline e-diary followed by visit 3/baseline.

If a subject is suffering from a symptomatic urinary tract infection (UTI) at visit 1/screening or is diagnosed with one between visit 1/screening and visit 3/baseline, the UTI should be treated successfully (clinical recovery) prior to baseline. If a symptomatic UTI is present at or just before visit 3/baseline, all baseline assessments should be postponed with a maximum of 7 days until the UTI is successfully treated (clinical recovery). The 7-day baseline e-diary does not have to be repeated if at least the 2-day weekend e-diary and 1 day of the weekday e-diary were completed while the subject did not suffer from a symptomatic UTI.

Subjects will enter the efficacy treatment period if they meet the eligibility criteria and satisfactorily complete the pretreatment period (ability to complete bladder e-diary, catheterized volumes, questionnaires and self blood pressure measurement [SBPM]).

# Efficacy Treatment Period: From the first dose the day after baseline measurements visit 3/baseline to visit 8/week 24

Study drug administration will begin the day after the baseline visit (i.e., on day 1). The initial dose of mirabegron will be based on the subject's weight and is predicted to achieve plasma concentrations equivalent to the steady state exposures expected with 25 mg mirabegron administered once daily in adults (PED25).

At visit 4/week 2, visit 5/week 4 and visit 6/week 8, subjects are expected to be up-titrated to the pediatric equivalent dose of 50 mg in adults (PED50), unless:

- The investigator considers the subject to be effectively treated with PED25, based on urodynamics and e-diary;
- 2. There are safety or tolerability issues with PED25.

Dose down-titration to PED25 can be performed at any time if there is a safety issue.

If a subject is suffering from a symptomatic UTI in the week prior to any (un)scheduled urodynamic investigation (e.g., visit 5/week 4, visit 8/week 24), the UTI should be treated successfully first (clinical recovery). To allow for treatment of the UTI, these visits may be postponed with an additional maximum of 7 days on top of the already existing visit window. The 7-day e-diary does not have to be repeated if at least the 2-day weekend e-diary and 1 day of the weekday e-diary were completed while the subject did not suffer from a symptomatic UTI.

If a subject suffers from a symptomatic UTI in the week prior to any other study visit, these visits do not need to be postponed and the 7-day e-diary does not have to be repeated.

### Long-term Safety Period: From visit 8/week 24 to visit 10/week 52 (EOT or EOT)

For long-term safety evaluation, following visit 8/week 24, subjects will stay on their individual dose level until visit 10/week 52 (EOT/EOS).

# 3.3 Assignment and Allocation

No randomization is performed for the study and all subjects will receive active mirabegron treatment (open-label).

Subject number assignment will be coordinated centrally by using an interactive response system. Subjects will be assigned a subject number at study entry. The full subject number will consist of 10 digits: 5 for the site number (provided by the Sponsor) and 5 for the consecutive subject number.

An enrolled subject who withdraws or discontinues before dosing will be considered a screening failure and will be replaced. If a subject discontinues treatment after dosing, this subject will be replaced at the discretion of the Sponsor.

### 4 SAMPLE SIZE

The primary endpoint will be the change from baseline in maximum cystometric capacity (MCC) after 24 weeks of mirabegron treatment. There are data from previous studies that indicate the effect size that can be expected as a result of the treatment with mirabegron. Franco et al. (2005) analyzed 2 age groups (1 to 5 years, and 6 to 15 years) and reported mean (SD) MCC changes from baseline of 71.5 (88) mL and 75.4 (102.7) mL respectively after 24 weeks treatment with oxybutynin. Goessl et al. (2000) reported an increase of 52.8 mL after 3 months treatment with tolterodine. Cartwright et al. (2009) reported an increase of 98 mL after 14 weeks treatment with oxybutynin and a corresponding SD of 87 mL.

A study with 44 evaluable subjects who have valid (as by the central reviewer's assessment) nonmissing MCC measurements at treatment week 24 and at baseline would have a 90 percent power to detect a statistical significant change from baseline, if the real change from baseline in the subject population is at least 52 mL and the real SD for change from baseline is  $\leq 103$  mL. The power calculation was done assuming a paired t-test with 2-sided significance level of 0.05.

Assuming 30% of enrolled subjects will discontinue or will not be evaluable for the primary endpoint, a total of approximately 63 subjects may need to be enrolled so that 44 subjects are evaluable in total.

These sample size considerations should allow sufficient precision for the assessment of the primary objective in this nonrandomized pediatric trial.

Detailed criteria for analysis sets will be laid out in Classification Specifications and the allocation of subjects to analysis sets will be determined prior to database hard-lock.

### 5 ANALYSIS SETS

In accordance with International Conference on Harmonization (ICH) recommendations in guidelines E3 and E9, the following analysis sets will be used for the analyses.

Detailed criteria for analysis sets will be laid out in Classification Specifications (CS) and the allocation of subjects to analysis sets will be determined prior to database hard lock.

### 5.1 All Screened Set

The All Screened Set will consist of all subjects for whom a valid informed consent/assent is available, as per applicable local law.

Three signatures might be available from the informed consent/assent. For calculations using the date of informed consent/assent the last available date will be used.

The All Screened Set will be used to summarize disposition of subjects who were screened.

### 5.2 All Allocated Set

The All Allocated Set will consist of all allocated subjects, i.e. all those subjects with a non-missing registration date at visit 3 (baseline).

This set will be used to summarize disposition of subjects who were allocated to mirabegron treatment.

### 5.3 Full Analysis Set (FAS)

The full analysis set (FAS) will consist of all subjects who:

- Took at least 1 dose of study drug, and
- Had a valid (as by the central reviewer's assessment) nonmissing MCC measurement at baseline and at a post-baseline visit for the primary efficacy endpoint.

The final selection of subjects for the FAS will be confirmed in the Analysis Set Classification Meeting (ASCM) based upon a review of all the pertinent data.

The FAS will be used for primary analyses of efficacy data, for sensitivity and subgroup analyses [Sections 7.4.1.2.5] and 7.8] and for summaries of some demographic and baseline characteristics.

# 5.4 Per Protocol Set (PPS)

The per protocol set (PPS) includes all subjects of the FAS who fulfill the protocol in terms of their eligibility, interventions and outcome assessments, and for whom valid MCC measurements at visit 3/baseline and at visit 8/week 24 are reported.

The list of the protocol deviations that may result in a subject in the FAS being excluded from the PPS is provided below (Section 5.4.1). The final selection of subjects for the PPS will be confirmed in the ASCM based upon a review of all the pertinent data.

The PPS will be used for secondary analyses of efficacy data. Also, selected demographic and baseline characteristics may also be summarized for the PPS.

### 5.4.1 Reasons for Exclusion From PPS

A subject may be excluded from the PPS if there has been a deviation from the protocol sufficient to affect the assessment of the efficacy of the study drug. Such deviations may include (but are not limited to) reasons why a subject was ineligible to have been included in the study, whether there were interventions that were prohibited by the protocol, or whether the subject did not adhere adequately to the study treatment or outcome assessments.

There will be no partial exclusion (e.g. of particular timepoints only) of a subject from the PPS; all of a subject's data will be excluded.

Some reasons for exclusion of a subject from the PPS are given below; however the final decision on whether or not a particular protocol deviation (see Section 7.2.2) requires the exclusion of a subject will be confirmed at the ASCM with all reasons for the decision documented in the meeting minutes.

### **Eligibility Deviations**

The inclusion and exclusion criteria for the study are detailed in Appendix 1: Inclusion and Exclusion Criteria These are all assessed at Visit 1/screening and Visit 3/baseline.

A subject will be excluded from the PPS if:

- Any of inclusion criteria 4 or 5 are not met.
- Any of exclusion criteria 1, 3, 4, 5, 6, 7, 8, 17, or 18 are met.

Violations of other inclusion and exclusion criteria may also result in exclusion of the PPS if it is considered that there is a risk that the violation affects the assessment of the efficacy of the study drug. All such violations will be considered on an individual basis at the ASCM.

#### NDO not confirmed

A subject will be excluded from the PPS if NDO cannot be confirmed by the expert review of the urodynamic traces recorded at visit 3/baseline, whether or not it is recorded that inclusion criterion 4 has been met. However, the decision for inclusion/exclusion of the subject from the PPS will be part of the Central Review Committee Data.

### **Prohibited medications**

A subject will be excluded from the PPS if he/she received prohibited medications from start of wash-out period (visit 2) to baseline and from visit 7 to visit 8. Except for Botox which is not allowed if taken from <4 months before screening and/or during the whole study period. These include, but are not limited to, the following (see Appendix 2 for a more complete list):

### Prohibited medications:

- Any medication, other than the study drug, used for the management of NDO;
- Any drugs that are sensitive cytochrome (CYP) 2D6 substrates with a narrow therapeutic index or sensitive P-glycoprotein (P-gp) substrates
- Any strong cytochrome P450 (CYP) 3A4 inhibitors if the subject has a mild to moderate renal impairment (eGFR 30 – 89 mL/min).

### Compliance to study medication

A subject will be excluded from the PPS for either of the reasons below based on compliance to the study medication (see Section 6.5.4 for details on the calculation of the compliance rate between study visits):

- Treatment stopped before the primary endpoint has been reached (MCC at visit 8/week 24);
- Treatment compliance of less than 80% between visit 7/week 12 and visit 8/week 24.

All evidence and reasons for determining a violation based on compliance to the study medication will be documented in the minutes of the ASCM.

### Missing primary efficacy endpoint

A subject will be excluded from the PPS if he/she does not have a valid baseline (visit 3) value and a valid visit 8 value (based on the week 24 efficacy visit windows [Day 99 to Day 237]— see Section 7.11.3] and not imputed from earlier weeks) of the primary efficacy variable (MCC).

### **Development of discontinuation criteria**

A subject may be excluded from PPS if they developed discontinuation criteria prior to visit 8/week 24 but were not withdrawn from the study. The decision for inclusion/exclusion of the subject from the PPS will be determined at the ASCM and documented in the minutes of this meeting.

# 5.5 Safety Analysis Set (SAF)

The safety analysis set (SAF) will consist of all subjects who took at least 1 dose of study drug.

The SAF will be used for summaries of demographic and baseline characteristics and all safety and tolerability related variables.

# 5.6 Pharmacokinetics Analysis Set (PKAS)

The Pharmacokinetics Analysis Set (PKAS) consists of the subset of subjects of the SAF for whom plasma concentration data are available to facilitate derivation of at least one PK parameter and for whom the time of last dose prior to sampling is known.

Additional subjects may be excluded from the PKAS at the discretion of the Global Clinical Modeling & Simulation Lead (GCMSL). Any formal definitions for exclusion of subjects or time-points from the PKAS will be documented in the Classification Specifications.

Since the actual bioanalytical results may only become available after the data review meeting, additional data points may be excluded at the time of pharmacokinetic analysis at the discretion of the GCMSL. These data points will be reported in the modeling report.

The PKAS is used for all tables and graphical summaries of the PK data.

# 5.7 Pharmacodynamic Analysis Set (PDAS)

The PDAS is not defined for this study.

### **6** ANALYSIS VARIABLES

## 6.1 Efficacy Endpoints

### **Urodynamic assessments:**

Urodynamic assessments will be performed at visit 3/baseline, visit 5/week 4, and visit 8/week 24. Additional urodynamic assessments can be performed at e.g. visit 10/week 52 (EOT/EOS), or at any other time point when deemed necessary by the investigator.

The following parameters will be determined:

- MCC at end of filling (mL)
- Bladder compliance
- Filling volume until first detrusor contraction (> 15 cm H<sub>2</sub>O)
- Filling volume at 20 cm, 30 cm and 40 cm H<sub>2</sub>O detrusor pressure (if reached)
- Number of overactive detrusor contractions (>15 cm H<sub>2</sub>O) until end of filling
- Detrusor pressure at end of filling
- MCC expressed as percentage of Expected Bladder Capacity (EBC)

Except for Bladder compliance and MCC expressed as % of EBC, the results of the urodynamic assessments will be entered in the eCRF. Bladder compliance will be calculated by external experts and will be obtained from an external database. MCC expressed as % of EBC will be calculated using EBC = 24.5 x age(years) + 62 (Palmer et al, 1997).

### **Bladder diary:**

The bladder diary is part of the subject's e-diary. After a successful visit 1/screening, all subjects should start with the completion of a 2-day weekend e-diary visit to get acquainted with the e-diary and the assessments. Completion of this diary should start in the weekend prior to visit 2.

The e-diary data is reviewed by the investigator prior to the start of visit 3 and discussed and confirmed with the subject or parent(s)/caregiver(s) during the (telephone) visit. If the investigator is under the impression that the subject and/or parent(s)/caregiver(s) can perform all the required assessments and are able to complete all required forms with credible data, completion is considered successful.

If completion is not considered successful, the investigator should counsel/re-train the subject or parent(s)/ caregiver(s) prior to the start of the 7-day baseline e-diary. In case the subject and/or parent(s)/caregiver(s) are still not able to complete the 7-day baseline e-diary satisfactorily, the subject should be excluded from further participation in the study.

If successful completion of the 2-day weekend e-diary is confirmed at visit 2:

- Subjects from group A start with collection of the 7-day baseline e-diary, followed by visit 3/baseline.
- Subjects in group B start with a 14-day washout. In the second week of the washout period collection of their 7-day baseline e-diary starts, followed by visit 3/baseline.

Subsequent bladder diaries will be completed by the subject or the subject's parent/caregiver in the week prior to visit 4/week 2, visit 5/week 4, visit 6/week 8, visit 7/week 12, visit 8/week 24, visit 9/week 36 and visit 10/week 52 (EOT/EOS). Completion of 7-day bladder diaries should start approximately 7 days prior to the indicated visit (or telephone contact).

The following information will be collected in the bladder diary:

Daily during the 7-day period:

- Time of CICs
- Presence of leakage between CICs
- Sleep time and wake-up time

On 2 consecutive weekend days within the 7-day period (weekend e-diary):

- Catheterized volume
- Grade of leakage between CICs
- Weight of diaper/pad (visit 3/baseline and visit 8/week 24)
- Number of Leakages between CICs
- Position of measure
- Urine weight

Results will be directly entered by the subject or subject's parent(s)/caregiver(s) in the ediary.

### **Questionnaires:**

The following questionnaires will be used:

- The PIN-Q [Appendix 4.1] will be completed on one weekend day preceding visit 3/baseline, visit 8/week 24 and visit 10/week 52 (EOT/EOS).
- The PGI-S [Appendix 4.2] will be completed on one weekend day preceding visit 3/baseline, visit 8/week 24 and visit 10/week 52 (EOT/EOS).
- The Acceptability Questionnaires [Appendix 4.3 and Appendix 4.4] will be completed on one weekend day preceding visit 5/week 4, visit 8/week 24 and visit 10/week 52 (EOT/EOS).
- The CGI-C [Appendix 4.5] will be completed at visit 8/week 24 and at visit 10/week 52 (EOT/EOS).

The PIN-Q with a Likert scale adopted for 20 measures is used. Questionnaires (i.e., PIN-Q, PGI-S and the Acceptability Questionnaires) will be provided via the e-diary. Results will be directly entered in the e-diary by the subject or subject's parent/caregiver. The CGI-C will be completed by the investigator and the results will be entered in the eCRF.

The primary and secondary variables will be calculated based on the following:

- <u>Valid</u> urodynamic assessments made at visit 3/baseline, visit 5/week 4 and visit 8/week 24,
- Diary data collected at each visit from Visit 3 to Visit 10/EOS. Only <u>valid diary days</u> from week end diary and/or week day diary as appropriate will be used.
- Quality of Life data (<u>valid PIN-Q</u> and PGI-S questionnaires) collected at Visits 3, 8 and 10/EOS (baseline, week 24, and week 52 respectively),
- Clinician reported Questionnaire (valid CGI-C) collected at Visit 8/Week 24 and Visit 10/Week 52).

A valid urodynamic assessment is an urodynamic assessment confirmed to be valid by central reviewers.

A valid bladder diary day in the <u>weekday diary</u> is any e-diary day for which at least 1 catheterization with complete date and time is recorded.

A valid bladder diary day in the <u>weekend diary</u> is any e-diary day for which at least one catheterized volume greater than 0 mL and complete date and time is recorded. See section 6.1.3.2 for calculating catheterized volume.

A valid PIN-Q questionnaire is a questionnaire with answers to at least 18 of the 20 individual items used to create the total score. A PGI-S questionnaire is considered valid when subject answer to the question "How did you feel about your bladder condition during the past 3 days?"

A CGI-C is considered valid when the physician rates the change in the subject's overall bladder symptoms.

Analysis windows will be used, as described in section 7.11.3

The efficacy endpoints are described in Table 2

A summary of the efficacy endpoints is presented in Table 3

ISN/Protocol 178-CL-206A

Table 2 **Efficacy Endpoints** 

| Endpoint | Endpoint Description |
|---|---|
| Number | * * |
| Primary Efficacy E | Endpoint based on Urodynamic Measures |
| 1 Change from baseline in MCC at visit 8/week 24 | |
| Secondary Efficacy Endpoints based on Urodynamic Measures | |
| 2 | Change from baseline in MCC at visit 5/week 4 |
| 3,4 Change from baseline in Bladder compliance $(\Delta V/\Delta P)$ at visit 5/w | |
| | and visit 8/week 24 |
| 5,6 | Change from baseline in number of overactive detrusor contractions |
| | (> 15 cm H <sub>2</sub> O) until end of filling at visit5/week 4 and visit 8/week 24 |
| 7,8 | Change from baseline in detrusor pressure at end of filling at visit 5/week |
| | 4 and visit 8/week 24 |
| 9,10 | Change from baseline in filling volume until first overactive detrusor |
| | contraction (> 15 cm H <sub>2</sub> O) at visit 5/week 4 and visit 8/week 24 |
| Secondary Efficacy | Endpoints: Bladder Volume and Leakage Measures based on 7-day diary |
| 11 | Change from baseline at visit 4/week 2, visit 5/week 4, visit 6/week 8, |
| | visit 7/week 12, visit 8/week 24, visit 9/week 36 and visit 10/week 52 |
| | (EOT/EOS) in average catheterized volume per catheterization |
| 12 | Change from baseline at visit 4/week 2, visit 5/week 4, visit 6/week 8, |
| | visit 7/week 12, visit 8/week 24, visit 9/week 36 and visit 10/week 52 |
| | (EOT/EOS) in maximum catheterized volume |
| 13 | Change from baseline at visit 4/week 2, visit 5/week 4, visit 6/week 8, |
| | visit 7/week 12, visit 8/week 24, visit 9/week 36 and visit 10/week 52 |
| | (EOT/EOS) in maximum catheterized daytime volume |
| 14 | Change from baseline at visit 4/week 2, visit 5/week 4, visit 6/week 8, |
| | visit 7/week 12, visit 8/week 24, visit 9/week 36 and visit 10/week 52 |
| | (EOT/EOS)) in average morning catheterized volume (based on first |
| 1.5 | catheterization after subject woke up) |
| 15 | Change from baseline at visit 4/week 2, visit 5/week 4, visit 6/week 8, |
| | visit 7/week 12, visit 8/week 24, visit 9/week 36 and visit 10/week 52 |
| | (EOT/EOS) in mean number of leakage episodes per day (day and night |
| 17 | time) Charge from baseling at visit 4/week 2 visit 5/week 4 visit 6/week 9 |
| 16 | Change from baseline at visit 4/week 2, visit 5/week 4, visit 6/week 8, |
| | visit 7/week 12, visit 8/week 24, visit 9/week 36 and visit 10/week 52 |
| | (EOT/EOS) in number of dry (leakage-free) days/7 days (day and night |
| Table continued a | time) |
| Table continued or | ri nexi page |

| Endpoint | Endpoint Description |
|---|---|
| Number | |
| Secondary Efficacy Endpoints: Subject- or Clinician reported Questionnaire Endpoints | |
| 17, 18 | Change from baseline at visit 8/week 24 and visit 10/week 52 |
| | (EOT/EOS) in PIN-Q |
| 19, 20 | Change from baseline at visit 8/week 24 and visit 10/week 52 |
| | (EOT/EOS) in PGI-S |
| 21, 22 | Clinician Global Impression of Change (CGI-C) at visit 8/week 24 and visit 10/week 52 (EOT/EOS) |
| 23, 24, 25 | Acceptability at visit 5/week 4, visit 8/week 24 and visit 10/week 52 (EOT/EOS) |
| <b>Exploratory Effica</b> | cy Endpoints based on Urodynamic Measures |
| 26, 27 | Change from baseline at visit 5/week 4 and visit 8/week 24 in filling |
| ŕ | volume at 20 cm, 30 cm and at 40 cm H <sub>2</sub> O detrusor pressure, given that |
| | those pressures are reached during the examination |
| 28, 29 | Change from baseline at visit 5/week 4 and visit 8/week 24 in MCC |
| 20, 25 | expressed as percentage of EBC |
| Exploratory Effica | cy Endpoints based on 7-day diary |
| 30 | Change from baseline at visit 4/week 2, visit 5/week 4, visit 6/week 8, |
| 30 | visit 7/week 12, visit 8/week 24, visit 9/week 36 and visit 10/week 52 |
| | (EOT/EOS) in mean grade of leakage |
| 31 | Change from baseline at visit 4/week 2, visit 5/week 4, visit 6/week 8, |
| J1 | visit 7/week 12, visit 8/week 24, visit 9/week 36 and visit 10/week 52 |
| | (EOT/EOS) in total catheterized volume per day |
| 32 | |
| 32 | Change from baseline at visit 4/week 2, visit 5/week 4, visit 6/week 8, |
| | visit 7/week 12, visit 8/week 24, visit 9/week 36 and visit 10/week 52 |
| 22 | (EOT/EOS) in number of CICs/day |
| 33 | Shift from baseline at visit 4/week 2, visit 5/week 4, visit 6/week 8, |
| | visit 7/week 12, visit 8/week 24, visit 9/week 36 and visit 10/week 52 |
| | (EOT/EOS) in Responder with respect to leakage (complete responder, |
| 2.4 | partial responder, non-responder) |
| 34 | For subjects with no leakage during the sleeping time: Change from |
| | baseline at visit 4/week 2, visit 5/week 4, visit 6/week 8, visit 7/week 12, |
| | visit 8/week 24, visit 9/week 36 and visit 10/week 52 (EOT/EOS) in |
| | average morning catheterized volume (based on first catheterization after |
| | subject woke up) |
| 35 | For subjects with leakage during the sleeping time: Change from baseline |
| | at visit 4/week 2, visit 5/week 4, visit 6/week 8, visit 7/week 12, visit |
| | 8/week 24, visit 9/week 36 and visit 10/week 52 (EOT/EOS) in average |
| | morning catheterized volume (based on first catheterization after subject |
| | woke up) |
| 36 | Change from baseline at visit 4/week 2, visit 5/week 4, visit 6/week 8, |
| | visit 7/week 12, visit 8/week 24, visit 9/week 36 and visit 10/week 52 |
| | (EOT/EOS) in percentage of catheterizations without intermittent leakage |
| | accident |

**Table 3 Summary of Efficacy Endpoints** 

| Variable | Outcome | Endpoints | | | | | | |
|---|---|---|---|---|---|---|---|---|
| | | Visit 4/ | Visit 5/ | Visit 6/ | Visit 7/ | Visit 8/ | Visit 9/ | Visit 10/ |
| | | week 2 | week 4 | week 8 | week 12 | week 24 | week 36 | week 52 (EOT/EOS) |
| Primary and secondary urodynamic | | | | | | | | |
| endpoints: | | | | | | | | |
| MCC | Change from baseline | | 2 | | | 1 | | |
| Bladder compliance | Change from baseline | | 3 | | | 4 | | |
| NODC* | Change from baseline | | 5 | | | 6 | | |
| Detrusor pressure | Change from baseline | | 7 | | | 8 | | |
| Filling volume | Change from baseline | | 9 | | | 10 | | |
| Secondary bladder volume and leakage | | | | | | | | |
| measures endpoints (7-day diary) | | | | | | | | |
| Average CV <sup>£</sup> | Change from baseline | 11 | | | | | | |
| Maximum CV <sup>£</sup> per day | Change from baseline | 12 | | | | | | |
| Maximum CV <sup>£</sup> (daytime) | Change from baseline | 13 | | | | | | |
| Average CV <sup>£</sup> (morning) | Change from baseline | 14 | | | | | | |
| Mean NLE <sup>&amp;</sup> per day (day and night time) | Change from baseline | 15 | | | | | | |
| Number of dry <sup>\$</sup> days/7 days (day and night | Change from baseline | 16 | | | | | | |
| time) | | | | | | | | |
| , | | | | | | | | |
| Secondary questionnaire endpoints | | | | | | | | |
| PIN-Q | Change from baseline | | | | | 17 | | 18 |
| PGI-S | Change from baseline | | | | | 19 | | 20 |
| CGI-C | N (%) | | | | | 21 | | 22 |
| Acceptability (tablets and oral suspension) | N (%) | | 23 | | | 24 | | 25 |
| Exploratory urodynamic and 7-day diary | | | | | | | | |
| endpoints | | | | | | | | |
| Filling volume (20, 30 and 40 cm H <sub>2</sub> O) | Change from baseline | | 26 | | | 27 | | |
| Table continued on next page | | | | | | | | |

# **Sponsor: Astellas Pharma Global Development, Inc.** ISN/Protocol 178-CL-206A

| Variable | Outcome | Endpoints | | | | | | |
|---|---|---|---|---|---|---|---|---|
| | | Visit 4/ | Visit 5/ | Visit 6/ | Visit 7/ | Visit 8/ | Visit 9/ | Visit 10/ |
| | | week 2 | week 4 | week 8 | week 12 | week 24 | week 36 | week 52 (EOT/EOS) |
| MCC expressed as % of EBC | Change from baseline | | 28 | | | 29 | | |
| Mean Grade of leakage | N(%) | 30 | | | | | | |
| Total CV <sup>£</sup> per 24 h | Change from baseline | 31 | | | | | | |
| No of CICs/day | Change from baseline | 32 | | | | | | |
| Responder with respect to leakage | Shift from baseline 33 | | | | | | | |
| Subjects with no leakage during the sleeping | | | | | | | | |
| time: Average CV <sup>£</sup> (morning) | By Visit 34 | | | | | | | |
| Subjects with leakage during the sleeping time: | | | | | | | | |
| Average CV <sup>£</sup> (morning) | By Visit 35 | | | | | | | |
| Reduction in percentage of Catheterizations | | | | | | | | |
| without intermittent leakage accident | Shift from Baseline 36 | | | | | | | |

<sup>\*</sup>Number of Overactive Detrusor Contractions (NODC); <sup>£</sup> Catheterized Volume (CV); <sup>&</sup> Number of Leakage Episodes (NLE), <sup>\$</sup> Leakage free

### 6.1.1 Primary Efficacy Endpoint

The primary efficacy endpoint will be the change from baseline in MCC at visit 8/week 24 (based on filling urodynamics).

### 6.1.1.1 Maximum Cystometric Capacity (MCC)

MCC (mL) is recorded in the "VOLUME" section of the "Urodynamic Testing" pages of the eCRF under "Volume at the end of filling".

Baseline MCC is the MCC recorded at the baseline visit. The change from baseline at visit 8/week 24 in MCC is the MCC at the week 24 visit minus the baseline MCC.

For the primary analysis no imputation of missing data will be performed, ie, only non-missing (week 24) data will be used for analysis.

In addition, MCC will be calculated using the last observation carried forward (LOCF) method (see section 7.11.1): ie, the latest available post-baseline value from before week 24 will be carried forward and used for analysis. To calculate the change from baseline, the baseline MCC must be available and at least the visit 5/week 4 MCC, any unscheduled visit MCC before week 24, or the visit 8/week 24 MCC, else the primary efficacy variable is missing. Missing values at visit 8/week 24 will be imputed from previous post-baseline values using the last observation carried forward (LOCF) method (see section 7.11.1).

In addition, the MCC will also be calculated without using the LOCF technique, ie., only non-missing data will be used for analysis.

### 6.1.2 Primary Estimand

The estimand of most clinical importance, following a hypothetical strategy, for this study is defined by the following 4 attributes:

- Target population: all subjects who took at least 1 dose of the study drug, and in whom a
  valid non-missing MCC measurement at baseline and after administration of the study
  drug is available;
- Outcome measurement: MCC at visit 8/week 24;
- Intercurrent event: had the subject not discontinued the study drug for any reason;
- Population-based summary: difference of MCC at visit 8/week 24 (or prior, due to study drug discontinuation) compared to baseline.

For a single arm baseline controlled study, this "de jure" estimand is considered the appropriate choice. As some effect is expected early in the study and with continued treatment could be expected to be maintained, it's considered appropriate to impute for subjects with missing values at visit 8/week 24 by their visit 5/week 4 value (if available).

A "de facto" estimand (treatment policy) was not chosen for this study. As this is a single arm treatment, a treatment policy estimand (which typically compares two randomized arms regardless of treatment changes) was not considered suitable for this type of study. A further reason against the use of the treatment policy estimand is the fact that subjects need to immediately start a different treatment after study drug discontinuation, which may differ

across different investigators, and is likely different from the treatment they took before entering this study. The impact of such a treatment mix on the effect of mirabegron would be difficult to interpret.

Difference of MCC at visit 8/week 24 (or prior, due to study drug discontinuation) compared to baseline is the primary estimator.

As a sensitivity analysis, Mixed-Effect Model Repeated Measure (MMRM) will be used to handle any missing endpoint at visit 8/week 24.

### 6.1.3 Secondary Efficacy Endpoints

Secondary efficacy endpoints are described in Table 2 and Table 3 above.

### **6.1.3.1** Urodynamic Measures

For each of these endpoints, the change from baseline at the post-baseline value is the value at the post-baseline visit minus the value at the baseline visit. If either the baseline value or the post-baseline visit value is missing, the change from baseline will be missing. No imputation will be done.

### 6.1.3.1.1 Overactive Detrusor Contractions (>15 cmH<sub>2</sub>O)

The volume (mL) of fluid instilled until the first detrusor contraction (>15 cm H<sub>2</sub>O) is recorded in the "VOLUME" section of the "Urodynamic Testing" pages of the eCRF. If no contraction occurred, the bladder volume will be missing in the eCRF and the MCC at that visit will be used.

# 6.1.3.1.2 Number of Overactive Detrusor Contractions and Detrusor Pressure at end of filling

The number of overactive detrusor contractions (>15 cm H<sub>2</sub>O) until end of filling is recorded in the same section as the Overactive Detrusor Contractions of the "Urodynamic Testing" pages of the eCRF. Detrusor pressure at end of filling (cm H<sub>2</sub>O) is recorded in the same section of the eCRF.

#### 6.1.3.1.3 Bladder Compliance

Bladder compliance ( $\Delta V/\Delta P$ det) will be assessed by the independent central reviewers and reported as annotations on the urodynamic trace and in an external database, not in the eCRF.

The calculation of the bladder compliance will be performed by the central reviewers. To standardize this calculation, the most linear part of the volume/pressure relationship will be isolated and used for calculating compliance. The values for V and P at the beginning and the end of this portion of the tracing are then used to calculate  $\Delta V/\Delta P$ det [Bauer, 2015].

### 6.1.3.2 Bladder Volume and Leakage Measures

For each of these endpoints (see Table 2 and Table 3), the change from baseline to the post-baseline value is the value at the post-baseline visit minus the value at the baseline visit. If either the baseline value or the post-baseline visit value is missing, the change from baseline will be missing. No imputation will be done.

The value calculated from the 7-day diary period before visit 3 will be regarded as the baseline value. Each post-baseline value will be calculated using the 7-day diary period before the post-baseline visit.

Catheterized volume per catheterization is not directly collected in the 7-day diary, instead the weight of the pee per catheterization is entered. If the subject recorded the presence of poo this measurement will be invalid and considered as missing for analysis purposes. Catheterized volume per catheterization [mL] will be calculated as weight of the pee per catheterization [mg], using the following conversion formula: 1 g = 1 mL.

### 6.1.3.2.1 Average catheterized volume per catheterization (weekend diary)

For each subject, the average catheterized volume per catheterization is calculated as the sum of all available (non-missing) catheterized volumes recorded <u>over both</u> of the 2 measuring days in the weekend diary, whether or not these 2 days are consecutive divided by the number of catheterizations with non-missing volumes.

If volumes are recorded on 1 single day of the weekend diary, then the average catheterized volume per catheterization is calculated using all available (non-missing) catheterized volumes recorded on that day.

If no volumes are recorded on any day of the weekend diary, then the average catheterized volume per catheterization will be missing.

### 6.1.3.2.2 Maximum catheterized volume per day (weekend diary)

For each subject, the maximum catheterized volume per day is calculated using all available (non-missing) catheterized volumes recorded for the 2 measuring days in the weekend ediary, whether or not these 2 days are consecutive. The maximum value will be calculated separately for each measuring day and the mean of these two values will be used.

If volumes are recorded on 1 single day of the weekend e-diary, then the maximum catheterized volume per day is calculated using all available (non-zero) catheterized volumes recorded on that day.

If no volumes are recorded on any day of the weekend e-diary, then the maximum catheterized volume per day will be missing.

### 6.1.3.2.3 Maximum catheterized daytime volume (weekend diary)

For each subject, the maximum catheterized daytime volume is calculated using all available (non-missing) catheterized daytime volumes for the 2 measuring days in the weekend e-diary, whether or not these 2 days are consecutive. The maximum value will be calculated separately for each measuring day and the mean of these two values will be used.

If volumes are recorded on 1 single day of the weekend e-diary, then the maximum catheterized daytime volume is calculated using all available (non-zero) catheterized daytime volumes recorded on that day.

If no volumes are recorded on any day of the weekend e-diary, then the maximum catheterized daytime volume will be missing.

Daytime is defined as the time between wake-up time (minus 30 min) and time to sleep (plus 29 minutes) recorded in the e-diary; e.g. if the wake-up time is HH:MM=08:30 and sleep time is HH:MM=22:00, then daytime is defined from 08.00 to 22.29.

If wake up time and/or time sleeps is missing imputation rules will be applied as per section 7.11.1.2

### 6.1.3.2.4 Average morning catheterized volume (weekend diary)

On a volume-measuring day in the e-diary, the first morning catheterized volume is the first recorded non-zero volume within or after the hour of the wake-up time, e.g. if the wake-up time is HH:MM=08:30, then the first non-zero volume recorded during the 8-9am hour period or later period is used. If the wake-up time is missing on a measuring day, the first non-zero recorded volume after 06:00 will be used. If no non-zero volume is recorded before 15:00 on a measuring day, the first morning catheterized volume will be missing for that e-diary day.

The average first morning catheterized volume is calculated as the average of the available first morning catheterized volumes recorded for the 2 measuring days in the weekend e-diary, whether or not these 2 days are consecutive.

If the first morning catheterized volume is recorded on 1 single day of the weekend e-diary, then the average morning catheterized is the first morning catheterized on that day.

If no first morning catheterized volumes are recorded on any day of the weekend e-diary, then the average first morning catheterized volume will be missing.

# 6.1.3.2.5 Mean number of leakage episodes per day (day and night time) (weekend diary)

For each subject, the mean number of leakage episodes per day (during day and night time) is calculated using all available (non-missing) number of leakage episodes for the 2 measuring days in the weekend diary during day and night time.

If the number of leakage episodes is recorded on 1 single day in the 7-day diary during day and night time, then the mean number of leakage episodes per day during day and night time is equal to the total number of leakage episodes recorded on that day during day and night time.

If no leakage episodes are recorded on any day of the weekend diary during day and night time, then the mean number of leakage episodes per day will be zero. If nothing is recorded, e.g., not completing the diary, the result is missing.

# 6.1.3.2.6 Number of dry (leakage-free) days per 7 days (day and night time) (7-day diary)

Let  $D_{dry}$  be the number of valid diary days where the response to the question 'Did you leak between this catheterization and the last one' is 'No' each time a new catheterization is entered during the day and night time period.

Let  $D_{wet}$  be the number of valid diary days where the response to the question 'Did you leak between this catheterization and the last one' is 'Yes' for at least one catheterization entered during the day and night time period.

If  $(D_{dry} + D_{wet}) > 3$ , then the number of dry days per 7 days is calculated as

$$\frac{D_{dry}}{\left(D_{dry} + D_{wet}\right)} \times 7$$

Otherwise its value is missing.

## 6.1.3.2.7 Number of dry (leakage -free) nights per 7 days

Let  $N_{dry}$  be the number of valid diary days where the response to the question 'Did you leak between this catheterization and the last one' is 'No' each time a new catheterization is entered during the night time period.

Let  $N_{wet}$  be the number of valid diary days where the response to the question 'Did you leak between this catheterization and the last one' is 'Yes' for at least one catheterization entered during the night time period.

If  $(N_{dry} + N_{wet}) > 3$ , then the number of dry nights per 7 days is calculated as

$$\frac{N_{dry}}{\left(N_{dry} + N_{wet}\right)} \times 7$$

Otherwise its value is missing.

### 6.1.3.2.8 Identification of leakage during sleeping time

For identification of a leakage during the sleeping time: since time for sleep and time for wake up are available, all leakages which occurred during this period are considered as 'Sleeping time Leakages'.

For identification, at a visit, of a leakage during the sleeping time all leakages which occurred during this period are considered as 'Sleeping time Leakages'. If there are:

- 0 leakages, the subject is considered as "Subject with no leakage" at that visit
- \ge 1 leakages, the subject is considered as "Subject with leakage" at the visit

### 6.1.3.3 Subject- or Clinician-reported Questionnaire

### 6.1.3.3.1 Pediatric Incontinence Questionnaire (PIN-Q)

The total PinQ score (Bower, 2006) is 20 multiplied by the average of the individual PinQ items where each of the 20 Likert scales have been converted to a score:

- For items 6 and 17; 0: "No" to 4: "Definitely" will be used; and
- For the other 18 items; 0: "No" to 4: "All the time" will be used.

It is expected that completed questionnaires will have at most a limited number of missing values; if the answers to more than two questions are missing, the total score will not be calculated and will be missing.

Individual item scores will not be directly imputed.

The change from baseline to each post-baseline visit in the total PinQ score is the value at the post-baseline visit minus the value at the baseline visit. If either the baseline value or the post-baseline visit value is missing, the change from baseline will be missing.

If change is:

- Less than 0, there is an improvement between the two time-points;
- Equal 0, there is no change between the two time-points;
- Greater than 0, there is a worsening between the two time-points.

### 6.1.3.3.2 Patient Global Impression of Severity Scale (PGI-S)

The Patient Global Impression of Severity Scale (PGI-S) is an answer of the question: "How did you feel about your bladder condition DURING THE PAST 3 DAYS?"

Subjects will evaluate their recent condition ticking one of the following categories: "Really Bad" (0), "Bad" (1), "Not Bad, Not Good" (2), "Good" (3) and "Really Good" (4).

PGI-S will be summarized as a continuous variable. The change from baseline to each post-baseline visit in the PGI-S score is the value at the post-baseline visit minus the value at the baseline visit. If either the baseline value or the post-baseline visit value is missing, the change from baseline will be missing.

A positive change indicates an improvement while a negative change indicates a worsening.

### 6.1.3.3.3 Clinician Global Impression of Change (CGI-C)

The Clinician Global Impression of Change (CGI-C) is a 7 point scale that requires the clinician to assess how much the subject's overall bladder symptoms since the start of the study on day 1 has improved or worsened and rated as: very much improved (1); much improved (2); minimally improved (3); no change (4); minimally worse (5); much worse (6); or very much worse (7).

CGI-C will be summarized as a categorical variable.

### 6.1.3.3.4 Acceptability (for tablets)

Subjects will evaluate the taste of the study medication ticking one of the following categories: "Really Bad" (0), "Bad" (1), "Not Bad, Not Good" (2), "Good" (3) and "Really Good" (4).

Subjects will evaluate the swallow of the study medication ticking one of the following categories: "Really Difficult" (0), "Difficult" (1), "Not Difficult, Not Easy" (2), "Easy" (3) and "Really Easy" (4).

Taste and swallow acceptability will be summarized as categorical variables.
### 6.1.3.3.5 Acceptability (for oral suspension)

Subjects will evaluate the taste of the study medication ticking one of the following categories: "Really Bad" (0), "Bad" (1), "Not Bad, Not Good" (2), "Good" (3) and "Really Good" (4).

Subjects will evaluate the smell of the study medication ticking one of the following categories: "Really Bad" (0), "Bad" (1), "Not Bad, Not Good" (2), "Good" (3) and "Really Good" (4).

Subjects will evaluate the consumption of the study medication ticking one of the following categories: "Really Difficult" (0), "Difficult" (1), "Not Difficult, Not Easy" (2), "Easy" (3) and "Really Easy" (4).

Subjects will evaluate the preparation of the study medication ticking one of the following categories: "Really Difficult" (0), "Difficult" (1), "Not Difficult, Not Easy" (2), "Easy" (3) and "Really Easy" (4).

Taste, smell, consumption and preparation acceptability will be summarized as categorical variables.

## **6.1.4** Exploratory Efficacy Endpoints

The exploratory efficacy endpoints are summarized in Table 2 and Table 3. No imputation will be done.

## 6.1.4.1 Exploratory efficacy endpoints based on urodynamic measures

### 6.1.4.1.1 Filling volume at 20 cm, 30 cm and at 40 cm H<sub>2</sub>O detrusor pressure

Bladder volumes at 20, 30 and 40 cm H<sub>2</sub>O detrusor pressure are recorded in the "VOLUME" section of the "Urodynamic Testing" pages of the eCRF. If detrusor pressure cannot be reached during the examination, the volume will be missing.

## 6.1.4.2 Exploratory efficacy endpoints based on 7-day diary

### 6.1.4.2.1 MCC expressed as percentage of EBC

MCC expressed as % of EBC will be as:

100% x MCC/EBC, where EBC = 24.5 x age(years) + 62.

## 6.1.4.2.2 Grade of leakage (weekend diary)

Grade of worst leakage will be assessed by answering to 1 of the 2 questions as appropriate: "How wet was your diaper/pad?" or "How wet were your clothes?".

Subjects will evaluate the grade of leakage by ticking one of the following categories: "Fully Wet" (0), "Quite Wet" (1), "Slightly Wet" (2).

If a subject experiences leakage episodes but there is no answer to the leakage question, the leakage grade will be missing.

## 6.1.4.2.3 Total catheterized volume per day (weekend diary)

The total catheterized volume per 24h is calculated using all available (non-missing) catheterized volumes recorded for the 2 measuring days in the diary, whether or not these 2 days are consecutive. The total value will be calculated separately for each measuring day and the mean of these two values will be used.

If no volumes are recorded on any day of the weekend diary, then the total catheterized volume per day will be missing.

## 6.1.4.2.4 Number of CICs/day (weekday diary)

The number of CICs per day will be calculated as the total number of CICs reported during valid diary days in the weekday diary divided by the total number of valid weekday diary days).

## 6.1.4.2.5 Responder in respect to leakage (weekend diary)

The percent change from baseline to a post-baseline visit in the number of leakage episodes during the weekend diary will be calculated as follows:

$$R_x = \frac{\textit{No.Leakage Epis. at Visit } x - \textit{No.Leakage Epis. at baseline}}{\textit{No.Leakage Epis. at baseline}} \times 100$$

A complete responder will be defined as a subject with a 100% improvement from baseline (i.e.  $R_X$ = -100%). A partial responder will be defined as a subject with a percent improvement from baseline  $\geq$ 50% and <100% (i.e. -100% <  $R_X$   $\leq$  -50%). A non-responder will be defined as a subject with an improvement from baseline <50% or a worsening from baseline (i.e.  $R_X$  > -50%).

If the number of leakage episodes at baseline is equal to zero, a constant equal to 0.5 will be added to the baseline number of leakages to allow denominator calculation.

If the number of leakage episodes at baseline and/or at a post-baseline visit is missing then the response category in respect to leakage will be missing.

## 6.1.4.2.6 Percentage of Catheterizations without Intermittent Leakage Accident

For each visit the percentage of catheterizations without intermittent leakage accident is:

100% x (total number of catheterizations without intermittent leakage accident / total number of catheterizations).

For reporting 3 response criteria are defined:

- No response: <50% reduction from baseline:
- Partial response; 50-99% reduction from baseline; and
- Complete response; 100% reduction from baseline.

# 6.2 Safety Endpoints

The following safety endpoints will be assessed:

Table 4Safety Endpoints

| <b>Endpoint Number</b> | Endpoint Description |
|---|---|
| | Enupoint Description |
| Safety Endpoints† | In sidence and associate of tweeter out amount advance associate (TEAEs) |
| 2245 | Incidence and severity of treatment-emergent adverse events (TEAEs) |
| 2,3,4,5 | Change from baseline in vital signs (clinic measurements): systolic blood |
| | pressure, at visit 5/week 4, visit 7/week 12, visit 8/week 24 and visit 10/week |
| 6.700 | 52 (EOT/EOS) |
| 6,7,8,9 | Change from baseline in vital signs (clinic measurements): diastolic blood |
| | pressure at visit 5/week 4, visit 7/week 12, visit 8/week 24 and visit 10/week 52 (EOT/EOS) |
| 10,11,12,13 | Change from baseline in vital signs (clinic measurements): pulse rate at visit |
| | 5/week 4, visit 7/week 12, visit 8/week 24 and visit 10/week 52 (EOT/EOS) |
| 14,15,16,17 | Change from baseline in vital signs (clinic measurements): temperature at visit |
| | 5/week 4, visit 7/week 12, visit 8/week 24 and visit 10/week 52 (EOT/EOS) |
| 18,19,20,21,22,23,2 | Change from baseline in vital signs (self blood pressure measurement SBPM): |
| 4 | systolic blood pressure at visit 4/week 2, visit 5/week 4, visit 6/week 8, visit |
| | 7/week 12, visit 8/week 24, visit 9/week 36 and visit 10/week 52 (EOT/EOS) |
| | and on 2 consecutive days at around 1 and 2 weeks after start of dosing with |
| | PED25 (day 1) and after up titration to PED50 (visit 4/week 2, visit 5/week 4 |
| | or visit 6/week 8), if not already covered by the scheduled visit 4/week 2 |
| | and/or visit 5/week 4 SBPM. |
| 25,26,27,28,29,30,3 | Change from baseline in vital signs (SBPM): diastolic blood pressure at visit |
| 1 | 4/week 2, visit 5/week 4, visit 6/week 8, visit 7/week 12, visit 8/week 24, visit |
| | 9/week 36 and visit 10/week 52 (EOT/EOS) and on 2 consecutive days at |
| | around 1 and 2 weeks after start of dosing with PED25 (day 1) and after up |
| | titration to PED50 (visit 4/week 2, visit 5/week 4 or visit 6/week 8), if not |
| | already covered by the scheduled visit 4/week 2 and/or visit 5/week 4 SBPM. |
| 32,33,34,35,36,37,3 | Change from baseline in vital signs (SBPM): pulse rate at visit 4/week 2, visit |
| 8 | 5/week 4, visit 6/week 8, visit 7/week 12, visit 8/week 24, visit 9/week 36 and |
| | visit 10/week 52 (EOT/EOS) and on 2 consecutive days at around 1 and 2 |
| | weeks after start of dosing with PED25 (day 1) and after up titration to PED50 |
| | (visit 4/week 2, visit 5/week 4 or visit 6/week 8), if not already covered by the |
| | scheduled visit 4/week 2 and/or visit 5/week 4 SBPM. |
| 39,40 | Change from baseline in hematology and biochemistry tests at visit 7/week 12 |
| | and visit 10/week 52 (EOT/EOS) |
| 41,42,43,44 | Change from baseline in urinalysis tests at visit 5/week 4, visit 7/week 12, visit |
| | 8/week 24 and visit 10/week 52 (EOT/EOS) |
| 45,46,47,48 | Change and categorized shift from baseline in ECG parameters at visit 5/week |
| | 4, visit 7/week 12, visit 8/week 24 and visit 10/week 52 (EOT/EOS) |
| 49 | Categorized shift summary from baseline to visit 10/week 52 (EOT/EOS) in |
| | upper urinary tract ultrasound assessment |
| 50,51 | Change from baseline in eGFR at visit 7/week 12 and visit 10/week 52 |
| | (EOT/EOS) |
| Exploratory Safety | |
| 52,53 | Change from baseline in body height and weight at visit 8/week 24 and visit |
| | 10/week 52 (EOT/EOS) |

<sup>†</sup> Physical Examination will be analyzed as part of subject medical history or AEs depending on the time of the finding.

**Table 5 Summary of Safety Endpoints** 

| Variable | Endpoints | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| | | Week 2 | Week 4 | Week 8 | Week 12 | Week 24 | Week 36 | Week 52 |
| TEAE | N (%) | | | | 1 | | | |
| $\mathrm{SBP}^{\mathrm{CM}}$ | Change from baseline | | 2 | | 3 | 4 | | 5 |
| $\mathrm{DBP}^{\mathrm{CM}}$ | Change from baseline | | 6 | | 7 | 8 | | 9 |
| PR <sup>CM</sup> | Change from baseline | | 10 | | 11 | 12 | | 13 |
| Body Temperature <sup>CM</sup> | Change from baseline | | 14 | | 15 | 16 | | 17 |
| $SBP^{SM}$ | Change from baseline | 18 | 19 | 20 | 21 | 22 | 23 | 24 |
| $DBP^{SM}$ | Change from baseline | 25 | 26 | 27 | 28 | 29 | 30 | 31 |
| $PR^{SM}$ | Change from baseline | 32 | 33 | 34 | 35 | 36 | 37 | 38 |
| Hamatalass, and his shamistm. | Change from baseline | | | | 39 | | | 40 |
| Hematology and biochemistry | Categorized shift from baseline | | | | 39 | | | 40 |
| Urinalysis | Change from baseline | | 41 | | 42 | 43 | | 44 |
| Officiallysis | Categorized shift from baseline | | | | 42 | 43 | | 44 |
| ECC | Change from baseline | | 45 | | 46 | | 47 | 48 |
| ECG Categorized shift from baseline | | | 43 | | 46 | | 4/ | 48 |
| Upper Urinary Tract Ultrasound | Categorized shift from baseline | | | | | | | 49 |
| eGFR# | Change from baseline | | | | 50 | | | 51 |
| Height and Weight | Change from baseline | | | | | 52 | | 53 |

<sup>&</sup>lt;sup>CM</sup> Clinic Measurements

SM Self Measurements

<sup>#</sup> will be calculated according to the Larson Formula (Larson et al, 2004], and the modified Schwartz 2009 (for children < 12 years old) and the Cockcroft-Gault equation (for adolescents) formulas

## 6.2.1 Vital signs

## **6.2.1.1** Clinic Measurement of Vital Signs

Triplicate blood pressure and pulse measurements and single body temperature measurements (ear thermometer) will be performed at visit 1/screening, visit 3/baseline, and on visit 5/week 4, visit 7/week 12, visit 8/week 24 and visit 10/week 52 (EOT/EOS). Clinic measurements of vital signs at visit 1/screening and visit 3/baseline will be used to assess eligibility.

The measurements will be per standard clinic practices and should be consistent for all visits. For each subject the correct size of the blood pressure cuff must be determined and used when assessing blood pressures. Blood pressure and pulse will be measured with approximately 2-minute intervals, after the subject has been calm and without distress for at least 5 minutes.

The subject should be seated with the back supported, feet on the floor and right arm supported, legs uncrossed and the cubital fossa at heart level. If sitting is not possible, supine is allowed, but measurements should always be taken in the same position. The subject should not move and should remain silent during the reading, as moving and talking can affect the reading.

The right arm is preferred in repeated measures of blood pressure for consistency and comparison to standard tables. The same arm should be used throughout the study whenever possible. Vital sign measurements should be performed prior to blood sampling.

For the purpose of the analyses of vital signs, the average per visit for vital signs measured at the clinic will be calculated as follows:

- If three or more measurements are reported, the average of all values will be used.
- If only two measurements are reported, the average of the two values will be used.
- If only one measurement is reported, it will be displayed for the average.
- If all measurements are missing, then the average will be missing.

The method of body temperature measurement is via an ear thermometer and should be consistent for all visits.

Clinically relevant adverse changes in vital signs will be recorded as an AE [Section 6.2.3]

### **6.2.1.2** Self Measurement of Vital Signs

Triplicate SBPM (blood pressure and pulse rate) will be performed on the 2 weekend days prior to each visit. Additional SBPM will be done on 2 consecutive days at around 1 and 2 weeks after start of dosing with PED25 (day 1) and after up-titration to PED50 (visit 4/week 2, visit 5/week 4 or visit 6/week 8), if not already covered by the scheduled visit 4/week 2 and/or visit 5/week 4 SBPM.

Following successful completion of the first 2-day weekend e-diary, confirmed at visit 2, subsequent measurements will be performed in the weekend preceding visit 3/baseline,

visit 4/week 2, visit 5/week 4, visit 6/week 8, visit 7/week 12, visit 8/week 24, visit 9/week 36 and visit 10/week 52 (EOT/EOS).

Devices for measuring blood pressure and pulse rate will be provided to subjects for home measurements. Detailed on-site training to use the SBPM device and a booklet with operating instructions in local language will be provided to the subject and parent(s)/caregiver(s).

For each subject the correct cuff size will be determined by the investigator by measuring the circumference of the subject's upper arm in order to give the subject the device with the best cuff type. Ideally, the bladder length of the cuff should be 80% to 100% of the arm's circumference and the width of the bladder approximately 40% (the bladder is the inflatable part of the cuff). The cuff should be put on according to the instructions given by investigator.

Morning measurements should be taken after waking up, before breakfast and before study drug intake, evening measurements should be taken prior to bedtime. If deemed necessary by the Investigator, subjects may be asked to perform additional measurements.

Self-measurements should, where possible, be performed in the same position as the clinic measurements for vital signs.

Results will be directly entered by the subject or subject's parent/caregiver in the e-diary.

For the purpose of the analyses, the average self-measurement vital signs will be calculated using all values from the 2-days diary collection separately for the regular measurements and the extra measurements. If all measurements are missing, then the average will be missing. However, if the extra measurements are not performed because they are covered by the regular ones, the regular measurements values will be duplicated so that they are included in both the regular and the extra analyses.

### **6.2.1.3** Conversion of Blood Pressure to Percentiles

Both the systolic and diastolic blood pressure site measurements will additionally be converted to percentiles specific to the age (years), sex and height (cm) of the subject using the following steps [NIH, 2005]:

- The height of a subject is measured at Visits 1, 3, 8, 10/EOS and, if applicable, at the Early Discontinuation Visit. As the children and adolescents in this study may be expected to increase in height during the course of the study, the height of the child at a study visit will be imputed by linearly interpolating between Visit 3 and a post-baseline visit as follow:
  - Let D<sub>visit</sub> be the date of the study visit, H<sub>1</sub> be the most recent height measurement at or prior to the study visit, D<sub>1</sub> be the date of H<sub>1</sub>, H<sub>2</sub> be the earliest height measurement at or after the study visit, and D<sub>2</sub> be the date of H<sub>2</sub>.

The height at 
$$D_{visit}$$
 is estimated as:  $H_{visit} = H_1 + \left(\frac{D_{visit} - D_1}{D_2 - D_1}\right) (H_2 - H_1)$ 

- Let Z = the z-score (i.e. the number of standard deviations above or below the mean) of the height (cm) of the subject at the study visit relative to healthy subjects of the same age and gender using CDC growth charts [CDC, 2000]. The formula and example SAS code to calculate this are given in Appendix 12
- Let BP = the blood pressure (mmHg) that is being converted (either systolic or diastolic) and Y=the age of the child in years.
- Taking the coefficients from the appropriate column in Table 6 below, compute  $Z_{BP}$ , the Z-score for the blood pressure:

$$Z_{BP} = \left[ BP - \alpha - \sum_{j=1}^{4} \beta_{j} (Y - 10)^{j} - \sum_{k=1}^{4} \gamma_{k} Z^{k} \right] / \sigma$$

- If  $\Phi$ (.) is the area under the standard normal curve to the left of Z, calculate P, the gender, age and height specific percentile of the blood pressure as  $P=\Phi(Z_{BP})*100\%$ .
- The exact age at a visit will be calculated as:

$$Age = \frac{(D_V - D_B + 1)}{365.25}$$

where  $D_v$  is the visit date and  $D_B$  is the subject's date of birth. When the exact age at a visit is missing and cannot be calculated because of a missing date of birth, but where the age entered at screening is known only to be Y years (an integer), the percentile will be calculated for age=Y+0.5.

Table 6 Coefficients for Conversion of Blood Pressure to Percentiles

| | | | Systo | olic BP | Diasto | lic BP |
|---|---|---|---|---|---|---|
| Variable | | Symbol | Male | Female | Male | Female |
| Intercept | | A | 102.19768 | 102.01027 | 61.01217 | 60.50510 |
| Age | (Age-10) | $\beta_1$ | 1.82416 | 1.94397 | 0.68314 | 1.01301 |
| | $(Age-10)^2$ | $\beta_2$ | 0.12776 | .00598 | -0.09835 | 0.01157 |
| | $(Age-10)^3$ | $\beta_3$ | 0.00249 | -0.00789 | 0.01711 | 0.00424 |
| | $(Age-10)^4$ | $\beta_4$ | -0.00135 | -0.00059 | 0.00045 | -0.00137 |
| Height | Z | $\gamma_1$ | 2.73157 | 2.03526 | 1.46993 | 1.16641 |
| Z-Score | $Z^2$ | $\gamma_2$ | -0.19618 | 0.02534 | -0.07849 | 0.12795 |
| | $\mathbb{Z}^3$ | γ <sub>3</sub> | -0.04659 | -0.01884 | -0.03144 | -0.03869 |
| | $\mathbf{Z}^4$ | γ <sub>4</sub> | 0.00947 | 0.00121 | 0.00967 | -0.00079 |
| Standard Deviat | ion | σ | 10.7128 | 10.4855 | 11.6032 | 10.9573 |

To illustrate, a boy born on 1<sup>st</sup> January 2001 comes for a study visit on 13<sup>th</sup> January 2013. His height is measured as 159 cm and his systolic blood pressure (the mean of the triplicate) is 120 mmHg. In Appendix 12 the z-score for the boy's height is worked through as an example and Z is found to equal 1.2836. The coefficients for the conversion of the blood pressure are taken from the appropriate column (systolic BP, Male) of Table 6 The value of

**Sponsor: Astellas Pharma Global Development, Inc.** ISN/Protocol 178-CL-206A

 $Z_{BP}$  is found to equal 0.97623 which equates to the 83.6<sup>th</sup> percentile of the standard normal curve.

## 6.2.1.4 Pulse Rate in Relation to Age

Resting pulse rate will be compared to age-related norms [Fleming et al., 2011] according to the percentiles shown in Table 7

Table 7 Percentiles for Resting Pulse Rate in Relation to Age and Gender

| | Percentile | | | | | | |
|---|---|---|---|---|---|---|---|
| Age | 1 <sup>st</sup> | 10 <sup>th</sup> | 25 <sup>th</sup> | 50 <sup>th</sup> | 75 <sup>th</sup> | 90 <sup>th</sup> | 99 <sup>th</sup> |
| 3-4y | 70 | 86 | 94 | 104 | 113 | 123 | 136 |
| 4-6y | 65 | 81 | 89 | 98 | 108 | 117 | 131 |
| 6-8y | 59 | 74 | 82 | 91 | 101 | 111 | 123 |
| 8-12y | 52 | 67 | 75 | 84 | 93 | 103 | 115 |
| 12-15y | 47 | 62 | 69 | 78 | 87 | 96 | 108 |
| 15-18y | 43 | 58 | 65 | 73 | 83 | 92 | 104 |

Each value of pulse rate will be categorized as either being above the age-specific 99<sup>th</sup> percentile or below the 1<sup>st</sup> percentile.

## **6.2.1.5** Body Temperature

Body Temperature will be compared to a reference range of 35.4 to 37.7 degrees [Kliegman et al, 2007].

### **6.2.2** Adverse Events

Collection of details of adverse events will begin at visit 1 after the signing of informed consent and will continue for all subsequent study visits. Adverse events will be evaluated during the telephone assessments at visit 2/wash-out period, visit 4/week 2, visit 6/week 8 and visit 9/week 36 and at each time the subject visits the clinic in person.

An AE with an onset date prior to the first dose of study drug is not considered treatmentemergent but rather as part of the <u>baseline signs and symptoms</u> of the study. These AEs will be listed in the AE listing.

A treatment-emergent adverse event (TEAE) is defined as an adverse event with date of onset occurring on or after the first dose of study medication and up to the end of study. If the adverse event occurs on Day 1 and the onset check box is marked "Onset after first dose of study drug" or the onset check box is left blank, then the adverse event will be considered treatment emergent. If the adverse event occurs on Day 1 and the onset check box is marked "Onset before first dose of study drug", then the adverse event will not be considered treatment emergent. If a subject experiences an event both before and after the first dose of study drug, the event will be considered a TEAE only if it has worsened in severity (i.e. it is reported with a new start date). All adverse events collected that begin within 7 days after taking the last dose of study drug will also be counted as a TEAE and for Serious Adverse Events (SAE) the follow-up period will be until the end of the study.

All AEs will be compared with a list of AEs that Astellas considers to be "Always Serious" and those AEs that are on the list will be upgraded to "Serious".

A drug-related TEAE is defined as any TEAE with at least a possible relationship to study treatment as assessed by the investigator or with a missing assessment of the causal relationship.

Common TEAEs are defined as preferred terms (PTs) that have been reported by at least 5% of the subjects.

When an AE start or stop date is missing, the date will be imputed using the rules in Section 7.11.1.3

Adverse events of interest are:

- CV
  - Increased blood pressure
  - QT prolongation
  - o Increased heart rate, tachycardia, atrial fibrillation, or palpitations (Note: these 3 CV events will be analyzed combined and separately)
- Urinary Tract Infection (UTI)
- Hypersensitivity reactions
- Urinary retention
- Neoplasm
- Seizure
- Syncope
- Fetal disorders after exposure during pregnancy
- Concomitant treatment with cytochrome P450 (CYP) 2D6 substrates with narrow therapeutic indices or individually dose-titrated.

AEs of interest will be identified using Standardized MedDRA queries (SMQ), version 16.0, see Table 8, or sponsor-defined list of search terms, see Appendix 3.

Table 8 Standardized MedDRA Queries, Version 16.0

| Hypertension SMQ – Narrow search |
|----------------------------------------------|
| Torsade de pointes/QT prolongation SMQ – |
| Broad search |
| Arrhythmia related investigations signs and |
| symptoms SMQ – Broad search, |
| Supraventricular tachyarrhythmias (SMQ) |
| Broad search, |
| Tachyarrhythmia terms nonspecific (SMQ) |
| – Narrow search, |
| Ventricular tachyarrhythmias (SMQ) - |
| narrow search plus Ventricular tachycardia |
| Hypersensitivity SMQ – Narrow search |
| Neoplasm SMQ – Narrow search |
| Lower Level Term 10039906 |
| Syncope SMQ – Narrow search (also |
| included as part of the CV - Increased heart |
| rate, tachycardia, atrial fibrillation, and |
| palpitations) |
| PT 10042772 |
| Congenital, familial and genetic disorders - |
| SMQ Narrow |
| Fetal disorders – SMQ Broad search |
| Neonatal disorders – SMQ Broad search |
| PT Drug interaction |
| PT Potentiating drug interaction |

## 6.2.3 Clinical Laboratory Variables

Hematology and biochemistry assessments will be taken at visit 1/screening, visit 7/week 12 and visit 10/week 52 (EOT/EOS). In the event that an AE related to hematology/biochemistry parameters is found at visit 1/screening, an additional hematology/biochemistry assessment is to be taken at visit 3/baseline.

Urinalysis is to be assessed at visit 1/screening, at visit 3/baseline, and at visit 5/week 4, visit 7/week 12, visit 8/week 24 and visit 10/week 52 (EOT/EOS).

To allow for an early DSMB safety assessment, the first 5-10 subjects who reach study visit 5/week 4 will have an additional blood draw at this visit [see Table 1]. These data will be summarized in a table.

All safety laboratory assessments will be performed at a central laboratory, except for urine pregnancy testing, which is done locally. Pregnancy test in female subjects of childbearing

potential will be performed in serum (if blood is drawn for hematology/biochemistry) or urine (at the other visits).

The investigator may decide to repeat the safety laboratory assessments, should the results be important for safety reasons and considered clinically relevant. Repeating safety laboratory assessments for re-screening is not allowed. The clinical significance of out-of-range laboratory findings is to be determined and documented by the investigator/sub-investigator who is a qualified physician. Clinically significant adverse changes will be recorded as an AE [Section 5.5.1 of the protocol].

The laboratory parameters that will be assessed during the conduct of the study are listed in Table 9

Table 9 Laboratory Assessments

| | By Central Laboratory | |
|---|---|---|
| Assessment | Collecting tube | Parameters to be analyzed |
| Hematology | EDTA tube | HbA1c |
| | | Hemoglobin |
| | | Hematocrit |
| | | Platelets |
| | | Red blood cells |
| | | White blood cells |
| | | Differential white blood cell count |
| Biochemistry | Serum tube | Alanine aminotransferase |
| | | Albumin |
| | | Alkaline phosphatase |
| | | Aspartate aminotransferase |
| | | Calcium |
| | | Chloride |
| | | Creatine phosphokinase |
| | | Creatinine |
| | | Cystatin C |
| | | Estimated glomerular filtration rate |
| | | (Larsson, modified Schwartz and Cockcroft- |
| | | Gault) |
| | | Gamma-glutamyl transaminase |
| | | Glucose |
| | | hCG † |
| | | Lactate dehydrogenase |
| | | Potassium |
| | | Sodium |
| | | Total bilirubin |
| | | Total protein |
| | | Urea |
| | | Uric acid |
| Table continued on next page | | • |

| | By Central Lab | oratory |
|------------|--------------------|---------------------------|
| Assessment | Collecting tube | Parameters to be analyzed |
| Urinalysis | Dipstick | Protein |
| | | Glucose |
| | | pН |
| | Polypropylene tube | Urobilinogen |
| | | Bilirubin |
| | | Ketones |
| | | Nitrite |
| | | Casts |
| | | Crystals |
| | | Bacteria |
| | | Epithelial cells |
| | | Small round cells |
| | | Yeasts |
| | | Red blood cells |
| | | White blood cells ‡ |
| | Done Local | lly |
| Pregnancy | Urine | hCG † |

HbA1c: glycosylated hemoglobin A1c; hCG: human chorionic gonadotropin;

Blood samples for evaluation of hematology and biochemistry assessments (including liver function tests) are collected at visit 1/screening, visit 3/baseline<sup>#</sup>, visit 5/week 4<sup>\$</sup>, visit 7/week 12 and at the EOS (Visit 10).

The value of each hematology and biochemistry parameter will be compared to its normal range and classified as High, Low or Normal. Urinalysis parameters will be similarly classified as either Normal or Abnormal.

When calculating changes or shifts in a result from baseline, the value from Visit 1 will be used as baseline. If the Visit 1 value is missing, the latest pre-baseline value will be used (i.e. from Visit 1 or any unscheduled visit conducted between Visit 1 and 3).

### 6.2.4 Physical Examinations

Physical examinations will be performed at visit 1/screening and visit 10/week 52 (EoS) and will include assessments of the main body systems.

<sup>†</sup> Only in female subjects of childbearing potential

 $<sup>\</sup>ddagger$  If white blood cell count is >100/ $\mu$ L (or '++' for semi-quantitative results) a urine culture will be done including an antibiotic sensitivity test.

<sup>#</sup> Additional hematology/biochemistry will be taken at baseline only if an AE related to hematology/biochemistry parameters occurred between visit 1/screening and visit 3/baseline.

<sup>\$</sup> The first group of subjects (minimum of 5, maximum of 10) who reach study visit 5/week 4 will have an additional blood draw for a DSMB-mandated interim safety check at this visit.

The physical examination will be performed per clinic standards and clinically significant findings at screening will be recorded as part of the subject's medical history. Clinically significant findings discovered after visit 1/screening will be recorded as an AE.

## 6.2.5 12-lead Electrocardiogram (ECG)

A 12-lead ECG will be performed in triplicate one minute apart at visit 1/screening, visit 3/baseline, visit 5/week 4, visit 7/week 12, visit 8/week 24 and at visit 10/week 52 (EOT/EOS). The ECGs will be taken with the subject in the supine position, after the subject has been lying quietly for at least 5 minutes. ECG traces will be evaluated by the investigator who will give an overall interpretation and may leave a qualifying comment in the eCRF. The overall interpretation will be recorded as

- Normal, or
- Abnormal not clinically significant, or
- Abnormal clinically significant

All ECGs will be further evaluated by a cardiologist at the central laboratory. When the central laboratory cardiologist's overall interpretation is abnormal, an applicable abnormality code will be assigned. ECG abnormalities are coded for the particular class of abnormality (rhythm, QT interval, etc.) as well as the specific abnormality within each class. Details of this coding are given in Appendix 13: ECG Abnormality Codes

As well as the overall interpretation, the following ECG variables will be supplied by the central laboratory: PR Interval (msec), RR Interval (msec), QRS Duration (msec), QT Interval (msec), QTcF interval (msec) and Heart rate (HR) (beats/min). QT with Bazett correction range (QTcB interval<=450 ms, all ages) will be only used for the inclusion criteria evaluation and won't be presented.

The mean of each triplicate of ECG measurements recorded during the study will be used for each ECG variable. If fewer or more than 3 results are recorded the mean of all available values will be used.

Let  $M_1$  and  $M_3$  equal the means of a continuous ECG variable at Visit 1 and Visit 3, respectively. The baseline value of the variable, used to assess study eligibility and all changes from baseline during the study, will equal  $(M_1+M_3)/2$ .

## 6.2.6 Estimated Glomerular Filtration Rate and Upper Urinary Tract Ultrasound

Renal function will be assessed via monitoring plasma creatinine and cystatin C levels at visit 1/screening, visit 7/week 12 and visit 10/week 52 (EOT/EOS). In addition, the estimated glomerular filtration rate (eGFR) will be calculated by the central laboratory using the Larsson formula [Larsson et al, 2004]:

$$eGFR = 94.577 * [Cys C (mg/L)]^1.2623$$

In addition, BARC will calculate the eGFR using the modified Schwartz 2009 (for children < 12 years old) and the Cockcroft-Gault equation (for adolescents) formulas.-

The presence or absence of structural abnormalities of the urinary tract, upper tract dilation, vesicoureteral reflux, or obstruction at the ureterovesical or ureteropelvic junction will be assessed with an ultrasound of the upper urinary tract at visit 3/baseline, and at visit 10/week 52 (EOT/EOS).

For the first group of subjects (minimum of 5, maximum of 10) who reach study visit 5/week 4, the renal function will also be determined at visit 5/week 4 to allow for the early DSMB safety assessment.

## 6.2.7 Height, Weight and BMI

Height and weight will be recorded at visit 1/screening, visit 3/baseline, visit 8/week 24 and at visit 10/week 52 (EOT/EOS).

As the study subjects are children and adolescents who are still growing, assessment of any effect of treatment on height and weight will be based on comparison with age (at screening) and gender norms from growth charts supplied by the Centers for Disease Control and Prevention. These charts enable the calculation of z-scores for height and weight based on the age (in months) and sex for children, adolescents and young adults up to the age of 20 years [Kuczmarski et al, 2002]. The formulae and example SAS code for the calculation of these Z-scores are given in Appendix 12

The change from baseline in the z-score for height and the z-score for weight will be calculated as the value at the relevant visit minus the baseline value. If either of these values is missing, the change from baseline will be missing.

## 6.3 Pharmacokinetic Variables

Samples of venous blood for pharmacokinetic assessments will be taken when the subject has reached steady state at the optimal dose (considered to be reached after 10 days of daily dosing). A total of 4 pharmacokinetic samples will be collected, divided over 2 sampling days. These 2 days can be selected from the options given in the schedule of assessments (i.e., on visit 5/week 4, visit 6/week 8, visit 7/week 12, visit 8/week 24, visit 9/week 36 or visit 10/week 52) and do not have to be in a specific (consecutive) order:

- Sampling day 1: 1 trough sample (i.e., pre-dose sample).
- Sampling day 2: 1 trough and 2 post-dose samples taken between 2h and 5h post-dose, with at least 1 hour in between the samples.

On visit days where a pharmacokinetic sample is planned in the clinic, completion of breakfast and study drug dosing should occur in the clinic. Dosing on a sampling day with post-dose samples must occur within 1 hour after completion of breakfast.

In addition to the dosing time, the time of completion of breakfast, and type of breakfast will be collected in the eCRF on this sampling day.

The following plasma pharmacokinetic parameters will be calculated for each subject:

- Maximum concentration (C<sub>max</sub>) at steady state
- Time to attain  $C_{max}$  ( $t_{max}$ )

- Area under the plasma concentration—time curve (AUC) for a dose interval (AUC<sub>24</sub>)
- Plasma concentration before drug administration (C<sub>trough</sub>) at steady state
- Terminal elimination half-life  $(t_{1/2})$
- Apparent oral clearance (CL/F)
- Apparent volume of distribution (Vz/F).

Additional pharmacokinetic parameters may be calculated based on the model used.

Further details of the derivation of the pharmacokinetic parameters are given in the pharmacokinetics data analysis plan (PKDAP).

# 6.4 Pharmacodynamic Variables

There are no pharmacodynamic variables in this study.

### 6.5 Other Variables

### **6.5.1** Baseline Characteristics

Baseline characteristics and other variables that will be collected or derived are:

- Informed consent/assent (collected at screening);
- Demographic characteristics (collected at screening);
- Inclusion/Exclusion (collected at screening and baseline);
- Medical history (collected at screening), including a detailed NDO history;
- Current NDO medications (collected at screening and start of washout);
- Antimuscarinics medication stopped for lack of efficacy prior to start of treatment (yes/no).

If  $D_{diag}$  is the date of diagnosis and  $D_{Scr}$  is the date of last informed consent given at Screening, the years since diagnosis of NDO at Screening is

$$Y_{Diag} = \frac{\left(D_{Scr} - D_{Diag} + 1\right)}{365.25}$$

When one of these dates is partial, the rules in Section 7.11.1.2 will be used to impute it.

If D<sub>B</sub> is the subject's date of birth, the age at Screening is

$$Age_{Scr} = \frac{(D_{Scr} - D_B + 1)}{365.25}$$

If the date of birth is not given, the age at Screening will be equal to the value recorded on the demographics page of the eCRF (an integer number of years) plus 0.5. e.g. if the age is given as 12 years in the eCRF, a value of 12.5 will be used in calculations/statistical analyses involving age (an exception to this rule is given for the conversion of blood pressure values to percentiles; see Section 6.2.1.3).

# 6.5.2 Previous and Concomitant Medications and Therapies

All treatments, both drug and non-drug therapies, whether prescribed, over the counter (OTC) or "alternative" that are used during the study will be recorded on the case report

form. Details include generic and/or brand names of medications, reason for use, route, dose, and start and end dates. This also includes drugs used on a chronic or as-needed basis.

Previous medication is defined as medication with at least one dose taken before the date of the first dose of the study drug.

Concomitant medication is defined as medication with at least one dose taken between the date of first dose (inclusive) and the date of last dose (inclusive) of the study drug.

A list of prohibited medications is given in Appendix 2: List of Excluded Concomitant Medications

When the start and stop dates of a medication or therapy are partial/missing, the dates will be imputed using the rules in Section 7.11.1.5

## 6.5.3 Exposure to Study Drug

The duration of exposure to each dose of study drug (PED25 and PED50) by visit and for the whole period will also be calculated using the following information that is recorded in the eCRF:

- Overall start date and stop date of the study medication.
   The first dose of study drug is to be administered on Day 1, the day after the baseline visit (Visit 3). The initial dose will be PED25 for all subjects. The last dose of treatment is to be taken in the morning of Visit 10.
- Start date and new dose of study drug at each titration step.
   At Visits 4, 5 and 6 the dose may be up-titrated, down-titrated, or may remain the same.
- Start date and new dose of study drug after each unscheduled dose change.
- At any time during the treatment period, the subject may have an unscheduled dose interruption or reduction. At each unscheduled change in dose, the new dose, start date and reason are recorded. Dose increasing is scheduled only during time window between Visit 4/Week 2 and Visit 6/Week 8.

In addition, the return date of study medication is assumed to be the date of clinical visit.

In all cases where there is a dose change, either because of dose titration or an unscheduled dose interruption, reduction or increase, the last dose of the medication at the old level will be assumed to be the day before the given date of first dose at the new level. In this way, the subject's dosing history can be reduced to a series of unbroken intervals within each of which, the dose level is constant. From these, the subject's exposure at each dose can be calculated.

To illustrate, consider a subject with the following dose information on the eCRF:

- The dates of the very first and very last dose of the study medication given as D1=1st July 2016, Dlast=24th September 2016.
- Up-titration to PED50 at Visit 4. The first dose at the new level is given as D2=15th July 2016.

- Study drug interrupted at an unscheduled visit. The date of last dose at the PED 50 level is given as D3=18th July 2016
- Study drug re-started at PED25 at an unscheduled visit. The first dose at the new level is given as D4=22 July 2016.
- Remains at PED25 at Visit 5 (D5=29th July 2016). Up-titration to PED50 at Visit 6. First dose at the new level is given as D6=29thAugust 2016.

From these dates we calculate the following:

- The duration of exposure to the treatment can be calculated as ETOT=Dlast-D1+1-(D4-D3-1)=83 days.
- Between Visits 3 and 4, the subject is on PED25. The last dose at PED25 is given on D2-1, the day before the subject has the first dose at the new level PED50. The exposure at PED25 between Visits 3 and 4 is, therefore, (D2-1)-D1+1=14 days
- Between Visits 4 and 5, the study drug is temporarily suspended and then restarted at a new level. The subject will be considered to be exposed to the PED50 dose from D2 until D3, i.e. D3-D2+1=4 days.
- For the calculation of the exposure, suspension of the study drug is not ignored. The dose will be considered interrupted between D3 to D4-1, i.e. (D4-1-D3)=3 days.
- The study drug is at PED25 from D4 to D6-1, the date of the last dose prior to Visit 6, i.e. (D6-1)-D4+1=38 days.
- Subject is on PED50 from D6 to Dlast, a total of Dlast-D6+1=27 days.
- The total exposure at PED50 is EPED50=31 days, at PED25 is EPED25=52 days
- The total exposure between Visits 3 and 4 is E1=14 days, between Visits 4 and 5 is E2=11 days, between Visits 5 and 6 is E3=31 days and between Visits 6 and 7 is E4=27 days.

## 6.5.4 Compliance to Study Drug

### **Tablet compliance**

Compliance will be calculated according to the number of tablets of study medication dispensed, the number of kits used and the duration of exposure between the applicable visits and overall.

Each kit of study medication contains 35 tablets. At each dispensing visit, subjects will receive an adequate number of kits of both PED25 and PED50 as follows:

- At Visit 3, 1 kit of 25 mg and 1 kit of 50 mg will be dispensed
- At Visit 5, 2 kits of 25 mg and 2 kits of 50 mg will be dispensed
- At Visit 7, 3 kits of 25 mg or 3 kits of 50 mg will be dispensed
- At Visit 8, 7 kits of 25 mg or 7 kits of 50 mg will be dispensed

The total number of tablets used between Visits i and j (i < j) is calculated as:

N<sub>used</sub> = Total number of tablets dispensed at Visit i - Total number of tablets returned at Visit j

When a kit is not returned it will be assumed that all the medication from this kit was not used.

When a kit is returned late, it will be assumed that the medication was used during the study period that it was dispensed for, e.g. all the medication used from a kit dispensed at Visit 3 and returned at Visit 5 will be assumed to have been used between Visits 3 and 5.

The amount of expected study drug intake depends on the number of days of study drug treatment and the number of prescribed daily tablets. Since subjects are supposed to take 1 tablet per day, the total number of expected tablets to be used between Visits i and j is calculated as follows:

 $N_{prescribed}$  = (Number of Exposure Days between Visit\_i and Visit\_j) x 1 tablet, where Number of Exposure Days is calculated as: (Return date – Dispense date ) + 1. Between Visits i and j the compliance to study medication will be calculated as follows:

Compliance = 
$$(N_{used} / N_{prescribed}) \times 100\%$$
.

To illustrate, at Visit 3 a subject was dispensed 1 kit of 25 mg and 1 kit of 50 mg. The date of first dose was 1<sup>st</sup> July 2016. When the subject returned at Visit 4 (18<sup>th</sup> July 2016), the 25 mg kit contained 20 tablets and the 50 mg kit was full (35 tablets).

$$N_{used} = (35-20) + (35-35) = 15 \text{ tablets}$$
 Number of exposure days =  $(18Jul2016 - 01Jul2016) + 1day = 18 days$ , Hence,  $N_{prescribed} = 18 \text{ tablets}$  Compliance between Visits 3 and 4 =  $(15/18) \times 100\% = 83.3\%$ .

For the whole study period, the total amount of study drug used (TOTN $_{used}$ ) is equal to the sum of the values of N $_{used}$  at each applicable visit. Similarly, the total amount of study drug prescribed (TOTN $_{prescribed}$ ) is equal to the sum of the values of N $_{prescribed}$  at each applicable visit. Using these total values, the subject's compliance over the whole study period can be calculated as 100% x (TOTN $_{used}$ / TOTN $_{prescribed}$ ).

### **Suspension Compliance**

Compliance for suspension will be calculated according to:

- Number of bottles dispensed at each visit (see <u>Table 10</u>);
- Weight of the bottles returned to the site; and
- Duration of exposure between the applicable visits and overall.

Number of Kits to be Dispensed at each Visit

| | | Number of kits | | | | |
|---|---|---|---|---|---|---|
| Dose Level | Weight | Visit 3 /<br>Baseline | Visit 5 /<br>Week 4 | Visit 7 /<br>Week 12 | Visit 8 /<br>Week 24 | Visit 9 /<br>Week 36 |
| PED25 | <22 kg | 4 | 6 | 5 | 6 | 7 |
| | 22 - <35 kg | 5 | 8 | 6 | 7 | 8 |
| | ≥ 35 kg | 6 | 10 | 8 | 9 | 11 |
| PED50 | <22 kg | NA | 6 | 8 | 9 | 11 |
| | 22 - <35 kg | NA | 8 | 11 | 11 | 14 |
| | > 35 kg | NA | 10 | 14 | 15 | 19 |

NA: Not Applicable

Table 10

Each kit of study medication contains a bottle with mirabegron granules. After filling the bottle containing the granules with 100 mL drinking water, the weight of the bottle with content should be 137 g.

Doses are calculated weight-based, see Table 11 The body weight at Visit 3/baseline determines the weight range for the starting dose (PED25) and the up-titration dose (PED50) to be used.

Table 11 Weight based Doses for Suspension

| Dose Level | Weight Range | Suspension Volume † |
|------------|--------------|---------------------|
| PED25 | 11 - < 22 kg | 3 mL |
| | 22 - < 35 kg | 4 mL |
| | ≥ 35 kg | 6 mL |
| PED50 | 11 - < 22 kg | 6 mL |
| | 22 - < 35 kg | 8 mL |
| | ≥ 35 kg | 11 mL |

PED25: Pediatric equivalent dose 25 mg; PED50: Pediatric equivalent dose 50 mg † Suspension strength: 8 mg/mL

At each dispensing visit, subjects will receive an adequate number of kits of both PED25 and PED50 following the same procedure as descripted above for tablets.

The total dose of suspension used between Visits i and Visit j ( $i \le j$ ) is calculated as:

 $W_{used}$  = Total weight of bottles dispensed at Visit i - Total weight of bottles returned at Visit j, and taking into account the suspension strength of 8 mg/mL.

#### where:

- Total weight dispensed = Number of kits dispensed at the Visit i x 137; and
- Total weight returned = Sum of the unused amount of study medication in each kit returned at Visit j.

When a kit is not returned it will be assumed that all the medication from this kit was not used.

When a kit is returned late, it will be assumed that the medication was used during the study

period that it was dispensed for, e.g. all the medication used from a kit dispensed at Visit 3 and returned at Visit 5 will be assumed to have been used between Visits 3 and 5.

The amount of expected study drug intake depends on the number of days of study drug treatment and the number of prescribed daily suspension pouches. Since subjects are supposed to administer 1 dose per day, the total amount of expected suspension to be used between Visit i and Visit j is calculated as follows:

W<sub>prescribed</sub> = Duration in days between Visit i and Visit j times the subject's specific dose, see Table 11

The weight of the subject's specific dose is determined by using a conversion factor of 1 mL corresponds to 1.0216 g.

The compliance to study medication between Visits i and j will be calculated as follows:

Compliance = 
$$(W_{used} / W_{prescribed}) \times 100\%$$
.

To illustrate, a subject, who weighted 25 kg and with dose level PED25, was dispensed with 5 kits at Visit 3. The date of first dose was 1<sup>st</sup> July 2016. When the subject returned at Visit 4 (31<sup>th</sup> July 2016), 3 kits were not used and the weight of the 2 used kits was: 32 and 124 g.

## Compliance calculation:

- 1. Total amount of reconstituted study drug administered was resolved in (137-32) + (137-124) = 118 g of suspension, which is equal to 118/1.0216 mL = 115.5 mL.
- 2. Given that the solution strength is 8 mg/mL this means that in total 115.5 mL x 8 mg/mL = 924 mg of study drug was administered to the subject.
- 3. Duration was 31 days (= 31 July 1 July +1), hence expected amount of study drug to be administered is 31 x 4 mL = 124 mL (based on the weight of the subject the suspension volume is 4 mL, see Table 11). This results in 124 mL x 8 mg/mL = 992 mg of study drug.
- 4. Compliance between Visits 3 and  $4 = (924/992) \times 100\% = 93.15\%$ .

For the whole study period, the total amount of study drug used (TOTW<sub>used</sub>) is equal to the sum of the values of  $W_{used}$  at each applicable visit. Similarly, the total amount of study drug prescribed (TOTW<sub>prescribed</sub>) is equal to the sum of the values of  $W_{prescribed}$  at each applicable visit. Using these total values, the subject's compliance over the whole study period can be calculated as  $100\%*TOTW_{used}/TOTW_{prescribed}$ .

## 7 STATISTICAL METHODOLOGY

## 7.1 General Considerations

All statistical analyses and summary information are to be generated according to this analysis plan. Any deviation from this plan will be documented in the final study report.

For continuous variables, descriptive statistics will include the number of subjects (n), mean, standard deviation, median, minimum and maximum. When needed, the use of other percentiles (e.g.10%, 25%, 75% and 90%) will be mentioned in the relevant section. Frequencies and percentages will be displayed for categorical data. Percentages by categories will be based on the number of subjects with no missing data, i.e. will add up to 100%.

Subjects who were screening failures or who were treated but withdrew from the study will be counted only once in summary tables. Information from both screening numbers will be shown in the individual subject listings.

Listings will be produced separately for children and adolescents, unless specified otherwise.

All statistical comparisons will be made using 2-sided tests at the  $\alpha$ =0.05 significance level unless specifically stated otherwise. All summaries will be presented by age group and overall, unless specifically stated otherwise. All null hypotheses will be of no change from baseline, all alternative hypotheses will be 2-sided, unless specifically stated otherwise.

Missing primary efficacy endpoint values will be analyzed using the Last Observation Carried Forward (LOCF) method at Week 24. More details are provided in the relevant sections of this SAP.

All data processing, summaries, and analyses will be performed using SAS® Version 9.3 or higher on Unix. Specifications for table, figure, and data listing formats can be found in the TLF specifications for this study.

# 7.2 Study Population

## 7.2.1 Disposition of Subjects

The following subject data will be presented:

- Number and percentage of subjects who
  - were included in the All Screened Set (i.e. who gave informed consent/assent);
  - were a screening failure;
  - were eligible for study drug treatment.
- Number and percentage of subjects in the All Allocated Set, FAS, PPS, SAF and PKAS:
- Number and percentage of subjects in the All Screened Set who completed or discontinued pretreatment period, by the primary reason for screening status;
- Number and percentage of subjects who completed or discontinued treatment period, by the primary reason for discontinuation, for All Allocated Set, SAF, FAS, PPS and PKAS;

- Number and percentage of subjects who completed or discontinued end of study period, by the primary reason for discontinuation, for All Allocated Set, SAF, FAS, PPS and PKAS;
- Number and percentage of subjects in the FAS who were excluded from the PPS by reason for exclusion (defined in Section 5.4.1).

The number of subjects will be tabulated by protocol version for the All Subjects Screened.

A listing of all early withdrawals, subjects who withdraw within 7 days, will be presented irrespectively whether they were dosed or not. The reason for withdrawal will be included in this listing.

A listing of screen failure with the primary screen failure reason will be provided for the screening failure subjects. In addition, disposition will be listed for All Allocated Subjects with treatment and study discontinuations.

## 7.2.2 Protocol Deviations

Protocol deviations as defined in the study protocol (see Section 8.1.6 Protocol Deviations) will be assessed for All Allocated Set.

The number and percentage of subjects with any deviation criterion will be summarized for each criterion and overall, by age group as well as by study site. Subjects deviating from a criterion more than once will be counted once for the corresponding criterion. Any subjects who have more than one protocol deviation will be counted once in the overall summary. A data listing will be provided by site and subject for the All Allocated Set.

The protocol deviation criteria will be uniquely identified in the summary table and listing. The unique identifiers will be as follows:

- PD1 Entered into the study even though they did not satisfy entry criteria
- PD2 Developed withdrawal criteria during the study and was not withdrawn
- PD3 Received wrong treatment or incorrect dose
- PD4 Received excluded concomitant treatment
- † Subjects who are discontinued within the first 7 days of dosing, after the centrally read urodynamic trace or the ECG results from visit 3/baseline show the subject is no longer fulfilling the eligibility criteria, will not result in a protocol deviation.

A listing of inclusion and exclusion criteria, listing of first and last evaluations as well as a listing of subjects who were excluded from at least 1 analysis set will be provided for the All Allocated Set.

## 7.2.3 Demographic and Other Baseline Characteristics

Demographic and other baseline characteristics will be summarized by age category and overall.

Demographic and other baseline characteristics data will be provided in listing format by site and subject for the All Screened Set.

The number and percentage of subjects allocated to treatment in each region, country and site will be presented for the SAF.

Regions are defined as follows:

- Europe: Norway, Latvia, Lithuania, Denmark, Belgium, Poland, Slovakia, Romania and Serbia
- Asia and Pacific (APAC): Philippines, South Korea, Australia, Taiwan and Malaysia
- Middle East and North Africa (MENA): Turkey, Israel and Jordan
- Latin America (LatAm): Mexico and Colombia

The final list of participating/enrolling countries might be updated after end of recruitment when the list becomes final.

If sites in additional countries will be opened due to changes in recruitment strategy, these countries will be allocated respectively and reported in the CSR.

Descriptive statistics for age, height, weight, and BMI at screening will be presented as well as frequency tabulations for sex, ethnicity and race. In addition, summaries for height with respect to age- and sex-specific percentiles (Charts from the Centers for Disease Control and Prevention (CDC), See 10.6 and 10.7), and weight with respect to height- and sex- specific percentiles (CDC, See 10.8 and 10.9) will be provided. These summaries will be produced for the SAF, FAS and PPS.

Collection of date of birth depends on local regulations. Day of birth will be recorded in the eCRF as the first of the month when the day is not allowed to be collected. In cases where only year of birth is allowed to be collected, day and month will be recorded in the eCRF as the first of January. Age at Screening will be recalculated in SDTM and ADAM datasets.

Demographic characteristics of subjects on previous antimuscarinic treatment (oxybutynin at screening vs. other treatment from concomitant medications dataset) will be summarized for the FAS, PPS and SAF.

Medical history (NDO Medical History and Medical History Other than NDO) is coded in MedDRA and will be summarized by System Organ Class (SOC) and Preferred Term (PT) using SAF. Subjects will only be counted once per MedDRA level and the medical history will be sorted by descending incidence of the overall SOCs and within PTs.

The data on NDO diagnosis and history, including duration of NDO disease (at first dose of mirabegron), NDO medical condition(s), urethral sphincter activity, retardation, wheelchair bound, surgery (including for closure of spina bifida, shunt for hydrocephalus, other) and time since surgery (calculated in months) will be summarized with descriptive statistics and frequency tabulations as appropriate using SAF.

### 7.2.4 Previous and Concomitant Medications

Previous and concomitant medications (for NDO or other indications) will be coded with WHO-DD, and will be summarized by therapeutic subgroup (ATC 2nd level), chemical

subgroup (ATC 4th level) and preferred WHO name for the SAF. Subjects taking the same medication multiple times will be counted once per ATC level. A medication which can be classified into several chemical and/or therapeutic subgroups is presented in all chemical and therapeutic subgroups. Previous and concomitant medications will be sorted by alphabetical order by Therapeutic Subgroup and Chemical Subgroup and Preferred WHO Name.

A summary of all previous medications and concomitant medications will be produced for the NDO and non-NDO medications separately using SAF. Only the last NDO medication before start of study medication will be used for calculations.

Previous and concomitant NDO medications, non-NDO medications and non-NDO non-medication therapies will be listed using All Screened Subjects.

A listing of previous and concomitant NDO medications with ATC codes by WHO preferred name will be provided for All Screened Subjects.

# 7.3 Study Drugs

All summaries of this section will be presented by age group, dose group (see below) and overall, unless specifically stated otherwise.

## **7.3.1 Dosing**

As per study schedule (Table 1), all subjects will start with a PED equal to 25 mg of mirabegron (PED25). From visit 4/week 2 to visit 6/week 8 subjects can be:

- 1. up-titrated to PED50 at least once (dose group labelled "25/50") or,
- 2. maintained at PED25 for any reasons for the whole study (dose group labelled "25only").

These 2 dose groups are mutually exclusive and add up to the total number of subjects in the SAF population.

A subject who is up-titrated to PED50 can remain at that dose level, but can also experience a reduction, an interruption or a further increase of the dose. For these reasons, all subjects up-titrated to PED50 will also be categorized on the basis of the duration of their exposure to PED50 (see Section 6.5.3 for more details).

In particular, the following 2 dose groups (within the dose group "25/50") are of interest:

- a. Subjects up-titrated to PED50 for at least of 4 weeks (28 days) [dose group labelled "50min4w"],
- b. Subjects up-titrated to PED50 for at least 2 weeks (14 days) [dose group labelled "50min2w"].

These two groups are <u>not mutually</u> exclusive and do not add up to the total number of subjects in the "25/50" dose group.

The following information on the study drug dose titration will be presented for the SAF:

• Number and percent of subjects in each dose group ("25/50", "25only", "50min4w" and "50min2w") at each follow-up visit (Visits 4, 5, 6, 7, 8, 9 and 10),

- Number and percent of subjects with dose increases, decreases or no changes at each titration step (from Visit 4 to 6),
- Unscheduled dose changes and interruptions (will be listed only).

Details of dose calculation and drug dispensing will be listed for each subject at each visit.

## 7.3.2 Exposure

The following information on drug exposure will be presented for the SAF:

 Descriptive statistics for cumulative amount of the drug subject was exposed to and average daily dose; and

Duration of exposure will be summarized in the following ways.

- Descriptive statistics
- Exposure time will be categorized according to the following categories for both the titration period and the fixed dose period:
  - o less than 14 days
  - o at least 14 days, less than 28 days
  - o at least 28 days, less than 56 days
  - o at least 56 days
  - Unknown

and by the following categories for the whole treatment period:

- less than 84 days
- o at least 84 days, less than 168 days
- o at least 168 days, less than 252 days
- o at least 252 days, less than 364 days
- o at least 364 days
- Unknown

Counts and percentages of subjects in each of these categories will be summarized for each dose group and overall for the SAF.

## 7.3.3 Treatment Compliance

Compliance with the dosing schedule will be summarized for subjects in the SAF.

The following summaries will be produced separately for the titration period (Visit 3 to Visit 7)<sup>18</sup>, for the period between Visit 7 and Visit 8, and for the whole treatment period:

- Descriptive statistics
- Percent compliance will be categorized according to the following categories:
  - o less than 70%
  - o at least 70%, less than 80%
  - o at least 80%, less than 120%

<sup>\*</sup> Period from Visit 3 to Visit 7 was chosen because no drug dispensing and collecting data is obtained at Visit 4 and Visit 6.

- o at least 120%, less than 130%
- o at least 130%
- Unknown.

A subject will be considered compliant if the calculated compliance over the whole treatment period is at least 70% and is additionally at least 80% between Visit 7 and Visit 8.

Treatment compliance details, including all data relevant to the calculation, will be listed by for each subject by study visit and overall.

## 7.4 Analysis of Efficacy

Efficacy data will be summarized for the FAS and the PPS for all visits.

Baseline for efficacy variables is the last assessment made prior to the first intake of study drug at visit 3 (day -1).

Visit windows will be applied as defined in Section 7.11

## 7.4.1 Analysis of Primary Endpoint

## 7.4.1.1 Primary Analysis of Primary Endpoint/Estimand

The primary efficacy variable is the change from baseline in MCC at visit 8/week 24.

MCC and change from baseline in MCC at visit 8/week 24 will be summarized using descriptive statistics for continuous variable (n, mean, SD, min, median, and max) for the FAS. Missing MCC observations at visit 8/week 24 will be imputed using the Last Observation Carried Forward (LOCF) method.

In accordance with the definition of the estimand, the change from baseline in MCC at visit 8/week 24 will be analyzed using a paired t-test. The following hypotheses will be tested at the 2-sided significance level 0.05:

- H<sub>0</sub>: Mean change from baseline in MCC at visit 8/ week 24 is equal to zero
- H<sub>1</sub>: Mean change from baseline in MCC at visit 8/ week 24 in MCC is not equal to zero

The mean change from baseline estimate in MCC at visit 8/week 24, together with two-sided 95% CI and the t-test p-value will be provided using the UNIVARIATE procedure in SAS.

Example SAS code is as follows:

```
proc univariate;
    class time;
    var chgebc;
run;
```

In addition to the test of the null hypothesis, it will be assessed whether the lower bound of the two-sided 95% CI excludes 0 mL. No adjustment for multiplicity will be made.

MCC at each visit and change from baseline in MCC at visit 8/week 24 (without LOCF) will be also plotted and listed for SAF and PPS.

## 7.4.1.2 Secondary Analyses of Primary Endpoint

The following secondary analyses of the primary endpoint will be produced.

## 7.4.1.2.1 Analysis without LOCF

The same analysis described in Section 7.4.1.1 will be repeated both for FAS without imputing for missing data and for PPS.

## 7.4.1.2.2 Analysis using Baseline Value Carried Forward

For cases were the MCC value is non-missing at baseline but missing at visit 8/week 24, the same analysis as described in Section 7.4.1.1 will be performed using a Baseline Observation Carried Forward (BOCF) approach. For this analysis the baseline value will be imputed for the missing value at Visit 8/week 24.

This analysis will be performed for the All Enrolled Subjects.

## 7.4.1.2.3 Analysis using Repeated Measures ANCOVA

A repeated measures ANCOVA will be performed considering the change from baseline (without LOCF) and baseline MCC. This analysis will serve as a sensitivity analysis to the LOCF method used in the primary model to assess the robustness of the findings. Data obtained at baseline (visit 3), at visit 5/week 4 and at visit 8/week 24 will be used. Since there are only 2 post-baseline time points in a 24 week period, the model will assume an unstructured covariance among the within subject repeated measurements. If there is a convergence problem due to the unstructured covariance matrix, the unstructured covariance matrix will be replaced by the compound symmetry covariance matrix. This analysis will be performed both for FAS and PPS.

Example SAS code is as follows:

```
proc mixed;
    class subject agegroup visit;
    model change = visit agegroup agegroup*visit MCC_baseline;
    repeated visit / subject=subject type=un;
    lsmeans visit agegroup*visit / diff cl alpha=0.05;
run;
```

In this code the LSMEANS statement will produce least squares mean (LS mean) estimates for both age groups combined and also within each age group using a single analysis of covariance (ANCOVA) model.

Model fitting will be visually assessed. A scatter plot of residuals versus predicted values, along with histogram and normal probability plots will be produced.

## 7.4.1.2.4 Effect of age and gender

The p-value of the change from baseline to week 24 (with and without LOCF) will be assessed using an ANCOVA model including gender, age group and a gender by age group interaction as fixed effects and the baseline MCC as a covariate.

LS mean estimates, together with 95% CIs, will be provided.

Example SAS code is as follows:

```
proc mixed;
   class agegroup gender;
   model change = agegroup gender agegroup*gender
   MCC baseline;
   lsmeans gender agegroup*gender / diff cl alpha=0.05;
run;
```

In this code the LSMEANS statement will produce LS mean estimates for both age groups combined and also within each age group using a single ANCOVA model.

## 7.4.1.2.5 Nonparametric Analysis of Primary Endpoint

A Wilcoxon signed-rank test will be used as a sensitivity analysis. This test is produced by the UNIVARIATE procedure in SAS and ranks the absolute values of the differences between the paired data and calculates a statistic on the number of negative and positive differences. Analysis will be done on the FAS, with (LOCF) and without imputation.

Example SAS code is as follows:

```
proc univariate;
    var chg;
run;
```

Box-Whisker plots of the change from baseline data will be presented for getting insight into the distribution of the data.

### 7.4.1.2.6 Overall Impact on Primary Endpoint

For the MCC, the 95% CI will be calculated for mean change from baseline per age group, per formulation, and per dosing regimen (with and without LOCF), using an ANCOVA model.

In addition to the hypothesis testing test, it will be assessed whether the lower bound of the two-sided 95% CI excludes 0 mL.

In addition, the nonparametric Wilcoxon signed-rank test on change from baseline data will be performed. Only statistical hypothesis testing (p-values) will be performed.

Analyses will be performed on the FAS, with (LOCF) and without imputation.

## 7.4.1.2.7 Sensitivity Analysis of the Primary Estimand

As a sensitivity analysis for the estimand, the change from baseline to weeks 4 and 24 in MCC will be analyzed using a mixed-effect model repeated measures (MMRM) with week as fixed effect and baseline value and week by baseline interaction as covariates. The contrast between baseline and week 24 will be the primary statistical inference obtained from this model.

<sup>&</sup>lt;sup>†</sup> Dosing regimen here refers to whether the subjects had been up-titrated to PED50 at least once or maintained at PED25 for safety reasons at least until visit 8/week 24.

The MMRM analysis will present the least square (LS) mean estimate, standard error (SE), and 2-sided 90% CI for change from baseline to each treatment week. The differences in the LS mean estimates will be used to obtain 1-sided P values for MCC at week 24 versus MCC at baseline.

Since there are only 2 post-baseline time points in a 24 week period, the model will assume unstructured covariance among the within subject repeated measurements. If this is not feasible, an additional covariance structure will be considered the compound symmetry covariance matrix.

## 7.4.2 Analysis of Secondary Endpoints

Each of the secondary efficacy endpoints will be summarized with descriptive statistics (n, mean, SD, min, median, max for continuous variables; frequency and percentage for categorical variables) at each visit and for change from baseline at each visit when applicable. Each of the secondary efficacy endpoints will be plotted by visit change from baseline will also be plotted at each visit, if applicable.

The change from baseline for each continuous secondary efficacy endpoint (without LOCF) will be summarized and analyzed using the same t-test (see section 7.4.1.1) as for the primary efficacy endpoint. The mean change from baseline estimate together with 95% CI and the relative p-value will be provided using the UNIVARIATE procedure in SAS.

For the analysis of Bladder Volume until first detrusor contraction (>15 cm H<sub>2</sub>O mL) expressed as MCC, a Wilcoxon signed-rank test will be used to compare Change from Baseline at Week 4 and at Week 24 (without LOCF) with 0.

The following hypotheses will be tested:

H<sub>0</sub>: Medians of bladder volumes expressed as MCC are equal at Baseline and Week 24 (Change from Baseline=0)

H<sub>1</sub>: Medians of bladder volumes expressed as MCC differ at Baseline and Week 24 (Change from Baseline differs from 0)

The Wilcoxon signed-rank test p-value will be provided.

Example SAS code is as follows:

```
proc univariate;
    class time;
    var chgebc;
run;
```

The medians (with first and third quartiles) of the Bladder Volumes as MCC will be presented for Baseline and Week 24. Furthermore, Box-whisker plots will be presented.

Additionally, a graph will present the Bladder Volumes as MCC (on the horizontal axis) using Detrusor Contraction as event indicator variable. The percentage of subjects will be shown on the vertical axis. Baseline and week 24 values will be overlaid on the same graph.

Example SAS code is as follows (where 'Status'=0 if the value is censored, and 1 otherwise):

```
ods trace on/listing;
ods output ProductLimitEstimates= RisKNumbers;
proc lifetest data=km atrisk plots=survival(cb=hw atrisk) outsurv=s1;
    time change * Status(0);
    strata visit;
run;
ods trace off;
```

Separate analyses will be performed including and excluding subjects who had censored change from baseline.

All analyses of secondary endpoints will be produced for subjects in the FAS.

CGI-C and acceptability results will be tabulated per time point of assessment.

## 7.4.3 Analysis of Exploratory Endpoints

Each of the exploratory efficacy endpoints and changes from baseline will be summarized and plotted by visit.

The change from baseline for each continuous exploratory endpoint (without LOCF) will be summarized and analyzed using the same t-test (see section 7.4.1.1) as for the primary efficacy endpoint.

All analyses of exploratory endpoints will be produced for subjects in the FAS.

The data will be summarized with descriptive statistics according to the nature of variables (n, mean, SD, SEM, 95% CI, min, median, max for continuous; frequency and percentage for categorical) at each visit and for change from baseline.

A listing will be presented for subjects with a filling volume of >40 cm H<sub>2</sub>O detrusor pressure at week 24. Listing will, among other, present the MCC and MCC expressed as % of EBC.

## 7.4.4 Analysis of Other Variables

There are no other efficacy endpoints in this study.

## 7.4.5 Sensitivity Analysis

Due to measurement mistakes it was found that for some assessments negative values were recorded in e-diary for the weight of urine. This affected the following parameters:

- Average catheterized volume per catheterization
- Maximum catheterized volume
- Maximum catheterized daytime volume
- Average morning catheterized volume (based on first catheterization after subject woke up)
- Total catheterized volume per day

- Average morning catheterized volume for subjects with no leakage during the sleeping time (based on first catheterization after subject woke up)
- Average morning catheterized volume for subjects with leakage during the sleeping time (based on first catheterization after subject woke up)

As a consequence of this measurement mistake a sensitivity analysis will be performed for these parameters, which will exclude all subjects with at least 1 negative value.

For each visit, the change from baseline for each efficacy endpoints will be summarized and analyzed using the same t-test (see section 7.4.1.1) as for the primary efficacy endpoint. The mean change from baseline estimate together with 95% CI and the relative p-value will be provided using the UNIVARIATE procedure in SAS.

# 7.5 Analysis of Safety

Unless specified otherwise, safety data will be summarized for the SAF.

Safety parameters such as vital signs and weight will also be summarized with respect to height- and sex-specific percentiles. Height will also be summarized with respect to age- and sex-specific percentiles.

Subgroup presentations regarding age (children and adolescents), formulation (tablets and suspension) and dosing regimen (PED25 and PED50) will be tabulated for the following parameters: AEs, vital signs and ECGs. For any of the subgroups specified, at least 10 subjects by stratum are required.

Summaries will be provided for the SAF unless otherwise specified, whereas listings will be provided for the All Allocated Set. Visit windows will be applied to all data except AEs, as defined in Section 7.11.3

Summaries and listings of SAEs and Serious TEAEs include SAEs upgraded by the sponsor based on review of the Sponsor's list of Always Serious terms if any upgrade was done.

#### 7.5.1 Adverse Events

The MedDRA coding dictionary will be used to summarize the AEs in this study by SOC, HLT and PT.

An overview table will include the following details:

- Number of TEAEs and number and percentage of subjects with TEAEs
- Number of drug-related TEAEs and number and percentage of subjects with drugrelated TEAEs
- Number of serious TEAEs and number and percentage of subjects with serious TEAEs
- Number of serious drug-related AEs and number and percentage of subjects with serious drug-related AEs
- Number of TEAEs leading to permanent discontinuation of study drug and number and percentage of subjects with TEAEs leading to permanent discontinuation of study drug.

- Number of drug-related TEAEs leading to permanent discontinuation of study drug and number and percentage of subjects with drug-related TEAEs leading to permanent discontinuation of study drug,
- Number of TEAEs leading to death and number and percentage of subjects with TEAEs leading to death,
- Number of drug-related TEAEs leading the death and number and percentage of subjects with TEAEs leading to death
- Number and percentage of subjects who died.

The number and percentage of AEs which started after Visit 1 and before the first dose of study drug will be summarized by SOC, HLT (only for the table presenting TEAEs) and PT, as well as by worst intensity (mild, moderate or severe) using SAF.

All summaries will be sorted alphabetically by SOC and within SOC by descending frequency of PT for all subjects combined (overall), or alphabetically by SOC and within SOC by HLT (descending frequency) and within HLT by descending frequency of PT for all subjects combined (overall), the latter only for the table presenting TEAEs.

The number and percentage of subjects with TEAEs, as classified by SOC and PT will be summarized using SAF. Summaries will be provided for:

- TEAEs (by SOC, HLT and PT)
- Drug-related TEAEs
- Serious TEAEs
- Drug-related serious TEAEs
- TEAEs leading to permanent discontinuation of study drug
- Drug-related TEAEs leading to permanent discontinuation of study drug
- TEAEs leading to death
- Drug-related TEAEs leading to death
- TEAEs excluding serious adverse events that equal or exceed a threshold of 5.0%, regardless of dose
- TEAEs including serious adverse events that equal or exceed a threshold of 2.0%, regardless of dose

The number of TEAEs and the number and percentage of subjects with TEAEs as classified by SOC and PT will also be summarized by worst severity (mild, moderate, severe), by worst relationship to study drug (not related, possibly related, probably related) and by time intervals categories. In the subject count, if a subject has multiple TEAEs with the same SOC or PT, but with differing severity, then the subject will be counted only once with the worst severity, however, if any of the severity values are missing then the subject will be counted only once with missing severity. Similarly, in the subject count, if a subject has multiple TEAEs with the same SOC or PT, but with differing relationship, then the subject will be counted only once with the highest degree of relationship, however, if any of the relationship values are missing then the subject will be counted only once with missing relationship. If category for the same AE is missing, missing should be used, else use maximum relationship.

Time intervals are based on time from first dose of study drug and will be categorized according to the following categories:

- less than 2 weeks (i.e. less than 14 days);
- at least 2 weeks, less than 4 weeks (i.e. at least 14 days and less than 28 days);
- at least 4 weeks, less than 8 weeks (i.e. at least 28 days and less than 56 days);
- at least 8 weeks, less than 12 weeks (i.e. at least 56 days and less than 84 days);
- at least 12 weeks, less than 24 weeks (i.e. at least 84 days and less than 168 days);
- at least 24 weeks, less than 36 weeks (i.e. at least 168 days and less than 252 days);
- at least 36 weeks, less than 52 weeks (i.e. at least 252 days and less than 364 days); and
- at least 52 weeks (i.e. at least 364 days).

At risk denominators for summaries by time interval for onset and by time interval for prevalence will be the same across all AE categories (Overall, SOC and PT), i.e. a subject is at risk in all time period denominators up to EOS.

At risk denominators for summary by time intervals for first onset will depend on AE category and time interval according to the following algorithm:

- For each subject, day of first AE onset is determined for each AE category (Overall, SOC and PT).
- Within each AE category, a subject is at risk in all time intervals denominators up to the first AE onset.

If there is no first AE then the subject will be included in all time intervals up to EOS.

Drug related TEAEs will be presented in a similar way.

AEs of interest are described in Section 6.2.2 and will be summarized for PT only (no SOC).

#### 7.5.1.1 Adverse Events of Interest

For each of the TEAEs of interest, the frequency of TEAEs will be summarized by PT.

## 7.5.2 Clinical Laboratory Evaluation

All laboratory data will be summarized using SAF.

The baseline visit is the last measurement taken prior to initial study drug administration.

Quantitative clinical laboratory variables, i.e. hematology, biochemistry, and urinalysis will be summarized separately using mean, standard deviation, minimum, maximum and median at each visit. Additionally, a within-subject change will be calculated as the post-baseline measurement minus the baseline measurement and summarized in the same way.

Values lower than the limit of quantification (LOQ) for laboratory parameters will be set to 0 for the calculation of descriptive statistics.

Each laboratory result will be classified as low (L), normal (N), or high (H) at each visit according to the laboratory supplied reference ranges. The number and percentage of subjects

below and above reference range will be summarized at each visit according to the laboratory supplied reference ranges.

Frequency tabulations of qualitative clinical laboratory variables (urinalysis) will be presented at each visit.

Hematology and biochemistry results will be collected at visit 1/screening, visit 3/baseline, visit 7/week 12 and visit 10/EoT visit. Shifts from Baseline to Week 12 and EoT will be summarized by two types of shift tables:

- Shift tables of reference range (low, normal, high) changes from baseline to Week 12 and EOT, and.
- Summary shifts of reference range changes from baseline to Week 12 and EOT. These shifts are categorized as:
  - o "Shift to Low": shift from normal or high to low
  - o "Shift to High": shift from normal or low to high
  - "Categorized Increase": shift from low to normal or from normal to high
  - o "Categorized No Change": value stays in the same reference range
  - o "Categorized Decrease": shift from high to normal or from normal to low.

All clinical laboratory data collected during the study and variables derived from it will be listed using SAF.

#### 7.5.2.1 Liver function tests

The following potentially clinically significant criteria for liver tests – defined as Alkaline Phosphatase (ALP), Alanine Transaminase (ALT), total bilirubin, Aspartate Transaminase (AST) and their combination are defined. The subject's highest value during the investigational period will be used.

| <u>Parameter</u> | Criteria |
|---|---|
| ALT | > 3xULN |
| | > 5xULN |
| | > 10xULN |
| | > 20xULN |
| AST | > 3xULN |
| | > 5xULN |
| | > 10xULN |
| | > 20xULN |
| ALT or AST | > 3xULN |
| Total Bilirubin | > 2xULN |
| ALP | > 1.5xULN |
| ALT and/or AST AND Total Bilirubin * | (ALT and/or AST $> 3xULN$ ) and |
| | total bilirubin > 2xULN |
| ALT and/or AST AND Alkaline Phosphatase | ALT and/or AST $> 3xULN$ AND Alkaline |
| AND Total Bilirubin * | Phosphatase < 2xULN AND Total Bilirubin |
| | > 2xULN |

The number and percentage of subjects with potentially clinically significant values in liver enzyme and total bilirubin tests during the investigational period will be presented

## 7.5.3 Vital Signs

#### 7.5.3.1 Clinic Measurement

Values and changes from baseline for vital signs (SBP, DBP, pulse rate and measurement for temperature) and percentiles of SBP, DBP and Pulse Rate compared to age and height norms (see section 10.6 and 10.7 for Blood Pressures and section 10.5 for Pulse Rate) will be listed and summarized at each scheduled visit using mean, standard deviation, minimum, maximum and median. The number and percentage of subjects outside reference ranges will be shown.

For shifts from baseline to each post-baseline visit the categories used for presentation were obtained from the Fourth Report (NIH, 2005), considered primary presentation, and from the 2017 (American Academy of Pediatric) Clinical Practice Guidelines, considered supportive presentation.

## Using data from Fourth Report

For each scheduled post-baseline visit, shift tables from baseline to each post-baseline visit will be created with respect to the changes from normal blood pressure ( $<90^{th}$  percentile): to prehypertension (for children between  $90^{th}$  to  $95^{th}$  percentile, or for adolescents if  $\ge 120/80$  mmHg, but less than the  $95^{th}$  percentile); to stage 1 ( $95^{th}$  to  $99^{th}$  percentile + 5 mmHg); and to stage 2 ( $>99^{th}$  percentile + 5 mmHg), using cut-points reported by the Fourth ( $4^{th}$ ) Report (NIH, 2005). For the cut-off points ( $90^{th}$ ,  $95^{th}$  and  $99^{th}$  percentiles) see Appendix 10.1 and Appendix11.1.

## **Using data from 2017 Clinical Practice Guidelines**

For each scheduled post-baseline visit, shift tables from baseline to each post-baseline visit will be presented with respect to the changes from normal blood pressure to elevated blood pressure; stage 1 HTN, or stage 2 HTN, see Table 12 For the cut-off points (90<sup>th</sup>, and 95<sup>th</sup> percentiles) see Appendix 10.2 and Appendix 11.2.

 Table 12
 Definitions of Blood Pressure Categories and Stages

| Children Aged 1-<13 years | Adolescents Aged ≥13 years |
|---|---|
| Normal BP: <90th percentile | Normal BP: <120/<80 mm Hg |
| Elevated BP: ≥90th percentile to <95th | Elevated BP: 120/<80 to 129/<80 mmHg |
| percentile or 120/80 mmHg to <95th percentile | |
| (whichever is lower) | |
| Stage 1 HTN: ≥95th percentile to <95th | Stage 1 HTN: 130/80 to 139/89 mmHg |
| percentile + 12 mmHg, or 130/80 to 139/89 | |
| mmHg (whichever is lower) | |
| Stage 2 HTN: ≥95th percentile + 12 mmHg, or | Stage 2 HTN: ≥140/90 mmHg |
| ≥140/90 mmHg (whichever is lower) | |

Table obtained from: 2017 American Academy of Pediatric Clinical Practice Guidelines, Table 3

Note: the age classification into children and adolescents in the Clinical Practice Guidelines (2017) differs from the definition used in the protocol

Summaries will be presented for SBP and DBP separately, overall and by age group. See further details in see Section 6.2.1.3 Conversion of Blood Pressure to Percentiles.

In addition, PR measurements will be compared to age-related norms [Fleming et al, 2011] according to the percentiles shown in Table 13 Each PR value will be categorized as either below the 1<sup>st</sup> percentile, between the 1<sup>st</sup> and 99<sup>th</sup> percentile (limits included) or above the 99<sup>th</sup> percentile. Summaries will be presented overall and by age group.

For the number of subjects with PR values below and above the normal range, the normal range is defined as:  $1^{st} - 99^{th}$  percentile

Table 13 Percentiles for Pulse Rate in Relation to Age

| | | Percentile | | | | | |
|--------|-----|------------|------|------|------|------|------|
| Age | 1st | 10th | 25th | 50th | 75th | 90th | 99th |
| 3-4y | 70 | 86 | 94 | 104 | 113 | 123 | 136 |
| 4-6y | 65 | 81 | 89 | 98 | 108 | 117 | 131 |
| 6-8y | 59 | 74 | 82 | 91 | 101 | 111 | 123 |
| 8-12y | 52 | 67 | 75 | 84 | 93 | 103 | 115 |
| 12-15y | 47 | 62 | 69 | 78 | 87 | 96 | 108 |
| 15-18y | 43 | 58 | 65 | 73 | 83 | 92 | 104 |

Source: web appendix to the Fleming et al article (web table 5)

## Potentially Clinically Relevant (PCR)




#### 7.5.3.2 Self-Measurements

Similarly to the clinic vital signs measurements (section 7.5.3.1), values and changes from baseline for self vital signs measurements (SBP, DBP, pulse rate) and percentiles of self-measurements SBP and DBP compared to age and gender norms will be listed and summarized at each visit using mean, standard deviation, minimum, maximum and median. The number and percentage of subjects outside reference ranges will be shown.

For shifts from baseline to each post-baseline visit the categories used for presentation were obtained from Stergiou [2007], considered primary presentation, and from the 2017 (American Academy of Pediatric) Clinical Practice Guidelines, considered supportive presentation.

#### Using data from Stergiou [2007]

For each scheduled post-baseline visit, shift tables from baseline to each post-baseline visit will be created with respect to the changes from normal blood pressure (≤95<sup>th</sup> percentile) to abnormal blood pressure (>95<sup>th</sup> percentile), using cut-points reported in Table 14

 Table 14
 Systolic and Diastolic Home Blood Pressure Values

| Height | | Boys | | | Girls | |
|---|---|---|---|---|---|---|
| (cm) | n | 50 <sup>th a</sup> | 95 <sup>th a</sup> | n | 50 <sup>th a</sup> | 95 <sup>th a</sup> |
| 120–129 | 23 | 105/64 | 119/76 | 36 | 101/64 | 119/74 |
| 130–139 | 51 | 108/64 | 121/77 | 51 | 103/64 | 120/76 |
| 140-149 | 39 | 110/65 | 125/77 | 61 | 105/65 | 122/77 |
| 150–159 | 41 | 112/65 | 126/78 | 71 | 108/66 | 123/77 |
| 160–169 | 45 | 115/65 | 128/78 | 148 | 110/66 | 124/78 |
| 170–179 | 91 | 117/66 | 132/78 | 46 | 112/66 | 125/79 |
| 180–189 | 57 | 121/67 | 134/79 | 7 | 114/67 | 128/80 |

<sup>&</sup>lt;sup>a</sup> Values are systolic/diastolic blood pressure (Stergiou, 2007)

#### **Using data from Clinical Practice Guidelines [2017]**

For each scheduled post-baseline visit, shift tables from baseline to each post-baseline visit will be presented with respect to the changes from normal blood pressure to elevated blood

pressure; stage 1 HTN, or stage 2 HTN, see Table 12 For the cut-off points (90<sup>th</sup>, and 95<sup>th</sup> percentiles) see Appendix 10.2 and Appendix 11.2.

#### **Potentially Clinically Relevant (PCR)**



#### 7.5.4 Height and Weight

Height, weight and BMI, and in addition, z-scores and percentiles compared to age and sex norms, will be listed and summarized overall for the SAF for each visit using mean, SD, 95% CI of the mean, median, minimum, and maximum.

The change from baseline to EoT in the z-score will additionally be summarized by displaying the number and percentage of subjects with changes in each of the following categories: <-1.0, >=-1.0 to <-0.5, >=-0.5 to <=0.5, >0.5 to <=1.0, >1.0.

The summary statistics for percentiles will be calculated by transforming the relevant z-score statistic to a percentile of the standard normal curve, e.g. the mean percentile will be the transformed mean z-score, rather than the mean of the individual percentiles. No estimate of SD will be calculated for the percentiles, and no summary statistics will be generated for the change from baseline in percentile.

#### 7.5.5 Electrocardiograms (ECGs)

ECG variables (QT, QTcF, HR, PR, QRS and RR) will be listed and summarized using mean, standard deviation, minimum, maximum and median at each treatment visit, including changes from baseline.

For categorical ECG variables reported by the local investigator, the worst non-missing value among the assessments will be used in the analyses. Number and percentage of subjects with normal, not clinically significant abnormal and clinically significant abnormal results as assessed by the local investigator for the 12 lead ECG will be tabulated at each visit. Abnormal results will be presented for a certain visit if abnormal interpretation was recorded for at least one of the ECGs taken during the measurements for the particular visit.

All abnormalities will be listed together with the respective abnormality code and description.

For categorical ECG variables reported by the central laboratory, the worst non-missing value among the assessments will be used in the analysis. Number and percentage of subjects with abnormalities and number and percentage of subjects with normal and abnormal results as assessed by the central laboratory will be tabulated at each visit. Abnormal results will be presented for a certain visit if abnormal interpretation was recorded for at least one of the ECGs taken during the measurements for the particular visit.

Shift tables will be presented for changes from baseline at each visit including local interpretation categories. Shift tables will also be presented as above from baseline to worst post-baseline value during the treatment period. Similar shift tables will summarize Central Reader interpretation categories.

The corrected QT interval (i.e. QTcF) will be summarized for at each visit showing the number and percentage of subjects with a mean of the triplicate QTc values (ms) in each of the following categories:

For the children category

 $\bullet$  > 440 ms

For the male adolescents category

- $\bullet$  > 450 ms
- $\bullet$  > 500 ms

For the female adolescents category

- $\bullet$  > 480 ms
- $\bullet$  > 500 ms

Note that these categories are cumulative in that subjects satisfying criterion for more extreme category will also be counted in each applicable less extreme category.

The corrected QT interval (i.e. QTcF) will also be summarized for each age group at each visit showing the frequencies of subjects with the following changes from baseline:  $<0, \ge 0$  and  $<30, \ge 30$  and <60,and  $\ge 60$  ms.

#### 7.5.6 Pregnancies

A detailed listing of all pregnancies will be provided if any occur using All Screened Set.

#### 7.5.7 Estimated Glomerular Filtration Rate and Upper Urinary Tract Ultrasound

Values and changes from baseline of plasma creatinine, plasma cystatin C and eGFR levels will be summarized together with the other Biochemistry variables (described in section 7.5.2). The eGFR results will be summarized based upon the Larsson, the modified Schwartz 2009 (for children < 12 years old) and the Cockcroft-Gault equation (for adolescents) using mean, standard deviation, minimum, maximum and median overall at each visit.

Number and percent of subjects with normal, not clinically significant abnormal and clinically significant abnormal ultrasound of the upper urinary tract results will be tabulated for overall at each visit. The results of the ultrasound of the upper urinary tract will be listed. Any clinically-significant abnormality should be recorded as an AE and will be included in the summaries of the AE tables.

# 7.6 Analysis of PK

#### 7.6.1 Estimation of Pharmacokinetic Parameters

| Pharmacokinetic data analysis will be performed by the GCMSL with mixed effects |
|---|
| modeling using NONMEM (version 7.3 or higher, |
| USA). For the analysis, actual sampling times will be used. |

Since the PK sampling is sparse and skewed towards the early phase of the profile with less information in the terminal phase, it is likely that the data from this study may be pooled with other pediatric pharmacokinetic data with richer sampling; this will support the model-based assessment of the following pharmacokinetic parameters for each subject:

$$\bullet \quad C_{max},\,t_{max},\,AUC_{24},\,C_{trough},\,CL/F,\,and\,\,V_z/F$$

Additional pharmacokinetic parameters may be calculated based on the model used. Further details of the derivation of the pharmacokinetic parameters are given in the PK DAP.

#### 7.6.2 Statistical Analysis

Descriptive statistics (n, mean, SD, minimum, median, maximum, coefficient of variation [%CV], and geometric means) will be calculated for all plasma concentrations of mirabegron. Plasma concentration values below the limit of quantification (LOQ, 0.2 ng/mL) will be set equal to 0 in the calculation of summary statistics.

Plasma concentration data in each time window (see <u>Table 15</u>) will be summarized by age category (children and adolescents) and the subjects' treatment dose of mirabegron (PED25, PED50) within the age category.

Table 15 Time Windows for Summary of Plasma Concentration Data

| Target time | Actual Time |
|---|---|
| 2 trough samples | Within 1 hour prior to dosing (on sampling day 1 and 2) |
| 2 samples between 2 h and 5 h post-dose | > 1 hour to 6 hours post-dose (with at least 1 hour in between the |
| 2 samples between 2 if and 5 if post-dose | samples, on sampling day 2) |

Note: Measurements from plasma concentrations outside the time windows will not be included in the summary of the plasma concentrations, but can still be considered for the derivation of pharmacokinetic parameters, which is based on the actual sampling time after study drug intake.

The following plots will be produced:

- Mean (+/-SD) plasma concentration-time profiles (normal scale)
- Mean plasma concentration-time profiles (semi-log scale)
- Box plots of plasma concentration-time profiles (normal scale and semi-log scale)
- Individual subject plasma concentration-time profiles (normal scale "spaghetti plots")
- Individual subject plasma concentration-time profiles (normal scale and semi-log scale plots)

The first two plots will be produced for the PK report.

Further details will be described in the TLF specifications.

The pharmacokinetic analysis and results will be provided in a separate PK modeling report, which will supplement the CSR.

# 7.7 Analysis of PD

There are no PD data to be analyzed in this study.

# 7.8 Subgroups of Interest

The primary efficacy endpoint will be summarized descriptively with and without LOCF (unless otherwise specified) using FAS for the following subgroups:

- Age group (children vs. adolescents);
- Racial subgroups;
- Ethnicity (Hispanic or Latino / Not Hispanic or Latino)
- Formulation (tablets vs. oral suspension);
- Dosing regimen ("25/50" group vs. "25 only", please refer to section 7.3.1
- NDO medication treatment received at screening/prior to start of washout (yes vs. no);
- Stop of antimuscarinics medication specifically intended for NDO treatment (prior to study treatment) for lack of efficacy (yes vs. no [i.e., use of antimuscarinics stopped but for other reasons than for lack of efficacy]), if there are sufficient subject numbers;

 Excluding those subjects who had a positive urine culture at visit 3/baseline, visit 5/week 4, and/or visit 8/week 24 (without LOCF only), if there are sufficient subject numbers.

In addition, selected safety variables (all TEAEs and drug related TEAEs, vital signs, height and weight) will be summarized descriptively using SAF for the same subgroups.

Moreover, the selected safety variables, except for TEAEs, will be summarized with respect to age and sex-specific percentiles.

## 7.9 Other Analyses

There are no other analyses of data in this study.

### 7.10 Interim Analysis (and Early Discontinuation of the Clinical Study)

No interim analysis of the data for this study is planned.

However, safety data will be reviewed by an independent Drug Safety and Monitoring Board (DSMB). Details are described in the DSMB charter and the corresponding DSMB analysis plan.

# 7.11 Handling of Missing Data, Outliers, Visit Windows, and Other Information

#### 7.11.1 Missing Data

Missing primary efficacy endpoint values will be handled by using the Last Observation Carried Forward (LOCF) method. No values at baseline and no data from more than 5 days after the last dose of study medication will be carried forward to post-baseline visits for the analysis of the primary efficacy endpoint on the FAS.

As a general principle, no imputation of missing data for other variables will be done. Exceptions are EoT values for certain safety variables (lab values, vital signs, and ECGs), the start and stop dates of AEs and concomitant treatments, the date of diagnosis of NDO, the diary dates and the times of wake up and go to bed. Listings will present the actual partial dates/times; imputed dates/times will not be shown but derived parameters (e.g. duration of an AE) will be flagged.

#### 7.11.1.1 Imputation Rules for Missing Safety Variables

In case subject safety data (lab values, vital signs, or ECGs) at EoT (visit 10/week 52) is missing, the LOCF method will be used for the summaries of shift from baseline to EoT only. No values at baseline and no data from more than 5 days after the last dose of study medication will be carried forward to post-baseline visits.

#### 7.11.1.2 Imputation Rules for Diary Dates

Each item of diary data is collected with the corresponding page number of the diary on which it was recorded. This page number will be used to match "day" pages of the diary with the corresponding "night" pages. When the date for one of the two pages is missing, it will be imputed with the date from the other page.

When the dates for both pages are missing, or when the dates are present but different, the dates will be queried prior to database hard lock.

The time of waking up and going-to-bed may be imputed when they are missing to enable categorization of hour periods as "day time" or "night time".

If the hour of the wake-up time is missing, the wake-up time will be imputed as occurring a little time prior to the first catheterization, e.g. if the first catheterization is recorded in the 09:00-10:00 hour-period, then the hour of the wake-up time will be imputed as being "09:00". If there is no catheterization before 12:00, then the wake-up time will not be imputed.

If the hour of going-to-bed time is missing, the going-to-bed time will be imputed as occurring a short time after the last catheterization, e.g. if the last catheterization is recorded in the 20:00-21:00 hour-period, then the hour of going-to-bed will be imputed as being "21:00". If there is no catheterization before 24:00, then the going-to-bed time will not be imputed.

If the minutes of the wake-up time or going-to-bed time are missing, they will be imputed as "00.30"

#### 7.11.1.3 Imputation Rules for Adverse Events

If there are missing or incomplete onset dates of AEs, then a worst case scenario will be used for the classification of AEs as TEAEs and for the calculation of the longest possible duration of the AE that is <u>consistent with available information</u>. The eCRF includes a checkbox that asks "If the onset date is the same day as study drug start date or if a complete onset date is unknown, please select one (of the following)" and the 2 options are:

- Onset before first dose of study drug
- 4. Onset after first dose of the study drug

Let these 2 answers be referred to as Onset=Pre and Onset=Post respectively and also consider that the question may be unanswered (i.e. Onset=Missing).

Let the date of the first dose of study medication (not imputed) be DATE<sub>POST</sub>, and the date of onset of the AE be DATE<sub>AE</sub>.

On the assumption that inconsistencies in the data (e.g. Onset=Post, yet the year of onset is too early for this to be possible) have already been corrected, the method for imputing missing parts of a partial AE start date is as follows:

- When Onset=Pre, there will be no imputation of the AE onset date and the AE is not considered a TEAE;
- When Onset=Post, a worst case scenario will impute DATE<sub>AE</sub> to be the <u>earliest</u> date on or after DATE<sub>POST</sub> which is compatible with the non-missing parts of the date;
- When Onset=Missing, a worst case scenario will impute DATE<sub>AE</sub> as though Onset=Post. If no such date is possible (e.g. the year of the AE or the AE stop date are given and either are earlier than any part of the treatment period) then the AE is not considered a TEAE and no further attempt will be made to impute it.

When imputing the missing parts of a partial AE stop date, the following steps will be followed in order:

- If the year is unknown, the date will not be imputed and will be assigned a missing value;
- If the month is unknown, then assign December;
- If the day is unknown, then assign the last day of the month.

Imputation of start and/stop date should not result in having start dates after stop dates. If start date is completely missing, set it to stop date, and vice-versa.

If the AE is ongoing, the stop date will remain missing.

### 7.11.1.4 Imputation Rules for NDO Diagnosis Onset Date

The following steps will be followed when the onset date of NDO diagnosis is partially missing:

- Missing year, whether day and month are present or not: No imputations will occur;
- Missing day, but month and year are present: the day will be imputed as the 15th day of the month;
- Missing day and month, but year is present: the day and month will be imputed as 30 June of the year;
- If any such imputed date falls after the informed consent date, then the onset date will be taken as equal to the earliest informed consent date.

# 7.11.1.5 Imputation Rules for Start and End Dates for Concomitant Medications and Non-Medication Therapies

Start and stop dates for all concomitant medications and non-medication therapies are collected on the CRF. However, in case of missing or partial information in these dates, the following rules will be used:

If the start date is missing or partial:

- If the entire date is missing, use the earliest date of informed consent;
- If the year is missing, use the year of informed consent. If this makes the imputed date beyond the last visit date, reduce the year by 1;
- If the month is missing, use January;
- If the day is missing, use the first day of the month under consideration.

If the stop date is missing or partial:

- If year or the entire date is missing, no imputation is performed;
- If month is missing, use December;
- If day is missing, use the last day of the month under consideration;

Imputation of start and/stop date should not result in having start dates after stop dates.

#### 7.11.2 Outliers

All values will be included in the planned analyses. A sensitivity analysis excluding outliers may be performed as an additional secondary analysis, if considered appropriate by the study statistician or the medical expert.

#### 7.11.3 Visit Windows

The study protocol gives the overall study schedule and the permissible intervals for these visits expressed as the number of days relative to Visit 3 (see Schedule of Assessments).

Analyses will not exclude subject data due to the subject's failure to comply with the visit schedule; all subjects' data will be listed.

Data from screening (Visit 1) and start of washout (Visit 2), will not be windowed but assigned to the nominal visit.

Except for study dosing data, data from efficacy and some safety parameters will be assigned to windows as shown in Table 16

Table 16 Visit Windows for Efficacy and Safety Parameters

| CRF visit | Target day relative to<br>Baseline (Visit 3, Day -1) | Visit Window | Analysis<br>visit |
|---|---|---|---|
| CGI-C | | | |
| | 1 <del></del> | | |
| Upper urinary | tract ultrasound | | • |
| | 1 <del></del> | | |
| Acceptability q | uestionnaires | | • |
| | 1 <del></del> | | |
| Height and wei | ght | | • |
| | <del></del> | | |
| PinQ, PGI-S | • | | - |
| Table continued | on next page | | <u> </u> |



# Day 1 data are assumed to be prior to first dose. For the continuous ECGs, the baseline value will equal (M2+M3)/2 where M2 and M3 equal the triplicate means of at Visit 2 and Visit 3. Visit 2 will windowed from Day -15 to Day -8.

\$ for hematology/biochemistry at screening. Additional hematology/biochemistry taken at baseline only if an AE related to hematology/biochemistry parameters occurred between visit 1/screening and visit 3/baseline.

For non-diary data, if a subject has more than one non-missing value in a visit window, the non-missing assessment which is closest to the target day within a window will be used. If two or more values are equally close and on different days, the latest non-missing value will be used. If two or more values are equally close and on the same day, the mean will be used for continuous variables or the worst observed case for categorical variables.

For diary data, the assessment date for the whole diary will be considered to be the date of the last valid day of the diary. If more than one diary has an assessment date within the same window, and if this results in more than one non-missing value of a diary variable, the non-missing value with the diary assessment day that is closest to the target day will be used. In case of ties on different days, the later non-missing value will be used. In case of ties located on the same side of the target day (i.e., more than one value for the same day), the mean of the values will be used for continuous variables and the worst value for categorical variables. For analyzing diary data the labels of the study visits will not be used, they will be assigned based on the dates of assessment.

A two-day window around the visit date will be applied for the assignment of study period for exposure data.

<sup>\*</sup> Visit 10 may occur earlier due to early discontinuation as it is the last scheduled study visit.

ISN/Protocol 178-CL-206A

#### **DOCUMENT REVISION HISTORY** 8

| Version | <u>Date</u> | Changes | Comment/rationale for change |
|---|---|---|---|
| Draft 0.1 | 25-MAR-2016 | NA | NA |
| Final 1.0 | 21-APR-2016 | Set version to Final 1.0 | Finalization of document |
| Final 2.0 | 04-May-2018 | Whole document | Minor textual updates/changes and typing |
| | | | errors are not mentioned |
| | | Whole document | SMIP is removed from the exploratory safety |
| | | | endpoints. All text related to SMIP is removed |
| | | | from the document |
| | | List of Tables | List of Tables was added |
| | | List of abbreviations | List is updated |
| | | Section 6.1.3.1.3 | The calculation of bladder compliance is |
| | | | updated according to the central reviewers' |
| | | | algorithm. |
| | | Sections 6.2.1.1 and | Calculations of average vital signs are updated |
| | | 6.2.1.2 | to align with the DSMB SAP. |
| | | Sections 7.5.3.1 and | Normal blood pressure ranges are updated to |
| | | 7.5.3.2 | align with DSMB SAP. |
| | | Section 1 | Text is updated to include CT206. |
| | | T 11 1 | Text on PK Analysis is updated. |
| | | Table 1 | Table 1 is updated according to protocol of |
| | | G .: 5.3 | CT206. |
| | | Section 5.3 | Second bullet updated: |
| | | | New text: |
| | | | Had a valid (as by the central reviewer's |
| | | | assessment) nonmissing MCC measurement at |
| | | | baseline and at a post-baseline visit for the |
| | | | primary efficacy endpoint. Old text: |
| | | | Provided both <u>valid</u> baseline and at least 1 |
| | | | postbaseline value for the primary efficacy |
| | | | endpoint (MCC) |
| | | Section 5.4.1 | Text on "Prohibited Medication" is updated |
| | | 500tion 5.1.1 | with respect to Botox. |
| | | | New text (added text in italic): |
| | | | "Except for Botox which is not allowed <i>if</i> |
| | | | taken from <4 months before screening |
| | | | and/or during the whole study period." |
| | | Section 5.4.1 | Eligibility Deviations: the 2 bullets are |
| | | | updated |
| | | Section 6.1 | Parameter "MCC expressed as percentage of |
| | | Urodynamic | Expected Bladder Capacity (EBC)"added plus |
| | | assessments | additional text to describe the parameter |
| | | Section 6.1 | Text from sentence below is deleted: "to be |
| | | Questionnaires | completed by the subject or the subject's |
| | | | parent/caregiver" |
| | | Section 6.1 | Text now reads: Questionnaires (i.e., PIN-Q, |
| | | Questionnaires | PGI-S and the Acceptability Questionnaires) |

| Version | <u>Date</u> | Changes | Comment/rationale for change |
|---|---|---|---|
| | | | will be provided via the e-diary. |
| | | Section 6.1 | Sentence "Clinically relevant adverse changes |
| | | Questionnaires | will be recorded as an AE." just above "The |
| | | | primary and secondary variables will be" |
| | | | is deleted |
| | | Section 6.1 | Table 2 and Table 3 are updated with respect |
| | | | to deleted and added variables. |
| | | Section 6.1.2 | Section on Estimand is added |
| | | Section 6.1.3.2.1 – | Text: |
| | | 6.1.3.2.4 | "2 days are concurrent" is replaced by |
| | | 011131211 | "2 days are consecutive" |
| | | | Note: in version 1.0 it was section 6.1.2.2.1 – |
| | | | 6.1.2.2.4 |
| | | Section 6.1.3.2.2 and | Text "An alternative version of this variable |
| | | 6.1.3.2.3 | will be calculated as the maximum of all the |
| | | | daytime values recorded over the two |
| | | | measuring days." is deleted. |
| | | | Note: In version 1.0 it was section 6.1.2.2.2 |
| | | | and 6.1.2.2.3 |
| | | Section 6.1.3.2.5 and | Section title now reads: Mean number of |
| | | 6.1.3.2.6 | leakage episodes per day (day and night time) |
| | | | (weekend diary) |
| | | | In title header "day and night time" is |
| | | | presented instead of "night time" |
| | | | Note in version 1.0 it was section 6.1.2.2.5 |
| | | | and 6.1.2.2.6 |
| | | Section 6.1.3.3.1 | Text on items of PIN-Q is updated |
| | | | Note in version 1.0 it was section 6.1.2.3.1 |
| | | Section <u>6.1.3.3.5</u> | Section on Acceptability (for oral suspension) |
| | | | is added |
| | | Section 6.1.4.2.1 | Section is added to describe MCC expressed |
| | | 0 ( (1.400 | as percentage EBC |
| | | Section <u>6.1.4.2.3</u> | Last sentence: "total catheterized volume" |
| | | | instead of "maximum catheterized volume" |
| | | 0 ( (1.40) | Note in version 1.0 it was section 6.1.3.2.2 |
| | | Section 6.1.4.2.6 | Section is added to describe "Percentage of |
| | | | Catheterizations without Intermittent Leakage |
| | | g .; [63] | Accident" |
| | | Section 6.2 | Table 5 footnote added |
| | | Section <u>6.2.1.2</u> | As second sentence added: "Additional SBPM |
| | | | will be done on 2 consecutive days at around |
| | | | 1 and 2 weeks after start of dosing with |
| | | | PED25 (day 1) and after up-titration to PED50 |
| | | | (visit 4/week 2, visit 5/week 4 or visit 6/week |
| | | | 8), if not already covered by the scheduled |
| | | g .: [65.1.1] | visit 4/week 2 and/or visit 5/week 4 SBPM." |
| | | Section <u>6.2.1.4</u> | Table 7 is updated, now based on Fleming et |
| | | | al. [2011], instead of on Ostchega et al. [2011] |
| | | Section 6.2.2 | Timeframe for defining a TEAE is clarified. |

| <b>X</b> 7. | D-4- | Classic | C |
|---|---|---|---|
| <u>Version</u> | <u>Date</u> | Changes | Comment/rationale for change |
| | | | AEs of interest: First bullet (CV), the |
| | | | following text is added for clarification: |
| | | | "(Note: these 3 CV events will be analyzed |
| | | | combined and separately)" |
| | | Section 6.2.3 | Table 9 |
| | | Section 0.2.5 | "Estimated glomerular filtration rate |
| | | | (Larsson)" is replaced by |
| | | | "Estimated glomerular filtration rate |
| | | | (Larsson, modified Schwartz and Cockcroft- |
| | | | Gault)" |
| | | Section 6.5.4 | Text on "Suspension Compliance" is added |
| | | Section 7.2.1 | Wash out failures summary is removed as |
| | | | washout failure is not defined in the protocol. |
| | | | Follow-up summary is replaced by end of |
| | | | treatment summary. |
| | | | Analysis Sets are added. |
| | | | Text added with respect to a listing of all early |
| | | | withdrawals and a listing of screen failures. |
| | | Section 7.2.3 | Updated countries participating in the study |
| | | | and added text below this paragraph to explain |
| | | | that countries may be added to the list |
| | | Section 7.4.1.1 | The following text is added at end of section: |
| | | Section 7.1.1.1 | "MCC at each visit and change from baseline |
| | | | in MCC at visit 8/week 24 (without LOCF) |
| | | | will be also plotted and listed for SAF and |
| | | | PPS." |
| | | Section 7.4.3 | The following text is added at end of section: |
| | | | "A listing will be presented for subjects with a |
| | | | filling volume of >40 cm H <sub>2</sub> O detrusor |
| | | | pressure at week 24. Listing will, among |
| | | | other, present the MCC and MCC expressed |
| | | | as % of EBC." |
| | | Section 7.4.5 | Section on "Sensitivity analysis" is added. |
| | | 200011 7.1.0 | Section was added to investigate the effect of |
| | | | the urine measurement mistakes made. |
| | | Section 75 | |
| | | Section 7.5 | SAEs upgraded by the Sponsor is added. This |
| | | | was an omission in the previous version. Text |
| | | | added with respect to summarizing safety |
| | | | parameters with respect to height- and sex- |
| | | | specific percentiles. Height will be |
| | | | summarized with respect to age- and sex- |
| | | | specific percentiles. |
| | | Section 7.5 | Text added: "Subgroup presentations |
| | | | regarding age (children and adolescents), |
| | | | formulation (tablets and suspension) and |
| | | | dosing regimen (PED25 and PED50) will be |
| | | | tabulated for a number of safety parameters. |
| | | | Added text at end of Section "For any of the |
| | | | subgroups specified, at least 10 subjects by |
| | | | stratum are required.". |
| | 1 | | Structure are required |

| Version | <u>Date</u> | Changes | Comment/rationale for change |
|---|---|---|---|
| | | Section 7.5.1 | Number and percentage of subjects who |
| | | | died" instead of "Number of Deaths". |
| | | Section 7.5.2.1 | Text on "Liver Function Tests" is updated |
| | | Sections 7.5.3.1 and | Text on PCR for SBP and for DBP is updated |
| | | 7.5.3.2 | Text on prehypertension is updated |
| | | Section 7.6.2 | Table 15 is updated to reflect the sampling |
| | | | strategy |
| | | Section 9 | List of References is updated. |
| | | Section 10.1 | List of In- and Exclusion criteria is updated |
| | | Section 10.1 | according to protocol of 206 study". |
| | | Section 10.14 | List of Key Contributors and Approvers is |
| | | Section 10.14 | updated |
| Final 3.0 | 21-May-2019 | Whole document | Typos were corrected |
| Tillal 3.0 | 21-Way-2017 | Introduction | Introduction was updated to reflect it is the |
| | | Introduction | SAP for 206A. Reference to EU PIP, EMEA |
| | | | Decision, and US Written Request was added. |
| | | Section 3.2 and 7.2.3 | Deleted reference to USA |
| | | Section 6.1 | Full + Empty Bladder Pressure is deleted |
| | | | Tables are updated to show that change from |
| | | Section 6.1, Table 2 and Table 3 | 1 |
| | | and Table 3 | baseline in MCC expressed as % of EBC is |
| | | Section 6.1.2 | analyzed at Week 4 and Week 24. |
| | | Section 6.1.2 | Title updated: Estimand instead of Estimator |
| | | | and 1 sentence added: "Difference of MCC at |
| | | | visit 8/week 24 (or prior, due to study drug |
| | | | discontinuation) compared to baseline is the |
| | | | primary estimator." |
| | | | Text was added why the "de facto" estimand |
| | | | was not chosen for this study. |
| | | | Last sentence of his section: to impute was |
| | | G 4: (1220) | changed by "to handle" |
| | | Section 6.1.3.2.8 (new) | Added section on identification of leakage |
| | | G .: (1220 | during sleeping time |
| | | Section 6.1.3.2.8 | New section added for clarification |
| | | | "Identification of leakage during sleeping |
| | | G .: (22 | time" |
| | | Section 6.2.2 | AEs of Interest: |
| | | | Deleted is: Thermogenesis (brown fat). |
| | | | Added are: Seizure: Syncope; Fetal disorders |
| | | | after exposure during pregnancy; and |
| | | | Concomitant treatment with cytochrome P450 |
| | | | (CYP) 2D6 substrates with narrow therapeutic |
| | | | indices or individually dose-titrated. |
| | | | Last sentence of Section 6.2.2: text "and AEs |
| | | | related to mirabegron" is deleted |
| | | Section 6.5.4 | Compliance text was updated |
| | | Section 7.2.1 | A table was added which presented the |
| | | | number of subjects screened under each |
| | | | protocol version |
| | | Section 7.2.2 | PD4: "excluded" instead of "prohibited" |

| <u>Version</u> | <u>Date</u> | Changes | Comment/rationale for change |
|---|---|---|---|
| | | | concomitant medication |
| | | Section 7.2.3 | Added Analysis Set (SAF) for summary of |
| | | | Medical History data. |
| | | Section 7.3.3 | Titration period: Visit 3 to Visit 7 instead of |
| | | | Visit 4 to Visit 6 |
| | | Section 7.4.1.1 | SAS procedure TTEST was replaced by UNIVARIATE |
| | | Section 7.4.1.2.6 | Text was updated, no pooling of data from 206 and 206A and statistical method adapted. |
| | | Section 7.4.5 | Added to Average morning catheterized volume: once "for subjects with no leakage during the sleeping time" and "for subjects with leakage during the sleeping time" |
| | | Section 7.5.1 | AE will be summarized by SOC, HLT and PT instead of by SOC and PT for "All TEAEs" table only |
| | | Section 7.5.1.2 | Second paragraph is deleted |
| | | Section 7.5.2.1 | Old text replaced by standard text from SAP template |
| | | Section 7.5.3.1 | In addition to shift tables referencing to "Fourth Report" also shift table will be presented based on a more recent reference: "2017 American Academy of Pediatric Clinical Practice Guidelines", based on FDA request. |
| | | | Results based on Fourth Report are considered primary, results based on other reference are considered secondary. Additional table (Table 12) was inserted. Text updated for clinical measurements and home measurements (same lay-out for both) |
| | | Section 7.5.3.1 | For presenting the number of subjects with PR values below or above the normal range, the normal range is defined. Footnote was added to Table 12 to explain that the age classification into children and adolescents in the Clinical Practice Guidelines (2017) differs from the definition used in the protocol |
| | | Section 7.6.2 | Mean plasma concentration-time profiles only on semi-log scale. Added: Box plots of plasma concentration-time profiles (normal scale and semi-log scale). And text that "First 2 plots will be produced for PK report." |
| | | Section 7.8 | Ethnicity was added as subgroup based on request from FDA. Sentence "For any of these subgroups, at least |

| Version | <u>Date</u> | Changes | Comment/rationale for change |
|---|---|---|---|
| | | | 10 subjects by stratum are required." was |
| | | | deleted. |
| | | Section 7.11.3 | Title of table 16 was adapted and footnote was |
| | | | added to the table for clarification of visit 10. |
| | | | Two sentences were added at end of section: |
| | | | one to clarify that for the diary data the labels |
| | | | will not be used for analysis, and another one |
| | | | to explain for exposure data the assignment of |
| | | T. 11. 12. | study period |
| | | Table 13 (new) | Table is added with data from Stergiou 2007 reference |
| | | REFERENCES | Reference added: "2017 American Academy of Pediatric Clinical Practice Guidelines" |
| | | Section 10: | Numbering has changed |
| | | Appendices | |
| | | Section 10.1 | Exclusion criteria are re-numbered, starting |
| | | | now at 1. To be in line with numbering in |
| | | | Section 5.4.1 |
| | | Section 10.3, | Section is deleted |
| | | Appendix 3.2 | |
| | | Sections 10.10 and | Tables with results for males and females |
| | | 10.11 | from "2017 American Academy of Pediatric |
| | | | Clinical Practice Guidelines" reference are |
| | | | included |
| | | Section 10.14 | List of Key Contributors and Approvers is |
| | | | updated due to internal Astellas reorganization |

#### 9 REFERENCES

- 2017 American Academy of Pediatric Clinical Practice Guidelines (Flynn JT, Kaelber DC, Baker-Smith CM, et al. Clinical Practice Guideline for Screening and Management of High Blood Pressure in Children and Adolescents. Pediatrics.2017;140(3):e20171904)
- Bauer SB et al. *International Children's Continence Society standardization report on urodynamic studies of the lower urinary tract in children*. Neurourol Urodyn. 2015 May 21. doi:10.1002/nau.22783.
- Bower W.F. et al. *PinQ: A valid, reliable and reproducible quality-of-life measure in children with bladder dysfunction*, Journal of Pediatric Urology (2006) 2, 185-189
- Cartwright PC, Coplen DE, Kogan BA, et al. *Efficacy and safety of transdermal and oral oxybutynin in children with neurogenic detrusor overactivity*. J Urol 2009;82:1548-54.
- Cockcroft DW, Gault MH (1976). *Prediction of creatinine clearance from serum creatinine*. Nephron. 16 (1): 31–41. doi:10.1159/000180580. PMID 1244564.
- Fleming S, Thompson M, Stevens R, Heneghan C, Plüddemann A, Maconochie I, et al. *Normal ranges of heart rate and respiratory rate in children from birth to 18 years of age: a systematic review of observational studies.* Lancet. 2011;377:1011-18.
- Franco I, et al. *Efficacy and safety of oxybutynin in children with detrusor hyperreflexia secondary to neurogenic bladder dysfunction.* J Urol 2005;173:221-25.
- Goessl C, Sauter T, Michael T, et al. *Efficacy and tolerability of tolterodine in children with detrusor hyperreflexia*. Urology 2000;55:414-18.
- ICH Harmonized Tripartite Guideline E 3. Structure and Content of Clinical Study Reports, November 1995. (www.ich.org; Guidelines; "Efficacy" Topics)
- ICH Harmonized Tripartite Guideline E 9. Statistical Principles for Clinical Trials, February 1998. (www.ich.org; Guidelines; "Efficacy" Topics)
- Kliegman RM, Stanton BMD, St. Geme J, Schor NF, Behrman RE. Nelson Textbook of Pediatrics, 19<sup>th</sup> edition. Elsevier Science Health 2007
- Kuczmarski RJ, Ogden CL, Guo SS, et al. 2000 CDC growth charts for the United States: Method and development. National Center for Health Statistics. Vital Health Stat 11(246). 2002
- Larsson A, Malm J, Grubb A, Hansson LO. *Calculation of glomerular filtration rate expressed in ml/min from plasma cystatin C values in mg/L*. Scand J Clin Lab Invest 2004; 64:25-30
- Ostchega Y, Porter KS, Hughes J, Dillon CF, Nwankwo T. Resting pulse rate reference data for children, adolescents and adults: United states, 1999-2008. National Health Statistics Report No.41 (August 2011)
- Palmer LS, Richards I and Kaplan WE. Age related bladder capacity and bladder capacity growth in children with myelomeningocele. J Urol 1997;158: 1261.r

- Schwartz GJ, Muñoz A, Schneider MF, Mak RH, Kaskel F, Warady BA, et al. New Equations to Estimate GFR in Children with CKD. J Am Soc Nephrol. 2009;20:629–37.
- Stergiou G, Yiannes N, Rarra V and Panagiotakos D. *Home blood pressure normalcy in children and adolescents: the Arsakeion School study.* J Hypertens 2007, 25:1375–1379
- Temple R. Hy's law: Predicting Serious Hepatotoxicity. Pharmacoepidemiol Drug Saf. 2006 April;15(Suppl 4):241-3.
- The Fourth Report on the diagnosis, evaluation, and treatment of high blood pressure in children and adolescents. 2005. U.S. Department of Health and Human Services, National Institutes of Health National Heart, Lung, and Blood Institute. NIH Publication No. 05-5267. Originally printed September 1996 (96-3790) Revised May 2005.

  Available from: https://www.nhlbi.nih.gov/files/docs/resources/heart/hbp\_ped.pdf

#### 10 APPENDICES

## 10.1 Appendix 1: Inclusion and Exclusion Criteria

#### **Inclusion criteria:**

Subject is eligible for the study if all of the following apply:

- 1. Independent Ethics Committee (IEC)/Institutional Review Board (IRB)-approved written Informed Consent and privacy language as per national regulations must be obtained from the subject and/or from the subject's parent(s) or legal guardian(s) prior to any study-related procedures (including discontinuation of prohibited medication, if applicable); assent by the subject is given as required by local law.
- 2. Subject is male or female from 3 to less than 18 years of age.
- 3. Subject has a body weight of  $\geq 11$  kg.
- 4. Subject suffers from NDO confirmed by urodynamic investigation at baseline. The diagnosis of NDO must be confirmed by the presence of at least 1 involuntary detrusor contraction > 15 cm H<sub>2</sub>O from baseline detrusor pressure, and/or a decrease in compliance leading to an increase in baseline detrusor pressure of > 20 cm H<sub>2</sub>O.
- 5. Subject is exclusively using CIC (no voluntary voiding), starting at least 4 weeks prior to visit 1/screening
- 6. Subject has a current indication for drug therapy to manage NDO.
- 7. Subject is able to take the study drug in accordance with the protocol.
- 8. Female subject must either:
  - Be of nonchildbearing potential:
    - Clearly premenarchal or in the judgment of the Investigator is premenarchal,
    - o Documented surgically sterile,
  - Or, if of childbearing potential:
    - Agree not to try to become pregnant during the study and for 28 days after the final study drug administration,
    - And have a negative pregnancy test at visit 1/screening and at baseline,
    - O And, if sexually active must agree to use a highly effective method of birth control, which includes established use of oral, injected or implanted hormonal methods of contraception, OR placement of an intrauterine device (IUD) or intrauterine system (IUS). Birth control must be practiced from visit 1/screening and continuing throughout the study period, and for 28 days after the final study drug administration.
- 9. Male subject and their female spouse/partner who are of childbearing potential must be using a highly effective method of birth control, which includes established use of oral, injected or implanted hormonal methods of contraception, placement of an IUD or IUS.

- Birth control must be practiced from visit 1/screening and continuing throughout the study period, and for 28 days after the final study drug administration.
- 10. Female subject must not be breastfeeding from visit 1/screening until 28 days after last study drug administration.
- 11. Subject and subject's parent(s)/legal guardian(s) agree that the subject will not participate in another interventional study while participating in the study.
- 12. Subject and subject's parent(s)/legal guardian(s) are willing and able to comply with the study requirements and with the concomitant medication restrictions.

Waivers to the inclusion criteria are NOT allowed.

#### **Exclusion Criteria:**

Subject are excluded from participation if any of the following apply:

- 1. Subject has a known genitourinary condition (other than NDO) that may cause overactive contractions or incontinence (e.g., bladder extrophy, urinary tract obstruction, urethral diverticulum or fistula) or kidney/bladder stones or another persistent local pathology that may cause urinary symptoms.
- 2. Subject has one of the following gastrointestinal problems: partial or complete obstruction, decreased motility such as paralytic ileus, subjects at risk of gastric retention.
- 3. Subject has a urinary indwelling catheter within 4 weeks prior to or during the pretreatment period
- 4. Subject has a surgically treated underactive urethral sphincter
- 5. Subject has vesico-ureteral reflux grade 3 to 5.
- 6. Subject has undergone bladder augmentation surgery.
- 7. Subject receives electrostimulation therapy, if started within 30 days before visit 1/screening or is expected to start during the study period. Subjects who are on an established regimen may remain on this for the duration of the study.
- 8. Subject suffers from a symptomatic UTI at baseline (symptomatic is defined as pain, fever, hematuria, new onset foul-smelling urine). If present at visit 1/screening or diagnosed between visit 1/screening and visit 3/baseline, the UTI should be treated successfully (clinical recovery) prior to baseline. If a symptomatic UTI is present at baseline, all baseline assessments should be postponed for a maximum of 7 days until the UTI is successfully treated (clinical recovery).
- 9. Subject has a (mean) resting pulse rate > 99<sup>th</sup> percentile [Fleming et al, 2011].
- 10. Subject has an established hypertension and a systolic or diastolic blood pressure higher than 5 mmHg above the 99<sup>th</sup> percentile (stage 2 hypertension) or subject has a systolic or diastolic blood pressure that ranges from the 95<sup>th</sup> percentile to 5mmHg above the 99<sup>th</sup>

- percentile (stage 1 hypertension) which is not well-controlled. Percentiles are determined by sex, age, and height [The Fourth Report, 2005].
- 11. Subject has a risk of QT prolongation (e.g., hypokalemia, long QT syndrome [LQTS]; or family history of LQTS, exercise-induced syncope).
- 12. Subject has severe renal impairment (eGFR according to Larsson equation < 30 mL/min).
- 13. Subject's AST or ALT is greater than or equal to 2 times the upper limit of normal (ULN) or total bilirubin (TBL) greater than or equal to 1.5 times the ULN according to age and sex.
- 14. Subject has a history or presence of any malignancy prior to visit 1/screening.
- 15. Subject has known or suspected hypersensitivity to mirabegron, any of the excipients used in the current formulations or previous severe hypersensitivity to any drug.
- 16. Subject has participated in another clinical trial (and/or has taken an investigational drug) within 30 days (or 5 half-lives of the drug, or the limit set by national law, whichever is longer) prior to visit 1/screening.
- 17. Subject uses any of the following prohibited medications (after start of washout):
  - Any medication, other than the study drug used, for the management of NDO;
  - Any drugs that are sensitive CYP2D6 substrates with a narrow therapeutic index or individually dose-titrated, or sensitive P-glycoprotein (P-gp) substrates
  - Any strong CYP3A4 inhibitors if the subject has a mild to moderate renal impairment (eGFR 30 89 mL/min).
- 18. Subject has been administered intravesical botulinum toxin; except if given > 4 months prior to visit 1/screening and the subject experiences symptoms comparable to those existing prior to the botulinum toxin injections.
- 19. Subject has any other condition, which in the opinion of the Investigator, precludes the subject's participation in the study.
- 20. Subject's parent/legal guardian is an employee of the Astellas Group, the Contract Research Organization (CRO) involved, or the Investigator site executing the study.

Waivers to the exclusion criteria are NOT allowed.

### 10.2 Appendix 2: List of Excluded Concomitant Medications

Any medication used for the management of NDO (including tricyclic antidepressants, 1<sup>st</sup> generation H1-antagonists and alpha-blockers) and any drugs that are sensitive CYP2D6 substrates with a narrow therapeutic index and sensitive P-gp substrates.

Strong CYP3A4 inhibitors are excluded for subjects with mild to moderate renal impairment (mild: eGFR 60 to 89 mL/min; moderate: eGFR 30 to 59 mL/min).

Use of these medications is not permitted during the study phase. This list is <u>not exhaustive</u>. In case of doubt, the investigator should contact the local study monitor.

| Anticholinergics/ | Tricyclic antidepressants | 1st generation H1-antagonists |
|---|---|---|
| antimuscarinics | | Ť |
| Darifenacin | Alimemazine / Trimipramine | Tripelennamine |
| Dicyclomine/Dicycloverine | Amitriptyline | Dimenhydrinate |
| Fesoterodine | Amoxapine | Clemastine |
| Flavoxate | Clomipramine | Bromazine |
| Isopropamide | Desipramine | Orphenadrine |
| Oxybutynin | Dosulepin/ Dothiepin | Doxylamine |
| Oxyphencyclimine | Doxepine | Carbinoxamine |
| Propantheline | Imipramine | Diphenhydramine |
| Propiverine | Lofepramine | Cyclizine |
| Tolterodine | Maprotiline | Chlorcyclizine |
| Trospium | Mianserin | Hydroxyzine |
| Solifenacin | Mirtazapine | Meclizine |
| | Nortriptyline | |
| | Protriptyline | |
| Alpha-blockers | CYP2D6 with narrow | Sensitive P-gp substrates |
| | therapeutic index | |
| Tamsulosin | Thioridazine | Digoxin |
| Alfuzosin | Flecainide | Dabigatran |
| Doxazosin | Propafenone | |
| Terazosin | Imipramine | |
| Silodosin | Desipramine | |
| Strong CYP3A4 inhibitors | Other | |
| Itraconazole | Mirabegron (except for study dr | ug) |
| Ketoconazole | Botulinum toxin | |
| Ritonavir | | |
| Clarthromycin | | |

<sup>†</sup> Incidental use for motion sickness is accepted.

# 10.3 Appendix 3: AEs of Interest not covered by Standard MedDRA SMQs V16.0

The following is a list of AE terms to programmatically flag subjects with AE's of interest (see Section 7.5.1.1).

| Type | Term | Code | AE of Interest | MedDRA 16.0 Search Criteria |
|---|---|---|---|---|
| | Acute retention of urine | 10001055 | Acute urinary retention | Selected LLT (non-SMQ) |
| PT | Residual urine volume | 10050832 | Urinary retention | Selected PT's (non-SMQ) |
| PT | Residual urine volume increased | 10067758 | Urinary retention | Selected PT's (non-SMQ) |
| PT | Urinary retention | 10046555 | Urinary retention | Selected PT's (non-SMQ) |
| PT | Pyelonephritis<br>mycoplasmal | 10037603 | Urinary tract infection | Selected PT's (non-SMQ) |
| PT | Pyelonephritis viral | 10065213 | Urinary tract infection | Selected PT's (non-SMQ) |
| PT | Pyonephrosis | 10037653 | Urinary tract infection | Selected PT's (non-SMQ) |
| PT | Renal abscess | 10038351 | Urinary tract infection | Selected PT's (non-SMQ) |
| PT | Renal syphilis | 10038530 | Urinary tract infection | Selected PT's (non-SMQ) |
| PT | Renal tuberculosis | 10038534 | Urinary tract infection | Selected PT's (non-SMQ) |
| PT | Urethral abscess | 10046424 | Urinary tract infection | Selected PT's (non-SMQ) |
| PT | Urethral carbuncle | 10052299 | Urinary tract infection | Selected PT's (non-SMQ) |
| PT | Urethritis | 10046480 | Urinary tract infection | Selected PT's (non-SMQ) |
| PT | Urethritis chlamydial | 10046482 | Urinary tract infection | Selected PT's (non-SMQ) |
| PT | Urethritis gonococcal | 10046483 | Urinary tract infection | Selected PT's (non-SMQ) |
| PT | Urethritis trichomonal | 10046489 | Urinary tract infection | Selected PT's (non-SMQ) |
| PT | Urethritis ureaplasmal | 10046490 | Urinary tract infection | Selected PT's (non-SMQ) |

# 10.4 Appendix 4: Questionnaires

# **Appendix 4.1** Pediatric Incontinence Questionnaire

| 1. I get shy because of my bladder problem |
|---|
| □ No □ Hardly ever □ Sometimes □ Often □ All the time |
| 2. People in my family treat me in a different way because of my bladder problem |
| □ No □ Hardly ever □ Sometimes □ Often □ All the time |
| 3. I am worried that people might think my clothes smell of wee |
| □ No □ Hardly ever □ Sometimes □ Often □ All the time |
| 4. I think that my bladder problem won't get better |
| □ No □ Hardly ever □ Sometimes □ Often □ All the time |
| 5. Mum and Dad worry about me because of my bladder problem |
| □ No □ Hardly ever □ Sometimes □ Often □ All the time |
| 6. I would feel better about myself if I didn't have a bladder problem |
| □ No □ Maybe □ Probably □ Yes □ Definitely |
| 7. My bladder problem makes me feel nervous |
| □ No □ Hardly ever □ Sometimes □ Often □ All the time |
| 8. Mum or Dad sometimes seem a bit cranky because of my bladder problem |
| □ No □ Hardly ever □ Sometimes □ Often □ All the time |
| 9. My bladder problem stops me going on sleepovers or holidays □ No □ Hardly ever □ Sometimes □ Often □ All the time |
| 10. My bladder problem makes me feel bad about myself |
| □ No □ Hardly ever □ Sometimes □ Often □ All the time |
| 11. I wake up during my sleep because of my bladder problem |
| □ No □ Hardly ever □ Sometimes □ Often □ All the time |
| 12. I miss out on doing things because of my bladder problem |
| □ No □ Hardly ever □ Sometimes □ Often □ All the time |
| 13. I feel unhappy because of my bladder problem |
| □ No □ Hardly ever □ Sometimes □ Often □ All the time |
| 14. My bladder problem makes me feel sad |
| □ No □ Hardly ever □ Sometimes □ Often □ All the time |
| 15. I think about my bladder problem when choosing which sport to play |
| □ No □ Hardly ever □ Sometimes □ Often □ All the time |
| 16. I have to go to the toilet when I'm watching a movie |
| □ No □ Hardly ever □ Sometimes □ Often □ All the time |
| 17. If my bladder problem was fixed I would invite more friends to my house |
| □ No □ Maybe □ Probably □ Yes □ Definitely |
| 18. I choose hobbies that won't be spoiled by stopping to go to the toilet |
| □ No □ Hardly ever □ Sometimes □ Often □ All the time |
| 19. My bladder problem makes me feel different to other people |
| □ No □ Hardly ever □ Sometimes □ Often □ All the time |
| 20. I miss out on being with friends because of my bladder problem |
| □ No □ Hardly ever □ Sometimes □ Often □ All the time |

PINQ (UK-English) Astellas Pharma Europe Ltd FINAL V1 Oxford, Version 30NOV2011

Appendix 4.2 Patient Global Impression of Severity Scale

| How did you feel | about your bladd | er condition <u>DUR</u> | ING THE PAST 3 | B DAYS? |
|---|---|---|---|---|
| 0 | 0 1 2 3 4 | | | |
| | | | | $\odot$ |
| Really bad | Bad | Not bad, not good | Good | Really good |

# Appendix 4.3 Acceptability Questionnaire for Tablets

| | | Questions | | |
|---|---|---|---|---|
| 1. How was the <u>TASTE</u> of the study medication? | | | | |
| 0 | 0 1 2 3 4 | | | |
| | | | | $\odot$ |
| Really bad | Bad | Not bad, not | Good | Really good |
| | | good | | |
| 2. How was i | t to <u>SWALLOW</u> | the study medica | ation? | |
| 0 | 1 | 2 | 3 | 4 |
| 0 | | 2 | 3 | 4 |
| 0 Really difficult | 1<br>Difficult | Not difficult, not easy | 3<br>Easy | 4 Really easy |

Appendix 4.4 Acceptability Questionnaire for Oral Suspension

| | | Questions | | |
|---|---|---|---|---|
| 1. How was t | he <u>TASTE</u> of the | e study drug? | | |
| 0 | 1 | 2 | 3 | 4 |
| Really bad | Bad | Not bad, not<br>good | Good | Really good |
| 2. How was t | he <u>SMELL</u> of th | e study drug? | | |
| 0 | 1 | 2 | 3 | 4 |
| | | | $\odot$ | |
| Really bad | Bad | Not bad, not<br>good | Good | Really Good |
| 3. How was it | t to <u>TAKE</u> the st | udy drug? | | |
| 0 | 1 | 2 | 3 | 4 |
| Really difficult | Difficult | Not difficult, not easy | Easy | Really easy |

| 4. How was i | 4. How was it to PREPARE the study drug? | | | |
|---|---|---|---|---|
| 0 | 0 1 2 3 4 | | | |
| | | | $\odot$ | |
| Really difficult | Difficult | Not difficult,<br>not easy | Easy | Really easy |

# Appendix 4.5 Clinical Global Impression of Change Scale

| Clinical Global Impression of Change Scale |
|---|
| Please rate the degree of change in the subject's overall bladder symptoms since the start of the study on day 1 (tick 1 box) |
| Very much improved |
| Much improved |
| Minimally improved |
| No change |
| Minimally worse |
| Much worse |
| Very much worse |

# 10.5 Appendix 5 Centiles of heart rate for normal children from birth to 18 years of age [Fleming et al, 2011]



# 10.6 Appendix 6 CDC Data Table of Stature-for-age Chart for Males

## Males, Stature, Ages 2-20 Years

| Age (in<br>months) | 3rd<br>Percentile<br>Stature (in<br>centimeters) | 5th<br>Percentile<br>Stature (in<br>centimeters) | 10th<br>Percentile<br>Stature (in<br>centimeters) | 25th<br>Percentile<br>Stature (in<br>centimeters) | 50th<br>Percentile<br>Stature (in<br>centimeters) | 75th<br>Percentile<br>Stature (in<br>centimeters) | 90th<br>Percentile<br>Stature (in<br>centimeters) | 95th<br>Percentile<br>Stature (in<br>centimeters) | 97th<br>Percentile<br>Stature (in<br>centimeters) |
|---|---|---|---|---|---|---|---|---|---|
| 24 | 79.91084 | 80.72977 | 81.99171 | 84.10289 | 86.4522 | 88.80525 | 90.92619 | 92.19688 | 93.02265 |
| 24.5 | 80.26037 | 81.08868 | 82.36401 | 84.49471 | 86.86161 | 89.22805 | 91.35753 | 92.63177 | 93.45923 |
| 25.5 | 81.00529 | 81.83445 | 83.11387 | 85.25888 | 87.65247 | 90.05675 | 92.22966 | 93.53407 | 94.38278 |
| 26.5 | 81.73416 | 82.56406 | 83.84716 | 86.00517 | 88.42326 | 90.8626 | 93.07608 | 94.40885 | 95.27762 |
| 27.5 | 82.44846 | 83.27899 | 84.56534 | 86.73507 | 89.17549 | 91.64711 | 93.89827 | 95.25754 | 96.14512 |
| 28.5 | 83.14945 | 83.98045 | 85.26962 | 87.44977 | 89.91041 | 92.41159 | 94.69757 | 96.08149 | 96.98663 |
| 29.5 | 83.83819 | 84.66948 | 85.96098 | 88.15028 | 90.62908 | 93.15719 | 95.47522 | 96.88198 | 97.80345 |
| 30.5 | 84.51558 | 85.34694 | 86.64027 | 88.83745 | 91.33242 | 93.88496 | 96.23239 | 97.66027 | 98.59691 |
| 31.5 | 85.18238 | 86.01357 | 87.3082 | 89.51202 | 92.02127 | 94.59585 | 96.97022 | 98.41758 | 99.36828 |
| 32.5 | 85.83925 | 86.66999 | 87.9654 | 90.17464 | 92.69638 | 95.2908 | 97.68978 | 99.15514 | 100.1189 |
| 33.5 | 86.48678 | 87.3168 | 88.61244 | 90.82592 | 93.35847 | 95.97068 | 98.39218 | 99.87416 | 100.8501 |
| 34.5 | 87.12552 | 87.95452 | 89.24986 | 91.46645 | 94.00823 | 96.63637 | 99.07848 | 100.5759 | 101.5631 |
| 35.5 | 87.75597 | 88.58366 | 89.87816 | 92.0968 | 94.64637 | 97.28875 | 99.74979 | 101.2615 | 102.2593 |
| 36.5 | 88.37864 | 89.20473 | 90.49789 | 92.71756 | 95.27359 | 97.9287 | 100.4072 | 101.9324 | 102.9402 |
| 37.5 | 88.93297 | 89.77301 | 91.08608 | 93.3344 | 95.91475 | 98.58525 | 101.069 | 102.593 | 103.5983 |
| 38.5 | 89.47916 | 90.33306 | 91.66589 | 93.94268 | 96.54734 | 99.23358 | 101.7234 | 103.247 | 104.2503 |
| 39.5 | 90.01766 | 90.88532 | 92.23779 | 94.54291 | 97.17191 | 99.87426 | 102.3709 | 103.8948 | 104.8967 |
| 40.5 | 90.54891 | 91.43025 | 92.80225 | 95.13557 | 97.78898 | 100.5078 | 103.012 | 104.537 | 105.538 |
| 41.5 | 91.07337 | 91.96832 | 93.35972 | 95.72115 | 98.39903 | 101.1348 | 103.6473 | 105.1739 | 106.1747 |
| 42.5 | 91.59152 | 92.49999 | 93.91068 | 96.30009 | 99.00254 | 101.7556 | 104.2771 | 105.8061 | 106.8071 |
| 43.5 | 92.10382 | 93.0257 | 94.45556 | 96.87286 | 99.59998 | 102.3708 | 104.9021 | 106.434 | 107.4357 |
| 44.5 | 92.61073 | 93.54592 | 94.99482 | 97.43989 | 100.1918 | 102.9807 | 105.5225 | 107.0579 | 108.0609 |
| 45.5 | 93.11271 | 94.06109 | 95.52888 | 98.00159 | 100.7783 | 103.5858 | 106.1387 | 107.6784 | 108.683 |
| 46.5 | 93.61022 | 94.57166 | 96.05817 | 98.55838 | 101.36 | 104.1865 | 106.7513 | 108.2956 | 109.3024 |
| 47.5 | 94.10371 | 95.07806 | 96.5831 | 99.11064 | 101.9373 | 104.7831 | 107.3604 | 108.9101 | 109.9193 |
| 48.5 | 94.59361 | 95.5807 | 97.10407 | 99.65875 | 102.5105 | 105.3759 | 107.9665 | 109.522 | 110.5342 |
| 49.5 | 95.08035 | 96.08 | 97.62147 | 100.2031 | 103.0799 | 105.9654 | 108.5698 | 110.1317 | 111.1473 |
| 50.5 | 95.56435 | 96.57635 | 98.13566 | 100.7439 | 103.6459 | 106.5518 | 109.1706 | 110.7394 | 111.7588 |
| 51.5 | 96.046 | 97.07013 | 98.64701 | 101.2817 | 104.2087 | 107.1354 | 109.7693 | 111.3454 | 112.369 |
| 52.5 | 96.52568 | 97.5617 | 99.15585 | 101.8166 | 104.7687 | 107.7165 | 110.366 | 111.95 | 112.9781 |
| 53.5 | 97.00376 | 98.05141 | 99.6625 | 102.3491 | 105.3262 | 108.2953 | 110.9609 | 112.5533 | 113.5863 |
| 54.5 | 97.48058 | 98.53958 | 100.1673 | 102.8792 | 105.8813 | 108.872 | 111.5543 | 113.1555 | 114.1937 |
| 55.5 | 97.95648 | 99.02654 | 100.6705 | 103.4074 | 106.4343 | 109.4469 | 112.1464 | 113.7568 | 114.8006 |

Males, Stature, Ages 2-20 Years

| Age (in<br>months) | 3rd<br>Percentile<br>Stature (in<br>centimeters) | 5th<br>Percentile<br>Stature (in<br>centimeters) | 10th<br>Percentile<br>Stature (in<br>centimeters) | 25th<br>Percentile<br>Stature (in<br>centimeters) | 50th<br>Percentile<br>Stature (in<br>centimeters) | 75th<br>Percentile<br>Stature (in<br>centimeters) | 90th<br>Percentile<br>Stature (in<br>centimeters) | 95th<br>Percentile<br>Stature (in<br>centimeters) | 97th<br>Percentile<br>Stature (in<br>centimeters) |
|---|---|---|---|---|---|---|---|---|---|
| 56.5 | 98.43175 | 99.51256 | 101.1723 | 103.9339 | 106.9855 | 110.0201 | 112.7374 | 114.3574 | 115.4072 |
| 57.5 | 98.90667 | 99.99791 | 101.6731 | 104.4588 | 107.535 | 110.5919 | 113.3273 | 114.9575 | 116.0134 |
| 58.5 | 99.38151 | 100.4828 | 102.173 | 104.9825 | 108.083 | 111.1623 | 113.9164 | 115.557 | 116.6194 |
| 59.5 | 99.8565 | 100.9676 | 102.6723 | 105.505 | 108.6296 | 111.7316 | 114.5047 | 116.1561 | 117.2254 |
| 60.5 | 100.3318 | 101.4523 | 103.1712 | 106.0265 | 109.1751 | 112.2998 | 115.0924 | 116.755 | 117.8314 |
| 61.5 | 100.8077 | 101.9372 | 103.6697 | 106.5472 | 109.7196 | 112.8671 | 115.6795 | 117.3536 | 118.4374 |
| 62.5 | 101.2843 | 102.4225 | 104.1682 | 107.0673 | 110.2631 | 113.4335 | 116.2661 | 117.9521 | 119.0435 |
| 63.5 | 101.7618 | 102.9082 | 104.6666 | 107.5868 | 110.8058 | 113.9992 | 116.8522 | 118.5505 | 119.6498 |
| 64.5 | 102.2401 | 103.3945 | 105.1651 | 108.1058 | 111.3477 | 114.5641 | 117.438 | 119.1487 | 120.2562 |
| 65.5 | 102.7195 | 103.8814 | 105.6638 | 108.6244 | 111.889 | 115.1284 | 118.0234 | 119.7469 | 120.8627 |
| 66.5 | 103.2 | 104.369 | 106.1627 | 109.1427 | 112.4296 | 115.6921 | 118.6084 | 120.345 | 121.4694 |
| 67.5 | 103.6815 | 104.8574 | 106.6619 | 109.6607 | 112.9696 | 116.2551 | 119.1931 | 120.943 | 122.0761 |
| 68.5 | 104.1642 | 105.3466 | 107.1614 | 110.1785 | 113.509 | 116.8176 | 119.7774 | 121.5408 | 122.6829 |
| 69.5 | 104.6479 | 105.8364 | 107.6611 | 110.696 | 114.0479 | 117.3794 | 120.3613 | 122.1384 | 123.2897 |
| 70.5 | 105.1326 | 106.327 | 108.1612 | 111.2132 | 114.5861 | 117.9407 | 120.9447 | 122.7359 | 123.8965 |
| 71.5 | 105.6183 | 106.8182 | 108.6614 | 111.7302 | 115.1238 | 118.5012 | 121.5277 | 123.333 | 124.5031 |
| 72.5 | 106.1048 | 107.3099 | 109.1619 | 112.2469 | 115.6609 | 119.0611 | 122.1101 | 123.9297 | 125.1095 |
| 73.5 | 106.5921 | 107.8021 | 109.6624 | 112.7631 | 116.1973 | 119.6203 | 122.6918 | 124.526 | 125.7156 |
| 74.5 | 107.0799 | 108.2946 | 110.1629 | 113.2789 | 116.7329 | 120.1786 | 123.2729 | 125.1217 | 126.3212 |
| 75.5 | 107.5682 | 108.7873 | 110.6633 | 113.7942 | 117.2678 | 120.7361 | 123.8532 | 125.7168 | 126.9263 |
| 76.5 | 108.0566 | 109.2801 | 111.1634 | 114.3089 | 117.8018 | 121.2926 | 124.4327 | 126.3111 | 127.5307 |
| 77.5 | 108.5451 | 109.7727 | 111.6631 | 114.8229 | 118.3348 | 121.848 | 125.0111 | 126.9045 | 128.1344 |
| 78.5 | 109.0335 | 110.2649 | 112.1623 | 115.336 | 118.8668 | 122.4024 | 125.5884 | 127.4969 | 128.7371 |
| 79.5 | 109.5214 | 110.7566 | 112.6608 | 115.8481 | 119.3977 | 122.9555 | 126.1646 | 128.0882 | 129.3387 |
| 80.5 | 110.0086 | 111.2476 | 113.1583 | 116.3592 | 119.9272 | 123.5073 | 126.7394 | 128.6782 | 129.9391 |
| 81.5 | 110.495 | 111.7375 | 113.6548 | 116.869 | 120.4554 | 124.0576 | 127.3128 | 129.2668 | 130.5381 |
| 82.5 | 110.9801 | 112.2263 | 114.1499 | 117.3774 | 120.9821 | 124.6064 | 127.8846 | 129.8538 | 131.1356 |
| 83.5 | 111.4638 | 112.7135 | 114.6436 | 117.8842 | 121.5072 | 125.1535 | 128.4547 | 130.4392 | 131.7314 |
| 84.5 | 111.9459 | 113.1991 | 115.1356 | 118.3893 | 122.0305 | 125.6987 | 129.023 | 131.0226 | 132.3253 |
| 85.5 | 112.4259 | 113.6827 | 115.6257 | 118.8926 | 122.552 | 126.2421 | 129.5893 | 131.6041 | 132.9172 |
| 86.5 | 112.9036 | 114.1642 | 116.1136 | 119.3938 | 123.0714 | 126.7834 | 130.1535 | 132.1834 | 133.507 |
| 87.5 | 113.3789 | 114.6431 | 116.5992 | 119.8927 | 123.5886 | 127.3225 | 130.7154 | 132.7605 | 134.0943 |
| 88.5 | 113.8513 | 115.1194 | 117.0822 | 120.3893 | 124.1035 | 127.8594 | 131.275 | 133.335 | 134.6792 |


## Males, Stature, Ages 2-20 Years

| Age (in<br>months) | 3rd<br>Percentile<br>Stature (in<br>centimeters) | 5th<br>Percentile<br>Stature (in<br>centimeters) | 10th<br>Percentile<br>Stature (in<br>centimeters) | 25th<br>Percentile<br>Stature (in<br>centimeters) | 50th<br>Percentile<br>Stature (in<br>centimeters) | 75th<br>Percentile<br>Stature (in<br>centimeters) | 90th<br>Percentile<br>Stature (in<br>centimeters) | 95th<br>Percentile<br>Stature (in<br>centimeters) | 97th<br>Percentile<br>Stature (in<br>centimeters) |
|---|---|---|---|---|---|---|---|---|---|
| 89.5 | 114.3206 | 115.5927 | 117.5625 | 120.8833 | 124.616 | 128.3937 | 131.8321 | 133.907 | 135.2615 |
| 90.5 | 114.7867 | 116.0629 | 118.0398 | 121.3746 | 125.1259 | 128.9256 | 132.3865 | 134.4763 | 135.8409 |
| 91.5 | 115.2491 | 116.5297 | 118.5139 | 121.863 | 125.6331 | 129.4547 | 132.9381 | 135.0426 | 136.4173 |
| 92.5 | 115.7077 | 116.9928 | 118.9847 | 122.3483 | 126.1374 | 129.981 | 133.4868 | 135.606 | 136.9906 |
| 93.5 | 116.1623 | 117.4521 | 119.4519 | 122.8305 | 126.6388 | 130.5044 | 134.0325 | 136.1662 | 137.5607 |
| 94.5 | 116.6127 | 117.9074 | 119.9153 | 123.3092 | 127.137 | 131.0247 | 134.5751 | 136.7231 | 138.1274 |
| 95.5 | 117.0587 | 118.3585 | 120.3749 | 123.7845 | 127.632 | 131.5419 | 135.1144 | 137.2767 | 138.6906 |
| 96.5 | 117.5 | 118.8053 | 120.8305 | 124.2562 | 128.1237 | 132.0559 | 135.6504 | 137.8267 | 139.2502 |
| 97.5 | 117.9366 | 119.2475 | 121.2819 | 124.7242 | 128.6119 | 132.5664 | 136.1829 | 138.3731 | 139.806 |
| 98.5 | 118.3683 | 119.6851 | 121.729 | 125.1882 | 129.0966 | 133.0736 | 136.7118 | 138.9159 | 140.358 |
| 99.5 | 118.7949 | 120.1179 | 122.1716 | 125.6484 | 129.5777 | 133.5771 | 137.2371 | 139.4548 | 140.9062 |
| 100.5 | 119.2165 | 120.5459 | 122.6099 | 126.1045 | 130.055 | 134.0771 | 137.7587 | 139.9899 | 141.4503 |
| 101.5 | 119.633 | 120.969 | 123.0435 | 126.5565 | 130.5286 | 134.5734 | 138.2765 | 140.5211 | 141.9904 |
| 102.5 | 120.0442 | 121.3872 | 123.4726 | 127.0044 | 130.9983 | 135.066 | 138.7905 | 141.0484 | 142.5263 |
| 103.5 | 120.4502 | 121.8004 | 123.897 | 127.4481 | 131.4641 | 135.5548 | 139.3006 | 141.5716 | 143.0582 |
| 104.5 | 120.851 | 122.2086 | 124.3168 | 127.8876 | 131.926 | 136.0397 | 139.8069 | 142.0908 | 143.586 |
| 105.5 | 121.2467 | 122.6119 | 124.7319 | 128.3228 | 132.384 | 136.5209 | 140.3093 | 142.6061 | 144.1096 |
| 106.5 | 121.6372 | 123.0103 | 125.1425 | 128.7539 | 132.8381 | 136.9982 | 140.8077 | 143.1173 | 144.6291 |
| 107.5 | 122.0228 | 123.4039 | 125.5485 | 129.1807 | 133.2882 | 137.4717 | 141.3023 | 143.6245 | 145.1445 |
| 108.5 | 122.4034 | 123.7928 | 125.9501 | 129.6035 | 133.7345 | 137.9414 | 141.793 | 144.1278 | 145.656 |
| 109.5 | 122.7793 | 124.1771 | 126.3473 | 130.0222 | 134.1769 | 138.4073 | 142.28 | 144.6272 | 146.1634 |
| 110.5 | 123.1506 | 124.5569 | 126.7402 | 130.4369 | 134.6155 | 138.8696 | 142.7632 | 145.1228 | 146.6671 |
| 111.5 | 123.5175 | 124.9325 | 127.1291 | 130.8477 | 135.0504 | 139.3282 | 143.2428 | 145.6148 | 147.167 |
| 112.5 | 123.8803 | 125.304 | 127.514 | 131.2548 | 135.4818 | 139.7833 | 143.7188 | 146.1032 | 147.6633 |
| 113.5 | 124.2391 | 125.6717 | 127.8953 | 131.6584 | 135.9097 | 140.235 | 144.1915 | 146.5882 | 148.1562 |
| 114.5 | 124.5943 | 126.0358 | 128.273 | 132.0585 | 136.3343 | 140.6835 | 144.661 | 147.0699 | 148.6459 |
| 115.5 | 124.9462 | 126.3966 | 128.6474 | 132.4555 | 136.7557 | 141.1289 | 145.1273 | 147.5486 | 149.1325 |
| 116.5 | 125.295 | 126.7544 | 129.0189 | 132.8495 | 137.1742 | 141.5713 | 145.5909 | 148.0245 | 149.6163 |
| 117.5 | 125.6413 | 127.1096 | 129.3876 | 133.2407 | 137.5899 | 142.0111 | 146.0518 | 148.4979 | 150.0977 |
| 118.5 | 125.9852 | 127.4624 | 129.754 | 133.6295 | 138.0032 | 142.4484 | 146.5103 | 148.9689 | 150.5767 |
| 119.5 | 126.3272 | 127.8132 | 130.1183 | 134.0161 | 138.4143 | 142.8835 | 146.9668 | 149.438 | 151.0539 |
| 120.5 | 126.6678 | 128.1625 | 130.4809 | 134.4008 | 138.8234 | 143.3168 | 147.4214 | 149.9053 | 151.5294 |
| 121.5 | 127.0073 | 128.5106 | 130.8422 | 134.7841 | 139.231 | 143.7484 | 147.8747 | 150.3714 | 152.0038 |

http://www.cdc.gov/growthcharts/html charts/statage.htm/#males


Males, Stature, Ages 2-20 Years

| Age (in<br>months) | 3rd<br>Percentile<br>Stature (in<br>centimeters) | 5th<br>Percentile<br>Stature (in<br>centimeters) | 10th<br>Percentile<br>Stature (in<br>centimeters) | 25th<br>Percentile<br>Stature (in<br>centimeters) | 50th<br>Percentile<br>Stature (in<br>centimeters) | 75th<br>Percentile<br>Stature (in<br>centimeters) | 90th<br>Percentile<br>Stature (in<br>centimeters) | 95th<br>Percentile<br>Stature (in<br>centimeters) | 97th<br>Percentile<br>Stature (in<br>centimeters) |
|---|---|---|---|---|---|---|---|---|---|
| 122.5 | 127.3462 | 128.8579 | 131.2026 | 135.1663 | 139.6373 | 144.1789 | 148.3268 | 150.8365 | 152.4773 |
| 123.5 | 127.6851 | 129.2051 | 131.5625 | 135.5477 | 140.0427 | 144.6085 | 148.7782 | 151.301 | 152.9504 |
| 124.5 | 128.0243 | 129.5524 | 131.9224 | 135.9288 | 140.4477 | 145.0377 | 149.2294 | 151.7655 | 153.4235 |
| 125.5 | 128.3643 | 129.9004 | 132.2828 | 136.3101 | 140.8527 | 145.4669 | 149.6808 | 152.2303 | 153.8972 |
| 126.5 | 128.7058 | 130.2496 | 132.6441 | 136.692 | 141.2582 | 145.8965 | 150.1329 | 152.696 | 154.3718 |
| 127.5 | 129.0491 | 130.6005 | 133.0068 | 137.075 | 141.6646 | 146.3272 | 150.5861 | 153.1631 | 154.848 |
| 128.5 | 129.3949 | 130.9536 | 133.3714 | 137.4597 | 142.0725 | 146.7593 | 151.041 | 153.6321 | 155.3263 |
| 129.5 | 129.7436 | 131.3094 | 133.7386 | 137.8466 | 142.4824 | 147.1936 | 151.4982 | 154.1035 | 155.8072 |
| 130.5 | 130.0958 | 131.6686 | 134.1089 | 138.2362 | 142.8949 | 147.6305 | 151.9583 | 154.578 | 156.2913 |
| 131.5 | 130.452 | 132.0316 | 134.4828 | 138.6292 | 143.3107 | 148.0707 | 152.4218 | 155.0562 | 156.7792 |
| 132.5 | 130.8127 | 132.399 | 134.8608 | 139.0262 | 143.7304 | 148.5147 | 152.8894 | 155.5386 | 157.2715 |
| 133.5 | 131.1785 | 132.7714 | 135.2437 | 139.4278 | 144.1545 | 148.9633 | 153.3617 | 156.0258 | 157.7688 |
| 134.5 | 131.5498 | 133.1491 | 135.6318 | 139.8346 | 144.5838 | 149.4172 | 153.8394 | 156.5186 | 158.2717 |
| 135.5 | 131.9272 | 133.5329 | 136.026 | 140.2472 | 145.019 | 149.8769 | 154.323 | 157.0174 | 158.7806 |
| 136.5 | 132.311 | 133.9232 | 136.4266 | 140.6664 | 145.4607 | 150.3433 | 154.8133 | 157.5229 | 159.2964 |
| 137.5 | 132.7018 | 134.3205 | 136.8343 | 141.0928 | 145.9097 | 150.8169 | 155.3109 | 158.0356 | 159.8193 |
| 138.5 | 133.1 | 134.7252 | 137.2496 | 141.5269 | 146.3665 | 151.2984 | 155.8164 | 158.5562 | 160.35 |
| 139.5 | 133.5059 | 135.1378 | 137.673 | 141.9694 | 146.832 | 151.7885 | 156.3303 | 159.0851 | 160.889 |
| 140.5 | 133.9199 | 135.5588 | 138.105 | 142.4209 | 147.3066 | 152.2878 | 156.8532 | 159.6228 | 161.4365 |
| 141.5 | 134.3423 | 135.9885 | 138.5461 | 142.882 | 147.7911 | 152.7969 | 157.3857 | 160.1697 | 161.993 |
| 142.5 | 134.7733 | 136.4271 | 138.9968 | 143.3532 | 148.2859 | 153.3164 | 157.928 | 160.7262 | 162.5588 |
| 143.5 | 135.2132 | 136.8751 | 139.4573 | 143.835 | 148.7917 | 153.8466 | 158.4807 | 161.2924 | 163.1339 |
| 144.5 | 135.6621 | 137.3326 | 139.928 | 144.3277 | 149.3088 | 154.3881 | 159.0439 | 161.8686 | 163.7185 |
| 145.5 | 136.1202 | 137.7998 | 140.4091 | 144.8317 | 149.8376 | 154.941 | 159.6179 | 162.4549 | 164.3126 |
| 146.5 | 136.5875 | 138.2769 | 140.9009 | 145.3473 | 150.3784 | 155.5056 | 160.2026 | 163.0511 | 164.916 |
| 147.5 | 137.064 | 138.7638 | 141.4034 | 145.8746 | 150.9313 | 156.0819 | 160.7981 | 163.6571 | 165.5285 |
| 148.5 | 137.5496 | 139.2605 | 141.9167 | 146.4137 | 151.4964 | 156.6699 | 161.4041 | 164.2726 | 166.1497 |
| 149.5 | 138.0442 | 139.767 | 142.4407 | 146.9645 | 152.0735 | 157.2694 | 162.0203 | 164.8972 | 166.7791 |
| 150.5 | 138.5477 | 140.2831 | 142.9752 | 147.5269 | 152.6624 | 157.88 | 162.6462 | 165.5302 | 167.416 |
| 151.5 | 139.0597 | 140.8085 | 143.52 | 148.1005 | 153.2627 | 158.5012 | 163.2811 | 166.1711 | 168.0596 |
| 152.5 | 139.5799 | 141.3429 | 144.0746 | 148.6849 | 153.8738 | 159.1324 | 163.9243 | 166.8187 | 168.7091 |
| 153.5 | 140.108 | 141.8859 | 144.6388 | 149.2795 | 154.4951 | 159.7725 | 164.5748 | 167.4723 | 169.3634 |
| 154.5 | 140.6435 | 142.4369 | 145.2117 | 149.8836 | 155.1255 | 160.4207 | 165.2314 | 168.1305 | 170.0213 |


Males, Stature, Ages 2-20 Years

| Age (in<br>months) | 3rd<br>Percentile<br>Stature (in<br>centimeters) | 5th<br>Percentile<br>Stature (in<br>centimeters) | 10th<br>Percentile<br>Stature (in<br>centimeters) | 25th<br>Percentile<br>Stature (in<br>centimeters) | 50th<br>Percentile<br>Stature (in<br>centimeters) | 75th<br>Percentile<br>Stature (in<br>centimeters) | 90th<br>Percentile<br>Stature (in<br>centimeters) | 95th<br>Percentile<br>Stature (in<br>centimeters) | 97th<br>Percentile<br>Stature (in<br>centimeters) |
|---|---|---|---|---|---|---|---|---|---|
| 155.5 | 141.1858 | 142.9955 | 145.7928 | 150.4962 | 155.7642 | 161.0758 | 165.893 | 168.7923 | 170.6817 |
| 156.5 | 141.7345 | 143.5608 | 146.3813 | 151.1165 | 156.4099 | 161.7364 | 166.5581 | 169.4561 | 171.343 |
| 157.5 | 142.2889 | 144.1322 | 146.9763 | 151.7433 | 157.0612 | 162.401 | 167.2253 | 170.1205 | 172.004 |
| 158.5 | 142.8482 | 144.7089 | 147.5767 | 152.3754 | 157.7168 | 163.0682 | 167.8929 | 170.784 | 172.663 |
| 159.5 | 143.4118 | 145.29 | 148.1815 | 153.0113 | 158.3751 | 163.7363 | 168.5594 | 171.445 | 173.3186 |
| 160.5 | 143.9788 | 145.8746 | 148.7896 | 153.6498 | 159.0344 | 164.4035 | 169.2231 | 172.1018 | 173.9691 |
| 161.5 | 144.5483 | 146.4615 | 149.3998 | 154.2892 | 159.6931 | 165.0681 | 169.8822 | 172.7528 | 174.6131 |
| 162.5 | 145.1196 | 147.0498 | 150.0107 | 154.928 | 160.3493 | 165.7283 | 170.535 | 173.3965 | 175.249 |
| 163.5 | 145.6915 | 147.6385 | 150.621 | 155.5647 | 161.0015 | 166.3823 | 171.1798 | 174.0312 | 175.8753 |
| 164.5 | 146.2633 | 148.2262 | 151.2295 | 156.1977 | 161.6478 | 167.0284 | 171.8151 | 174.6554 | 176.4906 |
| 165.5 | 146.8339 | 148.812 | 151.8348 | 156.8253 | 162.2865 | 167.665 | 172.4393 | 175.2677 | 177.0935 |
| 166.5 | 147.4023 | 149.3947 | 152.4355 | 157.4462 | 162.9161 | 168.2905 | 173.0509 | 175.8668 | 177.6829 |
| 167.5 | 147.9674 | 149.9731 | 153.0304 | 158.0587 | 163.535 | 168.9033 | 173.6486 | 176.4515 | 178.2575 |
| 168.5 | 148.5284 | 150.5461 | 153.6181 | 158.6615 | 164.1418 | 169.5022 | 174.2313 | 177.0206 | 178.8165 |
| 169.5 | 149.0842 | 151.1127 | 154.1975 | 159.2532 | 164.7352 | 170.0859 | 174.7978 | 177.5733 | 179.3589 |
| 170.5 | 149.6338 | 151.6717 | 154.7674 | 159.8327 | 165.314 | 170.6535 | 175.3473 | 178.1088 | 179.884 |
| 171.5 | 150.1763 | 152.2221 | 155.3268 | 160.3988 | 165.8771 | 171.2039 | 175.879 | 178.6264 | 180.3913 |
| 172.5 | 150.7107 | 152.763 | 155.8746 | 160.9506 | 166.4236 | 171.7364 | 176.3923 | 179.1256 | 180.8804 |
| 173.5 | 151.2363 | 153.2935 | 156.4099 | 161.4872 | 166.9528 | 172.2504 | 176.8868 | 179.6061 | 181.3509 |
| 174.5 | 151.7521 | 153.8127 | 156.9319 | 162.0078 | 167.4641 | 172.7455 | 177.3622 | 180.0676 | 181.8027 |
| 175.5 | 152.2575 | 154.32 | 157.4399 | 162.5118 | 167.9571 | 173.2213 | 177.8183 | 180.5102 | 182.2358 |
| 176.5 | 152.7517 | 154.8147 | 157.9334 | 162.9988 | 168.4313 | 173.6778 | 178.2551 | 180.9338 | 182.6503 |
| 177.5 | 153.2342 | 155.2961 | 158.4118 | 163.4685 | 168.8867 | 174.1148 | 178.6727 | 181.3385 | 183.0463 |
| 178.5 | 153.7043 | 155.7638 | 158.8747 | 163.9205 | 169.3231 | 174.5324 | 179.0712 | 181.7247 | 183.4242 |
| 179.5 | 154.1615 | 156.2174 | 159.3218 | 164.3547 | 169.7405 | 174.9309 | 179.451 | 182.0927 | 183.7842 |
| 180.5 | 154.6056 | 156.6566 | 159.7529 | 164.7713 | 170.1393 | 175.3105 | 179.8124 | 182.4429 | 184.127 |
| 181.5 | 155.036 | 157.0811 | 160.168 | 165.1701 | 170.5195 | 175.6716 | 180.1559 | 182.7757 | 184.4528 |
| 182.5 | 155.4526 | 157.4907 | 160.5669 | 165.5514 | 170.8815 | 176.0146 | 180.482 | 183.0918 | 184.7624 |
| 183.5 | 155.8552 | 157.8853 | 160.9498 | 165.9154 | 171.2257 | 176.34 | 180.7912 | 183.3916 | 185.0562 |
| 184.5 | 156.2436 | 158.265 | 161.3167 | 166.2625 | 171.5525 | 176.6483 | 181.0841 | 183.6757 | 185.3349 |
| 185.5 | 156.6178 | 158.6298 | 161.6679 | 166.5929 | 171.8626 | 176.9402 | 181.3614 | 183.9449 | 185.599 |
| 186.5 | 156.9777 | 158.9798 | 162.0035 | 166.9072 | 172.1563 | 177.2163 | 181.6236 | 184.1997 | 185.8493 |
| 187.5 | 157.3235 | 159.315 | 162.3239 | 167.2057 | 172.4343 | 177.4771 | 181.8715 | 184.4408 | 186.0863 |


## Males, Stature, Ages 2-20 Years

| Age (in<br>months) | 3rd<br>Percentile<br>Stature (in<br>centimeters) | 5th<br>Percentile<br>Stature (in<br>centimeters) | 10th<br>Percentile<br>Stature (in<br>centimeters) | 25th<br>Percentile<br>Stature (in<br>centimeters) | 50th<br>Percentile<br>Stature (in<br>centimeters) | 75th<br>Percentile<br>Stature (in<br>centimeters) | 90th<br>Percentile<br>Stature (in<br>centimeters) | 95th<br>Percentile<br>Stature (in<br>centimeters) | 97th<br>Percentile<br>Stature (in<br>centimeters) |
|---|---|---|---|---|---|---|---|---|---|
| 188.5 | 157.6551 | 159.6359 | 162.6294 | 167.489 | 172.6972 | 177.7234 | 182.1056 | 184.6687 | 186.3107 |
| 189.5 | 157.9729 | 159.9425 | 162.9204 | 167.7576 | 172.9456 | 177.9558 | 182.3267 | 184.8843 | 186.5231 |
| 190.5 | 158.277 | 160.2352 | 163.1973 | 168.012 | 173.1801 | 178.175 | 182.5353 | 185.0879 | 186.724 |
| 191.5 | 158.5676 | 160.5143 | 163.4605 | 168.2528 | 173.4014 | 178.3815 | 182.7322 | 185.2804 | 186.9142 |
| 192.5 | 158.845 | 160.7802 | 163.7104 | 168.4805 | 173.6101 | 178.5762 | 182.9179 | 185.4623 | 187.0941 |
| 193.5 | 159.1095 | 161.0332 | 163.9476 | 168.6958 | 173.8067 | 178.7595 | 183.0931 | 185.6341 | 187.2643 |
| 194.5 | 159.3614 | 161.2738 | 164.1725 | 168.8991 | 173.992 | 178.9321 | 183.2583 | 185.7965 | 187.4254 |
| 195.5 | 159.6011 | 161.5023 | 164.3856 | 169.0911 | 174.1665 | 179.0946 | 183.414 | 185.9498 | 187.5779 |
| 196.5 | 159.829 | 161.7191 | 164.5873 | 169.2722 | 174.3308 | 179.2476 | 183.5609 | 186.0948 | 187.7222 |
| 197.5 | 160.0455 | 161.9247 | 164.7782 | 169.4431 | 174.4854 | 179.3915 | 183.6995 | 186.2318 | 187.8588 |
| 198.5 | 160.2508 | 162.1196 | 164.9587 | 169.6041 | 174.631 | 179.5271 | 183.8302 | 186.3613 | 187.9881 |
| 199.5 | 160.4456 | 162.3041 | 165.1292 | 169.756 | 174.768 | 179.6547 | 183.9535 | 186.4837 | 188.1106 |
| 200.5 | 160.63 | 162.4786 | 165.2903 | 169.8991 | 174.8969 | 179.7748 | 184.0699 | 186.5995 | 188.2267 |
| 201.5 | 160.8046 | 162.6437 | 165.4424 | 170.0339 | 175.0182 | 179.888 | 184.1797 | 186.7091 | 188.3368 |
| 202.5 | 160.9697 | 162.7997 | 165.586 | 170.1608 | 175.1323 | 179.9946 | 184.2835 | 186.8128 | 188.4411 |
| 203.5 | 161.1258 | 162.947 | 165.7214 | 170.2804 | 175.2398 | 180.095 | 184.3815 | 186.911 | 188.54 |
| 204.5 | 161.2733 | 163.086 | 165.8491 | 170.3931 | 175.341 | 180.1896 | 184.4741 | 187.004 | 188.6338 |
| 205.5 | 161.4125 | 163.2172 | 165.9694 | 170.4991 | 175.4362 | 180.2789 | 184.5617 | 187.0922 | 188.7229 |
| 206.5 | 161.5438 | 163.3409 | 166.0828 | 170.599 | 175.5259 | 180.3631 | 184.6446 | 187.1757 | 188.8075 |
| 207.5 | 161.6676 | 163.4575 | 166.1897 | 170.693 | 175.6104 | 180.4426 | 184.723 | 187.255 | 188.8878 |
| 208.5 | 161.7843 | 163.5673 | 166.2903 | 170.7816 | 175.6901 | 180.5176 | 184.7972 | 187.3302 | 188.9642 |
| 209.5 | 161.8942 | 163.6708 | 166.3851 | 170.865 | 175.7652 | 180.5885 | 184.8676 | 187.4016 | 189.0368 |
| 210.5 | 161.9977 | 163.7682 | 166.4743 | 170.9436 | 175.836 | 180.6555 | 184.9343 | 187.4694 | 189.1058 |
| 211.5 | 162.0951 | 163.8598 | 166.5583 | 171.0176 | 175.9028 | 180.7189 | 184.9975 | 187.5338 | 189.1715 |
| 212.5 | 162.1866 | 163.9461 | 166.6373 | 171.0873 | 175.9658 | 180.7789 | 185.0576 | 187.5951 | 189.234 |
| 213.5 | 162.2727 | 164.0272 | 166.7116 | 171.1529 | 176.0254 | 180.8357 | 185.1146 | 187.6534 | 189.2936 |
| 214.5 | 162.3537 | 164.1034 | 166.7816 | 171.2148 | 176.0816 | 180.8895 | 185.1687 | 187.7088 | 189.3503 |
| 215.5 | 162.4297 | 164.1751 | 166.8474 | 171.2732 | 176.1348 | 180.9405 | 185.2202 | 187.7617 | 189.4044 |
| 216.5 | 162.5011 | 164.2424 | 166.9094 | 171.3282 | 176.185 | 180.9889 | 185.2692 | 187.812 | 189.456 |
| 217.5 | 162.5681 | 164.3057 | 166.9676 | 171.3801 | 176.2326 | 181.0348 | 185.3159 | 187.86 | 189.5052 |
| 218.5 | 162.631 | 164.3651 | 167.0224 | 171.429 | 176.2776 | 181.0784 | 185.3603 | 187.9057 | 189.5522 |
| 219.5 | 162.69 | 164.4209 | 167.074 | 171.4752 | 176.3202 | 181.1199 | 185.4026 | 187.9494 | 189.5971 |
| 220.5 | 162.7453 | 164.4733 | 167.1224 | 171.5188 | 176.3606 | 181.1593 | 185.443 | 187.9911 | 189.6399 |


| Age (in<br>months) | 3rd<br>Percentile<br>Stature (in<br>centimeters) | 5th<br>Percentile<br>Stature (in<br>centimeters) | 10th<br>Percentile<br>Stature (in<br>centimeters) | 25th<br>Percentile<br>Stature (in<br>centimeters) | 50th<br>Percentile<br>Stature (in<br>centimeters) | 75th<br>Percentile<br>Stature (in<br>centimeters) | 90th<br>Percentile<br>Stature (in<br>centimeters) | 95th<br>Percentile<br>Stature (in<br>centimeters) | 97th<br>Percentile<br>Stature (in<br>centimeters) |
|---|---|---|---|---|---|---|---|---|---|
| | | | | S | | 3.4<br>(************************************ | | | |
| 221.5 | 162.7972 | 164.5224 | 167.168 | 171.5599 | 176.3989 | 181.1968 | 185.4815 | 188.0309 | 189.6809 |
| 222.5 | 162.8458 | 164.5686 | 167.2109 | 171.5988 | 176.4352 | 181.2325 | 185.5182 | 188.069 | 189.7201 |
| 223.5 | 162.8914 | 164.6119 | 167.2513 | 171.6355 | 176.4697 | 181.2666 | 185.5534 | 188.1054 | 189.7575 |
| 224.5 | 162.9341 | 164.6526 | 167.2892 | 171.6701 | 176.5024 | 181.299 | 185.5869 | 188.1402 | 189.7934 |
| 225.5 | 162.9741 | 164.6907 | 167.325 | 171.7029 | 176.5335 | 181.33 | 185.619 | 188.1736 | 189.8277 |
| 226.5 | 163.0115 | 164.7265 | 167.3585 | 171.7339 | 176.563 | 181.3595 | 185.6497 | 188.2055 | 189.8606 |
| 227.5 | 163.0465 | 164.76 | 167.3902 | 171.7632 | 176.5911 | 181.3877 | 185.6791 | 188.236 | 189.8922 |
| 228.5 | 163.0793 | 164.7915 | 167.4199 | 171.791 | 176.6179 | 181.4147 | 185.7073 | 188.2653 | 189.9224 |
| 229.5 | 163.11 | 164.821 | 167.4479 | 171.8172 | 176.6433 | 181.4405 | 185.7343 | 188.2934 | 189.9513 |
| 230.5 | 163.1387 | 164.8487 | 167.4742 | 171.8421 | 176.6676 | 181.4651 | 185.7601 | 188.3204 | 189.9791 |
| 231.5 | 163.1656 | 164.8746 | 167.499 | 171.8657 | 176.6907 | 181.4887 | 185.7849 | 188.3462 | 190.0058 |
| 232.5 | 163.1907 | 164.8989 | 167.5224 | 171.888 | 176.7127 | 181.5113 | 185.8087 | 188.3711 | 190.0314 |
| 233.5 | 163.2142 | 164.9217 | 167.5444 | 171.9091 | 176.7337 | 181.533 | 185.8316 | 188.3949 | 190.056 |
| 234.5 | 163.2361 | 164.9431 | 167.5651 | 171.9292 | 176.7538 | 181.5538 | 185.8535 | 188.4178 | 190.0797 |
| 235.5 | 163.2566 | 164.9631 | 167.5846 | 171.9483 | 176.773 | 181.5737 | 185.8746 | 188.4399 | 190.1024 |
| 236.5 | 163.2757 | 164.9819 | 167.6029 | 171.9663 | 176.7913 | 181.5928 | 185.8949 | 188.461 | 190.1242 |
| 237.5 | 163.2936 | 164.9995 | 167.6203 | 171.9835 | 176.8088 | 181.6111 | 185.9144 | 188.4814 | 190.1452 |
| 238.5 | 163.3103 | 165.016 | 167.6366 | 171.9998 | 176.8255 | 181.6287 | 185.9331 | 188.501 | 190.1654 |
| 239.5 | 163.3259 | 165.0315 | 167.6519 | 172.0153 | 176.8415 | 181.6456 | 185.9512 | 188.5198 | 190.1849 |
| 240 | 163.3333 | 165.0389 | 167.6593 | 172.0227 | 176.8492 | 181.6538 | 185.9599 | 188.529 | 190.1943 |
| 240 | 163.3333 | 165.0389 | 167.6593 | 172.0227 | 176.8492 | 181.6538 | 185.9599 | | 188.529 |

# 10.7 Appendix 7 CDC Data Table of Stature-for-age Chart for Females

### Females, Stature, Ages 2-20 Years

| Age (in<br>months) | 3rd<br>Percentile<br>Stature (in<br>centimeters) | 5th<br>Percentile<br>Stature (in<br>centimeters) | 10th<br>Percentile<br>Stature (in<br>centimeters) | 25th<br>Percentile<br>Stature (in<br>centimeters) | 50th<br>Percentile<br>Stature (in<br>centimeters) | 75th<br>Percentile<br>Stature (in<br>centimeters) | 90th<br>Percentile<br>Stature (in<br>centimeters) | 95th<br>Percentile<br>Stature (in<br>centimeters) | 97th<br>Percentile<br>Stature (in<br>centimeters) |
|---|---|---|---|---|---|---|---|---|---|
| 24 | 78.43754 | 79.25982 | 80.52476 | 82.63524 | 84.97556 | 87.31121 | 89.40951 | 90.66355 | 91.47729 |
| 24.5 | 78.82133 | 79.64777 | 80.91946 | 83.04213 | 85.39732 | 87.74918 | 89.86316 | 91.12707 | 91.94741 |
| 25.5 | 79.60198 | 80.44226 | 81.73541 | 83.8943 | 86.29026 | 88.68344 | 90.83505 | 92.12168 | 92.95685 |
| 26.5 | 80.37555 | 81.22666 | 82.53699 | 84.72592 | 87.15714 | 89.58751 | 91.77421 | 93.08254 | 93.93209 |
| 27.5 | 81.1357 | 81.9954 | 83.31968 | 85.53389 | 87.99602 | 90.46018 | 92.67969 | 94.00873 | 94.87215 |
| 28.5 | 81.87746 | 82.74411 | 84.07998 | 86.31589 | 88.80551 | 91.30065 | 93.55097 | 94.89974 | 95.77649 |
| 29.5 | 82.59712 | 83.46957 | 84.81532 | 87.07028 | 89.58477 | 92.10859 | 94.38793 | 95.75551 | 96.64505 |
| 30.5 | 83.29206 | 84.16953 | 85.52398 | 87.79609 | 90.33342 | 92.88403 | 95.19083 | 96.57635 | 97.47814 |
| 31.5 | 83.96065 | 84.84264 | 86.205 | 88.49291 | 91.05154 | 93.62741 | 95.9603 | 97.36295 | 98.27646 |
| 32.5 | 84.6021 | 85.4883 | 86.85807 | 89.16084 | 91.73964 | 94.33951 | 96.69729 | 98.11632 | 99.04107 |
| 33.5 | 85.2163 | 86.10656 | 87.48344 | 89.80045 | 92.39854 | 95.0214 | 97.40303 | 98.83778 | 99.77332 |
| 34.5 | 85.80379 | 86.69803 | 88.08186 | 90.4127 | 93.02945 | 95.67446 | 98.07904 | 99.52891 | 100.4748 |
| 35.5 | 86.36557 | 87.26379 | 88.6545 | 90.99891 | 93.63382 | 96.30029 | 98.72705 | 100.1915 | 101.1474 |
| 36.5 | 86.90307 | 87.80528 | 89.20285 | 91.56066 | 94.21336 | 96.90071 | 99.34899 | 100.8276 | 101.7931 |
| 37.5 | 87.43482 | 88.34236 | 89.74875 | 92.12298 | 94.79643 | 97.50724 | 99.97896 | 101.4726 | 102.4485 |
| 38.5 | 87.95945 | 88.87256 | 90.28811 | 92.67925 | 95.37392 | 98.10855 | 100.604 | 102.1129 | 103.0991 |
| 39.5 | 88.4785 | 89.39733 | 90.82228 | 93.2307 | 95.94693 | 98.70568 | 101.2251 | 102.7494 | 103.746 |
| 40.5 | 88.9933 | 89.91797 | 91.35246 | 93.7784 | 96.51645 | 99.29957 | 101.8432 | 103.383 | 104.3901 |
| 41.5 | 89.50502 | 90.43559 | 91.87972 | 94.32334 | 97.08337 | 99.89104 | 102.459 | 104.0144 | 105.032 |
| 42.5 | 90.01466 | 90.95115 | 92.40497 | 94.86634 | 97.64848 | 100.4808 | 103.0732 | 104.6444 | 105.6727 |
| 43.5 | 90.52307 | 91.46549 | 92.92901 | 95.40817 | 98.21247 | 101.0696 | 103.6866 | 105.2736 | 106.3126 |
| 44.5 | 91.031 | 91.97932 | 93.45252 | 95.94946 | 98.77593 | 101.6579 | 104.2996 | 105.9025 | 106.9523 |
| 45.5 | 91.53905 | 92.49325 | 93.97609 | 96.49076 | 99.3394 | 102.2462 | 104.9128 | 106.5316 | 107.5922 |
| 46.5 | 92.04774 | 93.00778 | 94.50021 | 97.03254 | 99.90331 | 102.835 | 105.5264 | 107.1613 | 108.2328 |
| 47.5 | 92.55748 | 93.52333 | 95.02528 | 97.57519 | 100.4681 | 103.4247 | 106.141 | 107.7919 | 108.8744 |
| 48.5 | 93.06862 | 94.04022 | 95.55164 | 98.11905 | 101.0339 | 104.0154 | 106.7567 | 108.4238 | 109.5172 |
| 49.5 | 93.58141 | 94.55872 | 96.07954 | 98.66436 | 101.6012 | 104.6075 | 107.3737 | 109.057 | 110.1614 |
| 50.5 | 94.09605 | 95.07903 | 96.60918 | 99.21132 | 102.17 | 105.2012 | 107.9924 | 109.6918 | 110.8073 |
| 51.5 | 94.61267 | 95.60128 | 97.14072 | 99.76009 | 102.7406 | 105.7965 | 108.6127 | 110.3283 | 111.4548 |
| 52.5 | 95.13134 | 96.12555 | 97.67423 | 100.3108 | 103.313 | 106.3936 | 109.2347 | 110.9665 | 112.1041 |
| 53.5 | 95.65211 | 96.65189 | 98.20976 | 100.8634 | 103.8873 | 106.9925 | 109.8585 | 111.6066 | 112.7552 |
| 54.5 | 96.17495 | 97.18029 | 98.74731 | 101.418 | 104.4635 | 107.5933 | 110.4841 | 112.2483 | 113.4079 |
| 55.5 | 96.69982 | 97.71069 | 99.28686 | 101.9745 | 105.0415 | 108.1958 | 111.1114 | 112.8917 | 114.0624 |

| Age (in<br>months) | 3rd<br>Percentile<br>Stature (in<br>centimeters) | 5th<br>Percentile<br>Stature (in<br>centimeters) | 10th<br>Percentile<br>Stature (in<br>centimeters) | 25th<br>Percentile<br>Stature (in<br>centimeters) | 50th<br>Percentile<br>Stature (in<br>centimeters) | 75th<br>Percentile<br>Stature (in<br>centimeters) | 90th<br>Percentile<br>Stature (in<br>centimeters) | 95th<br>Percentile<br>Stature (in<br>centimeters) | 97th<br>Percentile<br>Stature (in<br>centimeters) |
|---|---|---|---|---|---|---|---|---|---|
| 56.5 | 97.22663 | 98.24303 | 99.82832 | 102.5329 | 105.6213 | 108.8001 | 111.7404 | 113.5368 | 114.7184 |
| 57.5 | 97.75525 | 98.77719 | 100.3716 | 103.093 | 106.2029 | 109.406 | 112.3709 | 114.1833 | 115.3759 |
| 58.5 | 98.28555 | 99.31303 | 100.9165 | 103.6549 | 106.7861 | 110.0134 | 113.0028 | 114.8312 | 116.0347 |
| 59.5 | 98.81735 | 99.85039 | 101.463 | 104.2182 | 107.3707 | 110.6222 | 113.6359 | 115.4802 | 116.6945 |
| 60.5 | 99.35047 | 100.3891 | 102.0109 | 104.7829 | 107.9566 | 111.2321 | 114.2701 | 116.1301 | 117.3552 |
| 61.5 | 99.8847 | 100.9289 | 102.5599 | 105.3488 | 108.5436 | 111.8431 | 114.9052 | 116.7808 | 118.0166 |
| 62.5 | 100.4198 | 101.4696 | 103.1098 | 105.9156 | 109.1316 | 112.4548 | 115.5408 | 117.432 | 118.6783 |
| 63.5 | 100.9555 | 102.011 | 103.6604 | 106.4831 | 109.7202 | 113.0671 | 116.1768 | 118.0834 | 119.3402 |
| 64.5 | 101.4916 | 102.5529 | 104.2115 | 107.0512 | 110.3092 | 113.6797 | 116.813 | 118.7348 | 120.0019 |
| 65.5 | 102.0279 | 103.0948 | 104.7628 | 107.6194 | 110.8984 | 114.2923 | 117.449 | 119.3858 | 120.6632 |
| 66.5 | 102.564 | 103.6367 | 105.3141 | 108.1877 | 111.4876 | 114.9048 | 118.0845 | 120.0362 | 121.3238 |
| 67.5 | 103.0996 | 104.1782 | 105.865 | 108.7556 | 112.0764 | 115.5167 | 118.7193 | 120.6857 | 121.9832 |
| 68.5 | 103.6346 | 104.7191 | 106.4154 | 109.323 | 112.6646 | 116.1278 | 119.3531 | 121.334 | 122.6413 |
| 69.5 | 104.1685 | 105.259 | 106.9648 | 109.8895 | 113.2519 | 116.7379 | 119.9855 | 121.9807 | 123.2977 |
| 70.5 | 104.7012 | 105.7976 | 107.5131 | 110.4549 | 113.838 | 117.3466 | 120.6163 | 122.6256 | 123.9521 |
| 71.5 | 105.2323 | 106.3348 | 108.0599 | 111.0189 | 114.4226 | 117.9537 | 121.2452 | 123.2684 | 124.6042 |
| 72.5 | 105.7615 | 106.8701 | 108.605 | 111.5812 | 115.0055 | 118.5588 | 121.8718 | 123.9086 | 125.2536 |
| 73.5 | 106.2886 | 107.4033 | 109.148 | 112.1415 | 115.5863 | 119.1616 | 122.4959 | 124.5461 | 125.9 |
| 74.5 | 106.8132 | 107.9342 | 109.6888 | 112.6996 | 116.1648 | 119.7619 | 123.1171 | 125.1804 | 126.5432 |
| 75.5 | 107.3351 | 108.4624 | 110.227 | 113.255 | 116.7406 | 120.3594 | 123.7352 | 125.8114 | 127.1827 |
| 76.5 | 107.8541 | 108.9877 | 110.7623 | 113.8077 | 117.3136 | 120.9537 | 124.3499 | 126.4387 | 127.8184 |
| 77.5 | 108.3698 | 109.5099 | 111.2944 | 114.3572 | 117.8833 | 121.5447 | 124.9608 | 127.062 | 128.45 |
| 78.5 | 108.882 | 110.0285 | 111.8232 | 114.9034 | 118.4496 | 122.132 | 125.5678 | 127.6811 | 129.0771 |
| 79.5 | 109.3905 | 110.5435 | 112.3483 | 115.446 | 119.0123 | 122.7154 | 126.1705 | 128.2957 | 129.6996 |
| 80.5 | 109.8949 | 111.0545 | 112.8696 | 115.9847 | 119.571 | 123.2946 | 126.7688 | 128.9056 | 130.3171 |
| 81.5 | 110.3952 | 111.5613 | 113.3867 | 116.5193 | 120.1254 | 123.8695 | 127.3623 | 129.5105 | 130.9295 |
| 82.5 | 110.8909 | 112.0638 | 113.8995 | 117.0496 | 120.6755 | 124.4397 | 127.951 | 130.1103 | 131.5365 |
| 83.5 | 111.3821 | 112.5616 | 114.4077 | 117.5754 | 121.221 | 125.0051 | 128.5345 | 130.7047 | 132.138 |
| 84.5 | 111.8684 | 113.0546 | 114.9112 | 118.0964 | 121.7617 | 125.5655 | 129.1127 | 131.2936 | 132.7338 |
| 85.5 | 112.3496 | 113.5427 | 115.4097 | 118.6125 | 122.2974 | 126.1207 | 129.6855 | 131.8768 | 133.3238 |
| 86.5 | 112.8257 | 114.0256 | 115.9031 | 119.1235 | 122.8279 | 126.6706 | 130.2526 | 132.4542 | 133.9077 |
| 87.5 | 113.2963 | 114.5031 | 116.3913 | 119.6293 | 123.3531 | 127.215 | 130.814 | 133.0256 | 134.4857 |
| 88.5 | 113.7615 | 114.9752 | 116.874 | 120.1297 | 123.8728 | 127.7539 | 131.3696 | 133.5911 | 135.0574 |

http://www.cdc.gov/growthcharts/html\_charts/statage.htm/#females


| Age (in<br>months) | 3rd<br>Percentile<br>Stature (in<br>centimeters) | 5th<br>Percentile<br>Stature (in<br>centimeters) | 10th<br>Percentile<br>Stature (in<br>centimeters) | 25th<br>Percentile<br>Stature (in<br>centimeters) | 50th<br>Percentile<br>Stature (in<br>centimeters) | 75th<br>Percentile<br>Stature (in<br>centimeters) | 90th<br>Percentile<br>Stature (in<br>centimeters) | 95th<br>Percentile<br>Stature (in<br>centimeters) | 97th<br>Percentile<br>Stature (in<br>centimeters) |
|---|---|---|---|---|---|---|---|---|---|
| 89.5 | 114.2211 | 115.4418 | 117.3512 | 120.6246 | 124.387 | 128.287 | 131.9194 | 134.1505 | 135.623 |
| 90.5 | 114.6749 | 115.9026 | 117.8228 | 121.1138 | 124.8956 | 128.8144 | 132.4631 | 134.7038 | 136.1824 |
| 91.5 | 115.123 | 116.3577 | 118.2886 | 121.5974 | 125.3985 | 129.3359 | 133.0009 | 135.251 | 136.7356 |
| 92.5 | 115.5651 | 116.8069 | 118.7486 | 122.0753 | 125.8956 | 129.8516 | 133.5328 | 135.7922 | 137.2826 |
| 93.5 | 116.0012 | 117.2502 | 119.2028 | 122.5473 | 126.3869 | 130.3615 | 134.0587 | 136.3273 | 137.8236 |
| 94.5 | 116.4314 | 117.6875 | 119.6511 | 123.0135 | 126.8724 | 130.8656 | 134.5787 | 136.8565 | 138.3585 |
| 95.5 | 116.8555 | 118.1189 | 120.0935 | 123.4739 | 127.3522 | 131.364 | 135.093 | 137.3798 | 138.8876 |
| 96.5 | 117.2737 | 118.5443 | 120.53 | 123.9285 | 127.8263 | 131.8567 | 135.6015 | 137.8975 | 139.411 |
| 97.5 | 117.6858 | 118.9638 | 120.9607 | 124.3774 | 128.2947 | 132.3438 | 136.1046 | 138.4097 | 139.9289 |
| 98.5 | 118.092 | 119.3774 | 121.3855 | 124.8207 | 128.7576 | 132.8255 | 136.6024 | 138.9166 | 140.4415 |
| 99.5 | 118.4924 | 119.7852 | 121.8047 | 125.2584 | 129.2152 | 133.302 | 137.095 | 139.4184 | 140.9492 |
| 100.5 | 118.8869 | 120.1873 | 122.2182 | 125.6906 | 129.6675 | 133.7734 | 137.5828 | 139.9155 | 141.4521 |
| 101.5 | 119.2757 | 120.5838 | 122.6263 | 126.1177 | 130.1148 | 134.2401 | 138.066 | 140.4082 | 141.9507 |
| 102.5 | 119.659 | 120.9748 | 123.0291 | 126.5396 | 130.5574 | 134.7023 | 138.545 | 140.8968 | 142.4454 |
| 103.5 | 120.037 | 121.3606 | 123.4268 | 126.9568 | 130.9954 | 135.1604 | 139.0201 | 141.3817 | 142.9364 |
| 104.5 | 120.4097 | 121.7413 | 123.8196 | 127.3694 | 131.4293 | 135.6146 | 139.4918 | 141.8633 | 143.4244 |
| 105.5 | 120.7775 | 122.1171 | 124.2078 | 127.7777 | 131.8593 | 136.0654 | 139.9604 | 142.3422 | 143.9098 |
| 106.5 | 121.1405 | 122.4884 | 124.5916 | 128.1822 | 132.2859 | 136.5132 | 140.4265 | 142.8188 | 144.393 |
| 107.5 | 121.4991 | 122.8555 | 124.9715 | 128.5831 | 132.7094 | 136.9585 | 140.8906 | 143.2937 | 144.8747 |
| 108.5 | 121.8537 | 123.2186 | 125.3478 | 128.9808 | 133.1304 | 137.4018 | 141.3532 | 143.7674 | 145.3555 |
| 109.5 | 122.2044 | 123.5782 | 125.7208 | 129.3759 | 133.5493 | 137.8437 | 141.8149 | 144.2406 | 145.8359 |
| 110.5 | 122.5518 | 123.9347 | 126.0911 | 129.7689 | 133.9667 | 138.2847 | 142.2764 | 144.7139 | 146.3167 |
| 111.5 | 122.8963 | 124.2885 | 126.4592 | 130.1603 | 134.3832 | 138.7256 | 142.7382 | 145.1879 | 146.7984 |
| 112.5 | 123.2384 | 124.6402 | 126.8255 | 130.5506 | 134.7995 | 139.1669 | 143.2012 | 145.6634 | 147.2818 |
| 113.5 | 123.5785 | 124.9902 | 127.1907 | 130.9406 | 135.2163 | 139.6094 | 143.666 | 146.141 | 147.7676 |
| 114.5 | 123.9173 | 125.3393 | 127.5554 | 131.3309 | 135.6342 | 140.0538 | 144.1333 | 146.6215 | 148.2564 |
| 115.5 | 124.2553 | 125.688 | 127.9203 | 131.7223 | 136.054 | 140.501 | 144.6039 | 147.1056 | 148.7491 |
| 116.5 | 124.5933 | 126.0371 | 128.2861 | 132.1156 | 136.4766 | 140.9516 | 145.0785 | 147.594 | 149.2461 |
| 117.5 | 124.932 | 126.3872 | 128.6537 | 132.5115 | 136.9027 | 141.4065 | 145.5579 | 148.0874 | 149.7484 |
| 118.5 | 125.2721 | 126.7392 | 129.0238 | 132.9109 | 137.3333 | 141.8665 | 146.0429 | 148.5865 | 150.2564 |
| 119.5 | 125.6144 | 127.094 | 129.3973 | 133.3147 | 137.7691 | 142.3324 | 146.5341 | 149.092 | 150.7707 |
| 120.5 | 125.9599 | 127.4524 | 129.7752 | 133.7239 | 138.2112 | 142.8051 | 147.0322 | 149.6044 | 151.292 |
| 121.5 | 126.3095 | 127.8154 | 130.1584 | 134.1394 | 138.6602 | 143.2852 | 147.5379 | 150.1242 | 151.8205 |

http://www.cdc.gov/growthcharts/html\_charts/statage.htm/#females


| Age (in<br>months) | 3rd<br>Percentile<br>Stature (in<br>centimeters) | 5th<br>Percentile<br>Stature (in<br>centimeters) | 10th<br>Percentile<br>Stature (in<br>centimeters) | 25th<br>Percentile<br>Stature (in<br>centimeters) | 50th<br>Percentile<br>Stature (in<br>centimeters) | 75th<br>Percentile<br>Stature (in<br>centimeters) | 90th<br>Percentile<br>Stature (in<br>centimeters) | 95th<br>Percentile<br>Stature (in<br>centimeters) | 97th<br>Percentile<br>Stature (in<br>centimeters) |
|---|---|---|---|---|---|---|---|---|---|
| 122.5 | 126.6641 | 128.184 | 130.5479 | 134.562 | 139.1172 | 143.7735 | 148.0517 | 150.652 | 152.3568 |
| 123.5 | 127.0248 | 128.5591 | 130.9446 | 134.9929 | 139.5829 | 144.2707 | 148.5741 | 151.188 | 152.9011 |
| 124.5 | 127.3926 | 128.9419 | 131.3496 | 135.4328 | 140.0581 | 144.7773 | 149.1054 | 151.7325 | 153.4534 |
| 125.5 | 127.7687 | 129.3334 | 131.7639 | 135.8826 | 140.5435 | 145.2938 | 149.646 | 152.2856 | 154.0139 |
| 126.5 | 128.1541 | 129.7346 | 132.1885 | 136.3433 | 141.0397 | 145.8206 | 150.196 | 152.8473 | 154.5824 |
| 127.5 | 128.5499 | 130.1467 | 132.6243 | 136.8154 | 141.5472 | 146.3579 | 150.7552 | 153.4174 | 155.1586 |
| 128.5 | 128.9573 | 130.5705 | 133.0721 | 137.2997 | 142.0664 | 146.9059 | 151.3236 | 153.9955 | 155.742 |
| 129.5 | 129.3772 | 131.0071 | 133.5329 | 137.7967 | 142.5974 | 147.4643 | 151.9008 | 154.5812 | 156.3321 |
| 130.5 | 129.8106 | 131.4573 | 134.0072 | 138.3067 | 143.1404 | 148.0329 | 152.4861 | 155.1737 | 156.928 |
| 131.5 | 130.2585 | 131.9218 | 134.4955 | 138.83 | 143.695 | 148.6111 | 153.079 | 155.7721 | 157.5288 |
| 132.5 | 130.7217 | 132.4013 | 134.9983 | 139.3664 | 144.2609 | 149.1984 | 153.6783 | 156.3755 | 158.1335 |
| 133.5 | 131.2006 | 132.8962 | 135.5157 | 139.9157 | 144.8376 | 149.7937 | 154.283 | 156.9825 | 158.7407 |
| 134.5 | 131.6958 | 133.4067 | 136.0476 | 140.4775 | 145.424 | 150.3959 | 154.8918 | 157.5918 | 159.3491 |
| 135.5 | 132.2074 | 133.9328 | 136.5937 | 141.051 | 146.0192 | 151.0036 | 155.5032 | 158.202 | 159.9571 |
| 136.5 | 132.7354 | 134.4742 | 137.1534 | 141.6352 | 146.6217 | 151.6153 | 156.1156 | 158.8115 | 160.5633 |
| 137.5 | 133.2795 | 135.0304 | 137.7259 | 142.2288 | 147.23 | 152.2293 | 156.7273 | 159.4185 | 161.166 |
| 138.5 | 133.8388 | 135.6004 | 138.31 | 142.8304 | 147.8424 | 152.8438 | 157.3365 | 160.0213 | 161.7634 |
| 139.5 | 134.4125 | 136.1831 | 138.9043 | 143.4381 | 148.4569 | 153.4568 | 157.9413 | 160.6182 | 162.3541 |
| 140.5 | 134.9993 | 136.7769 | 139.507 | 144.0501 | 149.0714 | 154.0662 | 158.5398 | 161.2075 | 162.9363 |
| 141.5 | 135.5973 | 137.3801 | 140.1161 | 144.6641 | 149.6839 | 154.67 | 159.1302 | 161.7874 | 163.5084 |
| 142.5 | 136.2047 | 137.9905 | 140.7295 | 145.278 | 150.292 | 155.2663 | 159.7107 | 162.3564 | 164.069 |
| 143.5 | 136.8191 | 138.6058 | 141.3448 | 145.8893 | 150.8936 | 155.8529 | 160.2796 | 162.9129 | 164.6167 |
| 144.5 | 137.4381 | 139.2236 | 141.9594 | 146.4958 | 151.4866 | 156.428 | 160.8353 | 163.4555 | 165.1503 |
| 145.5 | 138.0588 | 139.841 | 142.5709 | 147.0949 | 152.0687 | 156.9899 | 161.3764 | 163.983 | 165.6685 |
| 146.5 | 138.6784 | 140.4554 | 143.1767 | 147.6845 | 152.6381 | 157.5369 | 161.9016 | 164.4943 | 166.1706 |
| 147.5 | 139.2941 | 141.064 | 143.7741 | 148.2623 | 153.193 | 158.0677 | 162.4097 | 164.9885 | 166.6555 |
| 148.5 | 139.9028 | 141.6641 | 144.3607 | 148.8263 | 153.7317 | 158.581 | 162.8999 | 165.4648 | 167.1228 |
| 149.5 | 140.5019 | 142.253 | 144.9342 | 149.3747 | 154.2529 | 159.0758 | 163.3715 | 165.9227 | 167.572 |
| 150.5 | 141.0885 | 142.8283 | 145.4925 | 149.9059 | 154.7555 | 159.5513 | 163.8239 | 166.3618 | 168.0027 |
| 151.5 | 141.6602 | 143.3877 | 146.0338 | 150.4184 | 155.2385 | 160.007 | 164.2568 | 166.7819 | 168.4147 |
| 152.5 | 142.2148 | 143.9294 | 146.5564 | 150.9113 | 155.7012 | 160.4425 | 164.6701 | 167.1829 | 168.808 |
| 153.5 | 142.7504 | 144.4516 | 147.059 | 151.3835 | 156.1432 | 160.8576 | 165.0637 | 167.5648 | 169.1827 |
| 154.5 | 143.2654 | 144.953 | 147.5405 | 151.8346 | 156.5643 | 161.2524 | 165.4378 | 167.9278 | 169.5391 |


| Age (in<br>months) | 3rd<br>Percentile<br>Stature (in<br>centimeters) | 5th<br>Percentile<br>Stature (in<br>centimeters) | 10th<br>Percentile<br>Stature (in<br>centimeters) | 25th<br>Percentile<br>Stature (in<br>centimeters) | 50th<br>Percentile<br>Stature (in<br>centimeters) | 75th<br>Percentile<br>Stature (in<br>centimeters) | 90th<br>Percentile<br>Stature (in<br>centimeters) | 95th<br>Percentile<br>Stature (in<br>centimeters) | 97th<br>Percentile<br>Stature (in<br>centimeters) |
|---|---|---|---|---|---|---|---|---|---|
| 155.5 | 143.7584 | 145.4325 | 148.0002 | 152.2642 | 156.9644 | 161.627 | 165.7928 | 168.2723 | 169.8773 |
| 156.5 | 144.2287 | 145.8894 | 148.4376 | 152.6721 | 157.3437 | 161.9818 | 166.1289 | 168.5987 | 170.1979 |
| 157.5 | 144.6756 | 146.3232 | 148.8525 | 153.0584 | 157.7025 | 162.3172 | 166.4466 | 168.9074 | 170.5013 |
| 158.5 | 145.0987 | 146.7338 | 149.2449 | 153.4234 | 158.0411 | 162.6338 | 166.7467 | 169.199 | 170.7881 |
| 159.5 | 145.4981 | 147.1213 | 149.615 | 153.7674 | 158.3603 | 162.9321 | 167.0296 | 169.4742 | 171.0587 |
| 160.5 | 145.874 | 147.4859 | 149.9633 | 154.0911 | 158.6606 | 163.2129 | 167.2961 | 169.7335 | 171.314 |
| 161.5 | 146.2269 | 147.8281 | 150.2902 | 154.3951 | 158.9427 | 163.477 | 167.5469 | 169.9777 | 171.5544 |
| 162.5 | 146.5573 | 148.1487 | 150.5966 | 154.6801 | 159.2075 | 163.725 | 167.7826 | 170.2074 | 171.7807 |
| 163.5 | 146.866 | 148.4483 | 150.8831 | 154.947 | 159.4557 | 163.9577 | 168.0042 | 170.4234 | 171.9935 |
| 164.5 | 147.1539 | 148.7279 | 151.1507 | 155.1966 | 159.6882 | 164.1761 | 168.2122 | 170.6263 | 172.1936 |
| 165.5 | 147.4219 | 148.9885 | 151.4003 | 155.4298 | 159.9058 | 164.3808 | 168.4075 | 170.817 | 172.3816 |
| 166.5 | 147.6712 | 149.2309 | 151.6329 | 155.6475 | 160.1094 | 164.5726 | 168.5907 | 170.9959 | 172.5582 |
| 167.5 | 147.9026 | 149.4562 | 151.8494 | 155.8507 | 160.2997 | 164.7523 | 168.7626 | 171.1639 | 172.7239 |
| 168.5 | 148.1173 | 149.6655 | 152.0508 | 156.0401 | 160.4777 | 164.9206 | 168.9239 | 171.3216 | 172.8796 |
| 169.5 | 148.3164 | 149.8598 | 152.2381 | 156.2167 | 160.6441 | 165.0783 | 169.0751 | 171.4696 | 173.0257 |
| 170.5 | 148.5009 | 150.04 | 152.4121 | 156.3813 | 160.7995 | 165.226 | 169.217 | 171.6085 | 173.1628 |
| 171.5 | 148.6717 | 150.2072 | 152.5738 | 156.5348 | 160.9449 | 165.3644 | 169.3501 | 171.7388 | 173.2915 |
| 172.5 | 148.8299 | 150.3621 | 152.7241 | 156.6778 | 161.0808 | 165.4941 | 169.4749 | 171.8611 | 173.4124 |
| 173.5 | 148.9764 | 150.5059 | 152.8638 | 156.8112 | 161.2079 | 165.6157 | 169.5921 | 171.976 | 173.5258 |
| 174.5 | 149.1121 | 150.6392 | 152.9936 | 156.9356 | 161.3268 | 165.7297 | 169.7022 | 172.0839 | 173.6324 |
| 175.5 | 149.2377 | 150.7629 | 153.1143 | 157.0517 | 161.4381 | 165.8366 | 169.8055 | 172.1853 | 173.7326 |
| 176.5 | 149.3542 | 150.8777 | 153.2266 | 157.16 | 161.5423 | 165.9369 | 169.9026 | 172.2806 | 173.8267 |
| 177.5 | 149.4622 | 150.9843 | 153.3312 | 157.2612 | 161.6399 | 166.0312 | 169.9939 | 172.3701 | 173.9152 |
| 178.5 | 149.5623 | 151.0833 | 153.4286 | 157.3558 | 161.7315 | 166.1197 | 170.0798 | 172.4544 | 173.9984 |
| 179.5 | 149.6553 | 151.1754 | 153.5193 | 157.4443 | 161.8174 | 166.2029 | 170.1606 | 172.5337 | 174.0768 |
| 180.5 | 149.7416 | 151.2611 | 153.604 | 157.5271 | 161.898 | 166.2812 | 170.2366 | 172.6084 | 174.1505 |
| 181.5 | 149.8219 | 151.341 | 153.683 | 157.6047 | 161.9738 | 166.3549 | 170.3083 | 172.6787 | 174.22 |
| 182.5 | 149.8967 | 151.4154 | 153.7569 | 157.6775 | 162.045 | 166.4244 | 170.3759 | 172.7451 | 174.2855 |
| 183.5 | 149.9663 | 151.4848 | 153.826 | 157.7458 | 162.112 | 166.4898 | 170.4396 | 172.8076 | 174.3472 |
| 184.5 | 150.0312 | 151.5497 | 153.8907 | 157.8099 | 162.1752 | 166.5516 | 170.4997 | 172.8667 | 174.4055 |
| 185.5 | 150.0918 | 151.6103 | 153.9513 | 157.8702 | 162.2347 | 166.6099 | 170.5566 | 172.9225 | 174.4606 |
| 186.5 | 150.1484 | 151.6671 | 154.0082 | 157.927 | 162.2908 | 166.6649 | 170.6103 | 172.9752 | 174.5125 |
| 187.5 | 150.2014 | 151.7203 | 154.0616 | 157.9804 | 162.3439 | 166.717 | 170.6611 | 173.025 | 174.5617 |


| Age (in<br>months) | 3rd<br>Percentile<br>Stature (in<br>centimeters) | 5th<br>Percentile<br>Stature (in<br>centimeters) | 10th<br>Percentile<br>Stature (in<br>centimeters) | 25th<br>Percentile<br>Stature (in<br>centimeters) | 50th<br>Percentile<br>Stature (in<br>centimeters) | 75th<br>Percentile<br>Stature (in<br>centimeters) | 90th<br>Percentile<br>Stature (in<br>centimeters) | 95th<br>Percentile<br>Stature (in<br>centimeters) | 97th<br>Percentile<br>Stature (in<br>centimeters) |
|---|---|---|---|---|---|---|---|---|---|
| 188.5 | 150.251 | 151.7702 | 154.1119 | 158.0308 | 162.394 | 166.7663 | 170.7091 | 173.0722 | 174.6082 |
| 189.5 | 150.2975 | 151.8171 | 154.1592 | 158.0784 | 162.4414 | 166.8129 | 170.7546 | 173.1168 | 174.6522 |
| 190.5 | 150.3412 | 151.8612 | 154.2037 | 158.1234 | 162.4862 | 166.8571 | 170.7978 | 173.1591 | 174.6938 |
| 191.5 | 150.3823 | 151.9027 | 154.2457 | 158.1659 | 162.5287 | 166.899 | 170.8387 | 173.1992 | 174.7333 |
| 192.5 | 150.4209 | 151.9418 | 154.2854 | 158.2061 | 162.569 | 166.9388 | 170.8775 | 173.2373 | 174.7708 |
| 193.5 | 150.4573 | 151.9787 | 154.3229 | 158.2442 | 162.6072 | 166.9766 | 170.9144 | 173.2734 | 174.8063 |
| 194.5 | 150.4917 | 152.0135 | 154.3584 | 158.2803 | 162.6435 | 167.0125 | 170.9494 | 173.3077 | 174.84 |
| 195.5 | 150.5241 | 152.0465 | 154.3919 | 158.3146 | 162.6781 | 167.0466 | 170.9827 | 173.3402 | 174.8721 |
| 196.5 | 150.5547 | 152.0776 | 154.4238 | 158.3472 | 162.7109 | 167.0791 | 171.0144 | 173.3712 | 174.9025 |
| 197.5 | 150.5837 | 152.1072 | 154.454 | 158.3782 | 162.7421 | 167.11 | 171.0446 | 173.4007 | 174.9314 |
| 198.5 | 150.6111 | 152.1352 | 154.4827 | 158.4077 | 162.7719 | 167.1395 | 171.0733 | 173.4288 | 174.959 |
| 199.5 | 150.6372 | 152.1617 | 154.51 | 158.4357 | 162.8002 | 167.1676 | 171.1007 | 173.4555 | 174.9852 |
| 200.5 | 150.6619 | 152.187 | 154.5359 | 158.4625 | 162.8273 | 167.1944 | 171.1268 | 173.481 | 175.0102 |
| 201.5 | 150.6854 | 152.211 | 154.5607 | 158.4879 | 162.8531 | 167.22 | 171.1517 | 173.5053 | 175.034 |
| 202.5 | 150.7077 | 152.2339 | 154.5842 | 158.5123 | 162.8778 | 167.2444 | 171.1754 | 173.5284 | 175.0567 |
| 203.5 | 150.7289 | 152.2556 | 154.6067 | 158.5355 | 162.9013 | 167.2677 | 171.1981 | 173.5505 | 175.0783 |
| 204.5 | 150.7491 | 152.2764 | 154.6281 | 158.5577 | 162.9238 | 167.29 | 171.2198 | 173.5716 | 175.099 |
| 205.5 | 150.7684 | 152.2962 | 154.6486 | 158.5789 | 162.9454 | 167.3114 | 171.2405 | 173.5918 | 175.1187 |
| 206.5 | 150.7868 | 152.3151 | 154.6681 | 158.5992 | 162.966 | 167.3318 | 171.2604 | 173.6111 | 175.1376 |
| 207.5 | 150.8044 | 152.3332 | 154.6868 | 158.6187 | 162.9858 | 167.3514 | 171.2793 | 173.6295 | 175.1556 |
| 208.5 | 150.8211 | 152.3504 | 154.7047 | 158.6373 | 163.0047 | 167.3701 | 171.2975 | 173.6471 | 175.1728 |
| 209.5 | 150.8372 | 152.3669 | 154.7218 | 158.6551 | 163.0228 | 167.3881 | 171.3149 | 173.664 | 175.1892 |
| 210.5 | 150.8525 | 152.3827 | 154.7382 | 158.6722 | 163.0402 | 167.4053 | 171.3315 | 173.6802 | 175.205 |
| 211.5 | 150.8672 | 152.3979 | 154.754 | 158.6886 | 163.0569 | 167.4218 | 171.3475 | 173.6956 | 175.2201 |
| 212.5 | 150.8812 | 152.4124 | 154.769 | 158.7043 | 163.0729 | 167.4376 | 171.3628 | 173.7104 | 175.2345 |
| 213.5 | 150.8947 | 152.4263 | 154.7835 | 158.7194 | 163.0882 | 167.4528 | 171.3775 | 173.7246 | 175.2483 |
| 214.5 | 150.9076 | 152.4396 | 154.7974 | 158.7339 | 163.103 | 167.4674 | 171.3915 | 173.7382 | 175.2616 |
| 215.5 | 150.92 | 152.4524 | 154.8107 | 158.7478 | 163.1172 | 167.4814 | 171.405 | 173.7513 | 175.2742 |
| 216.5 | 150.9319 | 152.4647 | 154.8235 | 158.7612 | 163.1308 | 167.4948 | 171.418 | 173.7638 | 175.2864 |
| 217.5 | 150.9433 | 152.4765 | 154.8358 | 158.774 | 163.1439 | 167.5078 | 171.4304 | 173.7758 | 175.2981 |
| 218.5 | 150.9542 | 152.4878 | 154.8476 | 158.7864 | 163.1565 | 167.5202 | 171.4424 | 173.7873 | 175.3093 |
| 219.5 | 150.9647 | 152.4987 | 154.859 | 158.7983 | 163.1686 | 167.5321 | 171.4538 | 173.7984 | 175.32 |
| 220.5 | 150.9749 | 152.5092 | 154.8699 | 158.8097 | 163.1802 | 167.5436 | 171.4649 | 173.809 | 175.3303 |


| Age (in<br>months) | 3rd<br>Percentile<br>Stature (in<br>centimeters) | 5th<br>Percentile<br>Stature (in<br>centimeters) | 10th<br>Percentile<br>Stature (in<br>centimeters) | 25th<br>Percentile<br>Stature (in<br>centimeters) | 50th<br>Percentile<br>Stature (in<br>centimeters) | 75th<br>Percentile<br>Stature (in<br>centimeters) | 90th<br>Percentile<br>Stature (in<br>centimeters) | 95th<br>Percentile<br>Stature (in<br>centimeters) | 97th<br>Percentile<br>Stature (in<br>centimeters) |
|---|---|---|---|---|---|---|---|---|---|
| 221.5 | 150.9846 | 152.5192 | 154.8804 | 158.8207 | 163.1914 | 167.5546 | 171.4755 | 173.8192 | 175.3402 |
| 222.5 | 150.9939 | 152.5289 | 154.8905 | 158.8313 | 163.2022 | 167.5653 | 171.4856 | 173.8192 | 175.3402 |
| | 151.0029 | 152.5382 | 154.9003 | 158.8415 | 163.2126 | 167.5755 | 171.4954 | 173.8384 | 175.3588 |
| | 151.0115 | 152.5472 | 154.9096 | 158.8514 | 163.2226 | 167.5853 | 171.5049 | 173.8474 | 175.3675 |
| 225.5 | 151.0198 | 152.5558 | 154.9187 | 158.8608 | 163.2322 | 167.5948 | 171.5139 | 173.8561 | 175.376 |
| 226.5 | 151.0279 | 152.5641 | 154.9273 | 158.8699 | 163.2415 | 167.6039 | 171.5226 | 173.8645 | 175.384 |
| 227.5 | 151.0356 | 152.5721 | 154.9357 | 158.8787 | 163.2504 | 167.6127 | 171.531 | 173.8725 | 175.3918 |
| 228.5 | 151.043 | 152.5798 | 154.9438 | 158.8872 | 163.259 | 167.6211 | 171.5391 | 173.8802 | 175.3993 |
| 229.5 | 151.0501 | 152.5873 | 154.9516 | 158.8953 | 163.2673 | 167.6293 | 171.5468 | 173.8877 | 175.4064 |
| 230.5 | 151.057 | 152.5944 | 154.959 | 158.9032 | 163.2753 | 167.6371 | 171.5543 | 173.8948 | 175.4133 |
| 231.5 | 151.0636 | 152.6013 | 154.9663 | 158.9107 | 163.283 | 167.6446 | 171.5615 | 173.9017 | 175.42 |
| 232.5 | 151.07 | 152.6079 | 154.9732 | 158.918 | 163.2904 | 167.6519 | 171.5684 | 173.9083 | 175.4264 |
| 233.5 | 151.0762 | 152.6143 | 154.9799 | 158.9251 | 163.2976 | 167.6589 | 171.5751 | 173.9147 | 175.4325 |
| 234.5 | 151.0821 | 152.6205 | 154.9864 | 158.9319 | 163.3045 | 167.6657 | 171.5815 | 173.9208 | 175.4384 |
| 235.5 | 151.0879 | 152.6265 | 154.9926 | 158.9384 | 163.3111 | 167.6722 | 171.5877 | 173.9267 | 175.4441 |
| 236.5 | 151.0934 | 152.6322 | 154.9986 | 158.9447 | 163.3175 | 167.6785 | 171.5937 | 173.9324 | 175.4496 |
| 237.5 | 151.0987 | 152.6377 | 155.0044 | 158.9508 | 163.3237 | 167.6845 | 171.5994 | 173.9379 | 175.4548 |
| 238.5 | 151.1038 | 152.6431 | 155.01 | 158.9567 | 163.3297 | 167.6904 | 171.6049 | 173.9432 | 175.4599 |
| 239.5 | 151.1088 | 152.6482 | 155.0154 | 158.9624 | 163.3354 | 167.696 | 171.6103 | 173.9482 | 175.4648 |
| 240 | 151.1112 | 152.6507 | 155.0181 | 158.9651 | 163.3383 | 167.6987 | 171.6129 | 173.9507 | 175.4671 |

# 10.8 Appendix 8 CDC Data Table of Weight-for-age Chart for Males

| | | | | | Trail | | | | 0=.1 |
|---|---|---|---|---|---|---|---|---|---|
| | 3rd<br>Percentile | 5th<br>Percentile | 10th<br>Percentile | 25th<br>Percentile | 50th<br>Percentile | 75th<br>Percentile | 90th<br>Percentile | 95th<br>Percentile | 97th<br>Percentile |
| 0 \ | | Weight (in | Weight (in | Weight (in | Weight (in | Weight (in | Weight (in | Weight (in | Weight (in |
| | kilograms) | kilograms) | kilograms) | kilograms) | kilograms) | kilograms) | kilograms) | kilograms) | kilograms) |
| 24 | 10.38209 | 10.64009 | 11.05266 | 11.78598 | 12.67076 | 13.63692 | 14.5834 | 15.18777 | 15.59648 |
| 24.5 | 10.44144 | 10.70051 | 11.1149 | 11.85182 | 12.74154 | 13.71386 | 14.66716 | 15.2763 | 15.68841 |
| 25.5 | 10.55847 | 10.81958 | 11.23747 | 11.98142 | 12.88102 | 13.8659 | 14.83332 | 15.45242 | 15.8717 |
| 26.5 | 10.6738 | 10.93681 | 11.35806 | 12.10889 | 13.01842 | 14.01623 | 14.99848 | 15.62819 | 16.05514 |
| 27.5 | 10.78798 | 11.0528 | 11.47728 | 12.23491 | 13.1545 | 14.16567 | 15.16351 | 15.8045 | 16.23967 |
| 28.5 | 10.90147 | 11.16803 | 11.59567 | 12.36007 | 13.2899 | 14.31493 | 15.32917 | 15.98214 | 16.42609 |
| 29.5 | 11.01466 | 11.28293 | 11.71368 | 12.4849 | 13.42519 | 14.46462 | 15.4961 | 16.16177 | 16.61508 |
| 30.5 | 11.12787 | 11.39782 | 11.8317 | 12.60983 | 13.56088 | 14.61527 | 15.66485 | 16.34395 | 16.8072 |
| 31.5 | 11.24135 | 11.513 | 11.95005 | 12.73523 | 13.69738 | 14.76732 | 15.83588 | 16.52915 | 17.00291 |
| 32.5 | 11.3553 | 11.62869 | 12.069 | 12.86144 | 13.83505 | 14.92117 | 16.00958 | 16.71773 | 17.2026 |
| 33.5 | 11.46988 | 11.74508 | 12.18875 | 12.9887 | 13.97418 | 15.07711 | 16.18624 | 16.91 | 17.40654 |
| 34.5 | 11.58521 | 11.8623 | 12.30948 | 13.11723 | 14.11503 | 15.23541 | 16.36612 | 17.10619 | 17.61495 |
| 35.5 | 11.70137 | 11.98046 | 12.43132 | 13.24721 | 14.2578 | 15.39628 | 16.5494 | 17.30646 | 17.82797 |
| 36.5 | 11.81842 | 12.09962 | 12.55436 | 13.37875 | 14.40263 | 15.55987 | 16.73623 | 17.51093 | 18.0457 |
| 37.5 | 11.93639 | 12.21984 | 12.67868 | 13.51197 | 14.54965 | 15.7263 | 16.9267 | 17.71965 | 18.26818 |
| 38.5 | 12.05529 | 12.34115 | 12.80431 | 13.64693 | 14.69893 | 15.89565 | 17.12085 | 17.93265 | 18.49539 |
| 39.5 | 12.17512 | 12.46354 | 12.93128 | 13.78366 | 14.85054 | 16.06797 | 17.3187 | 18.14992 | 18.72731 |
| 40.5 | 12.29587 | 12.58701 | 13.05959 | 13.92218 | 15.00449 | 16.24326 | 17.52025 | 18.37141 | 18.96385 |
| 41.5 | 12.41751 | 12.71154 | 13.18923 | 14.0625 | 15.16078 | 16.42153 | 17.72545 | 18.59705 | 19.20492 |
| 42.5 | 12.54001 | 12.8371 | 13.32017 | 14.20458 | 15.3194 | 16.60273 | 17.93424 | 18.82675 | 19.45041 |
| 43.5 | 12.66334 | 12.96366 | 13.45238 | 14.3484 | 15.4803 | 16.78682 | 18.14654 | 19.06041 | 19.70017 |
| 44.5 | 12.78746 | 13.09119 | 13.58581 | 14.49391 | 15.64343 | 16.97373 | 18.36226 | 19.29789 | 19.95407 |
| 45.5 | 12.91234 | 13.21963 | 13.72043 | 14.64105 | 15.80873 | 17.16336 | 18.58128 | 19.53907 | 20.21195 |
| 46.5 | 13.03792 | 13.34895 | 13.85618 | 14.78977 | 15.9761 | 17.35564 | 18.80348 | 19.78381 | 20.47366 |
| 47.5 | 13.16419 | 13.47911 | 13.99301 | 14.93998 | 16.14548 | 17.55044 | 19.02875 | 20.03197 | 20.73903 |
| 48.5 | 13.29111 | 13.61006 | 14.13086 | 15.09163 | 16.31677 | 17.74767 | 19.25695 | 20.28339 | 21.00793 |
| 49.5 | 13.41864 | 13.74176 | 14.26968 | 15.24463 | 16.48986 | 17.9472 | 19.48794 | 20.53795 | 21.28018 |
| 50.5 | 13.54675 | 13.87418 | 14.40943 | 15.39892 | 16.66468 | 18.14892 | 19.7216 | 20.79548 | 21.55565 |
| 51.5 | 13.67543 | 14.00727 | 14.55004 | 15.55441 | 16.8411 | 18.3527 | 19.95779 | 21.05586 | 21.83419 |
| 52.5 | 13.80466 | 14.14102 | 14.69148 | 15.71103 | 17.01904 | 18.55842 | 20.19637 | 21.31896 | 22.11568 |
| 53.5 | 13.93441 | 14.2754 | 14.8337 | 15.86872 | 17.19839 | 18.76598 | 20.43722 | 21.58464 | 22.39999 |
| 54.5 | 14.06467 | 14.41037 | 14.97666 | 16.0274 | 17.37906 | 18.97524 | 20.68022 | 21.8528 | 22.68702 |
| 55.5 | 14.19544 | 14.54593 | 15.12032 | 16.18701 | 17.56096 | 19.1861 | 20.92526 | 22.12331 | 22.97667 |
| 56.5 | 14.32672 | 14.68205 | 15.26465 | 16.34748 | 17.744 | 19.39846 | 21.17222 | 22.3961 | 23.26885 |
| 57.5 | 14.4585 | 14.81872 | 15.40962 | 16.50877 | 17.92809 | 19.6122 | 21.421 | 22.67106 | 23.56349 |
| 58.5 | 14.59079 | 14.95595 | 15.55521 | 16.67081 | 18.11316 | 19.82724 | 21.67152 | 22.94813 | 23.86054 |

| Age (in | Weight (in | 5th<br>Percentile<br>Weight (in<br>kilograms) | 10th<br>Percentile<br>Weight (in<br>kilograms) | 25th<br>Percentile<br>Weight (in<br>kilograms) | 50th<br>Percentile<br>Weight (in<br>kilograms) | 75th<br>Percentile<br>Weight (in<br>kilograms) | 90th<br>Percentile<br>Weight (in<br>kilograms) | 95th<br>Percentile<br>Weight (in<br>kilograms) | 97th<br>Percentile<br>Weight (in<br>kilograms) |
|---|---|---|---|---|---|---|---|---|---|
| 59.5 | 14.72359 | 15.09371 | 15.70139 | 16.83356 | 18.29912 | 20.04348 | 21.92369 | 23.22723 | 24.15995 |
| 60.5 | 14.85692 | 15.23202 | 15.84814 | 16.99698 | 18.48592 | 20.26086 | 22.17744 | 23.50833 | 24.46169 |
| 61.5 | 14.99078 | 15.37087 | 15.99546 | 17.16103 | 18.6735 | 20.47929 | 22.4327 | 23.79136 | 24.76575 |
| 62.5 | 15.1252 | 15.51027 | 16.14334 | 17.32567 | 18.8618 | 20.69871 | 22.68943 | 24.07632 | 25.07212 |
| 63.5 | 15.26018 | 15.65023 | 16.29176 | 17.49088 | 19.05077 | 20.91907 | 22.94758 | 24.36317 | 25.38081 |
| 64.5 | 15.39575 | 15.79076 | 16.44074 | 17.65664 | 19.24037 | 21.14031 | 23.20712 | 24.65192 | 25.69185 |
| 65.5 | 15.53193 | 15.93186 | 16.59026 | 17.82293 | 19.43058 | 21.36242 | 23.46802 | 24.94257 | 26.00527 |
| 66.5 | 15.66872 | 16.07356 | 16.74033 | 17.98974 | 19.62136 | 21.58534 | 23.73029 | 25.23514 | 26.32111 |
| 67.5 | 15.80617 | 16.21586 | 16.89096 | 18.15706 | 19.8127 | 21.80908 | 23.99391 | 25.52965 | 26.63944 |
| 68.5 | 15.94427 | 16.35879 | 17.04215 | 18.32489 | 20.00459 | 22.0336 | 24.2589 | 25.82615 | 26.96033 |
| 69.5 | 16.08306 | 16.50235 | 17.19393 | 18.49324 | 20.19703 | 22.25893 | 24.52527 | 26.12468 | 27.28386 |
| 70.5 | 16.22255 | 16.64657 | 17.34629 | 18.66211 | 20.39002 | 22.48505 | 24.79305 | 26.4253 | 27.6101 |
| 71.5 | 16.36276 | 16.79146 | 17.49926 | 18.83151 | 20.58357 | 22.712 | 25.06229 | 26.72807 | 27.93916 |
| 72.5 | 16.5037 | 16.93704 | 17.65285 | 19.00147 | 20.7777 | 22.93978 | 25.33302 | 27.03308 | 28.27115 |
| 73.5 | 16.64539 | 17.08332 | 17.80708 | 19.17199 | 20.97243 | 23.16845 | 25.6053 | 27.34039 | 28.60616 |
| 74.5 | 16.78785 | 17.23031 | 17.96197 | 19.34311 | 21.16779 | 23.39803 | 25.87919 | 27.6501 | 28.94432 |
| 75.5 | 16.93107 | 17.37804 | 18.11754 | 19.51485 | 21.36383 | 23.62858 | 26.15477 | 27.9623 | 29.28574 |
| 76.5 | 17.07507 | 17.52651 | 18.2738 | 19.68724 | 21.56058 | 23.86016 | 26.4321 | 28.27709 | 29.63055 |
| 77.5 | 17.21986 | 17.67574 | 18.43077 | 19.86032 | 21.75811 | 24.09284 | 26.71128 | 28.59457 | 29.97888 |
| 78.5 | 17.36543 | 17.82572 | 18.58848 | 20.03413 | 21.95645 | 24.32667 | 26.99239 | 28.91486 | 30.33083 |
| 79.5 | 17.5118 | 17.97649 | 18.74695 | 20.20871 | 22.15567 | 24.56175 | 27.27553 | 29.23806 | 30.68656 |
| 80.5 | 17.65895 | 18.12803 | 18.9062 | 20.38409 | 22.35584 | 24.79815 | 27.56081 | 29.56428 | 31.04617 |
| 81.5 | 17.80689 | 18.28036 | 19.06624 | 20.56032 | 22.55702 | 25.03598 | 27.84832 | 29.89365 | 31.4098 |
| 82.5 | 17.9556 | 18.43348 | 19.2271 | 20.73745 | 22.7593 | 25.27531 | 28.13817 | 30.22628 | 31.77756 |
| 83.5 | 18.10509 | 18.5874 | 19.3888 | 20.91553 | 22.96273 | 25.51626 | 28.43049 | 30.56228 | 32.14959 |
| 84.5 | 18.25535 | 18.74211 | 19.55136 | 21.0946 | 23.16742 | 25.75894 | 28.72538 | 30.90178 | 32.52599 |
| 85.5 | 18.40637 | 18.89763 | 19.71479 | 21.27471 | 23.37343 | 26.00344 | 29.02298 | 31.24489 | 32.90689 |
| 86.5 | 18.55813 | 19.05395 | 19.87913 | 21.45592 | 23.58086 | 26.24988 | 29.3234 | 31.59174 | 33.29238 |
| 87.5 | 18.71062 | 19.21107 | 20.04438 | 21.63828 | 23.78979 | 26.49839 | 29.62676 | 31.94243 | 33.68257 |
| 88.5 | 18.86385 | 19.369 | 20.21057 | 21.82185 | 24.00031 | 26.74907 | 29.9332 | 32.29708 | 34.07755 |
| 89.5 | 19.01778 | 19.52773 | 20.37771 | 22.00666 | 24.21251 | 27.00204 | 30.24283 | 32.65581 | 34.47742 |
| 90.5 | 19.17243 | 19.68727 | 20.54584 | 22.19278 | 24.42648 | 27.25743 | 30.55579 | 33.01871 | 34.88226 |
| 91.5 | 19.32776 | 19.84762 | 20.71496 | 22.38027 | 24.64231 | 27.51535 | 30.8722 | 33.38591 | 35.29215 |
| 92.5 | 19.48379 | 20.00878 | 20.88511 | 22.56917 | 24.8601 | 27.77593 | 31.19218 | 33.75749 | 35.70715 |
| 93.5 | 19.6405 | 20.17076 | 21.05629 | 22.75955 | 25.07992 | 28.03928 | 31.51586 | 34.13355 | 36.12732 |
| 94.5 | 19.79788 | 20.33357 | 21.22855 | 22.95145 | 25.30189 | 28.30554 | 31.84335 | 34.5142 | 36.55271 |
| 95.5 | 19.95594 | 20.4972 | 21.4019 | 23.14493 | 25.52607 | 28.5748 | 32.17478 | 34.8995 | 36.98338 |

| Age (in<br>months) | Percentile<br>Weight (in | 5th<br>Percentile<br>Weight (in<br>kilograms) | 10th<br>Percentile<br>Weight (in<br>kilograms) | 25th<br>Percentile<br>Weight (in<br>kilograms) | 50th<br>Percentile<br>Weight (in<br>kilograms) | 75th<br>Percentile<br>Weight (in<br>kilograms) | 90th<br>Percentile<br>Weight (in<br>kilograms) | | 97th<br>Percentile<br>Weight (in<br>kilograms) |
|---|---|---|---|---|---|---|---|---|---|
| 96.5 | 20.11467 | 20.66168 | 21.57637 | 23.34005 | 25.75257 | 28.84718 | 32.51025 | 35.28955 | 37.41935 |
| 97.5 | 20.27408 | 20.82702 | 21.75198 | 23.53686 | 25.98146 | 29.12281 | 32.84988 | 35.68443 | 37.86065 |
| 98.5 | 20.43418 | 20.99322 | 21.92878 | 23.73542 | 26.21284 | 29.40179 | 33.19377 | 36.08419 | 38.30731 |
| 99.5 | 20.59497 | 21.16032 | 22.10678 | 23.93579 | 26.44679 | 29.68422 | 33.54202 | 36.4889 | 38.75932 |
| 100.5 | 20.75647 | 21.32832 | 22.28602 | 24.13801 | 26.68339 | 29.97021 | 33.89472 | 36.89862 | 39.2167 |
| 101.5 | 20.91869 | 21.49726 | 22.46654 | 24.34216 | 26.92273 | 30.25986 | 34.25197 | 37.3134 | 39.67943 |
| 102.5 | 21.08166 | 21.66716 | 22.64838 | 24.54828 | 27.16489 | 30.55326 | 34.61384 | 37.73327 | 40.14749 |
| 103.5 | 21.2454 | 21.83805 | 22.83157 | 24.75645 | 27.40995 | 30.85051 | 34.98041 | 38.15826 | 40.62087 |
| 104.5 | 21.40994 | 22.00997 | 23.01617 | 24.9667 | 27.65797 | 31.15169 | 35.35176 | 38.58841 | 41.09952 |
| 105.5 | 21.57532 | 22.18296 | 23.20222 | 25.17912 | 27.90904 | 31.45689 | 35.72793 | 39.02372 | 41.5834 |
| 106.5 | 21.74156 | 22.35705 | 23.38976 | 25.39375 | 28.16324 | 31.76618 | 36.10899 | 39.46421 | 42.07247 |
| 107.5 | 21.90873 | 22.5323 | 23.57885 | 25.61067 | 28.42064 | 32.07964 | 36.49499 | 39.90987 | 42.56665 |
| 108.5 | 22.07685 | 22.70876 | 23.76955 | 25.82993 | 28.6813 | 32.39734 | 36.88596 | 40.36069 | 43.06589 |
| 109.5 | 22.24599 | 22.88648 | 23.96192 | 26.05161 | 28.9453 | 32.71933 | 37.28193 | 40.81665 | 43.5701 |
| 110.5 | 22.4162 | 23.06551 | 24.15601 | 26.27576 | 29.21271 | 33.04569 | 37.68294 | 41.27773 | 44.0792 |
| 111.5 | 22.58754 | 23.24593 | 24.35189 | 26.50246 | 29.48359 | 33.37646 | 38.08898 | 41.74388 | 44.5931 |
| 112.5 | 22.76008 | 23.42779 | 24.54962 | 26.73177 | 29.758 | 33.7117 | 38.50008 | 42.21507 | 45.11169 |
| 113.5 | 22.93388 | 23.61117 | 24.74929 | 26.96376 | 30.03602 | 34.05144 | 38.91622 | 42.69124 | 45.63487 |
| 114.5 | 23.10902 | 23.79613 | 24.95096 | 27.19851 | 30.3177 | 34.39573 | 39.33741 | 43.17232 | 46.16253 |
| 115.5 | 23.28558 | 23.98277 | 25.1547 | 27.43609 | 30.60311 | 34.7446 | 39.76363 | 43.65825 | 46.69454 |
| 116.5 | 23.46364 | 24.17115 | 25.3606 | 27.67657 | 30.8923 | 35.09808 | 40.19484 | 44.14895 | 47.23077 |
| 117.5 | 23.64329 | 24.36137 | 25.56874 | 27.92001 | 31.18533 | 35.4562 | 40.63103 | 44.64432 | 47.77109 |
| 118.5 | 23.8246 | 24.55351 | 25.77921 | 28.16651 | 31.48225 | 35.81896 | 41.07214 | 45.14428 | 48.31536 |
| 119.5 | 24.00769 | 24.74766 | 25.99208 | 28.41613 | 31.78312 | 36.1864 | 41.51813 | 45.64872 | 48.86343 |
| 120.5 | 24.19264 | 24.94392 | 26.20745 | 28.66894 | 32.08799 | 36.55851 | 41.96894 | 46.15753 | 49.41515 |
| 121.5 | 24.37956 | 25.14238 | 26.42541 | 28.92502 | 32.3969 | 36.93529 | 42.42452 | 46.6706 | 49.97037 |
| 122.5 | 24.56855 | 25.34314 | 26.64604 | 29.18446 | 32.70991 | 37.31675 | 42.88478 | 47.1878 | 50.52892 |
| 123.5 | 24.75971 | 25.54631 | 26.86945 | 29.44731 | 33.02704 | 37.70287 | 43.34967 | 47.70901 | 51.09064 |
| 124.5 | 24.95315 | 25.75198 | 27.09573 | 29.71365 | 33.34835 | 38.09365 | 43.81908 | 48.23408 | 51.65537 |
| 125.5 | 25.14898 | 25.96027 | 27.32496 | 29.98357 | 33.67387 | 38.48906 | 44.29292 | 48.76288 | 52.22293 |
| 126.5 | 25.34731 | 26.17126 | 27.55726 | 30.25713 | 34.00363 | 38.88907 | 44.77111 | 49.29526 | 52.79314 |
| 127.5 | 25.54826 | 26.38509 | 27.7927 | 30.53439 | 34.33766 | 39.29366 | 45.25354 | 49.83107 | 53.36584 |
| 128.5 | 25.75195 | 26.60184 | 28.0314 | 30.81543 | 34.67599 | 39.7028 | 45.7401 | 50.37016 | 53.94084 |
| 129.5 | 25.95847 | 26.82163 | 28.27343 | 31.10032 | 35.01864 | 40.11642 | 46.23066 | 50.91236 | 54.51797 |
| 130.5 | 26.16796 | 27.04457 | 28.51891 | 31.38912 | 35.36562 | 40.5345 | 46.72512 | 51.45752 | 55.09704 |
| 131.5 | 26.38051 | 27.27076 | 28.76791 | 31.68189 | 35.71695 | 40.95697 | 47.22334 | 52.00546 | 55.67787 |
| 132.5 | 26.59626 | 27.50031 | 29.02052 | 31.97868 | 36.07263 | 41.38377 | 47.72519 | 52.55602 | 56.26029 |

| Age (in | | 5th<br>Percentile<br>Weight (in<br>kilograms) | 10th<br>Percentile<br>Weight (in<br>kilograms) | 25th<br>Percentile<br>Weight (in<br>kilograms) | 50th<br>Percentile<br>Weight (in<br>kilograms) | 75th<br>Percentile<br>Weight (in<br>kilograms) | 90th<br>Percentile<br>Weight (in<br>kilograms) | 95th<br>Percentile<br>Weight (in<br>kilograms) | 97th<br>Percentile<br>Weight (in<br>kilograms) |
|---|---|---|---|---|---|---|---|---|---|
| 133.5 | 26.81531 | 27.73332 | 29.27685 | 32.27955 | 36.43266 | 41.81484 | 48.23054 | 53.10903 | 56.84411 |
| 134.5 | 27.03777 | 27.96989 | 29.53696 | 32.58454 | 36.79704 | 42.2501 | 48.73924 | 53.66432 | 57.42915 |
| 135.5 | 27.26376 | 28.21013 | 29.80095 | 32.89371 | 37.16577 | 42.68947 | 49.25114 | 54.22171 | 58.01524 |
| 136.5 | 27.49337 | 28.45412 | 30.06888 | 33.20709 | 37.53881 | 43.13287 | 49.76611 | 54.78102 | 58.60219 |
| 137.5 | 27.72672 | 28.70197 | 30.34084 | 33.52472 | 37.91616 | 43.5802 | 50.28397 | 55.34208 | 59.18983 |
| 138.5 | 27.9639 | 28.95376 | 30.61689 | 33.84662 | 38.29777 | 44.03137 | 50.80458 | 55.9047 | 59.77799 |
| 139.5 | 28.20501 | 29.20958 | 30.8971 | 34.17281 | 38.68361 | 44.48627 | 51.32778 | 56.46873 | 60.3665 |
| 140.5 | 28.45015 | 29.4695 | 31.18151 | 34.5033 | 39.07364 | 44.94478 | 51.85339 | 57.03397 | 60.95519 |
| 141.5 | 28.69939 | 29.7336 | 31.4702 | 34.83811 | 39.46781 | 45.40679 | 52.38125 | 57.60024 | 61.5439 |
| 142.5 | 28.95283 | 30.00195 | 31.76319 | 35.17724 | 39.86604 | 45.87218 | 52.91119 | 58.16739 | 62.13246 |
| 143.5 | 29.21053 | 30.2746 | 32.06052 | 35.52066 | 40.26828 | 46.3408 | 53.44304 | 58.73522 | 62.72072 |
| 144.5 | 29.47257 | 30.55162 | 32.36224 | 35.86837 | 40.67444 | 46.81253 | 53.97661 | 59.30357 | 63.30853 |
| 145.5 | 29.739 | 30.83304 | 32.66834 | 36.22034 | 41.08443 | 47.28721 | 54.51174 | 59.87226 | 63.89573 |
| 146.5 | 30.00988 | 31.11891 | 32.97885 | 36.57653 | 41.49817 | 47.7647 | 55.04825 | 60.44112 | 64.48219 |
| 147.5 | 30.28525 | 31.40925 | 33.29378 | 36.9369 | 41.91555 | 48.24483 | 55.58594 | 61.00999 | 65.06776 |
| 148.5 | 30.56516 | 31.70409 | 33.6131 | 37.30138 | 42.33644 | 48.72744 | 56.12464 | 61.57871 | 65.65231 |
| 149.5 | 30.84962 | 32.00343 | 33.93681 | 37.66991 | 42.76073 | 49.21236 | 56.66416 | 62.1471 | 66.2357 |
| 150.5 | 31.13865 | 32.30727 | 34.26488 | 38.04241 | 43.18828 | 49.6994 | 57.20431 | 62.715 | 66.81782 |
| 151.5 | 31.43227 | 32.61561 | 34.59726 | 38.4188 | 43.61896 | 50.18839 | 57.74492 | 63.28226 | 67.39854 |
| 152.5 | 31.73046 | 32.92842 | 34.93391 | 38.79897 | 44.05259 | 50.67913 | 58.28578 | 63.84873 | 67.97776 |
| 153.5 | 32.03321 | 33.24567 | 35.27477 | 39.18281 | 44.48903 | 51.17143 | 58.82671 | 64.41424 | 68.55535 |
| 154.5 | 32.3405 | 33.56731 | 35.61976 | 39.5702 | 44.92809 | 51.66508 | 59.36752 | 64.97865 | 69.13122 |
| 155.5 | 32.65229 | 33.89329 | 35.96879 | 39.96099 | 45.3696 | 52.15987 | 59.90801 | 65.54182 | 69.70526 |
| 156.5 | 32.96852 | 34.22353 | 36.32176 | 40.35506 | 45.81336 | 52.65558 | 60.448 | 66.10359 | 70.27738 |
| 157.5 | 33.28913 | 34.55796 | 36.67857 | 40.75222 | 46.25917 | 53.152 | 60.98729 | 66.66382 | 70.84748 |
| 158.5 | 33.61404 | 34.89647 | 37.03908 | 41.15232 | 46.70681 | 53.64889 | 61.52569 | 67.22238 | 71.41549 |
| 159.5 | 33.94317 | 35.23896 | 37.40317 | 41.55516 | 47.15606 | 54.14603 | 62.063 | 67.77913 | 71.98133 |
| 160.5 | 34.27642 | 35.58531 | 37.77067 | 41.96056 | 47.60669 | 54.64318 | 62.59903 | 68.33393 | 72.5449 |
| 161.5 | 34.61365 | 35.93538 | 38.14143 | 42.3683 | 48.05847 | 55.1401 | 63.13359 | 68.88665 | 73.10614 |
| 162.5 | 34.95475 | 36.28902 | 38.51526 | 42.77818 | 48.51113 | 55.63653 | 63.66648 | 69.43717 | 73.66498 |
| 163.5 | 35.29956 | 36.64606 | 38.89198 | 43.18995 | 48.96443 | 56.13224 | 64.1975 | 69.98535 | 74.22134 |
| 164.5 | 35.64794 | 37.00634 | 39.27138 | 43.60337 | 49.4181 | 56.62696 | 64.72647 | 70.53106 | 74.77517 |
| 165.5 | 35.99969 | 37.36965 | 39.65325 | 44.01821 | 49.87187 | 57.12044 | 65.25318 | 71.07419 | 75.32641 |
| 166.5 | 36.35464 | 37.7358 | 40.03736 | 44.43419 | 50.32546 | 57.61241 | 65.77745 | 71.61461 | 75.87498 |
| 167.5 | 36.71259 | 38.10456 | 40.42347 | 44.85104 | 50.77859 | 58.10262 | 66.29907 | 72.15219 | 76.42083 |
| 168.5 | 37.07331 | 38.47571 | 40.81133 | 45.26849 | 51.23096 | 58.5908 | 66.81785 | 72.68681 | 76.9639 |
| 169.5 | 37.43658 | 38.849 | 41.20067 | 45.68625 | 51.68229 | 59.07667 | 67.33359 | 73.21836 | 77.50413 |

| Age (in | 3rd<br>Percentile<br>Weight (in<br>kilograms) | 5th<br>Percentile<br>Weight (in<br>kilograms) | 10th<br>Percentile<br>Weight (in<br>kilograms) | 25th<br>Percentile<br>Weight (in<br>kilograms) | 50th<br>Percentile<br>Weight (in<br>kilograms) | 75th<br>Percentile<br>Weight (in<br>kilograms) | 90th<br>Percentile<br>Weight (in<br>kilograms) | 95th<br>Percentile<br>Weight (in<br>kilograms) | 97th<br>Percentile<br>Weight (in<br>kilograms) |
|---|---|---|---|---|---|---|---|---|---|
| 170.5 | 37.80215 | 39.22417 | 41.59121 | 46.10402 | 52.13226 | 59.55998 | 67.84611 | 73.7467 | 78.04146 |
| 171.5 | 38.16976 | 39.60097 | 41.98269 | 46.52151 | 52.58059 | 60.04046 | 68.3552 | 74.27172 | 78.57582 |
| 172.5 | 38.53916 | 39.97909 | 42.37479 | 46.9384 | 53.02696 | 60.51782 | 68.86067 | 74.7933 | 79.10716 |
| 173.5 | 38.91004 | 40.35826 | 42.76722 | 47.35437 | 53.47107 | 60.99182 | 69.36233 | 75.3113 | 79.63542 |
| 174.5 | 39.28212 | 40.73817 | 43.15967 | 47.76912 | 53.91261 | 61.46217 | 69.85999 | 75.82561 | 80.1605 |
| 175.5 | 39.65509 | 41.11851 | 43.55182 | 48.18232 | 54.35128 | 61.92862 | 70.35345 | 76.3361 | 80.68236 |
| 176.5 | 40.02863 | 41.49895 | 43.94334 | 48.59365 | 54.78677 | 62.3909 | 70.84252 | 76.84263 | 81.2009 |
| 177.5 | 40.40241 | 41.87917 | 44.3339 | 49.00279 | 55.21878 | 62.84876 | 71.32701 | 77.34509 | 81.71605 |
| 178.5 | 40.77608 | 42.25882 | 44.72317 | 49.40941 | 55.64701 | 63.30195 | 71.80674 | 77.84332 | 82.2277 |
| 179.5 | 41.14932 | 42.63757 | 45.1108 | 49.81318 | 56.07116 | 63.75019 | 72.2815 | 78.3372 | 82.73579 |
| 180.5 | 41.52175 | 43.01506 | 45.49646 | 50.21378 | 56.49096 | 64.19328 | 72.75113 | 78.82659 | 83.24017 |
| 181.5 | 41.89302 | 43.39093 | 45.8798 | 50.61091 | 56.90611 | 64.63096 | 73.21544 | 79.31134 | 83.74075 |
| 182.5 | 42.26275 | 43.76482 | 46.26048 | 51.00423 | 57.31634 | 65.063 | 73.67424 | 79.7913 | 84.23741 |
| 183.5 | 42.63058 | 44.13638 | 46.63815 | 51.39346 | 57.72139 | 65.48919 | 74.12736 | 80.26632 | 84.73 |
| 184.5 | 42.99612 | 44.50523 | 47.01247 | 51.77827 | 58.121 | 65.90932 | 74.57462 | 80.73625 | 85.21839 |
| 185.5 | 43.35899 | 44.87102 | 47.3831 | 52.15839 | 58.51492 | 66.32318 | 75.01586 | 81.20093 | 85.70242 |
| 186.5 | 43.71882 | 45.23338 | 47.74972 | 52.53352 | 58.90293 | 66.73059 | 75.4509 | 81.66019 | 86.18192 |
| 187.5 | 44.07523 | 45.59196 | 48.11199 | 52.90339 | 59.2848 | 67.13136 | 75.87959 | 82.11386 | 86.65673 |
| 188.5 | 44.42784 | 45.9464 | 48.46959 | 53.26773 | 59.66033 | 67.52534 | 76.30176 | 82.56177 | 87.12663 |
| 189.5 | 44.77629 | 46.29635 | 48.82222 | 53.6263 | 60.02932 | 67.91236 | 76.71726 | 83.00375 | 87.59143 |
| 190.5 | 45.1202 | 46.64147 | 49.16956 | 53.97886 | 60.39159 | 68.29229 | 77.12595 | 83.43962 | 88.05093 |
| 191.5 | 45.45922 | 46.98144 | 49.51134 | 54.32518 | 60.74699 | 68.665 | 77.52768 | 83.8692 | 88.50487 |
| 192.5 | 45.79301 | 47.31593 | 49.84727 | 54.66505 | 61.09537 | 69.03038 | 77.92233 | 84.29229 | 88.95303 |
| 193.5 | 46.12122 | 47.64464 | 50.17709 | 54.99828 | 61.4366 | 69.38833 | 78.30977 | 84.70871 | 89.39516 |
| 194.5 | 46.44354 | 47.96727 | 50.50055 | 55.3247 | 61.77057 | 69.73878 | 78.68987 | 85.11828 | 89.83098 |
| 195.5 | 46.75967 | 48.28356 | 50.81743 | 55.64414 | 62.09719 | 70.08164 | 79.06252 | 85.5208 | 90.26024 |
| 196.5 | 47.06932 | 48.59325 | 51.12752 | 55.95647 | 62.41639 | 70.41688 | 79.42763 | 85.91607 | 90.68264 |
| 197.5 | 47.37223 | 48.89609 | 51.43062 | 56.26158 | 62.72809 | 70.74445 | 79.78509 | 86.30392 | 91.0979 |
| 198.5 | 47.66815 | 49.19189 | 51.72656 | 56.55935 | 63.03228 | 71.06433 | 80.13483 | 86.68415 | 91.50571 |
| 199.5 | 47.95687 | 49.48044 | 52.0152 | 56.84971 | 63.32892 | 71.37652 | 80.47676 | 87.05657 | 91.90578 |
| 200.5 | 48.23819 | 49.76158 | 52.29642 | 57.13261 | 63.61802 | 71.68103 | 80.81082 | 87.42099 | 92.29779 |
| 201.5 | 48.51195 | 50.03518 | 52.57011 | 57.408 | 63.89959 | 71.97788 | 81.13696 | 87.77725 | 92.68144 |
| 202.5 | 48.778 | 50.30112 | 52.8362 | 57.67589 | 64.17367 | 72.26711 | 81.45512 | 88.12516 | 93.05643 |
| 203.5 | 49.03625 | 50.55931 | 53.09465 | 57.93627 | 64.44032 | 72.54879 | 81.76528 | 88.46456 | 93.42244 |
| 204.5 | 49.28662 | 50.80971 | 53.34544 | 58.18918 | 64.69961 | 72.82297 | 82.06741 | 88.79528 | 93.77917 |
| 205.5 | 49.52905 | 51.05229 | 53.58858 | 58.43468 | 64.95165 | 73.08975 | 82.3615 | 89.11718 | 94.12633 |
| 206.5 | 49.76354 | 51.28706 | 53.82409 | 58.67285 | 65.19653 | 73.34922 | 82.64755 | 89.43011 | 94.46364 |

| Age (in months) | • | 5th<br>Percentile<br>Weight (in<br>kilograms) | 10th<br>Percentile<br>Weight (in<br>kilograms) | 25th<br>Percentile<br>Weight (in<br>kilograms) | 50th<br>Percentile<br>Weight (in<br>kilograms) | 75th<br>Percentile<br>Weight (in<br>kilograms) | , | 95th<br>Percentile<br>Weight (in<br>kilograms) | 97th<br>Percentile<br>Weight (in<br>kilograms) |
|---|---|---|---|---|---|---|---|---|---|
| 207.5 | 49.9901 | 51.51404 | 54.05205 | 58.9038 | 65.4344 | 73.60152 | 82.92558 | 89.73396 | 94.79081 |
| 208.5 | 50.2088 | 51.73333 | 54.27255 | 59.12764 | 65.6654 | 73.84675 | 83.1956 | 90.02861 | 95.10761 |
| 209.5 | 50.4197 | 51.94499 | 54.4857 | 59.34454 | 65.8897 | 74.08507 | 83.45768 | 90.31396 | 95.41379 |
| 210.5 | 50.62293 | 52.14918 | 54.69165 | 59.55466 | 66.10749 | 74.31664 | 83.71185 | 90.58994 | 95.70913 |
| 211.5 | 50.81862 | 52.34603 | 54.89058 | 59.75819 | 66.31897 | 74.54164 | 83.9582 | 90.85649 | 95.99346 |
| 212.5 | 51.00695 | 52.53572 | 55.08267 | 59.95536 | 66.52437 | 74.76024 | 84.19682 | 91.11358 | 96.26661 |
| 213.5 | 51.18811 | 52.71847 | 55.26814 | 60.14639 | 66.7239 | 74.97267 | 84.42781 | 91.3612 | 96.52847 |
| 214.5 | 51.36232 | 52.8945 | 55.44723 | 60.33153 | 66.91784 | 75.17912 | 84.6513 | 91.59938 | 96.77894 |
| 215.5 | 51.52982 | 53.06406 | 55.6202 | 60.51105 | 67.10642 | 75.37983 | 84.86744 | 91.82817 | 97.01799 |
| 216.5 | 51.69086 | 53.2274 | 55.78731 | 60.68521 | 67.28993 | 75.57503 | 85.0764 | 92.04765 | 97.24564 |
| 217.5 | 51.84574 | 53.38481 | 55.94884 | 60.85431 | 67.46863 | 75.76499 | 85.27837 | 92.25795 | 97.46194 |
| 218.5 | 51.99472 | 53.53657 | 56.10508 | 61.01862 | 67.64281 | 75.94994 | 85.47356 | 92.45925 | 97.66704 |
| 219.5 | 52.13808 | 53.68296 | 56.25633 | 61.17846 | 67.81277 | 76.13018 | 85.66221 | 92.65175 | 97.86111 |
| 220.5 | 52.27612 | 53.82428 | 56.40286 | 61.33409 | 67.97877 | 76.30597 | 85.8446 | 92.83572 | 98.04443 |
| 221.5 | 52.40911 | 53.96079 | 56.54495 | 61.4858 | 68.14111 | 76.47759 | 86.02101 | 93.01148 | 98.21733 |
| 222.5 | 52.53731 | 54.09278 | 56.68288 | 61.63386 | 68.30005 | 76.64533 | 86.19177 | 93.17941 | 98.38026 |
| 223.5 | 52.66098 | 54.22046 | 56.81689 | 61.77851 | 68.45585 | 76.80948 | 86.35725 | 93.33994 | 98.53375 |
| 224.5 | 52.78032 | 54.34408 | 56.94719 | 61.91997 | 68.60872 | 76.97031 | 86.51781 | 93.49361 | 98.67844 |
| 225.5 | 52.89553 | 54.46381 | 57.07396 | 62.05842 | 68.75889 | 77.12809 | 86.6739 | 93.64099 | 98.81509 |
| 226.5 | 53.00674 | 54.57977 | 57.19732 | 62.19399 | 68.90653 | 77.2831 | 86.82597 | 93.78276 | 98.94455 |
| 227.5 | 53.11402 | 54.69205 | 57.31737 | 62.32678 | 69.05176 | 77.4356 | 86.97452 | 93.91968 | 99.06786 |
| 228.5 | 53.21739 | 54.80066 | 57.43409 | 62.4568 | 69.19467 | 77.5858 | 87.12008 | 94.05261 | 99.18615 |
| 229.5 | 53.31679 | 54.90552 | 57.54742 | 62.58399 | 69.33527 | 77.73392 | 87.26324 | 94.18252 | 99.30075 |
| 230.5 | 53.41207 | 55.00648 | 57.6572 | 62.70822 | 69.47351 | 77.88014 | 87.40462 | 94.31046 | 99.41315 |
| 231.5 | 53.50297 | 55.10328 | 57.76315 | 62.82922 | 69.60926 | 78.02461 | 87.54488 | 94.43765 | 99.52501 |
| 232.5 | 53.58913 | 55.19552 | 57.86488 | 62.94664 | 69.74228 | 78.16742 | 87.68474 | 94.5654 | 99.63819 |
| 233.5 | 53.67003 | 55.2827 | 57.96187 | 63.06 | 69.87224 | 78.30863 | 87.82495 | 94.69517 | 99.75477 |
| 234.5 | 53.74501 | 55.36413 | 58.05343 | 63.16863 | 69.99869 | 78.44824 | 87.96634 | 94.82857 | 99.87706 |
| 235.5 | 53.81325 | 55.43897 | 58.13869 | 63.27175 | 70.12104 | 78.58618 | 88.10976 | 94.96735 | 100.0076 |
| 236.5 | 53.87373 | 55.50617 | 58.21662 | 63.36835 | 70.23857 | 78.72234 | 88.25614 | 95.11344 | 100.1492 |
| 237.5 | 53.92519 | 55.56447 | 58.28594 | 63.45727 | 70.3504 | 78.8565 | 88.40645 | 95.26894 | 100.3048 |
| 238.5 | 53.96614 | 55.61236 | 58.34515 | 63.53709 | 70.45546 | 78.98839 | 88.56175 | 95.43613 | 100.4779 |
| 239.5 | 53.99482 | 55.64807 | 58.39247 | 63.60618 | 70.55252 | 79.11762 | 88.72311 | 95.61749 | 100.6721 |
| 240 | 54.00392 | 55.66071 | 58.41105 | 63.63611 | 70.59761 | 79.18111 | 88.80644 | 95.71431 | 100.7784 |

# 10.9 Appendix 9 CDC Data Table of Weight-for-age Chart for Females

| | 2.1 | <b>5</b> (1 | 10/1 | 254 | 504 | | | 1 | 05/1 |
|---|---|---|---|---|---|---|---|---|---|
| Age (in | 3rd<br>Percentile | 5th<br>Percentile | 10th<br>Percentile | 25th<br>Percentile | 50th<br>Percentile | 75th<br>Percentile | 90th<br>Percentile | 95th<br>Percentile | 97th<br>Percentile |
| months) | Weight (in | Weight (in | Weight (in | Weight (in | Weight (in | Weight (in | Weight (in | Weight (in | Weight (in |
| | kilograms) | kilograms) | kilograms) | kilograms) | kilograms) | kilograms) | kilograms) | kilograms) | kilograms) |
| 24 | 9.985668 | 10.21027 | 10.57373 | 11.23357 | 12.05504 | 12.98667 | 13.93766 | 14.56636 | 15.00156 |
| 24.5 | 10.04881 | 10.27483 | 10.64076 | 11.30567 | 12.13456 | 13.07613 | 14.03902 | 14.67659 | 15.11839 |
| 25.5 | 10.17173 | 10.40066 | 10.77167 | 11.44697 | 12.29102 | 13.25293 | 14.24017 | 14.89587 | 15.35122 |
| 26.5 | 10.29079 | 10.52274 | 10.89899 | 11.58501 | 12.44469 | 13.42753 | 14.43984 | 15.11428 | 15.58363 |
| 27.5 | 10.40664 | 10.64171 | 11.02338 | 11.72047 | 12.59622 | 13.60059 | 14.63873 | 15.33249 | 15.81632 |
| 28.5 | 10.5199 | 10.75819 | 11.14545 | 11.85392 | 12.74621 | 13.77271 | 14.83743 | 15.55113 | 16.0499 |
| 29.5 | 10.63112 | 10.87273 | 11.26575 | 11.98592 | 12.89517 | 13.9444 | 15.03646 | 15.7707 | 16.28491 |
| 30.5 | 10.74078 | 10.98581 | 11.38474 | 12.11692 | 13.04357 | 14.11611 | 15.23626 | 15.99164 | 16.52176 |
| 31.5 | 10.84935 | 11.09789 | 11.50288 | 12.24735 | 13.19181 | 14.28823 | 15.43719 | 16.21432 | 16.76085 |
| 32.5 | 10.95722 | 11.20934 | 11.62054 | 12.37757 | 13.34023 | 14.46106 | 15.63957 | 16.43904 | 17.00245 |
| 33.5 | 11.06475 | 11.32054 | 11.73806 | 12.50791 | 13.48913 | 14.63491 | 15.84365 | 16.66605 | 17.24681 |
| 34.5 | 11.17225 | 11.43177 | 11.85574 | 12.63865 | 13.63877 | 14.80998 | 16.04963 | 16.89553 | 17.49412 |
| 35.5 | 11.28 | 11.54332 | 11.97384 | 12.77001 | 13.78937 | 14.98647 | 16.25767 | 17.12762 | 17.7445 |
| 36.5 | 11.38824 | 11.65542 | 12.09259 | 12.90222 | 13.94108 | 15.16452 | 16.46789 | 17.36244 | 17.99807 |
| 37.5 | 11.49718 | 11.76826 | 12.21216 | 13.03542 | 14.09407 | 15.34425 | 16.68038 | 17.60006 | 18.25487 |
| 38.5 | 11.607 | 11.88202 | 12.33273 | 13.16977 | 14.24844 | 15.52574 | 16.89519 | 17.8405 | 18.51494 |
| 39.5 | 11.71783 | 11.99685 | 12.45442 | 13.30538 | 14.40429 | 15.70905 | 17.11235 | 18.08377 | 18.77826 |
| 40.5 | 11.82981 | 12.11284 | 12.57735 | 13.44234 | 14.56168 | 15.89422 | 17.33186 | 18.32988 | 19.04483 |
| 41.5 | 11.94304 | 12.23011 | 12.70158 | 13.58071 | 14.72064 | 16.08126 | 17.55371 | 18.57877 | 19.31458 |
| 42.5 | 12.05757 | 12.34871 | 12.8272 | 13.72054 | 14.88121 | 16.27016 | 17.77788 | 18.83042 | 19.58748 |
| 43.5 | 12.17348 | 12.4687 | 12.95423 | 13.86186 | 15.04341 | 16.46093 | 18.00432 | 19.08475 | 19.86343 |
| 44.5 | 12.2908 | 12.59011 | 13.08271 | 14.00469 | 15.20721 | 16.65353 | 18.23298 | 19.34169 | 20.14237 |
| 45.5 | 12.40954 | 12.71297 | 13.21265 | 14.14902 | 15.37263 | 16.84793 | 18.46379 | 19.60118 | 20.4242 |
| 46.5 | 12.52972 | 12.83726 | 13.34405 | 14.29485 | 15.53962 | 17.04408 | 18.69671 | 19.86313 | 20.70884 |
| 47.5 | 12.65132 | 12.96298 | 13.47689 | 14.44217 | 15.70817 | 17.24195 | 18.93166 | 20.12746 | 20.99619 |
| 48.5 | 12.77432 | 13.09012 | 13.61116 | 14.59093 | 15.87824 | 17.44149 | 19.16858 | 20.39409 | 21.28616 |
| 49.5 | 12.89869 | 13.21864 | 13.74682 | 14.74112 | 16.04978 | 17.64265 | 19.40739 | 20.66293 | 21.57866 |
| 50.5 | 13.02441 | 13.3485 | 13.88384 | 14.89269 | 16.22277 | 17.84537 | 19.64805 | 20.93393 | 21.8736 |
| 51.5 | 13.15141 | 13.47966 | 14.02217 | 15.0456 | 16.39715 | 18.04961 | 19.89048 | 21.20699 | 22.1709 |
| 52.5 | 13.27965 | 13.61206 | 14.16176 | 15.19981 | 16.57289 | 18.25533 | 20.13464 | 21.48207 | 22.4705 |
| 53.5 | 13.40907 | 13.74566 | 14.30257 | 15.35527 | 16.74994 | 18.46249 | 20.38048 | 21.7591 | 22.77232 |
| 54.5 | 13.53962 | 13.8804 | 14.44453 | 15.51193 | 16.92827 | 18.67105 | 20.62795 | 22.03803 | 23.07631 |
| 55.5 | 13.67121 | 14.01621 | 14.5876 | 15.66975 | 17.10783 | 18.88097 | 20.87704 | 22.31884 | 23.38243 |
| 56.5 | 13.80381 | 14.15303 | 14.73172 | 15.82868 | 17.28859 | 19.09224 | 21.1277 | 22.60148 | 23.69063 |
| 57.5 | 13.93732 | 14.29081 | 14.87683 | 15.98868 | 17.47052 | 19.30483 | 21.37993 | 22.88594 | 24.0009 |
| 58.5 | 14.0717 | 14.42947 | 15.02287 | 16.14971 | 17.65361 | 19.51874 | 21.63373 | 23.17222 | 24.31322 |

| Age (in | 3rd<br>Percentile | 5th<br>Percentile | 10th<br>Percentile | 25th<br>Percentile | 50th<br>Percentile | 75th<br>Percentile | 90th<br>Percentile | 95th<br>Percentile | 97th<br>Percentile |
|---|---|---|---|---|---|---|---|---|---|
| months) | Weight (in kilograms) | Weight (in kilograms) | Weight (in kilograms) | Weight (in kilograms) | Weight (in kilograms) | Weight (in kilograms) | Weight (in kilograms) | Weight (in kilograms) | Weight (in kilograms) |
| 59.5 | 14.20687 | 14.56897 | 15.16981 | 16.31173 | 17.83782 | 19.73395 | 21.88909 | 23.46031 | 24.62758 |
| 60.5 | 14.34277 | 14.70924 | 15.31758 | 16.47471 | 18.02314 | 19.95048 | 22.14604 | 23.75024 | 24.94401 |
| 61.5 | 14.47934 | 14.85022 | 15.46614 | 16.63861 | 18.20956 | 20.16834 | 22.4046 | 24.04202 | 25.26252 |
| 62.5 | 14.61652 | 14.99186 | 15.61545 | 16.80342 | 18.39709 | 20.38753 | 22.6648 | 24.3357 | 25.58315 |
| 63.5 | 14.75426 | 15.13412 | 15.76547 | 16.9691 | 18.58571 | 20.6081 | 22.92668 | 24.63133 | 25.90595 |
| 64.5 | 14.8925 | 15.27694 | 15.91616 | 17.13565 | 18.77545 | 20.83007 | 23.19031 | 24.92897 | 26.23096 |
| 65.5 | 15.03119 | 15.42029 | 16.06749 | 17.30305 | 18.96631 | 21.05349 | 23.45574 | 25.22868 | 26.55827 |
| 66.5 | 15.1703 | 15.56413 | 16.21943 | 17.4713 | 19.15831 | 21.2784 | 23.72305 | 25.53055 | 26.88796 |
| 67.5 | 15.30978 | 15.70843 | 16.37197 | 17.6404 | 19.35149 | 21.50486 | 23.99232 | 25.83467 | 27.2201 |
| 68.5 | 15.44961 | 15.85316 | 16.52509 | 17.81035 | 19.54588 | 21.73294 | 24.26364 | 26.14113 | 27.55481 |
| 69.5 | 15.58975 | 15.99831 | 16.67878 | 17.98118 | 19.74151 | 21.96271 | 24.5371 | 26.45005 | 27.8922 |
| 70.5 | 15.73018 | 16.14385 | 16.83304 | 18.15288 | 19.93843 | 22.19425 | 24.81282 | 26.76154 | 28.23237 |
| 71.5 | 15.87089 | 16.28977 | 16.98787 | 18.32549 | 20.1367 | 22.42763 | 25.09089 | 27.07573 | 28.57547 |
| 72.5 | 16.01186 | 16.43608 | 17.14327 | 18.49904 | 20.33636 | 22.66294 | 25.37145 | 27.39274 | 28.92162 |
| 73.5 | 16.1531 | 16.58277 | 17.29926 | 18.67356 | 20.53748 | 22.90029 | 25.65461 | 27.71272 | 29.27096 |
| 74.5 | 16.2946 | 16.72986 | 17.45586 | 18.84908 | 20.74013 | 23.13976 | 25.94051 | 28.0358 | 29.62364 |
| 75.5 | 16.43638 | 16.87736 | 17.61309 | 19.02566 | 20.94438 | 23.38146 | 26.22926 | 28.36213 | 29.97981 |
| 76.5 | 16.57843 | 17.02528 | 17.77097 | 19.20334 | 21.1503 | 23.6255 | 26.52102 | 28.69185 | 30.33962 |
| 77.5 | 16.7208 | 17.17365 | 17.92956 | 19.38217 | 21.35797 | 23.87199 | 26.81591 | 29.02513 | 30.70323 |
| 78.5 | 16.86349 | 17.3225 | 18.08887 | 19.56221 | 21.56748 | 24.12103 | 27.11407 | 29.36212 | 31.0708 |
| 79.5 | 17.00654 | 17.47187 | 18.24897 | 19.74353 | 21.77891 | 24.37274 | 27.41566 | 29.70296 | 31.44249 |
| 80.5 | 17.14998 | 17.6218 | 18.40989 | 19.9262 | 21.99235 | 24.62725 | 27.7208 | 30.04782 | 31.81846 |
| 81.5 | 17.29386 | 17.77232 | 18.5717 | 20.11027 | 22.20789 | 24.88466 | 28.02965 | 30.39685 | 32.19887 |
| 82.5 | 17.43821 | 17.9235 | 18.73445 | 20.29582 | 22.42562 | 25.14509 | 28.34233 | 30.75021 | 32.58389 |
| 83.5 | 17.5831 | 18.07539 | 18.89819 | 20.48293 | 22.64564 | 25.40866 | 28.659 | 31.10804 | 32.97366 |
| 84.5 | 17.72858 | 18.22805 | 19.063 | 20.67168 | 22.86804 | 25.67549 | 28.97979 | 31.47049 | 33.36833 |
| 85.5 | 17.8747 | 18.38153 | 19.22895 | 20.86215 | 23.09293 | 25.94569 | 29.30484 | 31.83771 | 33.76807 |
| 86.5 | 18.02152 | 18.53591 | 19.3961 | 21.05441 | 23.32039 | 26.21937 | 29.63426 | 32.20984 | 34.17302 |
| 87.5 | 18.16912 | 18.69124 | 19.56453 | 21.24855 | 23.55052 | 26.49666 | 29.9682 | 32.58701 | 34.5833 |
| 88.5 | 18.31757 | 18.84762 | 19.73432 | 21.44467 | 23.78342 | 26.77764 | 30.30677 | 32.96935 | 34.99906 |
| 89.5 | 18.46693 | 19.00511 | 19.90554 | 21.64283 | 24.01918 | 27.06244 | 30.65008 | 33.35698 | 35.42042 |
| 90.5 | 18.61729 | 19.16378 | 20.07828 | 21.84313 | 24.25789 | 27.35114 | 30.99825 | 33.75001 | 35.8475 |
| 91.5 | 18.76871 | 19.32373 | 20.25261 | 22.04564 | 24.49965 | 27.64385 | 31.35137 | 34.14856 | 36.2804 |
| 92.5 | 18.92129 | 19.48502 | 20.42863 | 22.25047 | 24.74454 | 27.94066 | 31.70954 | 34.55271 | 36.71922 |
| 93.5 | 19.07511 | 19.64775 | 20.6064 | 22.45768 | 24.99264 | 28.24165 | 32.07286 | 34.96256 | 37.16406 |
| 94.5 | 19.23024 | 19.81199 | 20.78601 | 22.66736 | 25.24403 | 28.54689 | 32.44138 | 35.37818 | 37.61498 |
| 95.5 | 19.38678 | 19.97783 | 20.96755 | 22.8796 | 25.4988 | 28.85648 | 32.8152 | 35.79964 | 38.07207 |

| A C . | 3rd | 5th | 10th | 25th | 50th | 75th | 90th | 95th | 97th |
|---|---|---|---|---|---|---|---|---|---|
| Age (in months) | Percentile Weight (in | Percentile<br>Weight (in | Percentile Weight (in | Percentile Weight (in | Percentile<br>Weight (in | Percentile<br>Weight (in | Percentile Weight (in | Percentile<br>Weight (in | Percentile<br>Weight (in |
| , | kilograms) | kilograms) | kilograms) | kilograms) | kilograms) | kilograms) | kilograms) | kilograms) | kilograms) |
| 96.5 | 19.54481 | 20.14535 | 21.15111 | 23.09446 | 25.75702 | 29.17046 | 33.19435 | 36.22699 | 38.53537 |
| 97.5 | 19.70442 | 20.31464 | 21.33675 | 23.31203 | 26.01874 | 29.4889 | 33.5789 | 36.66029 | 39.00492 |
| 98.5 | 19.86568 | 20.48579 | 21.52456 | 23.53237 | 26.28404 | 29.81185 | 33.96887 | 37.09956 | 39.48077 |
| 99.5 | 20.0287 | 20.65887 | 21.71462 | 23.75556 | 26.55298 | 30.13934 | 34.36431 | 37.54482 | 39.96292 |
| 100.5 | 20.19355 | 20.83397 | 21.907 | 23.98166 | 26.82559 | 30.47142 | 34.76522 | 37.99609 | 40.45138 |
| 101.5 | 20.36032 | 21.01117 | 22.10179 | 24.21073 | 27.10193 | 30.80811 | 35.17161 | 38.45335 | 40.94614 |
| 102.5 | 20.5291 | 21.19055 | 22.29905 | 24.44283 | 27.38203 | 31.14942 | 35.58347 | 38.91658 | 41.44718 |
| 103.5 | 20.69997 | 21.37219 | 22.49884 | 24.67802 | 27.66593 | 31.49536 | 36.00078 | 39.38577 | 41.95447 |
| 104.5 | 20.873 | 21.55616 | 22.70125 | 24.91634 | 27.95365 | 31.84592 | 36.42352 | 39.86086 | 42.46794 |
| 105.5 | 21.04828 | 21.74253 | 22.90633 | 25.15783 | 28.24521 | 32.20108 | 36.85164 | 40.34179 | 42.98755 |
| 106.5 | 21.22589 | 21.93138 | 23.11413 | 25.40252 | 28.5406 | 32.56084 | 37.28507 | 40.82849 | 43.5132 |
| 107.5 | 21.40589 | 22.12277 | 23.32471 | 25.65046 | 28.83984 | 32.92513 | 37.72376 | 41.32088 | 44.0448 |
| 108.5 | 21.58837 | 22.31677 | 23.53813 | 25.90167 | 29.14291 | 33.29393 | 38.16762 | 41.81885 | 44.58226 |
| 109.5 | 21.77338 | 22.51343 | 23.75442 | 26.15616 | 29.4498 | 33.66717 | 38.61656 | 42.32229 | 45.12543 |
| 110.5 | 21.96099 | 22.71282 | 23.97364 | 26.41394 | 29.76048 | 34.04479 | 39.07046 | 42.83107 | 45.67419 |
| 111.5 | 22.15126 | 22.91497 | 24.19581 | 26.67503 | 30.07493 34.4267 39.52921 | | 43.34505 | 46.22839 | |
| 112.5 | 22.34426 | 23.11994 | 24.42096 | 26.93942 | 30.39308 | 34.81282 39.99268 43.864 | | 43.86408 | 46.78786 |
| 113.5 | 22.54002 | 23.32778 | 24.64912 | 27.20709 | 30.7149 | 35.20305 | 40.46071 | 44.38798 | 47.35242 |
| 114.5 | 22.73861 | 23.53851 | 24.88031 | 27.47805 | 31.04032 | 35.59726 | 40.93316 | 44.91658 | 47.92187 |
| 115.5 | 22.94006 | 23.75217 | 25.11454 | 27.75225 | 31.36928 | 35.99535 | 41.40984 | 45.44968 | 48.49603 |
| 116.5 | 23.14441 | 23.96879 | 25.35181 | 28.02968 | 31.70168 | 36.39717 | 41.89057 | 45.98708 | 49.07465 |
| 117.5 | 23.3517 | 24.18838 | 25.59214 | 28.31029 | 32.03745 | 36.80259 | 42.37517 | 46.52854 | 49.65753 |
| 118.5 | 23.56195 | 24.41097 | 25.83551 | 28.59403 | 32.37649 | 37.21144 | 42.86342 | 47.07385 | 50.2444 |
| 119.5 | 23.77519 | 24.63656 | 26.08191 | 28.88087 | 32.71868 | 37.62356 | 43.35511 | 47.62276 | 50.83502 |
| 120.5 | 23.99143 | 24.86516 | 26.33132 | 29.17072 | 33.06392 | 38.03878 | 43.85001 | 48.17501 | 51.42913 |
| 121.5 | 24.21068 | 25.09677 | 26.58372 | 29.46353 | 33.41208 | 38.45691 | 44.34788 | 48.73033 | 52.02644 |
| 122.5 | 24.43296 | 25.33137 | 26.83907 | 29.75922 | 33.76303 | 38.87775 | 44.84847 | 49.28846 | 52.62666 |
| 123.5 | 24.65826 | 25.56895 | 27.09734 | 30.0577 | 34.11663 | 39.30111 | 45.35152 | 49.84911 | 53.22951 |
| 124.5 | 24.88657 | 25.80949 | 27.35848 | 30.35888 | 34.47272 | 39.72676 | 45.85676 | 50.41198 | 53.83467 |
| 125.5 | 25.11788 | 26.05297 | 27.62244 | 30.66267 | 34.83116 | 40.15449 | 46.36392 | 50.97677 | 54.44183 |
| 126.5 | 25.35217 | 26.29934 | 27.88915 | 30.96895 | 35.19176 | 40.58407 | 46.87271 | 51.54317 | 55.05067 |
| 127.5 | 25.58941 | 26.54856 | 28.15856 | 31.27762 | 35.55437 | 41.01526 | 47.38283 | 52.11086 | 55.66086 |
| 128.5 | 25.82958 | 26.8006 | 28.43059 | 31.58856 | 35.9188 | 41.44782 | 47.894 | 52.67951 | 56.27207 |
| 129.5 | 26.07263 | 27.05539 | 28.70516 | 31.90163 | 36.28486 | 41.88148 | 48.40589 | 53.2488 | 56.88395 |
| 130.5 | 26.31852 | 27.31287 | 28.98218 | 32.21671 | 36.65236 | 42.316 | 48.9182 | 53.81837 | 57.49615 |
| 131.5 | 26.56719 | 27.57298 | 29.26156 | 32.53364 | 37.02111 | 42.75111 | 49.43061 | 54.3879 | 58.10833 |
| 132.5 | 26.81859 | 27.83564 | 29.54321 | 32.8523 | 37.39089 | 43.18655 | 49.9428 | 54.95703 | 58.72013 |

| | 3rd | 5th | 10th | 25th | 50th | 75th | 90th | 95th | 97th |
|---|---|---|---|---|---|---|---|---|---|
| Age (in | Percentile | Percentile | Percentile | Percentile | Percentile | Percentile | Percentile | Percentile | Percentile |
| months) | Weight (in kilograms) | Weight (in kilograms) | Weight (in kilograms) | Weight (in kilograms) | Weight (in kilograms) | Weight (in kilograms) | Weight (in kilograms) | Weight (in kilograms) | Weight (in kilograms) |
| 133.5 | 27.07265 | 28.10077 | 29.827 | 33.17252 | 37.76149 | 43.62203 | 50.45443 | 55.52542 | 59.33118 |
| 134.5 | 27.3293 | 28.36829 | 30.11285 | 33.49415 | 38.1327 | 44.05728 | 50.96519 | 56.09271 | 59.94114 |
| 135.5 | 27.58846 | 28.63809 | 30.40062 | 33.81701 | 38.5043 | 44.49201 | 51.47473 | 56.65855 | 60.54964 |
| 136.5 | 27.85004 | 28.91009 | 30.69019 | 34.14096 | 38.87605 | 44.92595 | 51.98272 | 57.22257 | 61.15631 |
| 137.5 | 28.11395 | 29.18417 | 30.98143 | 34.4658 | 39.24775 | 45.3588 | 52.48882 | 57.78443 | 61.7608 |
| 138.5 | 28.38009 | 29.46022 | 31.27421 | 34.79137 | 39.61914 | 45.79028 | 52.9927 | 58.34376 | 62.36274 |
| 139.5 | 28.64837 | 29.73813 | 31.56838 | 35.11747 | 39.99 | 46.22009 | 53.49402 | 58.90022 | 62.96178 |
| 140.5 | 28.91866 | 30.01776 | 31.86381 | 35.44394 | 40.36009 | 46.64794 | 53.99244 | 59.45344 | 63.55756 |
| 141.5 | 29.19086 | 30.299 | 32.16034 | 35.77056 | 40.72918 | 47.07354 | 54.48762 | 60.00308 | 64.14972 |
| 142.5 | 29.46484 | 30.5817 | 32.45781 | 36.09716 | 41.09701 | 47.49661 | 54.97925 | 60.54878 | 64.73791 |
| 143.5 | 29.74046 | 30.86573 | 32.75608 | 36.42354 | 41.46336 | 47.91684 | 55.46697 | 61.0902 | 65.32179 |
| 144.5 | 30.0176 | 31.15094 | 33.05496 | 36.7495 | 41.82798 | 48.33396 | 55.95048 | 61.62701 | 65.90103 |
| 145.5 | 30.29612 | 31.43718 | 33.3543 | 37.07485 | 42.19063 | 48.74767 | 56.42944 | 62.15887 | 66.47528 |
| 146.5 | 30.57588 | 31.7243 | 33.65394 | 37.39937 | 42.55108 | 49.15771 | 56.90354 | 62.68544 | 67.04422 |
| 147.5 | 30.85671 | 32.01214 | 33.95368 | 37.72288 | 42.90909 | 49.56378 | 57.37247 | 63.20642 | 67.60754 |
| 148.5 | 31.13848 | 32.30053 | 34.25336 | 38.04517 | 43.26442 | 49.96562 | 57.83593 | 63.72148 | 68.16491 |
| 149.5 | 31.42101 | 32.58932 | 34.55281 | 38.36604 | 43.61683 | 1683 50.36297 58.29361 64.230 | | 64.23032 | 68.71605 |
| 150.5 | 31.70415 | 32.87832 | 34.85183 | 38.68529 | 43.96612 | 50.75555 | 58.74524 | 64.73264 | 69.26067 |
| 151.5 | 31.98774 | 33.16738 | 35.15025 | 39.00272 | 44.31204 | 51.14313 | 59.19053 | 65.22816 | 69.79847 |
| 152.5 | 32.27159 | 33.4563 | 35.44789 | 39.31812 | 44.65437 | 51.52544 | 59.62921 | 65.71661 | 70.32919 |
| 153.5 | 32.55554 | 33.74492 | 35.74455 | 39.63131 | 44.99291 | 51.90225 | 60.06103 | 66.19771 | 70.85258 |
| 154.5 | 32.8394 | 34.03306 | 36.04006 | 39.94209 | 45.32745 | 52.27334 | 60.48572 | 66.67121 | 71.36839 |
| 155.5 | 33.12301 | 34.32053 | 36.33424 | 40.25026 | 45.65777 | 52.63847 | 60.90306 | 67.13688 | 71.87638 |
| 156.5 | 33.40617 | 34.60715 | 36.62688 | 40.55564 | 45.98369 | 52.99745 | 61.31281 | 67.59448 | 72.37633 |
| 157.5 | 33.6887 | 34.89274 | 36.91782 | 40.85805 | 46.30501 | 53.35007 | 61.71477 | 68.04379 | 72.86804 |
| 158.5 | 33.97042 | 35.17711 | 37.20687 | 41.15729 | 46.62155 | 53.69614 | 62.10874 | 68.48463 | 73.35131 |
| 159.5 | 34.25114 | 35.46007 | 37.49385 | 41.45321 | 46.93314 | 54.03549 | 62.49452 | 68.91679 | 73.82597 |
| 160.5 | 34.53066 | 35.74145 | 37.77858 | 41.74562 | 47.23962 | 54.36794 | 62.87195 | 69.34011 | 74.29185 |
| 161.5 | 34.80881 | 36.02105 | 38.06087 | 42.03435 | 47.54083 | 54.69335 | 63.24088 | 69.75442 | 74.7488 |
| 162.5 | 35.08539 | 36.2987 | 38.34057 | 42.31926 | 47.83661 | 55.01159 | 63.60115 | 70.1596 | 75.19669 |
| 163.5 | 35.36022 | 36.57421 | 38.61748 | 42.60018 | 48.12685 | 55.32252 | 63.95264 | 70.5555 | 75.6354 |
| 164.5 | 35.63309 | 36.84739 | 38.89145 | 42.87697 | 48.41141 | 55.62603 | 64.29525 | 70.94203 | 76.06483 |
| 165.5 | 35.90384 | 37.11808 | 39.16232 | 43.14949 | 48.69018 | 55.92203 | 64.62889 | 71.31908 | 76.48488 |
| 166.5 | 36.17227 | 37.3861 | 39.42991 | 43.4176 | 48.96305 | 56.21044 | 64.95347 | 71.68659 | 76.89549 |
| 167.5 | 36.4382 | 37.65127 | 39.69408 | 43.68119 | 49.22993 | 56.49119 | 65.26895 | 72.04449 | 77.2966 |
| 168.5 | 36.70144 | 37.91342 | 39.95467 | 43.94012 | 49.49075 | 56.76423 | 65.57527 | 72.39275 | 77.68817 |
| 169.5 | 36.96182 | 38.17238 | 40.21154 | 44.1943 | 49.74544 | 57.02954 | 65.87243 | 72.73133 | 78.07017 |

| | 3rd | 5th | 10th | 25th | 50th | 75th | 90th | 95th | 97th |
|---|---|---|---|---|---|---|---|---|---|
| Age (in | Percentile | Percentile | Percentile | Percentile | Percentile | Percentile | Percentile | Percentile | Percentile |
| months) | Weight (in kilograms) | Weight (in kilograms) | Weight (in kilograms) | Weight (in kilograms) | Weight (in kilograms) | Weight (in kilograms) | Weight (in kilograms) | Weight (in kilograms) | Weight (in kilograms) |
| 170.5 | 37.21916 | 38.428 | 40.46454 | 44.44363 | 49.99394 | 57.28708 | 66.16042 | 73.06023 | 78.44259 |
| 171.5 | 37.4733 | 38.68012 | 40.71356 | 44.688 | 50.23621 | 57.53687 | 66.43925 | 73.37946 | 78.80544 |
| 172.5 | 37.72405 | 38.92858 | 40.95845 | 44.92735 | 50.47222 | 57.77893 | 66.70897 | 73.68906 | 79.15873 |
| 173.5 | 37.97127 | 39.17324 | 41.19909 | 45.1616 | 50.70196 | 58.01327 | 66.96961 | 73.98906 | 79.50251 |
| 174.5 | 38.21478 | 39.41396 | 41.43538 | 45.39069 | 50.92541 | 58.23994 | 67.22127 | 74.27953 | 79.83682 |
| 175.5 | 38.45445 | 39.6506 | 41.66721 | 45.61455 | 51.14259 | 58.45903 | 67.46402 | 74.56056 | 80.16173 |
| 176.5 | 38.69012 | 39.88303 | 41.89448 | 45.83316 | 51.35353 | 58.67061 | 67.69798 | 74.83223 | 80.4773 |
| 177.5 | 38.92165 | 40.11114 | 42.1171 | 46.04647 | 51.55825 | 58.87477 | 67.92327 | 75.09468 | 80.78364 |
| 178.5 | 39.14891 | 40.3348 | 42.33498 | 46.25446 | 51.75681 | 59.07164 | 68.14006 | 75.34802 | 81.08083 |
| 179.5 | 39.37177 | 40.55392 | 42.54806 | 46.45712 | 51.94926 | 59.26135 | 68.3485 | 75.59243 | 81.36901 |
| 180.5 | 39.59012 | 40.76839 | 42.75627 | 46.65445 | 52.13568 | 59.44404 | 68.54877 | 75.82805 | 81.6483 |
| 181.5 | 39.80385 | 40.97812 | 42.95955 | 46.84646 | 52.31616 | 59.61988 | 68.74109 | 76.05507 | 81.91883 |
| 182.5 | 40.01284 | 41.18304 | 43.15786 | 47.03316 | 52.4908 | 59.78905 | 68.92566 | 76.2737 | 82.18076 |
| 183.5 | 40.21702 | 41.38308 | 43.35116 | 47.21458 | 52.6597 | 59.95173 | 69.10273 | 76.48415 | 82.43425 |
| 184.5 | 40.4163 | 41.57816 | 43.53942 | 47.39077 | 52.82299 | 60.10814 | 69.27255 | 76.68664 | 82.67946 |
| 185.5 | 40.6106 | 41.76824 | 43.72263 | 47.56176 | 52.98079 | 60.2585 | 69.43538 | 76.88142 | 82.91657 |
| 186.5 | 40.79986 | 41.95328 | 43.90078 | 47.72763 | 53.13327 | 60.40303 | 69.59151 | 77.06875 | 83.14578 |
| 187.5 | 40.98403 | 42.13324 | 44.07388 | 47.88844 | 53.28056 | 60.54199 | 69.74124 | 77.2489 | 83.36727 |
| 188.5 | 41.16306 | 42.3081 | 44.24193 | 48.04426 | 53.42284 | 60.67562 | 69.88487 | 77.42214 | 83.58126 |
| 189.5 | 41.33692 | 42.47785 | 44.40496 | 48.1952 | 53.56028 | 60.8042 | 70.02272 | 77.58878 | 83.78795 |
| 190.5 | 41.50559 | 42.64249 | 44.563 | 48.34134 | 53.69307 | 60.928 | 70.15513 | 77.74911 | 83.98755 |
| 191.5 | 41.66907 | 42.80203 | 44.71609 | 48.48279 | 53.82138 | 61.04731 | 70.28244 | 77.90345 | 84.18029 |
| 192.5 | 41.82734 | 42.95649 | 44.8643 | 48.61968 | 53.94544 | 61.16241 | 70.40499 | 78.05211 | 84.36639 |
| 193.5 | 41.98043 | 43.1059 | 45.00768 | 48.75212 | 54.06543 | 61.2736 | 70.52314 | 78.19542 | 84.54608 |
| 194.5 | 42.12835 | 43.25031 | 45.14631 | 48.88026 | 54.18158 | 61.3812 | 70.63725 | 78.33372 | 84.7196 |
| 195.5 | 42.27115 | 43.38976 | 45.28027 | 49.00422 | 54.29411 | 61.48549 | 70.7477 | 78.46734 | 84.88718 |
| 196.5 | 42.40886 | 43.52432 | 45.40964 | 49.12417 | 54.40324 | 61.58681 | 70.85484 | 78.59661 | 85.04905 |
| 197.5 | 42.54155 | 43.65406 | 45.53455 | 49.24026 | 54.50921 | 61.68546 | 70.95905 | 78.72189 | 85.20546 |
| 198.5 | 42.66928 | 43.77907 | 45.65509 | 49.35265 | 54.61224 | 61.78176 | 71.06071 | 78.84351 | 85.35663 |
| 199.5 | 42.79212 | 43.89944 | 45.77138 | 49.46152 | 54.71257 | 61.87602 | 71.16017 | 78.96181 | 85.50282 |
| 200.5 | 42.91017 | 44.01527 | 45.88355 | 49.56702 | 54.81044 | 61.96856 | 71.2578 | 79.07713 | 85.64425 |
| 201.5 | 43.02352 | 44.12666 | 45.99174 | 49.66936 | 54.9061 | 62.05968 | 71.35395 | 79.18979 | 85.78117 |
| 202.5 | 43.13227 | 44.23375 | 46.09608 | 49.7687 | 54.99978 | 62.1497 | 71.44899 | 79.30012 | 85.91379 |
| 203.5 | 43.23654 | 44.33665 | 46.19672 | 49.86524 | 55.09172 | 62.23891 | 71.54326 | 79.40845 | 86.04235 |
| 204.5 | 43.33646 | 44.4355 | 46.29382 | 49.95916 | 55.18217 | 62.32761 | 71.63707 | 79.51506 | 86.16706 |
| 205.5 | 43.43215 | 44.53044 | 46.38753 | 50.05066 | 55.27135 | 62.41609 | 71.73076 | 79.62027 | 86.28815 |
| 206.5 | 43.52374 | 44.62161 | 46.47801 | 50.13993 | 55.35951 | 62.50462 | 71.82463 | 79.72434 | 86.40583 |

| | 3rd | 5th | 10th | 25th | 50th | 75th | 90th | 95th | 97th |
|---|---|---|---|---|---|---|---|---|---|
| Age (in | Percentile | Percentile | Percentile | Percentile | Percentile | Percentile | Percentile | Percentile | Percentile |
| months) | Weight (in kilograms) | Weight (in kilograms) | Weight (in kilograms) | Weight (in kilograms) | Weight (in kilograms) | Weight (in kilograms) | Weight (in | Weight (in kilograms) | Weight (in |
| | , | , | | | , | | kilograms) | | |
| 207.5 | 43.61137 | 44.70917 | 46.56543 | 50.22716 | 55.44686 | 62.59347 | 71.91896 | 79.82755 | 86.52029 |
| 208.5 | 43.69521 | 44.79326 | 46.64995 | 50.31253 | 55.53362 | 62.68289 | 72.01403 | 79.93015 | 86.63173 |
| 209.5 | 43.77538 | 44.87405 | 46.73174 | 50.39624 | 55.62001 | 62.77311 | 72.11008 | 80.03235 | 86.74034 |
| 210.5 | 43.85205 | 44.95168 | 46.81097 | 50.47847 | 55.70624 | 62.86437 | 72.20733 | 80.13439 | 86.84629 |
| 211.5 | 43.92537 | 45.02633 | 46.8878 | 50.5594 | 55.79248 | 62.95684 | 72.306 | 80.23643 | 86.94976 |
| 212.5 | 43.9955 | 45.09815 | 46.9624 | 50.63919 | 55.87892 | 63.05073 | 72.40626 | 80.33866 | 87.05088 |
| 213.5 | 44.06258 | 45.16729 | 47.03493 | 50.71802 | 55.96573 | 63.1462 | 72.50825 | 80.4412 | 87.14981 |
| 214.5 | 44.12679 | 45.23391 | 47.10554 | 50.79603 | 56.05305 | 63.24336 | 72.61209 | 80.54417 | 87.24667 |
| 215.5 | 44.18826 | 45.29817 | 47.17437 | 50.87336 | 56.141 | 63.34234 | 72.71787 | 80.64766 | 87.34157 |
| 216.5 | 44.24715 | 45.3602 | 47.24158 | 50.95014 | 56.2297 | 63.4432 | 72.82563 | 80.75172 | 87.43462 |
| 217.5 | 44.3036 | 45.42015 | 47.30728 | 51.02649 | 56.31922 | 63.546 | 72.9354 | 80.85638 | 87.5259 |
| 218.5 | 44.35775 | 45.47815 | 47.3716 | 51.10249 | 56.40963 | 63.65074 | 73.04714 | 80.96163 | 87.61548 |
| 219.5 | 44.40973 | 45.53431 | 47.43464 | 51.17823 | 56.50096 | 63.7574 | 73.1608 | 81.06744 | 87.70342 |
| 220.5 | 44.45965 | 45.58875 | 47.4965 | 51.25375 | 56.5932 | 63.86593 | 73.27626 | 81.17373 | 87.78975 |
| 221.5 | 44.50764 | 45.64157 | 47.55724 | 51.32908 | 56.68633 | 63.9762 | 73.39338 | 81.28039 | 87.87449 |
| 222.5 | 44.55377 | 45.69284 | 47.61693 | 51.40422 | 56.78026 | 64.08808 | 73.51197 | 81.3873 | 87.95764 |
| 223.5 | 44.59815 | 45.74262 | 47.67559 | 51.47916 | 56.8749 | 64.20136 | 73.63178 | 81.49427 | 88.03918 |
| 224.5 | 44.64082 | 45.79097 | 47.73323 | 51.55381 | 56.9701 | 64.3158 | 73.75253 | 81.60109 | 88.11907 |
| 225.5 | 44.68185 | 45.8379 | 47.78983 | 51.6281 | 57.06565 | 64.4311 | 73.87389 | 81.70752 | 88.19726 |
| 226.5 | 44.72126 | 45.88343 | 47.84535 | 51.70189 | 57.16132 | 64.54692 | 73.99546 | 81.81326 | 88.27366 |
| 227.5 | 44.75906 | 45.92751 | 47.89972 | 51.77499 | 57.2568 | 64.66283 | 74.1168 | 81.91801 | 88.34817 |
| 228.5 | 44.79521 | 45.97009 | 47.9528 | 51.8472 | 57.35176 | 64.77838 | 74.23744 | 82.02139 | 88.42066 |
| 229.5 | 44.82969 | 46.0111 | 48.00447 | 51.91825 | 57.44578 | 64.89303 | 74.35682 | 82.12303 | 88.491 |
| 230.5 | 44.8624 | 46.0504 | 48.05453 | 51.98781 | 57.5384 | 65.00619 | 74.47435 | 82.22248 | 88.55903 |
| 231.5 | 44.89324 | 46.08784 | 48.10274 | 52.05553 | 57.6291 | 65.1172 | 74.58939 | 82.31928 | 88.62455 |
| 232.5 | 44.92205 | 46.12322 | 48.14882 | 52.12097 | 57.71728 | 65.22534 | 74.70121 | 82.41292 | 88.68734 |
| 233.5 | 44.94866 | 46.1563 | 48.19244 | 52.18364 | 57.80227 | 65.32981 | 74.80907 | 82.50285 | 88.74718 |
| 234.5 | 44.97281 | 46.18678 | 48.23321 | 52.243 | 57.88334 | 65.42974 | 74.91215 | 82.58851 | 88.80382 |
| 235.5 | 44.99424 | 46.21432 | 48.27069 | 52.29842 | 57.95967 | 65.52419 | 75.00958 | 82.66927 | 88.85697 |
| 236.5 | 45.0126 | 46.23851 | 48.30438 | 52.34921 | 58.0304 | 65.61215 | 75.10041 | 82.74448 | 88.90635 |
| 237.5 | 45.02752 | 46.25891 | 48.3337 | 52.3946 | 58.09453 | 65.69252 | 75.18367 | 82.81345 | 88.95164 |
| 238.5 | 45.03852 | 46.27498 | 48.358 | 52.43376 | 58.15104 | 65.76413 | 75.25831 | 82.87546 | 88.99253 |
| 239.5 | 45.0451 | 46.28612 | 48.37657 | 52.46576 | 58.19877 | 65.82574 | 75.32321 | 82.92975 | 89.02867 |
| 240 | 45.04655 | 46.28963 | 48.38346 | 52.47876 | 58.21897 | 65.85238 | 75.35165 | 82.95375 | 89.04485 |

# 10.10 Blood Pressure Levels for Males by Age and Height Percentile

### **APPENDIX 10.1** Fourth (4th) Report

From Fourth (4<sup>th</sup>) Report, Males, see References

| | | | S | | Blood I<br>mmHg | Pressu | re | | | D | | : Blood<br>(mmHg | | ure | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Age | BP | | | | ercentil | | | | | | | ercenti | , | | |
| (years) | percentile | 5 <sup>th</sup> | 10 <sup>th</sup> | 25 <sup>th</sup> | 50 <sup>th</sup> | 75 <sup>th</sup> | 90 <sup>th</sup> | 95 <sup>th</sup> | 5 <sup>th</sup> | 10 <sup>th</sup> | 25 <sup>th</sup> | 50 <sup>th</sup> | 75 <sup>th</sup> | 90 <sup>th</sup> | 95 <sup>th</sup> |
| 3 | 90th | 100 | 101 | 103 | 105 | 107 | 108 | 109 | 59 | 59 | 60 | 61 | 62 | 63 | 63 |
| | 95th | 104 | 105 | 107 | 109 | 110 | 112 | 113 | 63 | 63 | 64 | 65 | 66 | 67 | 67 |
| | 99th | 111 | 112 | 114 | 116 | 118 | 119 | 120 | 71 | 71 | 72 | 73 | 74 | 75 | 75 |
| 4 | 90th | 102 | 103 | 105 | 107 | 109 | 110 | 111 | 62 | 63 | 64 | 65 | 66 | 66 | 67 |
| | 95th | 106 | 107 | 109 | 111 | 112 | 114 | 115 | 66 | 67 | 68 | 69 | 70 | 71 | 71 |
| | 99th | 113 | 114 | 116 | 118 | 120 | 121 | 122 | 74 | 75 | 76 | 77 | 78 | 78 | 79 |
| 5 | 90th | 104 | 105 | 106 | 108 | 110 | 111 | 112 | 65 | 66 | 67 | 68 | 69 | 69 | 70 |
| | 95th | 108 | 109 | 110 | 112 | 114 | 115 | 116 | 69 | 70 | 71 | 72 | 73 | 74 | 74 |
| | 99th | 115 | 116 | 118 | 120 | 121 | 123 | 123 | 77 | 78 | 79 | 80 | 81 | 81 | 82 |
| 6 | 90th | 105 | 106 | 108 | 110 | 111 | 113 | 113 | 68 | 68 | 69 | 70 | 71 | 72 | 72 |
| | 95th | 109 | 110 | 112 | 114 | 115 | 117 | 117 | 72 | 72 | 73 | 74 | 75 | 76 | 76 |
| | 99th | 116 | 117 | 119 | 121 | 123 | 124 | 125 | 80 | 80 | 81 | 82 | 83 | 84 | 84 |
| 7 | 90th | 106 | 107 | 109 | 111 | 113 | 114 | 115 | 70 | 70 | 71 | 72 | 73 | 74 | 74 |
| | 95th | 110 | 111 | 113 | 115 | 117 | 118 | 119 | 74 | 74 | 75 | 76 | 77 | 78 | 78 |
| | 99th | 117 | 118 | 120 | 122 | 124 | 125 | 126 | 82 | 82 | 83 | 84 | 85 | 86 | 86 |
| 8 | 90th | 107 | 109 | 110 | 112 | 114 | 115 | 116 | 71 | 72 | 72 | 73 | 74 | 75 | 76 |
| | 95th | 111 | 112 | 114 | 116 | 118 | 119 | 120 | 75 | 76 | 77 | 78 | 79 | 79 | 80 |
| | 99th | 119 | 120 | 122 | 123 | 125 | 127 | 127 | 83 | 84 | 85 | 86 | 87 | 87 | 88 |
| 9 | 90th | 109 | 110 | 112 | 114 | 115 | 117 | 118 | 72 | 73 | 74 | 75 | 76 | 76 | 77 |
| | 95th | 113 | 114 | 116 | 118 | 119 | 121 | 121 | 76 | 77 | 78 | 79 | 80 | 81 | 81 |
| | 99th | 120 | 121 | 123 | 125 | 127 | 128 | 129 | 84 | 85 | 86 | 87 | 88 | 88 | 89 |
| 10 | 90th | 111 | 112 | 114 | 115 | 117 | 119 | 119 | 73 | 73 | 74 | 75 | 76 | 77 | 78 |
| . • | 95th | 115 | 116 | 117 | 119 | 121 | 122 | 123 | 77 | 78 | 79 | 80 | 81 | 81 | 82 |
| | 99th | 122 | 123 | 125 | 127 | 128 | 130 | 130 | 85 | 86 | 86 | 88 | 88 | 89 | 90 |
| 11 | 90th | 113 | 114 | 115 | 117 | 119 | 120 | 121 | 74 | 74 | 75 | 76 | 77 | 78 | 78 |
| | 95th | 117 | 118 | 119 | 121 | 123 | 124 | 125 | 78 | 78 | 79 | 80 | 81 | 82 | 82 |
| | 99th | 124 | 125 | 127 | 129 | 130 | 132 | 132 | 86 | 86 | 87 | 88 | 89 | 90 | 90 |
| 12 | 90th | 115 | 116 | 118 | 120 | 121 | 123 | 123 | 74 | 75 | 75 | 76 | 77 | 78 | 79 |
| | 95th | 119 | 120 | 122 | 123 | 125 | 127 | 127 | 78 | 79 | 80 | 81 | 82 | 82 | 83 |
| | 99th | 126 | 127 | 129 | 131 | 133 | 134 | 135 | 86 | 87 | 88 | 89 | 90 | 90 | 91 |
| 13 | 90th | 117 | 118 | 120 | 122 | 124 | 125 | 126 | 75 | 75 | 76 | 77 | 78 | 79 | 79 |
| | 95th | 121 | 122 | 124 | 126 | 128 | 129 | 130 | 79 | 79 | 80 | 81 | 82 | 83 | 83 |
| | 99th | 128 | 130 | 131 | 133 | 135 | 136 | 137 | 87 | 87 | 88 | 89 | 90 | 91 | 91 |
| 14 | 90th | 120 | 121 | 123 | 125 | 126 | 128 | 128 | 75 | 76 | 77 | 78 | 79 | 79 | 80 |
| | 95th | 124 | 125 | 127 | 128 | 130 | 132 | 132 | 80 | 80 | 81 | 82 | 83 | 84 | 84 |
| | 99th | 131 | 132 | 134 | 136 | 138 | 139 | 140 | 87 | 88 | 89 | 90 | 91 | 92 | 92 |
| 15 | 90th | 122 | 124 | 125 | 127 | 129 | 130 | 131 | 76 | 77 | 78 | 79 | 80 | 80 | 81 |
| . • | 95th | 126 | 127 | 129 | 131 | 133 | 134 | 135 | 81 | 81 | 82 | 83 | 84 | 85 | 85 |
| | 99th | 134 | 135 | 136 | 138 | 140 | 142 | 142 | 88 | 89 | 90 | 91 | 92 | 93 | 93 |
| 16 | 90th | 125 | 126 | 128 | 130 | 131 | 133 | 134 | 78 | 78 | 79 | 80 | 81 | 82 | 82 |
| | 95th | 129 | 130 | 132 | 134 | 135 | 137 | 137 | 82 | 83 | 83 | 84 | 85 | 86 | 87 |
| | 99th | 136 | 137 | 139 | 141 | 143 | 144 | 145 | 90 | 90 | 91 | 92 | 93 | 94 | 94 |
| 17 | 90th | 127 | 128 | 130 | 132 | 134 | 135 | 136 | 80 | 80 | 81 | 82 | 83 | 84 | 84 |
| | 95th | 131 | 132 | 134 | 136 | 138 | 139 | 140 | 84 | 85 | 86 | 87 | 87 | 88 | 89 |
| | 99th | 139 | 140 | 141 | 143 | 145 | 146 | 147 | 92 | 93 | 93 | 94 | 95 | 96 | 97 |
| L | | | | | | | | | | | | | | | |

### **APPENDIX 10.2** 2017 Clinical Practice Guidelines

From 2017 (American Academy of Pediatric) Clinical Practice Guidelines, Table 4, Males, see References

| | | | Sys | tolic Blo | od Press | ure (mm | Hg) | | | Dias | stolic Blo | ood Press | sure (mm | Hg) | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Age | BP | | | | ercentile | | | | | | | ercentile | | | |
| (years) | Percentile | 5 <sup>th</sup> | 10 <sup>th</sup> | 25 <sup>th</sup> | 50 <sup>th</sup> | 75 <sup>th</sup> | 90 <sup>th</sup> | 95 <sup>th</sup> | 5 <sup>th</sup> | 10 <sup>th</sup> | 25 <sup>th</sup> | 50 <sup>th</sup> | 75 <sup>th</sup> | 90 <sup>th</sup> | 95 <sup>th</sup> |
| 3 | Height (cm) | 92.5 | 93.9 | 96.3 | 99 | 101.8 | 104.3 | 105.8 | 92.5 | 93.9 | 96.3 | 99 | 101.8 | 104.3 | 105.8 |
| | 90 <sup>th</sup> | 101 | 102 | 102 | 103 | 104 | 105 | 105 | 58 | 58 | 59 | 59 | 60 | 61 | 61 |
| | 95 <sup>th</sup> | 106 | 106 | 107 | 107 | 108 | 109 | 109 | 60 | 61 | 61 | 62 | 63 | 64 | 64 |
| | 95th+12mmHg | 118 | 118 | 119 | 119 | 120 | 121 | 121 | 72 | 73 | 73 | 74 | 75 | 76 | 76 |
| 4 | Height (cm) | 98.5 | 100.2 | 102.9 | 105.9 | 108.9 | 111.5 | 113.2 | 98.5 | 100.2 | 102.9 | 105.9 | 108.9 | 111.5 | 113.2 |
| | 90 <sup>th</sup> | 102 | 103 | 104 | 105 | 105 | 106 | 107 | 60 | 61 | 62 | 62 | 63 | 64 | 64 |
| | 95th | 107 | 107 | 108 | 108 | 109 | 110 | 110 | 63 | 64 | 65 | 66 | 67 | 67 | 68 |
| | 95th+12mmHg | 119 | 119 | 120 | 120 | 121 | 122 | 122 | 75 | 76 | 77 | 78 | 79 | 79 | 80 |
| 5 | Height (cm) | 104.4 | 106.2 | 109.1 | 112.4 | 115.7 | 118.6 | 120.3 | 104.4 | 106.2 | 109.1 | 112.4 | 115.7 | 118.6 | 120.3 |
| | 90 <sup>th</sup> | 103 | 104 | 105 | 106 | 107 | 108 | 108 | 63 | 64 | 65 | 65 | 66 | 67 | 67 |
| | 95 <sup>th</sup> | 107 | 108 | 109 | 109 | 110 | 111 | 112 | 66 | 67 | 68 | 69 | 70 | 70 | 71 |
| | 95th+12mmHg | 119 | 120 | 121 | 121 | 122 | 123 | 124 | 78 | 79 | 80 | 81 | 82 | 82 | 83 |
| 6 | Height (cm) | 110.3 | 112.2 | 115.3 | 118.9 | 122.4 | 125.6 | 127.5 | 110.3 | 112.2 | 115.3 | 118.9 | 122.4 | 125.6 | 127.5 |
| | 90 <sup>th</sup> | 105 | 105 | 106 | 107 | 109 | 110 | 110 | 66 | 66 | 67 | 68 | 68 | 69 | 69 |
| | 95 <sup>th</sup> | 108 | 109 | 110 | 111 | 112 | 113 | 114 | 69 | 70 | 70 | 71 | 72 | 72 | 73 |
| | 95th+12mmHg | 120 | 121 | 122 | 123 | 124 | 125 | 126 | 81 | 82 | 82 | 83 | 84 | 84 | 85 |
| 7 | Height (cm) | 116.1 | 118 | 121.4 | 125.1 | 128.9 | 132.4 | 134.5 | 116.1 | 118 | 121.4 | 125.1 | 128.9 | 132.4 | 134.5 |
| | 90 <sup>th</sup> | 106 | 107 | 108 | 109 | 110 | 111 | 111 | 68 | 68 | 69 | 70 | 70 | 71 | 71 |
| | 95 <sup>th</sup> | 110 | 110 | 111 | 112 | 114 | 115 | 116 | 71 | 71 | 72 | 73 | 73 | 74 | 74 |
| | 95th+12mmHg | 122 | 122 | 123 | 124 | 126 | 127 | 128 | 83 | 83 | 84 | 85 | 85 | 86 | 86 |
| 8 | Height (cm) | 121.4 | 123.5 | 127 | 131 | 135.1 | 138.8 | 141 | 121.4 | 123.5 | 127 | 131 | 135.1 | 138.8 | 141 |
| | 90 <sup>th</sup> | 107 | 108 | 109 | 110 | 111 | 112 | 112 | 69 | 70 | 70 | 71 | 72 | 72 | 73 |
| | 95 <sup>th</sup> | 111 | 112 | 112 | 114 | 115 | 116 | 117 | 72 | 73 | 73 | 74 | 75 | 75 | 75 |
| | 95th+12mmHg | 123 | 124 | 124 | 126 | 127 | 128 | 129 | 84 | 85 | 85 | 86 | 87 | 87 | 87 |
| 9 | Height (cm) | 126 | 128.3 | 132.1 | 136.3 | 140.7 | 144.7 | 147.1 | 126 | 128.3 | 132.1 | 136.3 | 140.7 | 144.7 | 147.1 |
| | 90 <sup>th</sup> | 107 | 108 | 109 | 110 | 112 | 113 | 114 | 70 | 71 | 72 | 73 | 74 | 74 | 74 |
| | 95 <sup>th</sup> | 112 | 112 | 113 | 115 | 116 | 118 | 119 | 74 | 74 | 75 | 76 | 76 | 77 | 77 |
| | 95th+12mmHg | 124 | 124 | 125 | 127 | 128 | 130 | 131 | 86 | 86 | 87 | 88 | 88 | 89 | 89 |
| 10 | Height (cm) | 130.2 | 132.7 | 136.7 | 141.3 | 146.9 | 150.1 | 152.7 | 130.2 | 132.7 | 136.7 | 141.3 | 146.9 | 150.1 | 152.7 |
| | 90 <sup>th</sup> | 108 | 109 | 111 | 112 | 113 | 115 | 116 | 72 | 73 | 74 | 74 | 75 | 75 | 76 |
| | 95 <sup>th</sup> | 112 | 113 | 114 | 116 | 118 | 120 | 121 | 76 | 76 | 77 | 77 | 78 | 78 | 78 |
| | 95th+12mmHg | 124 | 125 | 126 | 128 | 130 | 132 | 133 | 88 | 88 | 89 | 89 | 90 | 90 | 90 |
| 11 | Height (cm) | 134.7 | 137.3 | 141.5 | 145.4 | 151.3 | 155.8 | 158.5 | 134.7 | 137.3 | 141.5 | 145.4 | 151.3 | 155.8 | 158.5 |
| | 90 <sup>th</sup> | 110 | 111 | 112 | 114 | 116 | 117 | 118 | 74 | 74 | 75 | 75 | 75 | 76 | 76 |
| | 95 <sup>th</sup> | 114 | 114 | 116 | 118 | 120 | 123 | 124 | 77 | 78 | 78 | 78 | 78 | 78 | 78 |
| | 95th+12mmHg | 126 | 126 | 128 | 130 | 132 | 135 | 136 | 89 | 90 | 90 | 90 | 90 | 90 | 90 |
| 12 | Height (cm) | 140.3 | 143 | 147.5 | 152.7 | 157.9 | 162.6 | 165.5 | 140.3 | 143 | 147.5 | 152.7 | 157.9 | 152.6 | 165.5 |
| | 90th | 113 | 114 | 115 | 117 | 119 | 121 | 122 | 75 | 75 | 75 | 75 | 75 | 76 | 76 |
| | 95th | 116 | 117 | 118 | 121 | 124 | 126 | 128 | 78 | 78 | 78 | 78 | 78 | 79 | 79 |
| | 95th+12mmHg | 128 | 129 | 130 | 133 | 136 | 138 | 140 | 90 | 90 | 90 | 90 | 90 | 91 | 91 |

# 10.11 Blood Pressure Levels for Females by Age and Height Percentile

### **APPENDIX 11.1** Fourth (4th) Report

From Fourth (4<sup>th</sup>) Report, Females, see Reference.

| | | - | S | | | Pressu | re | | | D | | Blood | | ure | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | ( | mmHg | ) | | | | | | (mmHg | | | |
| Age | BP | | | | ercentil | | | | | | | ercenti | | | |
| (years) | percentile | 5 <sup>th</sup> | 10 <sup>th</sup> | 25 <sup>th</sup> | 50 <sup>th</sup> | 75 <sup>th</sup> | 90 <sup>th</sup> | 95 <sup>th</sup> | 5 <sup>th</sup> | 10 <sup>th</sup> | 25 <sup>th</sup> | 50 <sup>th</sup> | 75 <sup>th</sup> | 90 <sup>th</sup> | 95 <sup>th</sup> |
| 3 | 90th | 100 | 100 | 102 | 103 | 104 | 106 | 106 | 61 | 62 | 62 | 63 | 64 | 64 | 65 |
| | 95th | 104 | 104 | 105 | 107 | 108 | 109 | 110 | 65 | 66 | 66 | 67 | 68 | 68 | 69 |
| | 99th | 111 | 111 | 113 | 114 | 115 | 116 | 117 | 73 | 73 | 74 | 74 | 75 | 76 | 76 |
| 4 | 90th | 101 | 102 | 103 | 104 | 106 | 107 | 108 | 64 | 64 | 65 | 66 | 67 | 67 | 68 |
| | 95th | 105 | 106 | 107 | 108 | 110 | 111 | 112 | 68 | 68 | 69 | 70 | 71 | 71 | 72 |
| | 99th | 112 | 113 | 114 | 115 | 117 | 118 | 119 | 76 | 76 | 76 | 77 | 78 | 79 | 79 |
| 5 | 90th | 103 | 103 | 105 | 106 | 107 | 109 | 109 | 66 | 67 | 67 | 68 | 69 | 69 | 70 |
| | 95th | 107 | 107 | 108 | 110 | 111 | 112 | 113 | 70 | 71 | 71 | 72 | 73 | 73 | 74 |
| | 99th | 114 | 114 | 116 | 117 | 118 | 120 | 120 | 78 | 78 | 79 | 79 | 80 | 81 | 81 |
| 6 | 90th | 104 | 105 | 106 | 108 | 109 | 110 | 111 | 68 | 68 | 69 | 70 | 70 | 71 | 72 |
| | 95th | 108 | 109 | 110 | 111 | 113 | 114 | 115 | 72 | 72 | 73 | 74 | 74 | 75 | 76 |
| | 99th | 115 | 116 | 117 | 119 | 120 | 121 | 122 | 80 | 80 | 80 | 81 | 82 | 83 | 83 |
| 7 | 90th | 106 | 107 | 108 | 109 | 111 | 112 | 113 | 69 | 70 | 70 | 71 | 72 | 72 | 73 |
| | 95th | 110 | 111 | 112 | 113 | 115 | 116 | 116 | 73 | 74 | 74 | 75 | 76 | 76 | 77 |
| | 99th | 117 | 118 | 119 | 120 | 122 | 123 | 124 | 81 | 81 | 82 | 82 | 83 | 84 | 84 |
| 8 | 90th | 108 | 109 | 110 | 111 | 113 | 114 | 114 | 71 | 71 | 71 | 72 | 73 | 74 | 74 |
| | 95th | 112 | 112 | 114 | 115 | 116 | 118 | 118 | 75 | 75 | 75 | 76 | 77 | 78 | 78 |
| | 99th | 119 | 120 | 121 | 122 | 123 | 125 | 125 | 82 | 82 | 83 | 83 | 84 | 85 | 86 |
| 9 | 90th | 110 | 110 | 112 | 113 | 114 | 116 | 116 | 72 | 72 | 72 | 73 | 74 | 75 | 75 |
| | 95th | 114 | 114 | 115 | 117 | 118 | 119 | 120 | 76 | 76 | 76 | 77 | 78 | 79 | 79 |
| | 99th | 121 | 121 | 123 | 124 | 125 | 127 | 127 | 83 | 83 | 84 | 84 | 85 | 86 | 87 |
| 10 | 90th | 112 | 112 | 114 | 115 | 116 | 118 | 118 | 73 | 73 | 73 | 74 | 75 | 76 | 76 |
| | 95th | 116 | 116 | 117 | 119 | 120 | 121 | 122 | 77 | 77 | 77 | 78 | 79 | 80 | 80 |
| | 99th | 123 | 123 | 125 | 126 | 127 | 129 | 129 | 84 | 84 | 85 | 86 | 86 | 87 | 88 |
| 11 | 90th | 114 | 114 | 116 | 117 | 118 | 119 | 120 | 74 | 74 | 74 | 75 | 76 | 77 | 77 |
| | 95th | 118 | 118 | 119 | 121 | 122 | 123 | 124 | 78 | 78 | 78 | 79 | 80 | 81 | 81 |
| | 99th | 125 | 125 | 126 | 128 | 129 | 130 | 131 | 85 | 85 | 86 | 87 | 87 | 88 | 89 |
| 12 | 90th | 116 | 116 | 117 | 119 | 120 | 121 | 122 | 75 | 75 | 75 | 76 | 77 | 78 | 78 |
| | 95th | 119 | 120 | 121 | 123 | 124 | 125 | 126 | 79 | 79 | 79 | 80 | 81 | 82 | 82 |
| | 99th | 127 | 127 | 128 | 130 | 131 | 132 | 133 | 86 | 86 | 87 | 88 | 88 | 89 | 90 |
| 13 | 90th | 117 | 118 | 119 | 121 | 122 | 123 | 124 | 76 | 76 | 76 | 77 | 78 | 79 | 79 |
| | 95th | 121 | 122 | 123 | 124 | 126 | 127 | 128 | 80 | 80 | 80 | 81 | 82 | 83 | 83 |
| | 99th | 128 | 129 | 130 | 132 | 133 | 134 | 135 | 87 | 87 | 88 | 89 | 89 | 90 | 91 |
| 14 | 90th | 119 | 120 | 121 | 122 | 124 | 125 | 125 | 77 | 77 | 77 | 78 | 79 | 80 | 80 |
| | 95th | 123 | 123 | 125 | 126 | 127 | 129 | 129 | 81 | 81 | 81 | 82 | 83 | 84 | 84 |
| | 99th | 130 | 131 | 132 | 133 | 135 | 136 | 136 | 88 | 88 | 89 | 90 | 90 | 91 | 92 |
| 15 | 90th | 120 | 121 | 122 | 123 | 125 | 126 | 127 | 78 | 78 | 78 | 79 | 80 | 81 | 81 |
| | 95th | 124 | 125 | 126 | 127 | 129 | 130 | 131 | 82 | 82 | 82 | 83 | 84 | 85 | 85 |
| | 99th | 131 | 132 | 133 | 134 | 136 | 137 | 138 | 89 | 89 | 90 | 91 | 91 | 92 | 93 |
| 16 | 90th | 121 | 122 | 123 | 124 | 126 | 127 | 128 | 78 | 78 | 79 | 80 | 81 | 81 | 82 |
| | 95th | 125 | 126 | 127 | 128 | 130 | 131 | 132 | 82 | 82 | 83 | 84 | 85 | 85 | 86 |
| | 99th | 132 | 133 | 134 | 135 | 137 | 138 | 139 | 90 | 90 | 90 | 91 | 92 | 93 | 93 |
| 17 | 90th | 122 | 122 | 123 | 125 | 126 | 127 | 128 | 78 | 79 | 79 | 80 | 81 | 81 | 82 |
| | 95th | 125 | 126 | 127 | 129 | 130 | 131 | 132 | 82 | 83 | 83 | 84 | 85 | 85 | 86 |
| | 99th | 133 | 133 | 134 | 136 | 137 | 138 | 139 | 90 | 90 | 91 | 91 | 92 | 93 | 93 |

ISN/Protocol 178-CL-206A

### **APPENDIX 11.2** 2017 Clinical Practice Guidelines

From 2017 (American Academy of Pediatric) Clinical Practice Guidelines, Table 5, Females, see Reference

| | | | Sys | tolic Blo | od Press | ure (mm | Hg) | | Diastolic Blood Pressure (mmHg) | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Age | BP | | | | ercentile | | | | | | P | ercentile | es | | |
| (years) | Percentile | 5 <sup>th</sup> | $10^{th}$ | 25 <sup>th</sup> | 50 <sup>th</sup> | 75 <sup>th</sup> | 90 <sup>th</sup> | 95 <sup>th</sup> | 5 <sup>th</sup> | 10 <sup>th</sup> | 25 <sup>th</sup> | 50 <sup>th</sup> | 75 <sup>th</sup> | 90 <sup>th</sup> | 95 <sup>th</sup> |
| 3 | Height (cm) | 91 | 92.4 | 94.9 | 97.6 | 100.5 | 103.1 | 104.6 | 91 | 92.4 | 94.9 | 97.6 | 100.5 | 103.1 | 104.6 |
| | 90 <sup>th</sup> | 102 | 103 | 104 | 104 | 105 | 106 | 107 | 60 | 61 | 61 | 62 | 63 | 64 | 65 |
| | 95 <sup>th</sup> | 106 | 106 | 107 | 108 | 109 | 110 | 110 | 64 | 65 | 65 | 66 | 67 | 68 | 69 |
| | 95th+12mmHg | 118 | 118 | 119 | 120 | 121 | 122 | 122 | 76 | 77 | 77 | 78 | 79 | 80 | 81 |
| 4 | Height (cm) | 97.2 | 98.8 | 101.4 | 104.5 | 107.6 | 110.5 | 112.2 | 97.2 | 98.8 | 101.4 | 104.5 | 107.6 | 110.5 | 112.2 |
| | 90 <sup>th</sup> | 103 | 104 | 105 | 106 | 107 | 108 | 108 | 62 | 63 | 64 | 65 | 66 | 67 | 67 |
| | 95th | 107 | 108 | 109 | 109 | 110 | 111 | 112 | 66 | 67 | 68 | 69 | 70 | 70 | 71 |
| | 95th+12mmHg | 119 | 120 | 121 | 121 | 122 | 123 | 124 | 78 | 79 | 80 | 81 | 82 | 82 | 83 |
| 5 | Height (cm) | 103.6 | 105.3 | 108.2 | 111.5 | 114.9 | 118.1 | 120 | 103.6 | 105.3 | 108.2 | 111.5 | 114.9 | 118.1 | 120 |
| | 90 <sup>th</sup> | 104 | 105 | 106 | 107 | 108 | 109 | 110 | 64 | 65 | 66 | 67 | 68 | 69 | 70 |
| | 95 <sup>th</sup> | 108 | 109 | 109 | 110 | 111 | 112 | 113 | 68 | 69 | 70 | 71 | 72 | 73 | 73 |
| | 95th+12mmHg | 120 | 121 | 121 | 122 | 123 | 124 | 125 | 80 | 81 | 82 | 83 | 84 | 85 | 85 |
| 6 | Height (cm) | 110 | 111.8 | 114.9 | 118.4 | 122.1 | 125.6 | 127.7 | 110 | 111.8 | 114.9 | 118.4 | 122.1 | 125.6 | 127.7 |
| | 90 <sup>th</sup> | 105 | 106 | 107 | 108 | 109 | 110 | 111 | 67 | 67 | 68 | 69 | 70 | 71 | 71 |
| | 95 <sup>th</sup> | 109 | 109 | 110 | 111 | 112 | 113 | 114 | 70 | 71 | 72 | 72 | 73 | 74 | 74 |
| | 95th+12mmHg | 121 | 121 | 122 | 123 | 124 | 125 | 126 | 82 | 83 | 84 | 84 | 85 | 86 | 86 |
| 7 | Height (cm) | 115.9 | 117.8 | 121.1 | 124.9 | 128.8 | 132.5 | 134.7 | 115.9 | 117.8 | 121.1 | 124.9 | 128.8 | 132.5 | 134.7 |
| | 90th | 106 | 106 | 107 | 109 | 110 | 111 | 112 | 68 | 68 | 69 | 70 | 71 | 72 | 72 |
| | 95th | 109 | 110 | 111 | 112 | 113 | 114 | 115 | 72 | 72 | 73 | 73 | 74 | 74 | 75 |
| | 95th+12mmHg | 121 | 122 | 123 | 124 | 125 | 126 | 127 | 84 | 84 | 85 | 85 | 86 | 86 | 87 |
| 8 | Height (cm) | 121 | 123 | 126.5 | 130.6 | 134.7 | 138.5 | 140.9 | 121 | 123 | 126.5 | 130.6 | 134.7 | 138.5 | 140.9 |
| | 90 <sup>th</sup> | 107 | 107 | 108 | 110 | 111 | 112 | 113 | 69 | 70 | 71 | 72 | 72 | 73 | 73 |
| | 95 <sup>th</sup> | 110 | 111 | 112 | 113 | 115 | 116 | 117 | 72 | 73 | 74 | 74 | 75 | 75 | 75 |
| | 95th+12mmHg | 122 | 123 | 124 | 125 | 127 | 128 | 129 | 84 | 85 | 86 | 86 | 87 | 87 | 87 |
| 9 | Height (cm) | 125.3 | 127.6 | 131.3 | 135.6 | 140.1 | 144.1 | 146.6 | 125.3 | 127.6 | 131.3 | 135.6 | 140.1 | 144.1 | 146.6 |
| | 90 <sup>th</sup> | 108 | 108 | 109 | 111 | 112 | 113 | 114 | 71 | 71 | 72 | 73 | 73 | 73 | 73 |
| | 95 <sup>th</sup> | 112 | 112 | 113 | 114 | 116 | 117 | 118 | 74 | 74 | 75 | 75 | 75 | 75 | 75 |
| | 95th+12mmHg | 124 | 124 | 125 | 126 | 128 | 129 | 130 | 86 | 86 | 87 | 87 | 87 | 87 | 87 |
| 10 | Height (cm) | 129.7 | 132.2 | 136.3 | 141 | 145.8 | 150.2 | 152.8 | 129.7 | 132.2 | 136.3 | 141 | 145.8 | 150.2 | 152.8 |
| | 90 <sup>th</sup> | 109 | 110 | 111 | 112 | 113 | 115 | 116 | 72 | 73 | 73 | 73 | 73 | 73 | 73 |
| | 95 <sup>th</sup> | 113 | 114 | 114 | 116 | 117 | 119 | 120 | 75 | 75 | 76 | 76 | 76 | 76 | 76 |
| | 95th+12mmHg | 125 | 126 | 126 | 128 | 129 | 131 | 132 | 87 | 87 | 88 | 88 | 88 | 88 | 88 |
| 11 | Height (cm) | 135.6 | 138.3 | 142.8 | 147.8 | 152.8 | 157.3 | 160 | 135.6 | 138.3 | 142.8 | 147.8 | 152.8 | 157.3 | 160 |
| | 90 <sup>th</sup> | 111 | 112 | 113 | 114 | 116 | 118 | 120 | 74 | 74 | 74 | 74 | 74 | 75 | 75 |
| | 95 <sup>th</sup> | 115 | 116 | 117 | 118 | 120 | 123 | 124 | 76 | 77 | 77 | 77 | 77 | 77 | 77 |
| | 95th+12mmHg | 127 | 128 | 129 | 130 | 132 | 135 | 136 | 88 | 89 | 89 | 89 | 89 | 89 | 89 |
| 12 | Height (cm) | 142.8 | 145.5 | 149.9 | 154.8 | 159.6 | 163.8 | 166.4 | 142.8 | 145.5 | 149.9 | 154.8 | 159.6 | 163.8 | 166.4 |
| | 90th | 114 | 115 | 116 | 118 | 120 | 122 | 122 | 75 | 75 | 75 | 75 | 76 | 76 | 76 |
| | 95th | 118 | 119 | 120 | 122 | 124 | 125 | 126 | 78 | 78 | 78 | 78 | 79 | 79 | 79 |
| | 95th+12mmHg | 130 | 131 | 132 | 134 | 136 | 137 | 138 | 90 | 90 | 90 | 90 | 91 | 91 | 91 |

# 10.12 Appendix 12: Calculation of Z-Scores for Height, Weight and BMI for Age and Sex Norms

The Centers for Disease Control and Prevention have provided growth charts that enable the calculation of z-scores for height, weight and BMI based on the age (in months) and sex for children, adolescents and young adults upto the age of 20 years [Kuczmarski et al, 2002].

On the basis that a 12-month year consists of 365.25 days,  $A_m$ , the age in months of a child at a study visit, equals (date of visit – date of birth)/30.4375. This age should <u>not</u> be rounded to the nearest month in the calculation of the z-score.

For each gender, separate formulae for the height, weight and BMI norms curves are supplied for each month in a child's age with integer values of the age at the mid-point of each interval, e.g there are separate curves for 30.5-<31.5, 59.5-<60.5 months etc.

For a curve where the mid-point of the age interval is A whole months (e.g. for a child of 30.85 or 31.36 months, A=31), the formula of the curve relies on six constants,  $L_1$ ,  $M_1$ ,  $S_1$ ,  $L_2$ ,  $M_2$  and  $S_2$ .

For a child aged  $A_m$  months, the z-score (Z) for height can be derived as follows (z-scores for weight and BMI follow similar steps):

- Let  $r = (A_m A + 0.5)$
- Let  $L=L_1+(L_2-L_1)*r$ ,  $M=M_1+(M_2-M_1)*r$ , and  $S=S_1+(S_2-S_1)*r$

• If -0.01 < L < 0.01 then 
$$Z = \left(\frac{1}{S}\right) \log\left(\frac{height}{M}\right)$$

otherwise 
$$Z = \left(\frac{1}{LS}\right) \left(\frac{height}{M}\right)^{L} - 1$$

Formula are also given for if a z-score indicates a "biologically infeasible value" (BIV):

- Let  $LO = 0.5*(M M(1 2LS)^{\frac{1}{L}})$
- Let  $HI = 0.5*(M(1+2LS)^{\frac{1}{L}} M)$
- If height<M then flag=(height-M)/LO, otherwise flag=(height-M)/HI
- If flag<-5 or flag>3 then the height is a BIV.

To illustrate, a boy born on the 1<sup>st</sup> January 2001 comes for a visit on 13<sup>th</sup> January 2013 and his height is measured as 159 cm. The steps for calculating Z are as follows:

- The boy is 4395 days old at the visit, which gives  $A_m=4395/30.4375=144.3943$
- As 144.3943 is in the interval (143.5,144.5), A=144

- R=144.3943-144+0.5=0.8943
- The curve for A=144 has  $L_1$ =0.416777012,  $M_1$ =148.7917006,  $S_1$ =0.04987865,  $L_2$ =0.420919142,  $M_2$ =149.3088178 and  $S_2$ =0.049947823 (see example SAS code below).
- The values of L,M and S are calculated to be L=0.420481, M=149.254, and S=0.0499478.

• 
$$Z = \left(\frac{1}{0.420481*0.0499478}\right) \left(\left(\frac{159}{149.254}\right)^{0.420481} - 1\right) = 1.283576$$

LO=7.23925, HI=7.67069 and, as height>M, flag=(height-M)/HI=1.27053. This
does not represent a BIV

#### Example SAS code for the creation of the Z-Score and BIV flag is as follows:

```
*input dataset is called DATAIN and has at least the following variables;
*AGEMOS : Age in months;
       : 1=male, 2=female;
*HEIGHT : standing height in cm;
*WEIGHT : weight in kg;
       : BMI in kg/m^2;
**DATA FILE FOR HEIGHT-FOR-AGE;
data htcrv;
     infile cards pad;
     input sex age LH1 MH1 SH1 LH2 MH2 SH2;
1 24 0.875839864 86.042792680 0.040247430 1.007208070 86.861609340 0.040395626
1 25 1.007208070 86.861609340 0.040395626 0.837251351 87.652472820 0.040577525
1 26 0.837251351 87.652472820 0.040577525 0.681492975 88.423264340 0.040723122
1 27 0.681492975 88.423264340 0.040723122 0.538779654 89.175492280 0.040833194
1 28 0.538779654 89.175492280 0.040833194 0.407697153 89.910408530 0.040909059
1 29 0.407697153 89.910408530 0.040909059 0.286762453 90.629077620 0.040952433
1 30 0.286762453 90.629077620 0.040952433 0.174489485 91.332423790 0.040965330
1 31 0.174489485 91.332423790 0.040965330 0.069444521 92.021271670 0.040949976
 32 0.069444521 92.021271670 0.040949976 -0.029720564 92.696379460 0.040908737
1 33 -0.029720564 92.696379460 0.040908737 -0.124251789 93.358465460 0.040844062
1 34 -0.124251789 93.358465460 0.040844062 -0.215288396 94.008229230 0.040758431
1\ 35\ -0.215288396\ 94.008229230\ 0.040758431\ -0.303854340\ 94.646369810\ 0.040654312
1\ 36\ -0.303854340\ 94.646369810\ 0.040654312\ -0.390918369\ 95.273591060\ 0.040534120
1\ 37\ -0.390918369\ 95.273591060\ 0.040534120\ -0.254801167\ 95.914749290\ 0.040572876
1\ 38\ -0.254801167\ 95.914749290\ 0.040572876\ -0.125654535\ 96.547343280\ 0.040616910
 39 -0.125654535 96.547343280 0.040616910 -0.003167350 97.171913090 0.040666414
1 40 -0.003167350 97.171913090 0.040666414 0.112912210 97.788977270 0.040721467
1 41 0.112912210 97.788977270 0.040721467 0.222754969 98.399028300 0.040782045
1 42 0.222754969 98.399028300 0.040782045 0.326530126 99.002543380 0.040848042
1 43 0.326530126 99.002543380 0.040848042 0.424361560 99.599977000 0.040919281
1 44 0.424361560 99.599977000 0.040919281 0.516353108 100.191764000 0.040995524
1 45 0.516353108 100.191764000 0.040995524 0.602595306 100.778319800 0.041076485
 46 0.602595306 100.778319800 0.041076485 0.683170764 101.360041100 0.041161838
1 47 0.683170764 101.360041100 0.041161838 0.758158406 101.937305800 0.041251224
1 48 0.758158406 101.937305800 0.041251224 0.827636736 102.510473500 0.041344257
1\ 49\ 0.827636736\ 102.510473500\ 0.041344257\ 0.891686306\ 103.079885200\ 0.041440534
1 50 0.891686306 103.079885200 0.041440534 0.950391530 103.645864000 0.041539635
1 51 0.950391530 103.645864000 0.041539635 1.003830006 104.208713000 0.041641136
1 52 1.003830006 104.208713000 0.041641136 1.052135690 104.768725600 0.041744602
1 53 1.052135690 104.768725600 0.041744602 1.095366900 105.326163800 0.041849607
```

```
1 54 1.095366900 105.326163800 0.041849607 1.133652119 105.881282300 0.041955723
1 55 1.133652119 105.881282300 0.041955723 1.167104213 106.434314600 0.042062532
1 56 1.167104213 106.434314600 0.042062532 1.195845353 106.985476900 0.042169628
  57 1.195845353 106.985476900 0.042169628 1.220004233 107.534968000 0.042276619
1 58 1.220004233 107.534968000 0.042276619 1.239715856 108.082969500 0.042383129
1 59 1.239715856 108.082969500 0.042383129 1.255121285 108.629645700 0.042488804
 60 1.255121285 108.629645700 0.042488804 1.266367398 109.175144100 0.042593311
  61 1.266367398 109.175144100 0.042593311 1.273606657 109.719595400 0.042696342
1 62 1.273606657 109.719595400 0.042696342 1.276996893 110.263113600 0.042797615
1 63 1.276996893 110.263113600 0.042797615 1.276701119 110.805796700 0.042896877
  64 1.276701119 110.805796700 0.042896877 1.272887366 111.347726500 0.042993904
  65 1.272887366 111.347726500 0.042993904 1.265728536 111.888969400 0.043088503
1 66 1.265728536 111.888969400 0.043088503 1.255402281 112.429576100 0.043180513
 67 1.255402281 112.429576100 0.043180513 1.242090871 112.969582700 0.043269806
  68 1.242090871 112.969582700 0.043269806 1.225981067 113.509010800 0.043356287
1 69 1.225981067 113.509010800 0.043356287 1.207263978 114.047867800 0.043439893
1 70 1.207263978 114.047867800 0.043439893 1.186140222 114.586148600 0.043520597
  71 1.186140222 114.586148600 0.043520597 1.162796198 115.123831500 0.043598407
  72\ 1.162796198\ 115.123831500\ 0.043598407\ 1.137442868\ 115.660886200\ 0.043673359
 73 1.137442868 115.660886200 0.043673359 1.110286487 116.197269100 0.043745523
  74\ 1.110286487\ 116.197269100\ 0.043745523\ 1.081536236\ 116.732925000\ 0.043815003
  75 1.081536236 116.732925000 0.043815003 1.051403740 117.267787900 0.043881929
1 76 1.051403740 117.267787900 0.043881929 1.020102497 117.801781900 0.043946461
1\ 77\ 1.020102497\ 117.801781900\ 0.043946461\ 0.987847213\ 118.334821500\ 0.044008785
  78 0.987847213 118.334821500 0.044008785 0.954853043 118.866812300 0.044069112
  79 0.954853043 118.866812300 0.044069112 0.921334742 119.397652000 0.044127675
1 80 0.921334742 119.397652000 0.044127675 0.887505723 119.927230900 0.044184725
 81 0.887505723 119.927230900 0.044184725 0.853577030 120.455433000 0.044240532
  82 0.853577030 120.455433000 0.044240532 0.819756239 120.982136200 0.044295379
1 83 0.819756239 120.982136200 0.044295379 0.786246296 121.507213600 0.044349559
1 84 0.786246296 121.507213600 0.044349559 0.753244292 122.030534200 0.044403374
  85 0.753244292 122.030534200 0.044403374 0.720940222 122.551963400 0.044457130
1\ 86\ 0.720940222\ 122.551963400\ 0.044457130\ 0.689515708\ 123.071364500\ 0.044511135
1 87 0.689515708 123.071364500 0.044511135 0.659142731 123.588599000 0.044565693
1 88 0.659142731 123.588599000 0.044565693 0.629997853 124.103531200 0.044621104
  89 0.629997853 124.103531200 0.044621104 0.602203984 124.616016100 0.044677662
 90 0.602203984 124.616016100 0.044677662 0.575908038 125.125918200 0.044735646
  91\ \ 0.575908038\ \ 125.125918200\ \ 0.044735646\ \ 0.551231340\ \ 125.633101200\ \ 0.044795322
  92 0.551231340 125.633101200 0.044795322 0.528279901 126.137431900 0.044856941
 93 0.528279901 126.137431900 0.044856941 0.507143576 126.638780400 0.044920730
1 94 0.507143576 126.638780400 0.044920730 0.487895344 127.137021700 0.044986899
  95 \ \ 0.487895344 \ \ 127.137021700 \ \ 0.044986899 \ \ 0.470590753 \ \ 127.632036200 \ \ 0.045055632
  96 0.470590753 127.632036200 0.045055632 0.455267507 128.123710400 0.045127088
1 97 0.455267507 128.123710400 0.045127088 0.441945241 128.611938300 0.045201399
1\ 98\ 0.441945241\ 128.611938300\ 0.045201399\ 0.430625458\ 129.096622000\ 0.045278671
 99 0.430625458 129.096622000 0.045278671 0.421291648 129.577672300 0.045358979
1 100 0.421291648 129.577672300 0.045358979 0.413909588 130.055010100 0.045442372
1 101 0.413909588 130.055010100 0.045442372 0.408427813 130.528566900 0.045528869
1 102 0.408427813 130.528566900 0.045528869 0.404778262 130.998285700 0.045618459
 103 0.404778262 130.998285700 0.045618459 0.402877077 131.464121800 0.045711105
1 104 0.402877077 131.464121800 0.045711105 0.402625561 131.926043900 0.045806742
1 105 0.402625561 131.926043900 0.045806742 0.403911270 132.384034800 0.045905281
1 106 0.403911270 132.384034800 0.045905281 0.406609232 132.838092000 0.046006604
1 107 0.406609232 132.838092000 0.046006604 0.410583274 133.288229100 0.046110573
1 108 0.410583274 133.288229100 0.046110573 0.415687443 133.734475900 0.046217028
1 109 0.415687443 133.734475900 0.046217028 0.421767514 134.176880100 0.046325790
 110 0.421767514 134.176880100 0.046325790 0.428662551 134.615507600 0.046436662
1 111 0.428662551 134.615507600 0.046436662 0.436206531 135.050443300 0.046549430
1\ 112\ 0.436206531\ 135.050443300\ 0.046549430\ 0.444230000\ 135.481792500\ 0.046663871
1 113 0.444230000 135.481792500 0.046663871 0.452561760 135.909681300 0.046779748
 114 0.452561760 135.909681300 0.046779748 0.461030578 136.334257700 0.046896817
1 115 0.461030578 136.334257700 0.046896817 0.469466904 136.755692300 0.047014827
1 116 0.469466904 136.755692300 0.047014827 0.477704608 137.174179400 0.047133525
 117 0.477704608 137.174179400 0.047133525 0.485582720 137.589937800 0.047252654
1 118 0.485582720 137.589937800 0.047252654 0.492947182 138.003211400 0.047371961
1 119 0.492947182 138.003211400 0.047371961 0.499652617 138.414270300 0.047491194
1\ 120\ 0.499652617\ 138.414270300\ 0.047491194\ 0.505564115\ 138.823411400\ 0.047610108
1 121 0.505564115 138.823411400 0.047610108 0.510559047 139.230959200 0.047728463
1 122 0.510559047 139.230959200 0.047728463 0.514528903 139.637266300 0.047846030
1\ 123\ 0.514528903\ 139.637266300\ 0.047846030\ 0.517381177\ 140.042714000\ 0.047962592
1 124 0.517381177 140.042714000 0.047962592 0.519041285 140.447712700 0.048077942
```

```
1 125 0.519041285 140.447712700 0.048077942 0.519454524 140.852702200 0.048191889
1 126 0.519454524 140.852702200 0.048191889 0.518588072 141.258151500 0.048304259
1 127 0.518588072 141.258151500 0.048304259 0.516433004 141.664559200 0.048414893
1 128 0.516433004 141.664559200 0.048414893 0.513006312 142.072452000 0.048523648
1 129 0.513006312 142.072452000 0.048523648 0.508352901 142.482385200 0.048630402
1 130 0.508352901 142.482385200 0.048630402 0.502547502 142.894940300 0.048735050
 131 0.502547502 142.894940300 0.048735050 0.495696454 143.310724100 0.048837504
1 132 0.495696454 143.310724100 0.048837504 0.487939275 143.730366300 0.048937694
1 133 0.487939275 143.730366300 0.048937694 0.479449924 144.154516700 0.049035564
1 134 0.479449924 144.154516700 0.049035564 0.470437652 144.583841400 0.049131073
1 135 0.470437652 144.583841400 0.049131073 0.461147305 145.019019200 0.049224189
1 136 0.461147305 145.019019200 0.049224189 0.451858946 145.460735900 0.049314887
1 137 0.451858946 145.460735900 0.049314887 0.442886661 145.909678400 0.049403145
 138 0.442886661 145.909678400 0.049403145 0.434576385 146.366527800 0.049488934
 139 0.434576385 146.366527800 0.049488934 0.427302633 146.831951300 0.049572216
1 140 0.427302633 146.831951300 0.049572216 0.421464027 147.306592900 0.049652935
1 141 0.421464027 147.306592900 0.049652935 0.417477538 147.791063500 0.049731004
1 142 0.417477538 147.791063500 0.049731004 0.415771438 148.285929400 0.049806300
1\ 143\ 0.415771438\ 148.285929400\ 0.049806300\ 0.416777012\ 148.791700600\ 0.049878650
1 144 0.416777012 148.791700600 0.049878650 0.420919142 149.308817800 0.049947823
1 145 0.420919142 149.308817800 0.049947823 0.428606007 149.837639100 0.050013518
1 146 0.428606007 149.837639100 0.050013518 0.440218167 150.378426700 0.050075353
1 147 0.440218167 150.378426700 0.050075353 0.456097443 150.931333100 0.050132858
1 148 0.456097443 150.931333100 0.050132858 0.476536014 151.496388700 0.050185471
1 149 0.476536014 151.496388700 0.050185471 0.501766234 152.073489700 0.050232532
1 150 0.501766234 152.073489700 0.050232532 0.531951655 152.662387800 0.050273285
1 151 0.531951655 152.662387800 0.050273285 0.567179725 153.262681900 0.050306885
 152 0.567179725 153.262681900 0.050306885 0.607456565 153.873812400 0.050332406
 153 0.607456565 153.873812400 0.050332406 0.652704121 154.495058000 0.050348860
1 154 0.652704121 154.495058000 0.050348860 0.702759868 155.125536500 0.050355216
1 155 0.702759868 155.125536500 0.050355216 0.757379106 155.764208600 0.050350423
1 156 0.757379106 155.764208600 0.050350423 0.816239713 156.409885800 0.050333444
1 157 0.816239713 156.409885800 0.050333444 0.878947416 157.061241500 0.050303283
1 158 0.878947416 157.061241500 0.050303283 0.945053486 157.716828900 0.050259018
1 159 0.945053486 157.716828900 0.050259018 1.014046108 158.375092900 0.050199837
 160 1.014046108 158.375092900 0.050199837 1.085383319 159.034399000 0.050125062
1 161 1.085383319 159.034399000 0.050125062 1.158487278 159.693050100 0.050034180
1 162 1.158487278 159.693050100 0.050034180 1.232768816 160.349316800 0.049926861
1 163 1.232768816 160.349316800 0.049926861 1.307628899 161.001458600 0.049802977
1 164 1.307628899 161.001458600 0.049802977 1.382473225 161.647751500 0.049662610
1 165 1.382473225 161.647751500 0.049662610 1.456720479 162.286511900 0.049506051
1 166 1.456720479 162.286511900 0.049506051 1.529810247 162.916120200 0.049333801
 167 1.529810247 162.916120200 0.049333801 1.601219573 163.535045000 0.049146553
1 168 1.601219573 163.535045000 0.049146553 1.670433444 164.141848600 0.048945190
1 169 1.670433444 164.141848600 0.048945190 1.736995571 164.735219900 0.048730749
1 170 1.736995571 164.735219900 0.048730749 1.800483802 165.313975500 0.048504404
1 171 1.800483802 165.313975500 0.048504404 1.860518777 165.877071500 0.048267442
1 172 1.860518777 165.877071500 0.048267442 1.916765525 166.423608700 0.048021230
1 173 1.916765525 166.423608700 0.048021230 1.968934444 166.952835400 0.047767192
 174 1.968934444 166.952835400 0.047767192 2.016781776 167.464146600 0.047506783
1\ 175\ 2.016781776\ 167.464146600\ 0.047506783\ 2.060109658\ 167.957081400\ 0.047241456
1 176 2.060109658 167.957081400 0.047241456 2.098765817 168.431317500 0.046972650
1 177 2.098765817 168.431317500 0.046972650 2.132642948 168.886664400 0.046701759
1 178 2.132642948 168.886664400 0.046701759 2.161677790 169.323054800 0.046430122
1 179 2.161677790 169.323054800 0.046430122 2.185849904 169.740535100 0.046159004
1 180 2.185849904 169.740535100 0.046159004 2.205180153 170.139255000 0.045889585
 181 2.205180153 170.139255000 0.045889585 2.219728869 170.519456700 0.045622955
1 182 2.219728869 170.519456700 0.045622955 2.229593700 170.881464000 0.045360101
1 183 2.229593700 170.881464000 0.045360101 2.234907144 171.225671700 0.045101913
1 184 2.234907144 171.225671700 0.045101913 2.235833767 171.552534500 0.044849174
 185 2.235833767 171.552534500 0.044849174 2.232567138 171.862557600 0.044602566
1 186 2.232567138 171.862557600 0.044602566 2.225326500 172.156286500 0.044362674
1 187 2.225326500 172.156286500 0.044362674 2.214353232 172.434298300 0.044129985
 188 2.214353232 172.434298300 0.044129985 2.199905902 172.697193500 0.043904897
1 189 2.199905902 172.697193500 0.043904897 2.182262864 172.945589800 0.043687723
1 190 2.182262864 172.945589800 0.043687723 2.161704969 173.180112000 0.043478698
1 191 2.161704969 173.180112000 0.043478698 2.138524662 173.401389600 0.043277987
1 192 2.138524662 173.401389600 0.043277987 2.113023423 173.610051800 0.043085685
1 193 2.113023423 173.610051800 0.043085685 2.085490286 173.806717900 0.042901835
1 194 2.085490286 173.806717900 0.042901835 2.056219500 173.991999800 0.042726424
1 195 2.056219500 173.991999800 0.042726424 2.025496648 174.166495100 0.042559396
```

```
1 196 2.025496648 174.166495100 0.042559396 1.993598182 174.330785500 0.042400652
1 197 1.993598182 174.330785500 0.042400652 1.960789092 174.485434400 0.042250063
1 198 1.960789092 174.485434400 0.042250063 1.927320937 174.630985600 0.042107465
 199 1.927320937 174.630985600 0.042107465 1.893430240 174.767961700 0.041972676
1 200 1.893430240 174.767961700 0.041972676 1.859337259 174.896863400 0.041845488
1 201 1.859337259 174.896863400 0.041845488 1.825245107 175.018169100 0.041725679
1 202 1.825245107 175.018169100 0.041725679 1.791339209 175.132334500 0.041613015
1 203 1.791339209 175.132334500 0.041613015 1.757787065 175.239792600 0.041507249
1 204 1.757787065 175.239792600 0.041507249 1.724738292 175.340954000 0.041408129
1 205 1.724738292 175.340954000 0.041408129 1.692324905 175.436207100 0.041315398
 206 1.692324905 175.436207100 0.041315398 1.660661815 175.525919100 0.041228796
1 207 1.660661815 175.525919100 0.041228796 1.629847495 175.610435800 0.041148060
1 208 1.629847495 175.610435800 0.041148060 1.599964788 175.690083000 0.041072931
 209 1.599964788 175.690083000 0.041072931 1.571081817 175.765167100 0.041003150
  210 1.571081817 175.765167100 0.041003150 1.543252982 175.835975700 0.040938463
1 211 1.543252982 175.835975700 0.040938463 1.516519998 175.902778800 0.040878617
1 212 1.516519998 175.902778800 0.040878617 1.490912963 175.965829300 0.040823368
1 213 1.490912963 175.965829300 0.040823368 1.466451429 176.025364100 0.040772475
1 214 1.466451429 176.025364100 0.040772475 1.443145460 176.081605000 0.040725706
1 215 1.443145460 176.081605000 0.040725706 1.420996665 176.134759300 0.040682834
1 216 1.420996665 176.134759300 0.040682834 1.399999187 176.185020800 0.040643640
1 217 1.399999187 176.185020800 0.040643640 1.380140651 176.232570700 0.040607913
1 218 1.380140651 176.232570700 0.040607913 1.361403047 176.277578100 0.040575448
1 219 1.361403047 176.277578100 0.040575448 1.343763564 176.320200800 0.040546051
1 220 1.343763564 176.320200800 0.040546051 1.327195355 176.360586400 0.040519532
1 221 1.327195355 176.360586400 0.040519532 1.311668242 176.398872500 0.040495713
1 222 1.311668242 176.398872500 0.040495713 1.297149359 176.435187400 0.040474421
1 223 1.297149359 176.435187400 0.040474421 1.283603728 176.469651000 0.040455493
 224 1.283603728 176.469651000 0.040455493 1.270994782 176.502375100 0.040438773
1 225 1.270994782 176.502375100 0.040438773 1.259284830 176.533464000 0.040424111
1 226 1.259284830 176.533464000 0.040424111 1.248435461 176.563015300 0.040411366
1 227 1.248435461 176.563015300 0.040411366 1.238407910 176.591119700 0.040400405
1 228 1.238407910 176.591119700 0.040400405 1.229163362 176.617862100 0.040391101
1 229 1.229163362 176.617862100 0.040391101 1.220663228 176.643321900 0.040383334
1 230 1.220663228 176.643321900 0.040383334 1.212869374 176.667572900 0.040376990
 231 1.212869374 176.667572900 0.040376990 1.205744310 176.690684400 0.040371962
1 232 1.205744310 176.690684400 0.040371962 1.199251356 176.712721000 0.040368149
1 233 1.199251356 176.712721000 0.040368149 1.193354770 176.733743000 0.040365456
1 234 1.193354770 176.733743000 0.040365456 1.188019859 176.753807000 0.040363795
1 235 1.188019859 176.753807000 0.040363795 1.183213059 176.772965700 0.040363080
1 236 1.183213059 176.772965700 0.040363080 1.178901998 176.791268700 0.040363233
 237 1.178901998 176.791268700 0.040363233 1.175055543 176.808762200 0.040364179
  238 1.175055543 176.808762200 0.040364179 1.171643828 176.825489500 0.040365850
1 239 1.171643828 176.825489500 0.040365850 1.168638270 176.841491400 0.040368180
2 24 1.093625008 84.553793340 0.040723061 1.051272912 85.397316900 0.040859727
  25 1.051272912 85.397316900 0.040859727 1.041951175 86.290263180 0.041142161
  26 1.041951175 86.290263180 0.041142161 1.012592236 87.157141820 0.041349399
 27 1.012592236 87.157141820 0.041349399 0.970541909 87.996018400 0.041500428
  28 0.970541909 87.996018400 0.041500428 0.921129988 88.805511500 0.041610508
  29 0.921129988 88.805511500 0.041610508 0.868221392 89.584766890 0.041691761
  30\ 0.868221392\ 89.584766890\ 0.041691761\ 0.814544130\ 90.333417220\ 0.041753680
  31 0.814544130 90.333417220 0.041753680 0.761957977 91.051543600 0.041803562
  32 0.761957977 91.051543600 0.041803562 0.711660228 91.739635200 0.041846882
  33 0.711660228 91.739635200 0.041846882 0.664323379 92.398544290 0.041887626
  34 0.664323379 92.398544290 0.041887626 0.620285102 93.029453920 0.041928568
  35 0.620285102 93.029453920 0.041928568 0.579556310 93.633822780 0.041971514
  36 0.579556310 93.633822780 0.041971514 0.541980940 94.213357090 0.042017509
  37 0.541980940 94.213357090 0.042017509 0.511429832 94.796432390 0.042104522
  38 0.511429832 94.796432390 0.042104522 0.482799937 95.373919180 0.042199507
  39 0.482799937 95.373919180 0.042199507 0.455521041 95.946926770 0.042300333
  40 0.455521041 95.946926770 0.042300333 0.429150288 96.516449120 0.042405225
  41 0.429150288 96.516449120 0.042405225 0.403351725 97.083372110 0.042512706
  42 0.403351725 97.083372110 0.042512706 0.377878239 97.648480700 0.042621565
  43 0.377878239 97.648480700 0.042621565 0.352555862 98.212465790 0.042730809
  44 0.352555862 98.212465790 0.042730809 0.327270297 98.775930690 0.042839638
 45 0.327270297 98.775930690 0.042839638 0.301955463 99.339397350 0.042947412
  46 0.301955463 99.339397350 0.042947412 0.276583851 99.903312200 0.043053626
  47 0.276583851 99.903312200 0.043053626 0.251158446 100.468051600 0.043157889
 48 0.251158446 100.468051600 0.043157889 0.225705996 101.033927000 0.043259907
  49 0.225705996 101.033927000 0.043259907 0.200271450 101.601189800 0.043359463
 50 0.200271450 101.601189800 0.043359463 0.174913356 102.170035800 0.043456406
```

```
2 51 0.174913356 102.170035800 0.043456406 0.149700081 102.740609400 0.043550638
2 52 0.149700081 102.740609400 0.043550638 0.124706710 103.313007700 0.043642107
2 53 0.124706710 103.313007700 0.043642107 0.100012514 103.887283900 0.043730791
     54 0.100012514 103.887283900 0.043730791 0.075698881 104.463451100 0.043816701
    55 0.075698881 104.463451100 0.043816701 0.051847635 105.041485300 0.043899867
    56 0.051847635 105.041485300 0.043899867 0.028539670 105.621328700 0.043980337
    57 \ \ 0.028539670 \ \ 105.621328700 \ \ 0.043980337 \ \ 0.005853853 \ \ 106.202892100 \ \ 0.044058171
    58 0.005853853 106.202892100 0.044058171 -0.016133871 106.786058300 0.044133440
    59 -0.016133871 106.786058300 0.044133440 -0.037351181 107.370684100 0.044206218
    61 -0.057729947 107.956603100 0.044276588 -0.077206672 108.543627800 0.044344632
    62\; -0.077206672\; 108.543627800\; 0.044344632\; -0.095722830\; 109.131552100\; 0.044410436
    64 \ -0.113225128 \ 109.720153100 \ 0.044474084 \ -0.129665689 \ 110.309193400 \ 0.044535662
     65 -0.129665689 110.309193400 0.044535662 -0.145002179 110.898422800 0.044595254
    66 \;\; -0.145002179 \;\; 110.898422800 \;\; 0.044595254 \;\; -0.159197885 \;\; 111.487580600 \;\; 0.044652942 \;\; 0.04466294 \;\; 0.044664 \;\; 0.046664 \;\; 0.0466664 \;\; 0.046664 \;\; 0.0466664 \;\; 0.0
    67 -0.159197885 111.487580600 0.044652942 -0.172221748 112.076396700 0.044708809
    68 -0.172221748 112.076396700 0.044708809 -0.184048358 112.664594300 0.044762936
    69 \;\; -0.184048358 \;\; 112.664594300 \;\; 0.044762936 \;\; -0.194660215 \;\; 113.251890200 \;\; 0.04481540219 \;\; 0.0448119 \;\; 0
    70 -0.194660215 113.251890200 0.044815402 -0.204030559 113.838000600 0.044866288
    71 \;\; -0.204030559 \;\; 113.838000600 \;\; 0.044866288 \;\; -0.212174408 \;\; 114.422631700 \;\; 0.044915672 \;\; 0.04491672 \;
    72 -0.212174408 114.422631700 0.044915672 -0.219069129 115.005497800 0.044963636
    73 \;\; -0.219069129 \;\; 115.005497800 \;\; 0.044963636 \;\; -0.224722166 \;\; 115.586308900 \;\; 0.045010259
    74 \;\; -0.224722166 \;\; 115.586308900 \;\; 0.045010259 \;\; -0.229140412 \;\; 116.164778200 \;\; 0.045055624 \;\; 0.045010259 \;\; -0.045010259 \;\; -0.0450
     75 -0.229140412 116.164778200 0.045055624 -0.232335686 116.740622100 0.045099817
    76\;-0.232335686\;116.740622100\;0.045099817\;-0.234324563\;117.313562200\;0.045142924
    77 -0.234324563 117.313562200 0.045142924 -0.235128195 117.883325900 0.045185036
    79 -0.234772114 118.449648100 0.045226249 -0.233286033 119.012272200 0.045266662
2 80 -0.233286033 119.012272200 0.045266662 -0.230703633 119.570951300 0.045306383
2 81 -0.230703633 119.570951300 0.045306383 -0.227062344 120.125449500 0.045345524
    82 -0.227062344 120.125449500 0.045345524 -0.222403111 120.675542700 0.045384203
2 83 -0.222403111 120.675542700 0.045384203 -0.216770161 121.221020000 0.045422551
2 84 -0.216770161 121.221020000 0.045422551 -0.210210748 121.761684400 0.045460702
2 85 -0.210210748 121.761684400 0.045460702 -0.202774891 122.297354200 0.045498803
    86 -0.202774891 122.297354200 0.045498803 -0.194515104 122.827864000 0.045537012
2 87 -0.194515104 122.827864000 0.045537012 -0.185486099 123.353065200 0.045575495
   88 -0.185486099 123.353065200 0.045575495 -0.175744476 123.872827600 0.045614432
    89 -0.175744476 123.872827600 0.045614432 -0.165348396 124.387040000 0.045654016
    90 -0.165348396 124.387040000 0.045654016 -0.154357220 124.895611400 0.045694450
    91 -0.154357220 124.895611400 0.045694450 -0.142831123 125.398472000 0.045735953
    92 -0.142831123 125.398472000 0.045735953 -0.130830669 125.895574000 0.045778759
     93 -0.130830669 125.895574000 0.045778759 -0.118416354 126.386892900 0.045823114
    94 -0.118416354 126.386892900 0.045823114 -0.105648092 126.872428400 0.045869280
    95 -0.105648092 126.872428400 0.045869280 -0.092584657 127.352205600 0.045917535
    96 -0.092584657 127.352205600 0.045917535 -0.079283065 127.826275900 0.045968169
    97 -0.079283065 127.826275900 0.045968169 -0.065797888 128.294718700 0.046021490
   98 -0.065797888 128.294718700 0.046021490 -0.052180500 128.757642000 0.046077818
   99 -0.052180500 128.757642000 0.046077818 -0.038478250 129.215183900 0.046137487
    100 -0.038478250 129.215183900 0.046137487 -0.024733545 129.667514300 0.046200842
   101 -0.024733545 129.667514300 0.046200842 -0.010982868 130.114835400 0.046268240
   102 -0.010982868 130.114835400 0.046268240 0.002744306 130.557383900 0.046340046
    103 0.002744306 130.557383900 0.046340046 0.016426655 130.995432000 0.046416629
   104 0.016426655 130.995432000 0.046416629 0.030052231 131.429288700 0.046498361
2 105 0.030052231 131.429288700 0.046498361 0.043619747 131.859301500 0.046585611
    106 0.043619747 131.859301500 0.046585611 0.057139880 132.285857400 0.046678741
    107 0.057139880 132.285857400 0.046678741 0.070636605 132.709384500 0.046778099
2 108 0.070636605 132.709384500 0.046778099 0.084148480 133.130352700 0.046884010
2 109 0.084148480 133.130352700 0.046884010 0.097729873 133.549274900 0.046996769
   110 0.097729873 133.549274900 0.046996769 0.111452039 133.966707300 0.047116633
    111 0.111452039 133.966707300 0.047116633 0.125404005 134.383249900 0.047243801
2 112 0.125404005 134.383249900 0.047243801 0.139693160 134.799546300 0.047378413
   113 0.139693160 134.799546300 0.047378413 0.154445482 135.216282600 0.047520521
    114 0.154445482 135.216282600 0.047520521 0.169805275 135.634186000 0.047670085
2 115 0.169805275 135.634186000 0.047670085 0.185934346 136.054022300 0.047826946
2 116 0.185934346 136.054022300 0.047826946 0.203010488 136.476592500 0.047990810
   117 0.203010488 136.476592500 0.047990810 0.221225200 136.902728100 0.048161228
   118 0.221225200 136.902728100 0.048161228 0.240780542 137.333284600 0.048337570
   119 0.240780542 137.333284600 0.048337570 0.261885086 137.769133900 0.048519011
    120 0.261885086 137.769133900 0.048519011 0.284748919 138.211155200 0.048704503
   121 0.284748919 138.211155200 0.048704503 0.309577733 138.660222800 0.048892759
```

```
2 122 0.309577733 138.660222800 0.048892759 0.336566048 139.117193300 0.049082239
2 123 0.336566048 139.117193300 0.049082239 0.365889711 139.582889800 0.049271137
2 124 0.365889711 139.582889800 0.049271137 0.397699038 140.058084800 0.049457371
 125 0.397699038 140.058084800 0.049457371 0.432104409 140.543478700 0.049638596
2 126 0.432104409 140.543478700 0.049638596 0.469179930 141.039683200 0.049812203
2 127 0.469179930 141.039683200 0.049812203 0.508943272 141.547194500 0.049975355
 128 0.508943272 141.547194500 0.049975355 0.551354277 142.066373100 0.050125012
 129 0.551354277 142.066373100 0.050125012 0.596307363 142.597420000 0.050257992
2 130 0.596307363 142.597420000 0.050257992 0.643626542 143.140355300 0.050371024
 131 0.643626542 143.140355300 0.050371024 0.693062173 143.694998100 0.050460835
 132 0.693062173 143.694998100 0.050460835 0.744289752 144.260949700 0.050524236
 133 0.744289752 144.260949700 0.050524236 0.796910980 144.837580900 0.050558224
 134 0.796910980 144.837580900 0.050558224 0.850457280 145.424024600 0.050560083
 135 0.850457280 145.424024600 0.050560083 0.904395871 146.019174800 0.050527494
 136 0.904395871 146.019174800 0.050527494 0.958138449 146.621692000 0.050458634
2 137 0.958138449 146.621692000 0.050458634 1.011054559 147.230017700 0.050352269
2 138 1.011054559 147.230017700 0.050352269 1.062474568 147.842391800 0.050207825
 139 1.062474568 147.842391800 0.050207825 1.111727029 148.456887900 0.050025434
2 140 1.111727029 148.456887900 0.050025434 1.158135105 149.071441300 0.049805967
 141 1.158135105 149.071441300 0.049805967 1.201050821 149.683894300 0.049551023
 142 1.201050821 149.683894300 0.049551023 1.239852328 150.292032800 0.049262895
 143 1.239852328 150.292032800 0.049262895 1.274006058 150.893646900 0.048944504
2 144 1.274006058 150.893646900 0.048944504 1.303044695 151.486563600 0.048599314
2 145 1.303044695 151.486563600 0.048599314 1.326605954 152.068698500 0.048231224
 146 1.326605954 152.068698500 0.048231224 1.344443447 152.638095500 0.047844442
 147 1.344443447 152.638095500 0.047844442 1.356437773 153.192963100 0.047443362
 148 1.356437773 153.192963100 0.047443362 1.362602695 153.731703100 0.047032430
 149 1.362602695 153.731703100 0.047032430 1.363085725 154.252933200 0.046616026
 150 1.363085725 154.252933200 0.046616026 1.358162799 154.755501000 0.046198356
2 151 1.358162799 154.755501000 0.046198356 1.348227142 155.238490400 0.045783350
2 152 1.348227142 155.238490400 0.045783350 1.333772923 155.701221600 0.045374597
 153 1.333772923 155.701221600 0.045374597 1.315374704 156.143243800 0.044975281
 154 1.315374704 156.143243800 0.044975281 1.293664024 156.564323000 0.044588148
2 155 1.293664024 156.564323000 0.044588148 1.269304678 156.964425800 0.044215488
 156 1.269304678 156.964425800 0.044215488 1.242968236 157.343699500 0.043859135
 157 1.242968236 157.343699500 0.043859135 1.215311270 157.702450700 0.043520480
2 158 1.215311270 157.702450700 0.043520480 1.186955477 158.041123300 0.043200497
 159 1.186955477 158.041123300 0.043200497 1.158471522 158.360275600 0.042899776
 160 1.158471522 158.360275600 0.042899776 1.130367088 158.660558800 0.042618565
 161 1.130367088 158.660558800 0.042618565 1.103079209 158.942696400 0.042356812
2 162 1.103079209 158.942696400 0.042356812 1.076970655 159.207465400 0.042114211
 163 1.076970655 159.207465400 0.042114211 1.052329922 159.455679000 0.041890247
 164 1.052329922 159.455679000 0.041890247 1.029374161 159.688172000 0.041684240
2 165 1.029374161 159.688172000 0.041684240 1.008254396 159.905787100 0.041495379
2 166 1.008254396 159.905787100 0.041495379 0.989062282 160.109364700 0.041322765
 167 0.989062282 160.109364700 0.041322765 0.971837799 160.299733000 0.041165437
 168 0.971837799 160.299733000 0.041165437 0.956572150 160.477699600 0.041022401
 169 0.956572150 160.477699600 0.041022401 0.943242280 160.644052600 0.040892651
 170 0.943242280 160.644052600 0.040892651 0.931767062 160.799542800 0.040775193
 171 0.931767062 160.799542800 0.040775193 0.922058291 160.944891600 0.040669052
 172 0.922058291 160.944891600 0.040669052 0.914012643 161.080785700 0.040573288
 173 0.914012643 161.080785700 0.040573288 0.907516917 161.207875500 0.040487005
 174 0.907516917 161.207875500 0.040487005 0.902452436 161.326774400 0.040409354
 175 0.902452436 161.326774400 0.040409354 0.898698641 161.438059300 0.040339537
2 176 0.898698641 161.438059300 0.040339537 0.896143482 161.542272600 0.040276811
 177 0.896143482 161.542272600 0.040276811 0.894659668 161.639917000 0.040220488
 178 0.894659668 161.639917000 0.040220488 0.894138920 161.731464500 0.040169932
2 179 0.894138920 161.731464500 0.040169932 0.894475371 161.817353400 0.040124562
2 180 0.894475371 161.817353400 0.040124562 0.895569834 161.897991300 0.040083845
 181 0.895569834 161.897991300 0.040083845 0.897330209 161.973755800 0.040047295
 182 0.897330209 161.973755800 0.040047295 0.899671635 162.044996900 0.040014473
2 183 0.899671635 162.044996900 0.040014473 0.902516442 162.112038600 0.039984980
 184 0.902516442 162.112038600 0.039984980 0.905793969 162.175180000 0.039958458
 185 0.905793969 162.175180000 0.039958458 0.909440266 162.234697900 0.039934584
2 186 0.909440266 162.234697900 0.039934584 0.913397733 162.290847400 0.039913066
2 187 0.913397733 162.290847400 0.039913066 0.917614710 162.343864000 0.039893644
 188 0.917614710 162.343864000 0.039893644 0.922045055 162.393965200 0.039876087
 189 0.922045055 162.393965200 0.039876087 0.926647697 162.441351300 0.039860185
 190 0.926647697 162.441351300 0.039860185 0.931386217 162.486207100 0.039845754
 191 0.931386217 162.486207100 0.039845754 0.936228420 162.528702900 0.039832629
 192 0.936228420 162.528702900 0.039832629 0.941145943 162.568995800 0.039820663
```

```
2 193 0.941145943 162.568995800 0.039820663 0.946113880 162.607230900 0.039809725
2 194 0.946113880 162.607230900 0.039809725 0.951110430 162.643541800 0.039799700
2 195 0.951110430 162.643541800 0.039799700 0.956116576 162.678051900 0.039790485
 196 0.956116576 162.678051900 0.039790485 0.961115792 162.710875100 0.039781991
2 197 0.961115792 162.710875100 0.039781991 0.966093766 162.742116800 0.039774136
2 198 0.966093766 162.742116800 0.039774136 0.971038162 162.771874100 0.039766850
 199 0.971038162 162.771874100 0.039766850 0.975938391 162.800237100 0.039760070
 200 0.975938391 162.800237100 0.039760070 0.980785418 162.827288900 0.039753741
2 201 0.980785418 162.827288900 0.039753741 0.985571579 162.853106700 0.039747815
2 202 0.985571579 162.853106700 0.039747815 0.990290420 162.877761900 0.039742249
  203 0.990290420 162.877761900 0.039742249 0.994936555 162.901320800 0.039737004
2 204 0.994936555 162.901320800 0.039737004 0.999505539 162.923844900 0.039732048
2 205 0.999505539 162.923844900 0.039732048 1.003993753 162.945391200 0.039727352
 206 1.003993753 162.945391200 0.039727352 1.008398300 162.966013100 0.039722890
  207 1.008398300 162.966013100 0.039722890 1.012716921 162.985759900 0.039718640
 208 1.012716921 162.985759900 0.039718640 1.016947912 163.004677600 0.039714581
2 209 1.016947912 163.004677600 0.039714581 1.021090055 163.022809400 0.039710697
 210 1.021090055 163.022809400 0.039710697 1.025142554 163.040195300 0.039706971
2 211 1.025142554 163.040195300 0.039706971 1.029104983 163.056872700 0.039703391
2 212 1.029104983 163.056872700 0.039703391 1.032977233 163.072876800 0.039699945
 213 1.032977233 163.072876800 0.039699945 1.036759475 163.088240400 0.039696623
 214 1.036759475 163.088240400 0.039696623 1.040452117 163.102994300 0.039693415
2 215 1.040452117 163.102994300 0.039693415 1.044055774 163.117167300 0.039690313
2 216 1.044055774 163.117167300 0.039690313 1.047571238 163.130786600 0.039687311
 217 1.047571238 163.130786600 0.039687311 1.050999451 163.143877600 0.039684402
2 218 1.050999451 163.143877600 0.039684402 1.054341482 163.156464400 0.039681581
2 219 1.054341482 163.156464400 0.039681581 1.057598512 163.168569700 0.039678842
2 220 1.057598512 163.168569700 0.039678842 1.060771808 163.180214600 0.039676182
 221 1.060771808 163.180214600 0.039676182 1.063862715 163.191419400 0.039673596
2 222 1.063862715 163.191419400 0.039673596 1.066872639 163.202203000 0.039671082
2 223 1.066872639 163.202203000 0.039671082 1.069803036 163.212583500 0.039668635
 224 1.069803036 163.212583500 0.039668635 1.072655401 163.222577900 0.039666254
2 225 1.072655401 163.222577900 0.039666254 1.075431258 163.232202400 0.039663936
2 226 1.075431258 163.232202400 0.039663936 1.078132156 163.241472200 0.039661679
2 227 1.078132156 163.241472200 0.039661679 1.080759655 163.250401900 0.039659481
 228 1.080759655 163.250401900 0.039659481 1.083315329 163.259005200 0.039657339
2 229 1.083315329 163.259005200 0.039657339 1.085800751 163.267295400 0.039655252
 230 1.085800751 163.267295400 0.039655252 1.088217496 163.275284800 0.039653218
 231 1.088217496 163.275284800 0.039653218 1.090567133 163.282985400 0.039651237
2 232 1.090567133 163.282985400 0.039651237 1.092851222 163.290408600 0.039649306
2 233 1.092851222 163.290408600 0.039649306 1.095071313 163.297565000 0.039647424
 234 1.095071313 163.297565000 0.039647424 1.097228939 163.304465000 0.039645591
 235 1.097228939 163.304465000 0.039645591 1.099325619 163.311118500 0.039643804
2 236 1.099325619 163.311118500 0.039643804 1.101362852 163.317534900 0.039642063
2 237 1.101362852 163.317534900 0.039642063 1.103342119 163.323723100 0.039640367
 238 1.103342119 163.323723100 0.039640367 1.105264876 163.329691800 0.039638715
2 239 1.105264876 163.329691800 0.039638715 1.107132561 163.335449100 0.039637105
run;
**DATA FILE FOR WEIGHT-FOR-AGE;
data wtcrv;
     infile cards pad;
     input sex _age _LW1 _MW1 _SW1 _LW2 _MW2 _SW2;
cards;
1 24 -0.196701960 12.599134940 0.108095077 -0.216501213 12.741543960 0.108166006
1 25 -0.216501213 12.741543960 0.108166006 -0.239790488 12.881022760 0.108274706
1 26 -0.239790488 12.881022760 0.108274706 -0.266315853 13.018423820 0.108421025
1 27 -0.266315853 13.018423820 0.108421025 -0.295754969 13.154496600 0.108604770
1 28 -0.295754969 13.154496600 0.108604770 -0.327729368 13.289896670 0.108825681
1\ 29\ -0.327729368\ 13.289896670\ 0.108825681\ -0.361817468\ 13.425194080\ 0.109083424
 30 -0.361817468 13.425194080 0.109083424 -0.397568087 13.560881130 0.109377581
1 31 -0.397568087 13.560881130 0.109377581 -0.434520252 13.697378580 0.109707646
1 32 -0.434520252 13.697378580 0.109707646 -0.472188756 13.835046220 0.110073084
 33 -0.472188756 13.835046220 0.110073084 -0.510116627 13.974182990 0.110473254
1\ 34\ -0.510116627\ 13.974182990\ 0.110473254\ -0.547885579\ 14.115032400\ 0.110907400
1 35 -0.547885579 14.115032400 0.110907400 -0.585070110 14.257796180 0.111374787
1\ 36\ -0.585070110\ 14.257796180\ 0.111374787\ -0.621319726\ 14.402627490\ 0.111874514
1 37 -0.621319726 14.402627490 0.111874514 -0.656295986 14.549646140 0.112405687
1\ 38\ -0.656295986\ 14.549646140\ 0.112405687\ -0.689735029\ 14.698933260\ 0.112967254
1\ 39\ -0.689735029\ 14.698933260\ 0.112967254\ -0.721410388\ 14.850541510\ 0.113558110
1 40 -0.721410388 14.850541510 0.113558110 -0.751175223 15.004491430 0.114176956
```

```
1 41 -0.751175223 15.004491430 0.114176956 -0.778904279 15.160784540 0.114822482
1\ 42\ -0.778904279\ 15.160784540\ 0.114822482\ -0.804515498\ 15.319402460\ 0.115493292
1\ 43\ -0.804515498\ 15.319402460\ 0.115493292\ -0.828003255\ 15.480303130\ 0.116187777
1 44 -0.828003255 15.480303130 0.116187777 -0.849380372 15.643433090 0.116904306
1\ 45\ -0.849380372\ 15.643433090\ 0.116904306\ -0.868699650\ 15.808725350\ 0.117641148
1 46 -0.868699650 15.808725350 0.117641148 -0.886033992 15.976104560 0.118396541
1 47 -0.886033992 15.976104560 0.118396541 -0.901507878 16.145481940 0.119168555
1\ 48\ -0.901507878\ 16.145481940\ 0.119168555\ -0.915241589\ 16.316767270\ 0.119955320
1 49 -0.915241589 16.316767270 0.119955320 -0.927377772 16.489864600 0.120754916
1\ 50\ -0.927377772\ 16.489864600\ 0.120754916\ -0.938069819\ 16.664675290\ 0.121565421
1 51 -0.938069819 16.664675290 0.121565421 -0.947477940 16.841099480 0.122384927
1 52 -0.947477940 16.841099480 0.122384927 -0.955765694 17.019037460 0.123211562
1\ 53\ -0.955765694\ 17.019037460\ 0.123211562\ -0.963096972\ 17.198390800\ 0.124043503
1\ 54\ -0.963096972\ 17.198390800\ 0.124043503\ -0.969633434\ 17.379063410\ 0.124878992
  55 -0.969633434 17.379063410 0.124878992 -0.975532355 17.560962450 0.125716348
1\ 56\ -0.975532355\ 17.560962450\ 0.125716348\ -0.980937915\ 17.744000820\ 0.126554022
1 57 -0.980937915 17.744000820 0.126554022 -0.986006518 17.928091210 0.127390453
1\ 58\ -0.986006518\ 17.928091210\ 0.127390453\ -0.990866940\ 18.113156250\ 0.128224294
1 59 -0.990866940 18.113156250 0.128224294 -0.995644402 18.299122860 0.129054277
1 60 -0.995644402 18.299122860 0.129054277 -1.000453886 18.485924130 0.129879257
1 61 -1.000453886 18.485924130 0.129879257 -1.005399668 18.673499650 0.130698212
  62 \ -1.005399668 \ 18.673499650 \ 0.130698212 \ -1.010575003 \ 18.861795760 \ 0.131510245
1 63 -1.010575003 18.861795760 0.131510245 -1.016061941 19.050765790 0.132314586
1 64 -1.016061941 19.050765790 0.132314586 -1.021931241 19.240370190 0.133110593
  65 -1.021931241 19.240370190 0.133110593 -1.028242376 19.430576620 0.133897752
  66 -1.028242376 19.430576620 0.133897752 -1.035043608 19.621360070 0.134675673
1 67 -1.035043608 19.621360070 0.134675673 -1.042372125 19.812702800 0.135444090
  68 -1.042372125 19.812702800 0.135444090 -1.050254232 20.004594400 0.136202860
  69 -1.050254232 20.004594400 0.136202860 -1.058705595 20.197031710 0.136951959
1 70 -1.058705595 20.197031710 0.136951959 -1.067731529 20.390018720 0.137691478
1 71 -1.067731529 20.390018720 0.137691478 -1.077321193 20.583568620 0.138421673
  72 -1.077321193 20.583568620 0.138421673 -1.087471249 20.777695650 0.139142773
  73 -1.087471249 20.777695650 0.139142773 -1.098152984 20.972426310 0.139855242
 74 -1.098152984 20.972426310 0.139855242 -1.109334080 21.167791920 0.140559605
1 75 -1.109334080 21.167791920 0.140559605 -1.120974043 21.363830130 0.141256489
  76 -1.120974043 21.363830130 0.141256489 -1.133024799 21.560584670 0.141946613
1 77 -1.133024799 21.560584670 0.141946613 -1.145431351 21.758105060 0.142630785
1 78 -1.145431351 21.758105060 0.142630785 -1.158132499 21.956446270 0.143309898
1 79 -1.158132499 21.956446270 0.143309898 -1.171061612 22.155668420 0.143984924
1 80 -1.171061612 22.155668420 0.143984924 -1.184141975 22.355838620 0.144656953
1 81 -1.184141975 22.355838620 0.144656953 -1.197307185 22.557022680 0.145327009
1 82 -1.197307185 22.557022680 0.145327009 -1.210475099 22.759295580 0.145996289
1 83 -1.210475099 22.759295580 0.145996289 -1.223565263 22.962734400 0.146666000
1 84 -1.223565263 22.962734400 0.146666000 -1.236497304 23.167418880 0.147337375
1 85 -1.236497304 23.167418880 0.147337375 -1.249186293 23.373433410 0.148011715
1 86 -1.249186293 23.373433410 0.148011715 -1.261555446 23.580861450 0.148690256 1 87 -1.261555446 23.580861450 0.148690256 -1.273523619 23.789790960 0.149374297
1 88 -1.273523619 23.789790960 0.149374297 -1.285013783 24.000310640 0.150065107
1 89 -1.285013783 24.000310640 0.150065107 -1.295952066 24.212510280 0.150763933
  90 -1.295952066 24.212510280 0.150763933 -1.306268473 24.426480430 0.151471982
1 91 -1.306268473 24.426480430 0.151471982 -1.315897530 24.642312000 0.152190413
 92 -1.315897530 24.642312000 0.152190413 -1.324778843 24.860095960 0.152920322
1 93 -1.324778843 24.860095960 0.152920322 -1.332857581 25.079923030 0.153662731 1 94 -1.332857581 25.079923030 0.153662731 -1.340080195 25.301885840 0.154418635
1 95 -1.340080195 25.301885840 0.154418635 -1.346412105 25.526069770 0.155188768
 96 -1.346412105 25.526069770 0.155188768 -1.351813296 25.752565280 0.155973912
  97 -1.351813296 25.752565280 0.155973912 -1.356253969 25.981459900 0.156774684
1 98 -1.356253969 25.981459900 0.156774684 -1.359710858 26.212839900 0.157591579
1 99 -1.359710858 26.212839900 0.157591579 -1.362167159 26.446790270 0.158424964
1\ 100\ -1.362167159\ 26.446790270\ 0.158424964\ -1.363612378\ 26.683394570\ 0.159275071
 101 -1.363612378 26.683394570 0.159275071 -1.364042106 26.922734940 0.160141995
1 102 -1.364042106 26.922734940 0.160141995 -1.363457829 27.164891990 0.161025689
1 103 -1.363457829 27.164891990 0.161025689 -1.361865669 27.409945390 0.161925976
 104 -1.361865669 27.409945390 0.161925976 -1.359282610 27.657969780 0.162842452
1 105 -1.359282610 27.657969780 0.162842452 -1.355720571 27.909044330 0.163774719
1 106 -1.355720571 27.909044330 0.163774719 -1.351202536 28.163242640 0.164722138
1 107 -1.351202536 28.163242640 0.164722138 -1.345754408 28.420637440 0.165683945
1 108 -1.345754408 28.420637440 0.165683945 -1.339405453 28.681300050 0.166659247
1 109 -1.339405453 28.681300050 0.166659247 -1.332188093 28.945300290 0.167647017
1 110 -1.332188093 28.945300290 0.167647017 -1.324137479 29.212706450 0.168646104
1 111 -1.324137479 29.212706450 0.168646104 -1.315291073 29.483585270 0.169655235
```

```
1 112 -1.315291073 29.483585270 0.169655235 -1.305688240 29.758001980 0.170673022
1 113 -1.305688240 29.758001980 0.170673022 -1.295369867 30.036020210 0.171697970
1 114 -1.295369867 30.036020210 0.171697970 -1.284374967 30.317704170 0.172728540
1 115 -1.284374967 30.317704170 0.172728540 -1.272750864 30.603111070 0.173762961
1 116 -1.272750864 30.603111070 0.173762961 -1.260539193 30.892300720 0.174799493
1 117 -1.260539193 30.892300720 0.174799493 -1.247783611 31.185329840 0.175836284
1 118 -1.247783611 31.185329840 0.175836284 -1.234527763 31.482253150 0.176871417
1 119 -1.234527763 31.482253150 0.176871417 -1.220815047 31.783123290 0.177902912
1 120 -1.220815047 31.783123290 0.177902912 -1.206688407 32.087990620 0.178928740
1 121 -1.206688407 32.087990620 0.178928740 -1.192190150 32.396903130 0.179946830
1 122 -1.192190150 32.396903130 0.179946830 -1.177361786 32.709906200 0.180955078
1 123 -1.177361786 32.709906200 0.180955078 -1.162243894 33.027042440 0.181951361
1 124 -1.162243894 33.027042440 0.181951361 -1.146876007 33.348351480 0.182933537
1\ 125\ -1.146876007\ 33.348351480\ 0.182933537\ -1.131296524\ 33.673869730\ 0.183899465
 126 -1.131296524 33.673869730 0.183899465 -1.115542634 34.003630170 0.184847006
1 127 -1.115542634 34.003630170 0.184847006 -1.099650267 34.337662070 0.185774041
1 128 -1.099650267 34.337662070 0.185774041 -1.083654055 34.675990760 0.186678470
1 129 -1.083654055 34.675990760 0.186678470 -1.067587314 35.018637320 0.187558229
1 130 -1.067587314 35.018637320 0.187558229 -1.051482972 35.365617370 0.188411280
1 131 -1.051482972 35.365617370 0.188411280 -1.035367321 35.716947230 0.189235738
1 132 -1.035367321 35.716947230 0.189235738 -1.019277299 36.072625690 0.190029545
1 133 -1.019277299 36.072625690 0.190029545 -1.003235326 36.432659960 0.190790973
1 134 -1.003235326 36.432659960 0.190790973 -0.987269866 36.797043920 0.191518224
1\ 135\ -0.987269866\ 36.797043920\ 0.191518224\ -0.971406609\ 37.165767100\ 0.192209619
1 136 -0.971406609 37.165767100 0.192209619 -0.955670107 37.538812680 0.192863569
1 137 -0.955670107 37.538812680 0.192863569 -0.940083834 37.916157210 0.193478582
1\ 138\ -0.940083834\ 37.916157210\ 0.193478582\ -0.924670244\ 38.297770300\ 0.194053274
1 139 -0.924670244 38.297770300 0.194053274 -0.909450843 38.683614300 0.194586368
1 140 -0.909450843 38.683614300 0.194586368 -0.894446258 39.073644010 0.195076705
1 141 -0.894446258 39.073644010 0.195076705 -0.879676305 39.467806430 0.195523246
1 142 -0.879676305 39.467806430 0.195523246 -0.865160071 39.866040440 0.195925079
1 143 -0.865160071 39.866040440 0.195925079 -0.850915987 40.268276520 0.196281418
1\ 144\ -0.850915987\ 40.268276520\ 0.196281418\ -0.836961905\ 40.674436580\ 0.196591612
1 145 -0.836961905 40.674436580 0.196591612 -0.823315176 41.084433630 0.196855140
1 146 -0.823315176 41.084433630 0.196855140 -0.809992726 41.498171640 0.197071620
 147 -0.809992726 41.498171640 0.197071620 -0.797011132 41.915545280 0.197240806
1 148 -0.797011132 41.915545280 0.197240806 -0.784386693 42.336439780 0.197362591
1 149 -0.784386693 42.336439780 0.197362591 -0.772135506 42.760730780 0.197437004
1\ 150\ -0.772135506\ 42.760730780\ 0.197437004\ -0.760273528\ 43.188284190\ 0.197464210
1 151 -0.760273528 43.188284190 0.197464210 -0.748815968 43.618957030 0.197444522
1 152 -0.748815968 43.618957030 0.197444522 -0.737780398 44.052593100 0.197378345
1\ 153\ -0.737780398\ 44.052593100\ 0.197378345\ -0.727181568\ 44.489030270\ 0.197266263
 154 -0.727181568 44.489030270 0.197266263 -0.717035494 44.928094830 0.197108968
1\ 155\ -0.717035494\ 44.928094830\ 0.197108968\ -0.707358338\ 45.369603150\ 0.196907274
1\ 156\ -0.707358338\ 45.369603150\ 0.196907274\ -0.698166437\ 45.813361720\ 0.196662115
1 157 -0.698166437 45.813361720 0.196662115 -0.689476327 46.259167290 0.196374538
1\ 158\ -0.689476327\ 46.259167290\ 0.196374538\ -0.681304750\ 46.706807010\ 0.196045701
1 159 -0.681304750 46.706807010 0.196045701 -0.673668658 47.156058630 0.195676862
1 160 -0.673668658 47.156058630 0.195676862 -0.666585194 47.606690740 0.195269380
 161 -0.666585194 47.606690740 0.195269380 -0.660069969 48.058465720 0.194824730
1\ 162\ -0.660069969\ 48.058465720\ 0.194824730\ -0.654142602\ 48.511131380\ 0.194344410
1 163 -0.654142602 48.511131380 0.194344410 -0.648819666 48.964432240 0.193830046
1 164 -0.648819666 48.964432240 0.193830046 -0.644118611 49.418103740 0.193283319
1 165 -0.644118611 49.418103740 0.193283319 -0.640056805 49.871874090 0.192705974
1 166 -0.640056805 49.871874090 0.192705974 -0.636651424 50.325464780 0.192099812
1\ 167\ -0.636651424\ 50.325464780\ 0.192099812\ -0.633919328\ 50.778591210\ 0.191466681
 168 -0.633919328 50.778591210 0.191466681 -0.631876912 51.230963320 0.190808471
1 169 -0.631876912 51.230963320 0.190808471 -0.630539940 51.682286250 0.190127105
1 170 -0.630539940 51.682286250 0.190127105 -0.629923353 52.132261130 0.189424530
1 171 -0.629923353 52.132261130 0.189424530 -0.630041066 52.580585830 0.188702714
1\ 172\ -0.630041066\ 52.580585830\ 0.188702714\ -0.630905733\ 53.026955880\ 0.1879636368830
1 173 -0.630905733 53.026955880 0.187963636 -0.632528509 53.471065250 0.187209281
1 174 -0.632528509 53.471065250 0.187209281 -0.634918779 53.912607370 0.186441630
 175 -0.634918779 53.912607370 0.186441630 -0.638083884 54.351276080 0.185662657
1 176 -0.638083884 54.351276080 0.185662657 -0.642028835 54.786766590 0.184874323
1 177 -0.642028835 54.786766590 0.184874323 -0.646756013 55.218776570 0.184078567
1\ 178\ -0.646756013\ 55.218776570\ 0.184078567\ -0.652262297\ 55.647011310\ 0.183277339
1 179 -0.652262297 55.647011310 0.183277339 -0.658551638 56.071164070 0.182472427
1 180 -0.658551638 56.071164070 0.182472427 -0.665609025 56.490958620 0.181665781
1 181 -0.665609025 56.490958620 0.181665781 -0.673425951 56.906108860 0.180859180
1 182 -0.673425951 56.906108860 0.180859180 -0.681987284 57.316340590 0.180054395
```

```
1 183 -0.681987284 57.316340590 0.180054395 -0.691273614 57.721388460 0.179253153
1\ 184\ -0.691273614\ 57.721388460\ 0.179253153\ -0.701261055\ 58.120996960\ 0.178457127
1 185 -0.701261055 58.120996960 0.178457127 -0.711921092 58.514921430 0.177667942
1 186 -0.711921092 58.514921430 0.177667942 -0.723218488 58.902932080 0.176887192
1 187 -0.723218488 58.902932080 0.176887192 -0.735121189 59.284799480 0.176116307
1 188 -0.735121189 59.284799480 0.176116307 -0.747580416 59.660326260 0.175356814
1\ 189\ -0.747580416\ 59.660326260\ 0.175356814\ -0.760550666\ 60.029317040\ 0.174610071
1 190 -0.760550666 60.029317040 0.174610071 -0.773984558 60.391587210 0.173877336
1 191 -0.773984558 60.391587210 0.173877336 -0.787817728 60.746987850 0.173159953
1 192 -0.787817728 60.746987850 0.173159953 -0.801993069 61.095368470 0.172459052
1 193 -0.801993069 61.095368470 0.172459052 -0.816446409 61.436600770 0.171775726
1 194 -0.816446409 61.436600770 0.171775726 -0.831110299 61.770573720 0.171110986
1 195 -0.831110299 61.770573720 0.171110986 -0.845914498 62.097193990 0.170465756
1 196 -0.845914498 62.097193990 0.170465756 -0.860786514 62.416386280 0.169840869
  197 -0.860786514 62.416386280 0.169840869 -0.875652181 62.728093620 0.169237063
1 198 -0.875652181 62.728093620 0.169237063 -0.890436283 63.032277560 0.168654971
1 199 -0.890436283 63.032277560 0.168654971 -0.905063185 63.328918410 0.168095124
1 200 -0.905063185 63.328918410 0.168095124 -0.919457490 63.618015370 0.167557940
1 201 -0.919457490 63.618015370 0.167557940 -0.933544683 63.899586620 0.167043722
1 202 -0.933544683 63.899586620 0.167043722 -0.947251765 64.173669430 0.166552654
1 203 -0.947251765 64.173669430 0.166552654 -0.960507855 64.440320160 0.166084798
1 204 -0.960507855 64.440320160 0.166084798 -0.973244762 64.699614270 0.165640090
1 205 -0.973244762 64.699614270 0.165640090 -0.985397502 64.951646250 0.165218341
1 207 -0.996904762 65.196529500 0.164819236 -1.007705555 65.434401860 0.164442380
1 208 -1.007705555 65.434401860 0.164442380 -1.017756047 65.665400150 0.164087103
1 209 -1.017756047 65.665400150 0.164087103 -1.027002713 65.889701170 0.163752791
1 210 -1.027002713 65.889701170 0.163752791 -1.035402243 66.107491140 0.163438661
  211 -1.035402243 66.107491140 0.163438661 -1.042916356 66.318973110 0.163143825
1 212 -1.042916356 66.318973110 0.163143825 -1.049511871 66.524366180 0.162867311
1 213 -1.049511871 66.524366180 0.162867311 -1.055160732 66.723904430 0.162608072
1 214 -1.055160732 66.723904430 0.162608072 -1.059840019 66.917835630 0.162365006
1 215 -1.059840019 66.917835630 0.162365006 -1.063531973 67.106419560 0.162136973
1 216 -1.063531973 67.106419560 0.162136973 -1.066224038 67.289926030 0.161922819
1 217 -1.066224038 67.289926030 0.161922819 -1.067908908 67.468632550 0.161721398
1 218 -1.067908908 67.468632550 0.161721398 -1.068589885 67.642813780 0.161531530
1 219 -1.068589885 67.642813780 0.161531530 -1.068261146 67.812767500 0.161352313
1 220 -1.068261146 67.812767500 0.161352313 -1.066933756 67.978773310 0.161182785
1 221 -1.066933756 67.978773310 0.161182785 -1.064620976 68.141110220 0.161022184
1 222 -1.064620976 68.141110220 0.161022184 -1.061341755 68.300047410 0.160869943
1 223 -1.061341755 68.300047410 0.160869943 -1.057116957 68.455845400 0.160725793
1 224 -1.057116957 68.455845400 0.160725793 -1.051988979 68.608721740 0.160589574
  225 -1.051988979 68.608721740 0.160589574 -1.045990330 68.758892630 0.160461700
1 226 -1.045990330 68.758892630 0.160461700 -1.039168248 68.906530280 0.160342924
1 227 -1.039168248 68.906530280 0.160342924 -1.031579574 69.051764270 0.160234478
1 228 -1.031579574 69.051764270 0.160234478 -1.023291946 69.194672880 0.160138158
1 229 -1.023291946 69.194672880 0.160138158 -1.014385118 69.335273760 0.160056393
1 230 -1.014385118 69.335273760 0.160056393 -1.004952366 69.473513730 0.159992344
1 231 -1.004952366 69.473513730 0.159992344 -0.995101924 69.609257820 0.159949989
1 232 -0.995101924 69.609257820 0.159949989 -0.984958307 69.742277580 0.159934231
1\ 233\ -0.984958307\ 69.742277580\ 0.159934231\ -0.974663325\ 69.872238850\ 0.159951004
1 234 -0.974663325 69.872238850 0.159951004 -0.964376555 69.998688960 0.160007394
1 235 -0.964376555 69.998688960 0.160007394 -0.954274945 70.121043810 0.160111769
1 236 -0.954274945 70.121043810 0.160111769 -0.944551187 70.238574820 0.160273918
1 237 -0.944551187 70.238574820 0.160273918 -0.935410427 70.350396260 0.160505203
1\ 238\ -0.935410427\ 70.350396260\ 0.160505203\ -0.927059784\ 70.455461050\ 0.160818788
  239 -0.927059784 70.455461050 0.160818788 -0.919718461 70.552521270 0.161229617
2 24 -0.717882830 11.974537480 0.107078197 -0.752206570 12.134555230 0.107740345
  25 -0.752206570 12.134555230 0.107740345 -0.784233660 12.291024900 0.108477010
2\ 26\ -0.784233660\ 12.291024900\ 0.108477010\ -0.814095820\ 12.444692580\ 0.109280828
   27 -0.814095820 12.444692580 0.109280828 -0.841935504 12.596223350 0.110144488
  28 -0.841935504 12.596223350 0.110144488 -0.867889398 12.746209110 0.111060815
  29 -0.867889398 12.746209110 0.111060815 -0.892102647 12.895172180 0.112022759
   30 -0.892102647 12.895172180 0.112022759 -0.914718817 13.043571640 0.113023467
  31 \;\; -0.914718817 \;\; 13.043571640 \;\; 0.113023467 \;\; -0.935876584 \;\; 13.191808740 \;\; 0.114056328
  32 -0.935876584 13.191808740 0.114056328 -0.955723447 13.340229340 0.115114953
  33 \; -0.955723447 \; 13.340229340 \; 0.115114953 \; -0.974383363 \; 13.489133190 \; 0.116193327 \; 0.11619327 \; 0.11619327 \; 0.11619327 \; 0.11619327 \; 0.11619327 \; 0.1161927 \; 0.116197 \; 0.116197 \; 0.
  34 -0.974383363 13.489133190 0.116193327 -0.991980756 13.638774460 0.117285750
  35 -0.991980756 13.638774460 0.117285750 -1.008640742 13.789365470 0.118386848
  36 -1.008640742 13.789365470 0.118386848 -1.024471278 13.941083320 0.119491669
  37 -1.024471278 13.941083320 0.119491669 -1.039573604 14.094071750 0.120595658
```

```
2 38 -1.039573604 14.094071750 0.120595658 -1.054039479 14.248444980 0.121694676
2 39 -1.054039479 14.248444980 0.121694676 -1.067946784 14.404291690 0.122785030
2 40 -1.067946784 14.404291690 0.122785030 -1.081374153 14.561675290 0.123863400
   41 -1.081374153 14.561675290 0.123863400 -1.094381409 14.720640450 0.124926943
2 42 -1.094381409 14.720640450 0.124926943 -1.107021613 14.881213520 0.125973221
   43 -1.107021613 14.881213520 0.125973221 -1.119338692 15.043405530 0.127000212
   44 -1.119338692 15.043405530 0.127000212 -1.131367831 15.207214430 0.128006292
   45 -1.131367831 15.207214430 0.128006292 -1.143135936 15.372627290 0.128990225
   46 -1.143135936 15.372627290 0.128990225 -1.154662150 15.539622210 0.129951143
   47 -1.154662150 15.539622210 0.129951143 -1.165958392 15.708170170 0.130888527
   48 -1.165958392 15.708170170 0.130888527 -1.177029925 15.878236680 0.131802186
   49 -1.177029925 15.878236680 0.131802186 -1.187871001 16.049784520 0.132692269
   50 -1.187871001 16.049784520 0.132692269 -1.198484073 16.222770600 0.133559108
   51 \;\; -1.198484073 \;\; 16.222770600 \;\; 0.133559108 \;\; -1.208853947 \;\; 16.397153630 \;\; 0.134403386
   52 -1.208853947 16.397153630 0.134403386 -1.218965087 16.572891220 0.135225990
   53 -1.218965087 16.572891220 0.135225990 -1.228798212 16.749941870 0.136028014
   54 -1.228798212 16.749941870 0.136028014 -1.238330855 16.928265870 0.136810739
    55 -1.238330855 16.928265870 0.136810739 -1.247537914 17.107826150 0.137575606
   56 -1.247537914 17.107826150 0.137575606 -1.256392179 17.288588940 0.138324193
   57 -1.256392179 17.288588940 0.138324193 -1.264864846 17.470524440 0.139058192
   58 -1.264864846 17.470524440 0.139058192 -1.272926011 17.653607330 0.139779387
   59 -1.272926011 17.653607330 0.139779387 -1.280545140 17.837817220 0.140489635
   60 -1.280545140 17.837817220 0.140489635 -1.287691525 18.023139040 0.141190842
   61 \;\; -1.287691525 \;\; 18.023139040 \;\; 0.141190842 \;\; -1.294332076 \;\; 18.209564180 \;\; 0.141884974
    62 -1.294332076 18.209564180 0.141884974 -1.300441561 18.397087600 0.142573939
   63 -1.300441561 18.397087600 0.142573939 -1.305989011 18.585712430 0.143259709
   64 \ -1.305989011 \ 18.585712430 \ 0.143259709 \ -1.310946941 \ 18.775447280 \ 0.143944216
   65 \;\; -1.310946941 \;\; 18.775447280 \;\; 0.143944216 \;\; -1.315289534 \;\; 18.966307000 \;\; 0.144629359
    66 -1.315289534 18.966307000 0.144629359 -1.318992925 19.158312670 0.145316990
   67 -1.318992925 19.158312670 0.145316990 -1.322035315 19.351491630 0.146008903
   68 -1.322035315 19.351491630 0.146008903 -1.324398133 19.545877080 0.146706813
    69 -1.324398133 19.545877080 0.146706813 -1.326064539 19.741508540 0.147412363
    70 -1.326064539 19.741508540 0.147412363 -1.327020415 19.938431450 0.148127109
   71 \;\; -1.327020415 \;\; 19.938431450 \;\; 0.148127109 \;\; -1.327256387 \;\; 20.136696230 \;\; 0.148852482
   72 -1.327256387 20.136696230 0.148852482 -1.326763834 20.336359610 0.149589838
    73 -1.326763834 20.336359610 0.149589838 -1.325538668 20.537482980 0.150340400
   74 \;\; -1.325538668 \;\; 20.537482980 \;\; 0.150340400 \;\; -1.323579654 \;\; 20.740132770 \;\; 0.151105277 \;\; 0.15110527 \;\; 
   75 \;\; -1.323579654 \;\; 20.740132770 \;\; 0.151105277 \;\; -1.320888012 \;\; 20.944380280 \;\; 0.151885464
   76 \;\; -1.320888012 \;\; 20.944380280 \;\; 0.151885464 \;\; -1.317468695 \;\; 21.150300930 \;\; 0.1526818199 \;\; -1.320888012 \;\; -1.3208888012 \;\; -1.320888012 \;\; -1.3208888012 \;\; -1.320888012 \;\; -1.320888012 \;\; -1.320888012 \;\; -1.320888012 \;\; -1.320888012 \;\; -1.32
    77 -1.317468695 21.150300930 0.152681819 -1.313331446 21.357973320 0.153495050
   78 -1.313331446 21.357973320 0.153495050 -1.308487081 21.567480450 0.154325756
   79 -1.308487081 21.567480450 0.154325756 -1.302948173 21.778909020 0.155174414
    80 -1.302948173 21.778909020 0.155174414 -1.296733913 21.992346860 0.156041320
   81 -1.296733913 21.992346860 0.156041320 -1.289863329 22.207885410 0.156926667
   82 -1.289863329 22.207885410 0.156926667 -1.282358762 22.425617700 0.157830504
   83 -1.282358762 22.425617700 0.157830504 -1.274244931 22.645638240 0.158752743
   84 -1.274244931 22.645638240 0.158752743 -1.265548787 22.868042580 0.159693163
   85 -1.265548787 22.868042580 0.159693163 -1.256299378 23.092926790 0.160651410
   86 -1.256299378 23.092926790 0.160651410 -1.246530660 23.320385490 0.161626956
    87 -1.246530660 23.320385490 0.161626956 -1.236266832 23.550518710 0.162619308
2 88 -1.236266832 23.550518710 0.162619308 -1.225551344 23.783416520 0.163627600
   89 -1.225551344 23.783416520 0.163627600 -1.214410914 24.019177030 0.164651100
   90 -1.214410914 24.019177030 0.164651100 -1.202884389 24.257890740 0.165688808
   91 -1.202884389 24.257890740 0.165688808 -1.191007906 24.499647780 0.166739662
   92 -1.191007906 24.499647780 0.166739662 -1.178818621 24.744535360 0.167802495
   93 -1.178818621 24.744535360 0.167802495 -1.166354376 24.992637350 0.168876037
    94 -1.166354376 24.992637350 0.168876037 -1.153653688 25.244033710 0.169958922
   95 -1.153653688 25.244033710 0.169958922 -1.140751404 25.498802640 0.171049756
   96 -1.140751404 25.498802640 0.171049756 -1.127684095 25.757016800 0.172147043
   97 -1.127684095 25.757016800 0.172147043 -1.114490244 26.018742610 0.173249185
   98 -1.114490244 26.018742610 0.173249185 -1.101204848 26.284043120 0.174354569
   99 -1.101204848 26.284043120 0.174354569 -1.087863413 26.552975070 0.175461512
   100 -1.087863413 26.552975070 0.175461512 -1.074500927 26.825589040 0.176568284
   101 -1.074500927 26.825589040 0.176568284 -1.061151213 27.101929500 0.177673124
2 102 -1.061151213 27.101929500 0.177673124 -1.047847141 27.382034220 0.178774242
2 103 -1.047847141 27.382034220 0.178774242 -1.034620551 27.665934020 0.179869829
   104 -1.034620551 27.665934020 0.179869829 -1.021502197 27.953652400 0.180958063
   105 -1.021502197 27.953652400 0.180958063 -1.008521695 28.245205310 0.182037118
  106 -1.008521695 28.245205310 0.182037118 -0.995707494 28.540600850 0.183105172
   107 -0.995707494 28.540600850 0.183105172 -0.983086844 28.839839070 0.184160410
   108 -0.983086844 28.839839070 0.184160410 -0.970685789 29.142911710 0.185201039
```
```
2 109 -0.970685789 29.142911710 0.185201039 -0.958529157 29.449802080 0.186225287
2 110 -0.958529157 29.449802080 0.186225287 -0.946640568 29.760484790 0.187231416
2 111 -0.946640568 29.760484790 0.187231416 -0.935042447 30.074925700 0.188217723
 112 -0.935042447 30.074925700 0.188217723 -0.923756041 30.393081760 0.189182550
2 113 -0.923756041 30.393081760 0.189182550 -0.912801445 30.714900930 0.190124286
2 114 -0.912801445 30.714900930 0.190124286 -0.902197638 31.040322100 0.191041375
 115 -0.902197638 31.040322100 0.191041375 -0.891962513 31.369275060 0.191932319
 116 -0.891962513 31.369275060 0.191932319 -0.882112919 31.701680500 0.192795682
2 117 -0.882112919 31.701680500 0.192795682 -0.872664706 32.037449990 0.193630095
2 118 -0.872664706 32.037449990 0.193630095 -0.863632768 32.376486070 0.194434260
 119 -0.863632768 32.376486070 0.194434260 -0.855031092 32.718682250 0.195206948
2 120 -0.855031092 32.718682250 0.195206948 -0.846872805 33.063923180 0.195947008
2 121 -0.846872805 33.063923180 0.195947008 -0.839170224 33.412084700 0.196653365
 122 -0.839170224 33.412084700 0.196653365 -0.831934903 33.763034020 0.197325023
 123 -0.831934903 33.763034020 0.197325023 -0.825177688 34.116629900 0.197961065
2 124 -0.825177688 34.116629900 0.197961065 -0.818908758 34.472722830 0.198560655
2 125 -0.818908758 34.472722830 0.198560655 -0.813137675 34.831155240 0.199123037
 126 -0.813137675 34.831155240 0.199123037 -0.807873433 35.191761770 0.199647538
2 127 -0.807873433 35.191761770 0.199647538 -0.803122613 35.554371760 0.200133598
 128 -0.803122613 35.554371760 0.200133598 -0.798897710 35.918799760 0.200580618
 129 -0.798897710 35.918799760 0.200580618 -0.795203499 36.284861940 0.200988216
 130 -0.795203499 36.284861940 0.200988216 -0.792047959 36.652363650 0.201356017
2 131 -0.792047959 36.652363650 0.201356017 -0.789435274 37.021108180 0.201683791
2 132 -0.789435274 37.021108180 0.201683791 -0.787374433 37.390886680 0.201971282
 133 -0.787374433 37.390886680 0.201971282 -0.785870695 37.761489050 0.202218375
 134 -0.785870695 37.761489050 0.202218375 -0.784929893 38.132699100 0.202425006
2 135 -0.784929893 38.132699100 0.202425006 -0.784557605 38.504296030 0.202591183
 136 -0.784557605 38.504296030 0.202591183 -0.784759170 38.876054890 0.202716980
 137 -0.784759170 38.876054890 0.202716980 -0.785539703 39.247747070 0.202802535
2 138 -0.785539703 39.247747070 0.202802535 -0.786904102 39.619140760 0.202848049
2 139 -0.786904102 39.619140760 0.202848049 -0.788858208 39.989999940 0.202853758
 140 -0.788858208 39.989999940 0.202853758 -0.791403051 40.360092440 0.202820053
2\ 141\ -0.791403051\ 40.360092440\ 0.202820053\ -0.794546352\ 40.729175440\ 0.202747236
2 142 -0.794546352 40.729175440 0.202747236 -0.798291020 41.097010990 0.202635758
 143 -0.798291020 41.097010990 0.202635758 -0.802640891 41.463359070 0.202486098
  144 -0.802640891 41.463359070 0.202486098 -0.807599577 41.827979630 0.202298783
2 145 -0.807599577 41.827979630 0.202298783 -0.813170461 42.190633130 0.202074385
2 146 -0.813170461 42.190633130 0.202074385 -0.819356692 42.551081070 0.201813521
 147 -0.819356692 42.551081070 0.201813521 -0.826161176 42.909086530 0.201516851
 148 -0.826161176 42.909086530 0.201516851 -0.833586038 43.264415500 0.201185082
2 149 -0.833586038 43.264415500 0.201185082 -0.841634949 43.616834020 0.200818928
 150 -0.841634949 43.616834020 0.200818928 -0.850307441 43.966116900 0.200419208
 151 -0.850307441 43.966116900 0.200419208 -0.859607525 44.312035790 0.199986681
2 152 -0.859607525 44.312035790 0.199986681 -0.869534339 44.654373190 0.199522233
2 153 -0.869534339 44.654373190 0.199522233 -0.880088651 44.992913560 0.199026736
 154 -0.880088651 44.992913560 0.199026736 -0.891270585 45.327447040 0.198501096
2\ 155\ -0.891270585\ 45.327447040\ 0.198501096\ -0.903079458\ 45.657770130\ 0.197946255
2 156 -0.903079458 45.657770130 0.197946255 -0.915513542 45.983686560 0.197363191
 157 -0.915513542 45.983686560 0.197363191 -0.928569454 46.305008580 0.196752931
  158 -0.928569454 46.305008580 0.196752931 -0.942245864 46.621551830 0.196116472
2 159 -0.942245864 46.621551830 0.196116472 -0.956537923 46.933144040 0.195454890
2 160 -0.956537923 46.933144040 0.195454890 -0.971440492 47.239620580 0.194769279
 161 -0.971440492 47.239620580 0.194769279 -0.986947308 47.540826040 0.194060758
 162 -0.986947308 47.540826040 0.194060758 -1.003050887 47.836614660 0.193330477
2 163 -1.003050887 47.836614660 0.193330477 -1.019742425 48.126850820 0.192579614
 164 -1.019742425 48.126850820 0.192579614 -1.037011698 48.411409380 0.191809374
  165 -1.037011698 48.411409380 0.191809374 -1.054846957 48.690176130 0.191020995
2 166 -1.054846957 48.690176130 0.191020995 -1.073234825 48.963048100 0.190215739
2 167 -1.073234825 48.963048100 0.190215739 -1.092160195 49.229933910 0.189394901
2 168 -1.092160195 49.229933910 0.189394901 -1.111606122 49.490754090 0.188559804
 169 -1.111606122 49.490754090 0.188559804 -1.131553723 49.745441320 0.187711798
2 170 -1.131553723 49.745441320 0.187711798 -1.151982079 49.993940680 0.186852266
 171 -1.151982079 49.993940680 0.186852266 -1.172868141 50.236209850 0.185982617
  172 -1.172868141 50.236209850 0.185982617 -1.194184620 50.472222130 0.185104331
2 173 -1.194184620 50.472222130 0.185104331 -1.215907492 50.701955810 0.184218803
2 174 -1.215907492 50.701955810 0.184218803 -1.238005268 50.925409420 0.183327556
 175 -1.238005268 50.925409420 0.183327556 -1.260445591 51.142592290 0.182432113
 176 -1.260445591 51.142592290 0.182432113 -1.283193626 51.353526800 0.181534018
2 177 -1.283193626 51.353526800 0.181534018 -1.306212032 51.558248310 0.180634839
 178 -1.306212032 51.558248310 0.180634839 -1.329460945 51.756805130 0.179736168
 179 -1.329460945 51.756805130 0.179736168 -1.352897980 51.949258410 0.178839614
```

```
2 180 -1.352897980 51.949258410 0.178839614 -1.376478254 52.135681930 0.177946804
2 181 -1.376478254 52.135681930 0.177946804 -1.400154426 52.316161970 0.177059379
2 182 -1.400154426 52.316161970 0.177059379 -1.423876772 52.490797030 0.176178990
 183 -1.423876772 52.490797030 0.176178990 -1.447593267 52.659697570 0.175307296
2 184 -1.447593267 52.659697570 0.175307296 -1.471249702 52.822985720 0.174445958
2 185 -1.471249702 52.822985720 0.174445958 -1.494789826 52.980794900 0.173596636
 186 -1.494789826 52.980794900 0.173596636 -1.518155513 53.133269460 0.172760982
 187 -1.518155513 53.133269460 0.172760982 -1.541286949 53.280564250 0.171940640
2 188 -1.541286949 53.280564250 0.171940640 -1.564122852 53.422844170 0.171137232
2 189 -1.564122852 53.422844170 0.171137232 -1.586600712 53.560283700 0.170352363
 190 -1.586600712 53.560283700 0.170352363 -1.608657054 53.693066370 0.169587605
2 191 -1.608657054 53.693066370 0.169587605 -1.630227728 53.821384220 0.168844497
2 192 -1.630227728 53.821384220 0.168844497 -1.651248208 53.945437250 0.168124538
2 193 -1.651248208 53.945437250 0.168124538 -1.671653920 54.065432780 0.167429179
 194 -1.671653920 54.065432780 0.167429179 -1.691380583 54.181584860 0.166759816
2 195 -1.691380583 54.181584860 0.166759816 -1.710364557 54.294113560 0.166117788
2 196 -1.710364557 54.294113560 0.166117788 -1.728543207 54.403244310 0.165504365
 197 -1.728543207 54.403244310 0.165504365 -1.745855274 54.509207170 0.164920747
2\ 198\ -1.745855274\ 54.509207170\ 0.164920747\ -1.762241248\ 54.612236030\ 0.164368054
 199 -1.762241248 54.612236030 0.164368054 -1.777643747 54.712567870 0.163847320
2 200 -1.777643747 54.712567870 0.163847320 -1.792007891 54.810441840 0.163359491
 201 -1.792007891 54.810441840 0.163359491 -1.805281675 54.906098420 0.162905415
2 202 -1.805281675 54.906098420 0.162905415 -1.817416335 54.999778460 0.162485839
2 203 -1.817416335 54.999778460 0.162485839 -1.828366707 55.091722170 0.162101402
 204 -1.828366707 55.091722170 0.162101402 -1.838091576 55.182168110 0.161752634
 205 -1.838091576 55.182168110 0.161752634 -1.846554015 55.271352000 0.161439944
2 206 -1.846554015 55.271352000 0.161439944 -1.853721704 55.359505580 0.161163623
 207 -1.853721704 55.359505580 0.161163623 -1.859567242 55.446855310 0.160923833
 208 -1.859567242 55.446855310 0.160923833 -1.864068443 55.533621070 0.160720609
2 209 -1.864068443 55.533621070 0.160720609 -1.867208610 55.620014640 0.160553850
2 210 -1.867208610 55.620014640 0.160553850 -1.868976800 55.706238260 0.160423319
 211 -1.868976800 55.706238260 0.160423319 -1.869371157 55.792479390 0.160328578
2 212 -1.869371157 55.792479390 0.160328578 -1.868386498 55.878923560 0.160269232
2 213 -1.868386498 55.878923560 0.160269232 -1.866033924 55.965730220 0.160244549
2 214 -1.866033924 55.965730220 0.160244549 -1.862327775 56.053046010 0.160253714
 215 -1.862327775 56.053046010 0.160253714 -1.857289195 56.140998820 0.160295765
2 216 -1.857289195 56.140998820 0.160295765 -1.850946286 56.229695640 0.160369590
 217 -1.850946286 56.229695640 0.160369590 -1.843334250 56.319220300 0.160473930
2 218 -1.843334250 56.319220300 0.160473930 -1.834495505 56.409631050 0.160607377
2 219 -1.834495505 56.409631050 0.160607377 -1.824479785 56.500958110 0.160768380
2 220 -1.824479785 56.500958110 0.160768380 -1.813344222 56.593201070 0.160955249
2 221 -1.813344222 56.593201070 0.160955249 -1.801153404 56.686326190 0.161166157
 222 -1.801153404 56.686326190 0.161166157 -1.787979408 56.780263640 0.161399151
2 223 -1.787979408 56.780263640 0.161399151 -1.773901816 56.874904650 0.161652158
2 224 -1.773901816 56.874904650 0.161652158 -1.759007704 56.970098560 0.161922998
 225 -1.759007704 56.970098560 0.161922998 -1.743391606 57.065649890 0.162209399
2 226 -1.743391606 57.065649890 0.162209399 -1.727155460 57.161315280 0.162509006
2 227 -1.727155460 57.161315280 0.162509006 -1.710410733 57.256798210 0.162819353
2 228 -1.710410733 57.256798210 0.162819353 -1.693267093 57.351757920 0.163138124
 229 -1.693267093 57.351757920 0.163138124 -1.675854420 57.445781720 0.163462715
2 230 -1.675854420 57.445781720 0.163462715 -1.658302847 57.538404290 0.163790683
 231 -1.658302847 57.538404290 0.163790683 -1.640747464 57.629100940 0.164119574
2 232 -1.640747464 57.629100940 0.164119574 -1.623332891 57.717275800 0.164446997
2 233 -1.623332891 57.717275800 0.164446997 -1.606209374 57.802265530 0.164770638
2 234 -1.606209374 57.802265530 0.164770638 -1.589533346 57.883335020 0.165088289
 235 -1.589533346 57.883335020 0.165088289 -1.573467222 57.959674580 0.165397881
 236 -1.573467222 57.959674580 0.165397881 -1.558179166 58.030397300 0.165697507
2 237 -1.558179166 58.030397300 0.165697507 -1.543846192 58.094532090 0.165985386
2 238 -1.543846192 58.094532090 0.165985386 -1.530642461 58.151035750 0.166260109
2 239 -1.530642461 58.151035750 0.166260109 -1.518754013 58.198771400 0.166520370
run:
**DATA FILE FOR BMI-FOR-AGE;
data bmicrv;
     infile cards pad;
     input sex _age _LB1 _MB1 _SB1 _LB2 _MB2 _SB2;
1 24 -2.039988545 16.602280490 0.081057501 -1.982373595 16.547774870 0.080127429
1 25 -1.982373595 16.547774870 0.080127429 -1.924100169 16.494427630 0.079233994
```

```
1 26 -1.924100169 16.494427630 0.079233994 -1.865497930 16.442595520 0.078389356
1 27 -1.865497930 16.442595520 0.078389356 -1.807261899 16.392243400 0.077593501
1 28 -1.807261899 16.392243400 0.077593501 -1.750118905 16.343336540 0.076846462
1 29 -1.750118905 16.343336540 0.076846462 -1.694815840 16.295840970 0.076148308
1 30 -1.694815840 16.295840970 0.076148308 -1.642106779 16.249723710 0.075499126
1 31 -1.642106779 16.249723710 0.075499126 -1.592744414 16.204952680 0.074898994
 33 -1.547442391 16.161498710 0.074347997 -1.506902601 16.119332580 0.073846139
1 34 -1.506902601 16.119332580 0.073846139 -1.471770047 16.078427580 0.073393370
1\ 35\ -1.471770047\ 16.078427580\ 0.073393370\ -1.442628957\ 16.038758960\ 0.072989551
  36 -1.442628957 16.038758960 0.072989551 -1.419991255 16.000304010 0.072634432
 37 -1.419991255 16.000304010 0.072634432 -1.404277619 15.963042770 0.072327649
1\ 38\ -1.404277619\ 15.963042770\ 0.072327649\ -1.395863170\ 15.926954180\ 0.072068640
 39 -1.395863170 15.926954180 0.072068640 -1.394935252 15.892025820 0.071856805
  40 -1.394935252 15.892025820 0.071856805 -1.401671596 15.858240930 0.071691278
1 41 -1.401671596 15.858240930 0.071691278 -1.416100312 15.825588220 0.071571093
1 42 -1.416100312 15.825588220 0.071571093 -1.438164899 15.794057280 0.071495113
1\ 43\ -1.438164899\ 15.794057280\ 0.071495113\ -1.467669032\ 15.763642550\ 0.071462106
1\ 44\ -1.467669032\ 15.763642550\ 0.071462106\ -1.504376347\ 15.734336680\ 0.071470646
1\ 45\ -1.504376347\ 15.734336680\ 0.071470646\ -1.547942838\ 15.706135660\ 0.071519218
1 46 -1.547942838 15.706135660 0.071519218 -1.597896397 15.679040620 0.071606277
1 47 -1.597896397 15.679040620 0.071606277 -1.653732283 15.653051920 0.071730167
1 48 -1.653732283 15.653051920 0.071730167 -1.714869347 15.628172690 0.071889214
1 49 -1.714869347 15.628172690 0.071889214 -1.780673181 15.604408000 0.072081737
1 50 -1.780673181 15.604408000 0.072081737 -1.850468473 15.581764580 0.072306081
1 51 -1.850468473 15.581764580 0.072306081 -1.923551865 15.560250670 0.072560637
1 52 -1.923551865 15.560250670 0.072560637 -1.999220429 15.539874600 0.072843840
1\ 53\ -1.999220429\ 15.539874600\ 0.072843840\ -2.076707178\ 15.520649930\ 0.073154324
  54 -2.076707178 15.520649930 0.073154324 -2.155348017 15.502584270 0.073490667
1 55 -2.155348017 15.502584270 0.073490667 -2.234438552 15.485689730 0.073851672
1 56 -2.234438552 15.485689730 0.073851672 -2.313321723 15.469977180 0.074236235
 57 -2.313321723 15.469977180 0.074236235 -2.391381273 15.455456920 0.074643374
1 58 -2.391381273 15.455456920 0.074643374 -2.468032491 15.442139610 0.075072264
1 59 -2.468032491 15.442139610 0.075072264 -2.542781541 15.430032070 0.075522104
1 \ 60 \ -2.542781541 \ 15.430032070 \ 0.075522104 \ -2.615165950 \ 15.419141630 \ 0.075992250
  61\;\; -2.615165950\;\; 15.419141630\;\; 0.075992250\;\; -2.684789516\;\; 15.409473560\;\; 0.076482128
1\ 62\ -2.684789516\ 15.409473560\ 0.076482128\ -2.751316949\ 15.401031390\ 0.076991232
1\ 63\ -2.751316949\ 15.401031390\ 0.076991232\ -2.814459450\ 15.393817850\ 0.077519149
1\ 64\ -2.814459450\ 15.393817850\ 0.077519149\ -2.874024760\ 15.387830940\ 0.078065390
1\ 65\ -2.874024760\ 15.387830940\ 0.078065390\ -2.929840480\ 15.383069450\ 0.078629592
1 66 -2.929840480 15.383069450 0.078629592 -2.981796828 15.379529580 0.079211369
1\ 67\ -2.981796828\ 15.379529580\ 0.079211369\ -3.029831343\ 15.377205820\ 0.079810334
  68 -3.029831343 15.377205820 0.079810334 -3.073924224 15.376091070 0.080426086
1 69 -3.073924224 15.376091070 0.080426086 -3.114093476 15.376176770 0.081058206
1\ 70\ -3.114093476\ 15.376176770\ 0.081058206\ -3.150390040\ 15.377453040\ 0.081706249
  71 -3.150390040 15.377453040 0.081706249 -3.182893018 15.379908860 0.082369741
  72 \;\; -3.182893018 \;\; 15.379908860 \;\; 0.082369741 \;\; -3.211705110 \;\; 15.383532170 \;\; 0.083048178
 73 -3.211705110 15.383532170 0.083048178 -3.236948340 15.388310050 0.083741021
 74 -3.236948340 15.388310050 0.083741021 -3.258760110 15.394228830 0.084447700
  1 76 -3.277281546 15.401274960 0.085167651 -3.292683774 15.409432520 0.085900184
 77 -3.292683774 15.409432520 0.085900184 -3.305124073 15.418686910 0.086644667
1 78 -3.305124073 15.418686910 0.086644667 -3.314768951 15.429022730 0.087400421
1 79 -3.314768951 15.429022730 0.087400421 -3.321785992 15.440424390 0.088166744
1 80 -3.321785992 15.440424390 0.088166744 -3.326345795 15.452875810 0.088942897
1\ 81\ -3.326345795\ 15.452875810\ 0.088942897\ -3.328602731\ 15.466362180\ 0.089728202
 82 -3.328602731 15.466362180 0.089728202 -3.328725277 15.480867040 0.090521875
1 83 -3.328725277 15.480867040 0.090521875 -3.326870180 15.496374650 0.091323162
1 84 -3.326870180 15.496374650 0.091323162 -3.323188896 15.512869360 0.092131305
1\ 85\ -3.323188896\ 15.512869360\ 0.092131305\ -3.317827016\ 15.530335630\ 0.092945544
 86 -3.317827016 15.530335630 0.092945544 -3.310923871 15.548758070 0.093765118
1 87 -3.310923871 15.548758070 0.093765118 -3.302612272 15.568121430 0.094589270
1 88 -3.302612272 15.568121430 0.094589270 -3.293018361 15.588410650 0.095417247
  89 -3.293018361 15.588410650 0.095417247 -3.282260813 15.609611010 0.096248301
1 90 -3.282260813 15.609611010 0.096248301 -3.270454609 15.631707350 0.097081694
1 91 -3.270454609 15.631707350 0.097081694 -3.257703616 15.654685630 0.097916698
1 92 -3.257703616 15.654685630 0.097916698 -3.244108214 15.678531390 0.098752593
1 93 -3.244108214 15.678531390 0.098752593 -3.229761713 15.703230520 0.099588675
1 94 -3.229761713 15.703230520 0.099588675 -3.214751287 15.728769110 0.100424251
1\ 95\ -3.214751287\ 15.728769110\ 0.100424251\ -3.199158184\ 15.755133470\ 0.101258643
1 96 -3.199158184 15.755133470 0.101258643 -3.183057950 15.782310070 0.102091189
```

```
1 97 -3.183057950 15.782310070 0.102091189 -3.166520664 15.810285600 0.102921245
1 98 -3.166520664 15.810285600 0.102921245 -3.149610300 15.839047080 0.103748189
1 99 -3.149610300 15.839047080 0.103748189 -3.132389637 15.868581230 0.104571386
1 100 -3.132389637 15.868581230 0.104571386 -3.114911153 15.898875620 0.105390269
1 101 -3.114911153 15.898875620 0.105390269 -3.097226399 15.929917650 0.106204258
1 102 -3.097226399 15.929917650 0.106204258 -3.079383079 15.961694810 0.107012788
 103 -3.079383079 15.961694810 0.107012788 -3.061423765 15.994194890 0.107815327
1 104 -3.061423765 15.994194890 0.107815327 -3.043386071 16.027406070 0.108611374
1 105 -3.043386071 16.027406070 0.108611374 -3.025310003 16.061315900 0.109400388
1 106 -3.025310003 16.061315900 0.109400388 -3.007225737 16.095912920 0.110181915
 107 -3.007225737 16.095912920 0.110181915 -2.989164598 16.131185320 0.110955478
1 108 -2.989164598 16.131185320 0.110955478 -2.971148225 16.167122340 0.111720691
1 109 -2.971148225 16.167122340 0.111720691 -2.953208047 16.203711680 0.112477059
1 110 -2.953208047 16.203711680 0.112477059 -2.935363951 16.240942390 0.113224200
 111 -2.935363951 16.240942390 0.113224200 -2.917635157 16.278803460 0.113961734
1 112 -2.917635157 16.278803460 0.113961734 -2.900039803 16.317283850 0.114689291
1 113 -2.900039803 16.317283850 0.114689291 -2.882593796 16.356372670 0.115406523
1 114 -2.882593796 16.356372670 0.115406523 -2.865311266 16.396059160 0.116113097
1 115 -2.865311266 16.396059160 0.116113097 -2.848204697 16.436332650 0.116808702
1 116 -2.848204697 16.436332650 0.116808702 -2.831285052 16.477182560 0.117493042
1 117 -2.831285052 16.477182560 0.117493042 -2.814561890 16.518598430 0.118165840
1 118 -2.814561890 16.518598430 0.118165840 -2.798043470 16.560569870 0.118826835
1 119 -2.798043470 16.560569870 0.118826835 -2.781736856 16.603086610 0.119475785
1\ 120\ -2.781736856\ 16.603086610\ 0.119475785\ -2.765648008\ 16.646138440\ 0.120112464
1 121 -2.765648008 16.646138440 0.120112464 -2.749782197 16.689715180 0.120736656
1 122 -2.749782197 16.689715180 0.120736656 -2.734142443 16.733806950 0.121348181
1\ 123\ -2.734142443\ 16.733806950\ 0.121348181\ -2.718732873\ 16.778403630\ 0.121946849
1 124 -2.718732873 16.778403630 0.121946849 -2.703555506 16.823495380 0.122532501
1 125 -2.703555506 16.823495380 0.122532501 -2.688611957 16.869072380 0.123104991
1 126 -2.688611957 16.869072380 0.123104991 -2.673903164 16.915124870 0.123664186
1 127 -2.673903164 16.915124870 0.123664186 -2.659429443 16.961643170 0.124209969
1 128 -2.659429443 16.961643170 0.124209969 -2.645190534 17.008617660 0.124742239
1 129 -2.645190534 17.008617660 0.124742239 -2.631185649 17.056038790 0.125260905
1 130 -2.631185649 17.056038790 0.125260905 -2.617413511 17.103897050 0.125765895
1 131 -2.617413511 17.103897050 0.125765895 -2.603872392 17.152183020 0.126257147
 132 -2.603872392 17.152183020 0.126257147 -2.590560148 17.200887320 0.126734613
1 133 -2.590560148 17.200887320 0.126734613 -2.577474253 17.250000620 0.127198260
1 134 -2.577474253 17.250000620 0.127198260 -2.564611831 17.299513670 0.127648067
1 135 -2.564611831 17.299513670 0.127648067 -2.551969684 17.349417260 0.128084023
1 136 -2.551969684 17.349417260 0.128084023 -2.539539972 17.399703080 0.128506192
1 137 -2.539539972 17.399703080 0.128506192 -2.527325681 17.450360720 0.128914497
1 138 -2.527325681 17.450360720 0.128914497 -2.515320235 17.501381610 0.129309001
 139 -2.515320235 17.501381610 0.129309001 -2.503519447 17.552756740 0.129689741
1\ 140\ -2.503519447\ 17.552756740\ 0.129689741\ -2.491918934\ 17.604477140\ 0.130056765
1 141 -2.491918934 17.604477140 0.130056765 -2.480514136 17.656533900 0.130410133
1 142 -2.480514136 17.656533900 0.130410133 -2.469300331 17.708918110 0.130749913
1 143 -2.469300331 17.708918110 0.130749913 -2.458272656 17.761620940 0.131076187
1 144 -2.458272656 17.761620940 0.131076187 -2.447426113 17.814633590 0.131389042
1 145 -2.447426113 17.814633590 0.131389042 -2.436755595 17.867947290 0.131688579
 146 -2.436755595 17.867947290 0.131688579 -2.426255887 17.921553320 0.131974905
1 147 -2.426255887 17.921553320 0.131974905 -2.415921689 17.975442990 0.132248138
1 148 -2.415921689 17.975442990 0.132248138 -2.405747619 18.029607650 0.132508403
1 149 -2.405747619 18.029607650 0.132508403 -2.395728233 18.084038680 0.132755834
1 150 -2.395728233 18.084038680 0.132755834 -2.385858029 18.138727500 0.132990575
1 151 -2.385858029 18.138727500 0.132990575 -2.376131459 18.193665550 0.133212776
1 152 -2.376131459 18.193665550 0.133212776 -2.366542942 18.248844310 0.133422595
 153 -2.366542942 18.248844310 0.133422595 -2.357086871 18.304255300 0.133620197
1 154 -2.357086871 18.304255300 0.133620197 -2.347757625 18.359890030 0.133805756
1 155 -2.347757625 18.359890030 0.133805756 -2.338549576 18.415740090 0.133979452
1\ 156\ -2.338549576\ 18.415740090\ 0.133979452\ -2.329457100\ 18.471797060\ 0.134141470
 157 -2.329457100 18.471797060 0.134141470 -2.320474586 18.528052550 0.134292005
1 158 -2.320474586 18.528052550 0.134292005 -2.311596446 18.584498200 0.134431256
1 159 -2.311596446 18.584498200 0.134431256 -2.302817124 18.641125670 0.134559427
 160 -2.302817124 18.641125670 0.134559427 -2.294131107 18.697926630 0.134676731
1 161 -2.294131107 18.697926630 0.134676731 -2.285532933 18.754892780 0.134783385
1 162 -2.285532933 18.754892780 0.134783385 -2.277017201 18.812015840 0.134879611
1 163 -2.277017201 18.812015840 0.134879611 -2.268578584 18.869287530 0.134965637
1 164 -2.268578584 18.869287530 0.134965637 -2.260211837 18.926699590 0.135041695
1 165 -2.260211837 18.926699590 0.135041695 -2.251911809 18.984243780 0.135108024
1\ 166\ -2.251911809\ 18.984243780\ 0.135108024\ -2.243673453\ 19.041911850\ 0.1351648673453
1 167 -2.243673453 19.041911850 0.135164867 -2.235491842 19.099695570 0.135212469
```

```
1 168 -2.235491842 19.099695570 0.135212469 -2.227362173 19.157586720 0.135251083
1 169 -2.227362173 19.157586720 0.135251083 -2.219279790 19.215577070 0.135280963
1 170 -2.219279790 19.215577070 0.135280963 -2.211240187 19.273658390 0.135302371
1 171 -2.211240187 19.273658390 0.135302371 -2.203239029 19.331822470 0.135315568
1 172 -2.203239029 19.331822470 0.135315568 -2.195272161 19.390061060 0.135320824
1 173 -2.195272161 19.390061060 0.135320824 -2.187335625 19.448365940 0.135318407
1 174 -2.187335625 19.448365940 0.135318407 -2.179425674 19.506728850 0.135308594
1 175 -2.179425674 19.506728850 0.135308594 -2.171538789 19.565141530 0.135291662
1 176 -2.171538789 19.565141530 0.135291662 -2.163671689 19.623595710 0.135267891
1 177 -2.163671689 19.623595710 0.135267891 -2.155821357 19.682083100 0.135237567
1 178 -2.155821357 19.682083100 0.135237567 -2.147985046 19.740595380 0.135200976
1 179 -2.147985046 19.740595380 0.135200976 -2.140160305 19.799124200 0.135158409
1 180 -2.140160305 19.799124200 0.135158409 -2.132344989 19.857661210 0.135110159
1 181 -2.132344989 19.857661210 0.135110159 -2.124537282 19.916198000 0.135056522
 182 -2.124537282 19.916198000 0.135056522 -2.116735712 19.974726150 0.134997797
1 183 -2.116735712 19.974726150 0.134997797 -2.108939167 20.033237190 0.134934285
1 184 -2.108939167 20.033237190 0.134934285 -2.101146920 20.091722620 0.134866291
1 185 -2.101146920 20.091722620 0.134866291 -2.093358637 20.150173870 0.134794121
1\ 186\ -2.093358637\ 20.150173870\ 0.134794121\ -2.085574403\ 20.208582360\ 0.134718085
1 187 -2.085574403 20.208582360 0.134718085 -2.077794735 20.266939440 0.134638494
1 188 -2.077794735 20.266939440 0.134638494 -2.070020599 20.325236420 0.134555663
1 189 -2.070020599 20.325236420 0.134555663 -2.062253431 20.383464550 0.134469910
1 190 -2.062253431 20.383464550 0.134469910 -2.054495145 20.441615010 0.134381553
1\ 191\ -2.054495145\ 20.441615010\ 0.134381553\ -2.046748156\ 20.499678940\ 0.134290916
1 192 -2.046748156 20.499678940 0.134290916 -2.039015385 20.557647400 0.134198323
1 193 -2.039015385 20.557647400 0.134198323 -2.031300282 20.615511400 0.134104101
1 194 -2.031300282 20.615511400 0.134104101 -2.023606828 20.673261890 0.134008581
1 195 -2.023606828 20.673261890 0.134008581 -2.015942013 20.730889050 0.133912066
 196 -2.015942013 20.730889050 0.133912066 -2.008305745 20.788385100 0.133814954
1 197 -2.008305745 20.788385100 0.133814954 -2.000706389 20.845740030 0.133717552
1 198 -2.000706389 20.845740030 0.133717552 -1.993150137 20.902944490 0.133620200
1 199 -1.993150137 20.902944490 0.133620200 -1.985643741 20.959989090 0.133523244
1 200 -1.985643741 20.959989090 0.133523244 -1.978194510 21.016864330 0.133427032
1 201 -1.978194510 21.016864330 0.133427032 -1.970810308 21.073560670 0.133331914
1 202 -1.970810308 21.073560670 0.1333331914 -1.963499540 21.130068500 0.133238245
  203 -1.963499540 21.130068500 0.133238245 -1.956271141 21.186378130 0.133146383
1 204 -1.956271141 21.186378130 0.133146383 -1.949134561 21.242479820 0.133056690
1 205 -1.949134561 21.242479820 0.133056690 -1.942099744 21.298363760 0.132969531
1 206 -1.942099744 21.298363760 0.132969531 -1.935177101 21.354020090 0.132885274 1 207 -1.935177101 21.354020090 0.132885274 -1.928377480 21.409438910 0.132804292
1 208 -1.928377480 21.409438910 0.132804292 -1.921712136 21.464610260 0.132726962
1 209 -1.921712136 21.464610260 0.132726962 -1.915192685 21.519524140 0.132653664
 210 -1.915192685 21.519524140 0.132653664 -1.908831065 21.574170530 0.132584784
1 211 -1.908831065 21.574170530 0.132584784 -1.902639482 21.628539370 0.132520711
1 212 -1.902639482 21.628539370 0.132520711 -1.896630358 21.682620620 0.132461838
1 213 -1.896630358 21.682620620 0.132461838 -1.890816268 21.736404190 0.132408563
1 214 -1.890816268 21.736404190 0.132408563 -1.885209876 21.789880030 0.132361289
1 215 -1.885209876 21.789880030 0.132361289 -1.879823505 21.843038190 0.132320427
1 216 -1.879823505 21.843038190 0.132320427 -1.874670324 21.895868500 0.132286382
1 217 -1.874670324 21.895868500 0.132286382 -1.869760299 21.948361680 0.132259600
1 218 -1.869760299 21.948361680 0.132259600 -1.865113245 22.000505690 0.132240418
1 219 -1.865113245 22.000505690 0.132240418 -1.860734944 22.052292420 0.132229330
1 220 -1.860734944 22.052292420 0.132229330 -1.856633840 22.103713050 0.132226801
1 221 -1.856633840 22.103713050 0.132226801 -1.852827186 22.154756030 0.132233201
1 222 -1.852827186 22.154756030 0.132233201 -1.849323204 22.205412490 0.132248993
1 223 -1.849323204 22.205412490 0.132248993 -1.846131607 22.255673000 0.132274625
 224 -1.846131607 22.255673000 0.132274625 -1.843261294 22.305528310 0.132310549
1 225 -1.843261294 22.305528310 0.132310549 -1.840720248 22.354969300 0.132357221
1 226 -1.840720248 22.354969300 0.132357221 -1.838515440 22.403987060 0.132415103
1\ 227\ -1.838515440\ 22.403987060\ 0.132415103\ -1.836655860\ 22.452571820\ 0.132484631
1 228 -1.836655860 22.452571820 0.132484631 -1.835138046 22.500717780 0.132566359
1 229 -1.835138046 22.500717780 0.132566359 -1.833972004 22.548414370 0.132660699
1 230 -1.833972004 22.548414370 0.132660699 -1.833157751 22.595654220 0.132768153
1 231 -1.833157751 22.595654220 0.132768153 -1.832695620 22.642429560 0.132889211
1 232 -1.832695620 22.642429560 0.132889211 -1.832584342 22.688732920 0.133024368
1 233 -1.832584342 22.688732920 0.133024368 -1.832820974 22.734557130 0.133174129
1 234 -1.832820974 22.734557130 0.133174129 -1.833400825 22.779895300 0.133338999
1 235 -1.833400825 22.779895300 0.133338999 -1.834317405 22.824740870 0.133519496
1 236 -1.834317405 22.824740870 0.133519496 -1.835557520 22.869089120 0.133716192
1 237 -1.835557520 22.869089120 0.133716192 -1.837119466 22.912931510 0.133929525
1 238 -1.837119466 22.912931510 0.133929525 -1.838987063 22.956263730 0.134160073
```

```
1 239 -1.838987063 22.956263730 0.134160073 -1.841146139 22.999080620 0.134408381
2 24 -0.948720233 16.458752720 0.085877732 -1.024496827 16.388040560 0.085025838
2 25 -1.024496827 16.388040560 0.085025838 -1.102698353 16.318971900 0.084214052
  26 -1.102698353 16.318971900 0.084214052 -1.183966350 16.252079850 0.083455124
  27 -1.183966350 16.252079850 0.083455124 -1.268071036 16.187346690 0.082748284
 28 -1.268071036 16.187346690 0.082748284 -1.354751525 16.124754480 0.082092737
  29 -1.354751525 16.124754480 0.082092737 -1.443689692 16.064287620 0.081487717
  30 \;\; -1.443689692 \;\; 16.064287620 \;\; 0.081487717 \;\; -1.534541920 \;\; 16.005930010 \;\; 0.080932448 \\
  31 -1.534541920 16.005930010 0.080932448 -1.626928093 15.949666310 0.080426175
  32 -1.626928093 15.949666310 0.080426175 -1.720434829 15.895481970 0.079968176
  33 -1.720434829 15.895481970 0.079968176 -1.814635262 15.843361790 0.079557735
  34 -1.814635262 15.843361790 0.079557735 -1.909076262 15.793291460 0.079194187
  35 \;\; -1.909076262 \;\; 15.793291460 \;\; 0.079194187 \;\; -2.003296102 \;\; 15.745256400 \;\; 0.078876895
  36 \; -2.003296102 \; 15.745256400 \; 0.078876895 \; -2.096828937 \; 15.699241880 \; 0.078605255
  37 -2.096828937 15.699241880 0.078605255 -2.189211877 15.655232820 0.078378696
  38 -2.189211877 15.655232820 0.078378696 -2.279991982 15.613213710 0.078196674
  39 -2.279991982 15.613213710 0.078196674 -2.368732949 15.573168430 0.078058667
  40 -2.368732949 15.573168430 0.078058667 -2.455021314 15.535080190 0.077964169
  41 \;\; -2.455021314 \;\; 15.535080190 \;\; 0.077964169 \;\; -2.538471972 \;\; 15.498931450 \;\; 0.077912684
  42 -2.538471972 15.498931450 0.077912684 -2.618732901 15.464703840 0.077903716
  43 -2.618732901 15.464703840 0.077903716 -2.695488973 15.432378170 0.077936763
  44 -2.695488973 15.432378170 0.077936763 -2.768464816 15.401934360 0.078011309
  45 -2.768464816 15.401934360 0.078011309 -2.837426693 15.373351540 0.078126817
 46 -2.837426693 15.373351540 0.078126817 -2.902178205 15.346608420 0.078282739
  47 -2.902178205 15.346608420 0.078282739 -2.962580386 15.321681810 0.078478449
  48 -2.962580386 15.321681810 0.078478449 -3.018521987 15.298548970 0.078713325
  49 -3.018521987 15.298548970 0.078713325 -3.069936555 15.277186180 0.078986694
  50 \;\; -3.069936555 \;\; 15.277186180 \;\; 0.078986694 \;\; -3.116795864 \;\; 15.257569200 \;\; 0.079297841
  51 -3.116795864 15.257569200 0.079297841 -3.159107331 15.239673380 0.079646006
  52 \; -3.159107331 \; 15.239673380 \; 0.079646006 \; -3.196911083 \; 15.223473710 \; 0.080030389
  53 -3.196911083 15.223473710 0.080030389 -3.230276759 15.208944910 0.080450145
  54 -3.230276759 15.208944910 0.080450145 -3.259300182 15.196061520 0.080904391
  55 -3.259300182 15.196061520 0.080904391 -3.284099963 15.184797990 0.081392203
  56 -3.284099963 15.184797990 0.081392203 -3.304814150 15.175128710 0.081912623
  57 -3.304814150 15.175128710 0.081912623 -3.321596954 15.167028110 0.082464661
  58 \;\; -3.321596954 \;\; 15.167028110 \;\; 0.082464661 \;\; -3.334615646 \;\; 15.160470680 \;\; 0.083047295
  59 -3.334615646 15.160470680 0.083047295 -3.344047622 15.155431070 0.083659478
   60 \quad -3.344047622 \quad 15.155431070 \quad 0.083659478 \quad -3.350077710 \quad 15.151884050 \quad 0.084300139 
  61 \;\; -3.350077710 \;\; 15.151884050 \;\; 0.084300139 \;\; -3.352893805 \;\; 15.149804790 \;\; 0.084968200
  62 -3.352893805 15.149804790 0.084968200 -3.352691376 15.149168250 0.085662539
  63 -3.352691376 15.149168250 0.085662539 -3.349664380 15.149949840 0.086382035
  64 -3.349664380 15.149949840 0.086382035 -3.343998803 15.152125850 0.087125591
  65 -3.343998803 15.152125850 0.087125591 -3.335889574 15.155671860 0.087892047
  66 -3.335889574 15.155671860 0.087892047 -3.325522491 15.160564190 0.088680264
  67 \;\; \textbf{-3.325522491} \;\; 15.160564190 \;\; 0.088680264 \;\; \textbf{-3.313078460} \;\; 15.166779470 \;\; 0.089489106
  68 \;\; \textbf{-3.313078460} \;\; 15.166779470} \;\; 0.089489106 \;\; \textbf{-3.298732648} \;\; 15.174294640} \;\; 0.090317434
  69 -3.298732648 15.174294640 0.090317434 -3.282653831 15.183086940 0.091164117
  70 -3.282653831 15.183086940 0.091164117 -3.265003896 15.193133900 0.092028028
  71 -3.265003896 15.193133900 0.092028028 -3.245937506 15.204413350 0.092908048
  72 -3.245937506 15.204413350 0.092908048 -3.225606516 15.216902960 0.093803033
  73 \;\; -3.225606516 \;\; 15.216902960 \;\; 0.093803033 \;\; -3.204146115 \;\; 15.230581500 \;\; 0.094711916
  74 -3.204146115 15.230581500 0.094711916 -3.181690237 15.245427450 0.095633595
  75 -3.181690237 15.245427450 0.095633595 -3.158363475 15.261419660 0.096566992
  76 -3.158363475 15.261419660 0.096566992 -3.134282833 15.278537280 0.097511046
  77 -3.134282833 15.278537280 0.097511046 -3.109557879 15.296759670 0.098464710
  78 -3.109557879 15.296759670 0.098464710 -3.084290931 15.316066440 0.099426955
  79 -3.084290931 15.316066440 0.099426955 -3.058577292 15.336437450 0.100396769
  80 -3.058577292 15.336437450 0.100396769 -3.032505499 15.357852740 0.101373159
  81 -3.032505499 15.357852740 0.101373159 -3.006157600 15.380292610 0.102355150
  82 -3.006157600 15.380292610 0.102355150 -2.979609448 15.403737540 0.103341788
  83 \; -2.979609448 \; 15.403737540 \; 0.103341788 \; -2.952930993 \; 15.428168190 \; 0.104332139
  84 -2.952930993 15.428168190 0.104332139 -2.926186592 15.453565450 0.105325289
 85 -2.926186592 15.453565450 0.105325289 -2.899435307 15.479910370 0.106320346
  86 -2.899435307 15.479910370 0.106320346 -2.872731211 15.507184190 0.107316440
2 87 -2.872731211 15.507184190 0.107316440 -2.846123683 15.535368290 0.108312721
 88 -2.846123683 15.535368290 0.108312721 -2.819657704 15.564444260 0.109308364
  89 -2.819657704 15.564444260 0.109308364 -2.793374145 15.594393800 0.110302563
  90 -2.793374145 15.594393800 0.110302563 -2.767310047 15.625198800 0.111294537
  91 -2.767310047 15.625198800 0.111294537 -2.741498897 15.656841260 0.112283526
  92 -2.741498897 15.656841260 0.112283526 -2.715970894 15.689303330 0.113268793
  93 -2.715970894 15.689303330 0.113268793 -2.690753197 15.722567300 0.114249622
```

```
2 94 -2.690753197 15.722567300 0.114249622 -2.665870146 15.756615550 0.115225321
2 95 -2.665870146 15.756615550 0.115225321 -2.641343436 15.791430620 0.116195218
2 96 -2.641343436 15.791430620 0.116195218 -2.617192204 15.826995170 0.117158667
 97 -2.617192204 15.826995170 0.117158667 -2.593430614 15.863292410 0.118115073
2 98 -2.593430614 15.863292410 0.118115073 -2.570076037 15.900304840 0.119063807
 99 -2.570076037 15.900304840 0.119063807 -2.547141473 15.938015450 0.120004290
 100 -2.547141473 15.938015450 0.120004290 -2.524635245 15.976407870 0.120935994
 101 -2.524635245 15.976407870 0.120935994 -2.502569666 16.015464830 0.121858355
2 102 -2.502569666 16.015464830 0.121858355 -2.480951890 16.055169840 0.122770870
2 103 -2.480951890 16.055169840 0.122770870 -2.459785573 16.095506880 0.123673085
 104 -2.459785573 16.095506880 0.123673085 -2.439080117 16.136458810 0.124564484
 105 -2.439080117 16.136458810 0.124564484 -2.418838304 16.178009550 0.125444639
 106 -2.418838304 16.178009550 0.125444639 -2.399063683 16.220142810 0.126313121
 107 -2.399063683 16.220142810 0.126313121 -2.379756861 16.262842770 0.127169545
 108 -2.379756861 16.262842770 0.127169545 -2.360920527 16.306093160 0.128013515
2 109 -2.360920527 16.306093160 0.128013515 -2.342557728 16.349877590 0.128844639
2 110 -2.342557728 16.349877590 0.128844639 -2.324663326 16.394181180 0.129662637
 111 -2.324663326 16.394181180 0.129662637 -2.307240716 16.438987410 0.130467138
 112 -2.307240716 16.438987410 0.130467138 -2.290287663 16.484280820 0.131257852
 113 -2.290287663 16.484280820 0.131257852 -2.273803847 16.530045540 0.132034479
 114 -2.273803847 16.530045540 0.132034479 -2.257782149 16.576267130 0.132796819
 115 -2.257782149 16.576267130 0.132796819 -2.242227723 16.622928640 0.133544525
2 116 -2.242227723 16.622928640 0.133544525 -2.227132805 16.670015720 0.134277436
2 117 -2.227132805 16.670015720 0.134277436 -2.212495585 16.717512880 0.134995324
 118 -2.212495585 16.717512880 0.134995324 -2.198312750 16.765404960 0.135697996
 119 -2.198312750 16.765404960 0.135697996 -2.184580762 16.813676890 0.136385276
2 120 -2.184580762 16.813676890 0.136385276 -2.171295888 16.862313660 0.137057004
 121 -2.171295888 16.862313660 0.137057004 -2.158454232 16.911300360 0.137713039
 122 -2.158454232 16.911300360 0.137713039 -2.146051754 16.960622160 0.138353254
2 123 -2.146051754 16.960622160 0.138353254 -2.134084303 17.010264300 0.138977537
2 124 -2.134084303 17.010264300 0.138977537 -2.122547629 17.060212130 0.139585795
 125 -2.122547629 17.060212130 0.139585795 -2.111437411 17.110451060 0.140177947
2 126 -2.111437411 17.110451060 0.140177947 -2.100749266 17.160966560 0.140753927
2 127 -2.100749266 17.160966560 0.140753927 -2.090478774 17.211744240 0.141313686
2 128 -2.090478774 17.211744240 0.141313686 -2.080621484 17.262769730 0.141857186
 129 -2.080621484 17.262769730 0.141857186 -2.071172932 17.314028780 0.142384404
2 130 -2.071172932 17.314028780 0.142384404 -2.062128649 17.365507200 0.142895332
 131 -2.062128649 17.365507200 0.142895332 -2.053484173 17.417190900 0.143389972
 132 -2.053484173 17.417190900 0.143389972 -2.045235058 17.469065850 0.143868341
 133 -2.045235058 17.469065850 0.143868341 -2.037376880 17.521118110 0.144330469
2 134 -2.037376880 17.521118110 0.144330469 -2.029906684 17.5733333470 0.144776372
 135 -2.029906684 17.573333470 0.144776372 -2.022817914 17.625698690 0.145206138
 136 -2.022817914 17.625698690 0.145206138 -2.016107084 17.678199870 0.145619819
2 137 -2.016107084 17.678199870 0.145619819 -2.009769905 17.730823400 0.146017491
 138 -2.009769905 17.730823400 0.146017491 -2.003802134 17.783555750 0.146399239
 139 -2.003802134 17.783555750 0.146399239 -1.998199572 17.836383470 0.146765161
 140 -1.998199572 17.836383470 0.146765161 -1.992958064 17.889293210 0.147115364
 141 -1.992958064 17.889293210 0.147115364 -1.988073505 17.942271680 0.147449967
 142 -1.988073505 17.942271680 0.147449967 -1.983541835 17.995305700 0.147769097
 143 -1.983541835 17.995305700 0.147769097 -1.979359041 18.048382160 0.148072891
 144 -1.979359041 18.048382160 0.148072891 -1.975521156 18.101488040 0.148361495
2 145 -1.975521156 18.101488040 0.148361495 -1.972024258 18.154610390 0.148635067
 146 -1.972024258 18.154610390 0.148635067 -1.968864465 18.207736390 0.148893769
 147 -1.968864465 18.207736390 0.148893769 -1.966037938 18.260853250 0.149137776
2 148 -1.966037938 18.260853250 0.149137776 -1.963540872 18.313948320 0.149367270
 149 -1.963540872 18.313948320 0.149367270 -1.961369499 18.367009020 0.149582439
 150 -1.961369499 18.367009020 0.149582439 -1.959520079 18.420022840 0.149783482
2 151 -1.959520079 18.420022840 0.149783482 -1.957988900 18.472977390 0.149970604
2 152 -1.957988900 18.472977390 0.149970604 -1.956772271 18.525860350 0.150144020
 153 -1.956772271 18.525860350 0.150144020 -1.955866520 18.578659510 0.150303950
 154 -1.955866520 18.578659510 0.150303950 -1.955267984 18.631362750 0.150450621
2 155 -1.955267984 18.631362750 0.150450621 -1.954973011 18.683958010 0.150584270
 156 -1.954973011 18.683958010 0.150584270 -1.954977947 18.736433380 0.150705138
 157 -1.954977947 18.736433380 0.150705138 -1.955279136 18.788777000 0.150813475
2 158 -1.955279136 18.788777000 0.150813475 -1.955872909 18.840977130 0.150909535
2 159 -1.955872909 18.840977130 0.150909535 -1.956755579 18.893022120 0.150993582
 160 -1.956755579 18.893022120 0.150993582 -1.957923436 18.944900410 0.151065883
 161 -1.957923436 18.944900410 0.151065883 -1.959372737 18.996600550 0.151126714
 162 -1.959372737 18.996600550 0.151126714 -1.961099700 19.048111180 0.151176355
 163 -1.961099700 19.048111180 0.151176355 -1.963100496 19.099421050 0.151215094
 164 -1.963100496 19.099421050 0.151215094 -1.965371240 19.150518990 0.151243223
```

```
2 165 -1.965371240 19.150518990 0.151243223 -1.967907983 19.201393970 0.151261042
2 166 -1.967907983 19.201393970 0.151261042 -1.970706706 19.252035030 0.151268855
2 167 -1.970706706 19.252035030 0.151268855 -1.973763307 19.302431310 0.151266974
 168 -1.973763307 19.302431310 0.151266974 -1.977073595 19.352572090 0.151255713
2 169 -1.977073595 19.352572090 0.151255713 -1.980633277 19.402446710 0.151235395
 170 -1.980633277 19.402446710 0.151235395 -1.984437954 19.452044650 0.151206347
 171 -1.984437954 19.452044650 0.151206347 -1.988483106 19.501355480 0.151168902
 172 -1.988483106 19.501355480 0.151168902 -1.992764085 19.550368880 0.151123398
2 173 -1.992764085 19.550368880 0.151123398 -1.997276103 19.599074640 0.151070180
2 174 -1.997276103 19.599074640 0.151070180 -2.002014224 19.647462660 0.151009595
 175 -2.002014224 19.647462660 0.151009595 -2.006973350 19.695522940 0.150942000
 176 -2.006973350 19.695522940 0.150942000 -2.012148213 19.743245600 0.150867753
 177 -2.012148213 19.743245600 0.150867753 -2.017533363 19.790620860 0.150787221
 178 -2.017533363 19.790620860 0.150787221 -2.023123159 19.837639070 0.150700774
 179 -2.023123159 19.837639070 0.150700774 -2.028911755 19.884290660 0.150608788
2 180 -2.028911755 19.884290660 0.150608788 -2.034893091 19.930566200 0.150511645
2 181 -2.034893091 19.930566200 0.150511645 -2.041060881 19.976456360 0.150409731
 182 -2.041060881 19.976456360 0.150409731 -2.047408604 20.021951920 0.150303440
 183 -2.047408604 20.021951920 0.150303440 -2.053929490 20.067043770 0.150193169
 184 -2.053929490 20.067043770 0.150193169 -2.060616513 20.111722910 0.150079322
 185 -2.060616513 20.111722910 0.150079322 -2.067462375 20.155980470 0.149962308
 186 -2.067462375 20.155980470 0.149962308 -2.074459502 20.199807670 0.149842540
2 187 -2.074459502 20.199807670 0.149842540 -2.081600029 20.243195860 0.149720441
2 188 -2.081600029 20.243195860 0.149720441 -2.088875793 20.286136480 0.149596434
 189 -2.088875793 20.286136480 0.149596434 -2.096278323 20.328621090 0.149470953
 190 -2.096278323 20.328621090 0.149470953 -2.103798828 20.370641380 0.149344433
 191 -2.103798828 20.370641380 0.149344433 -2.111428194 20.412189110 0.149217319
 192 -2.111428194 20.412189110 0.149217319 -2.119156972 20.453256170 0.149090060
 193 -2.119156972 20.453256170 0.149090060 -2.126975375 20.493834570 0.148963110
2 194 -2.126975375 20.493834570 0.148963110 -2.134873266 20.533916400 0.148836931
2 195 -2.134873266 20.533916400 0.148836931 -2.142840157 20.573493870 0.148711989
 196 -2.142840157 20.573493870 0.148711989 -2.150865204 20.612559290 0.148588757
 197 -2.150865204 20.612559290 0.148588757 -2.158937201 20.651105060 0.148467715
 198 -2.158937201 20.651105060 0.148467715 -2.167044578 20.689123700 0.148349348
 199 -2.167044578 20.689123700 0.148349348 -2.175176987 20.726607280 0.148234120
 200 -2.175176987 20.726607280 0.148234120 -2.183317362 20.763550110 0.148122614
 201 -2.183317362 20.763550110 0.148122614 -2.191457792 20.799943370 0.148015249
 202 -2.191457792 20.799943370 0.148015249 -2.199583649 20.835780510 0.147912564
 203 -2.199583649 20.835780510 0.147912564 -2.207681525 20.871054490 0.147815078
 204 -2.207681525 20.871054490 0.147815078 -2.215737645 20.905758390 0.147723315
 205 -2.215737645 20.905758390 0.147723315 -2.223739902 20.939884770 0.147637768
 206 -2.223739902 20.939884770 0.147637768 -2.231667995 20.973428580 0.147559083
 207 -2.231667995 20.973428580 0.147559083 -2.239511942 21.006381710 0.147487716
 208 -2.239511942 21.006381710 0.147487716 -2.247257081 21.038737400 0.147424210
 209 -2.247257081 21.038737400 0.147424210 -2.254885145 21.070489960 0.147369174
 210 -2.254885145 21.070489960 0.147369174 -2.262382090 21.101632410 0.147323144
 211 -2.262382090 21.101632410 0.147323144 -2.269731517 21.132158450 0.147286698
 212 -2.269731517 21.132158450 0.147286698 -2.276917229 21.162061710 0.147260415
 213 -2.276917229 21.162061710 0.147260415 -2.283925442 21.191335100 0.147244828
 214 -2.283925442 21.191335100 0.147244828 -2.290731442 21.219974720 0.147240683
 215 -2.290731442 21.219974720 0.147240683 -2.297324270 21.247972620 0.147248467
 216 -2.297324270 21.247972620 0.147248467 -2.303687802 21.275322390 0.147268770
 217 -2.303687802 21.275322390 0.147268770 -2.309799971 21.302019330 0.147302299
 218 -2.309799971 21.302019330 0.147302299 -2.315651874 21.328054890 0.147349514
 219 -2.315651874 21.328054890 0.147349514 -2.321217310 21.353425630 0.147411215
 220 -2.321217310 21.353425630 0.147411215 -2.326481911 21.378124620 0.147487979
 221 -2.326481911 21.378124620 0.147487979 -2.331428139 21.402145890 0.147580453
2 222 -2.331428139 21.402145890 0.147580453 -2.336038473 21.425483510 0.147689289
 223 -2.336038473 21.425483510 0.147689289 -2.340295450 21.448131560 0.147815150
 224 -2.340295450 21.448131560 0.147815150 -2.344181703 21.470084120 0.147958706
 225 -2.344181703 21.470084120 0.147958706 -2.347680000 21.491335290 0.148120633
 226 -2.347680000 21.491335290 0.148120633 -2.350773286 21.511879180 0.148301619
 227 -2.350773286 21.511879180 0.148301619 -2.353444725 21.531709890 0.148502355
 228 -2.353444725 21.531709890 0.148502355 -2.355677743 21.550821550 0.148723546
 229 -2.355677743 21.550821550 0.148723546 -2.357456070 21.569208240 0.148965902
 230 -2.357456070 21.569208240 0.148965902 -2.358763788 21.586864060 0.149230142
 231 -2.358763788 21.586864060 0.149230142 -2.359585369 21.603783090 0.149516994
 232 -2.359585369 21.603783090 0.149516994 -2.359905726 21.619959390 0.149827195
 233 -2.359905726 21.619959390 0.149827195 -2.359710258 21.635387000 0.150161492
 234 -2.359710258 21.635387000 0.150161492 -2.358980464 21.650061260 0.150520734
 235 -2.358980464 21.650061260 0.150520734 -2.357714508 21.663972700 0.150905439
```

```
2 236 -2.357714508 21.663972700 0.150905439 -2.355892424 21.677117360 0.151316531
2 237 -2.355892424 21.677117360 0.151316531 -2.353501353 21.689489350 0.151754808
2 238 -2.353501353 21.689489350 0.151754808 -2.350528726 21.701082880 0.152221086
2 239 -2.350528726 21.701082880 0.152221086 -2.346962247 21.711892250 0.152716206
run;
data curves;
    merge htcrv wtcrv bmicrv;
           by sex _age;
run;
data test;
     set datain;
     _age=int(agemos+0.5);
                                                             *age rounded to nearest month;
     _id=_N_;
proc sort data=test out=test2;
   by sex _age _id;
run:
data test2;
     merge test2(in=a) curves(in=b);
          by sex _age;
     if a;
     if height lt 45 or height gt 300 then ht=.;
                                                             *implausible height;
     else ht=height;
     if weight lt 10 or weight gt 150 then _wt=.;
                                                             *implausible weight;
     else wt=weight;
     if bmi lt 10 or bmi gt 45 then bmi=.;
                                                             *implausible bmi;
     else bmi=bmi;
     r=(agemos-age+0.5);
      ***HEIGHT***;
     if _ht eq . then do;
         _ZH=.; _BIVH=.;
     end;
     else do;
       _{\rm LH} = _{\rm LH1+_r*(_LH2-_LH1)};
        MH = MH1+_r*(_MH2-_MH1);
SH = SH1+ r*(_SH2-_SH1);
       if ( LH gt -0.01 and LH lt 0.01) then ZH=log( ht/ MH)/ SH;
       else _ZH=((_ht/_Mh)**_LH-1)/(_LH*_SH);

_LOH=((_MH-_MH*(1-2*_LH*_SH)**(1/_LH))/2);

_HIH=((_MH*(1+2*_LH*_SH)**(1/_LH)-_MH)/2);
       if ht lt MH then flagH=( ht- MH) / LOH;
       else flagH=( ht- MH) / HIH;
       if flagH eq . then BIVH=.;
       else if flagH lt -5 then BIVH=1; *implausibly low value;
       else if flagH gt \bf 3 then _BIVH=\bf 2; *implausibly high value;
       else BIVH=0;
                                               *acceptable value;
     end;
     ***WEIGHT***;
     if \mbox{wt eq} . then do;
         ZW=.; BIVW=.;
     end;
     else do;
        LW = LW1+ r*(LW2-LW1);
       __MW = _MW1+_r*(_MW2-_MW1);
_SW = _SW1+_r*(_SW2-_SW1);
       if ( LW gt -0.01 and LW lt 0.01) then ZW=log( wt/ MW)/ SW;
       else ZW=(( wt/ MW) ** LW-1)/( LW* SW);
       _LOW=((_MW-_MW*(1-2*_LW*_SW)**(1/_LW))/2);
_HIW=((_MW*(1+2*_LW*_SW)**(1/_LW)-_MW)/2);
       if wt lt MW then flagW=(_wt-_MW)/_LOW;
       else flagW=( wt- MW)/ HIW;
       if flagW eq . then BIVW=.;
```

ISN/Protocol 178-CL-206A

```
else if flagW lt -5 then BIVW=1; *implausibly low value; else if flagW gt 5 then BIVW=2; *implausibly high value; else _BIVW=0; *acceptable value;
     end;
     ***BMI***;
     if \_bmi eq . then do;
         _ZB=.; _BIVB=.;
     end;
     else do;
                 LB1+ r*( LB2- LB1);
         LB =
        _____MB = __MB1+ r*(_MB2-_MB1);
SB = __SB1+ r*(_SB2-_SB1);
        if (_LB gt -0.01 and _LB lt 0.01) then _ZB=log(_bmi/_MB)/_SB; else ZB=(( bmi/ MB)** LB-1)/( LB* SB);
         LOB=(( MB- MB*(1-2* LB* SB)**(1/ LB))/2);
          _HIB=((_MB*(1+2*_LB*_SB)**(1/_LB)-_MB)/2);
       if _bmi lt _MB then flagB=(_bmi-_MB)/_LOB;
       else flagB=( bmi- MB)/ HIB;
       if flagB eq . then _{BIVB=.;}
       else if flagB lt -4 then BIVB=1; *implausibly low value;
       else if flagB gt 5 then _BIVB=2; *implausibly high value; else _BIVB=0; *acceptable value;
   end:
   keep _id _zh _bivh _zw _bivw _zb _bivb;
*output dataset contains original data plus Z scores and BIV flags for height, weight and
BMI;
proc sort data=test2;
     by _id;
data dataout(drop= id);
      merge test(drop=_age) test2;
             by _id;
run:
```

## 10.13 Appendix 13: ECG Abnormality Codes

ECG abnormalities are coded according to the class of the abnormality and specific type. Each type of abnormality is given a particular abnormality code. The classes of abnormality and the form of the abnormality codes for each class are as follows:

| Abnormality Class | Form of Abnormality Code |
|-------------------|--------------------------|
| Rhythm | 1xy or 1xy.z |
| PR Intervals | 3xy or 3xy.z |
| QT Intervals | 4xy or 4xy.z |
| P Wave | 6xy or 6xy.z |
| QRS Complex | 7xy or 7xy.z |
| ST Segment | 8xy or 8xy.z |
| T Wave | 90x or 90x.y |
| Other | 98x or 98x.y |

Specific abnormalities coded in each class are as follows:

#### Class: Rhythm

| Abnormality Text |
|-----------------------------------------------|
| Sinus Tachycardia |
| Sinus Bradycardia |
| Atrial Tachycardia - Without Block |
| Atrial Tachycardia - With Block |
| Atrial Flutter |
| Atrial Fibrillation |
| Ectopic Atrial Rhythm |
| PSVT(Paroxysmal Supraventricular Tachycardia) |
| Variable Atrial Pacemaker |
| Junctional Rhythm without Aberrancy |
| Junctional Rhythm with Aberrancy |
| Junctional Tachycardia |
| Junctional Rhythm |
| Ventricular Rhythm |
| Ventricular Tachycardia |
| Sustained Ventricular Tachycardia |
| Non-sustained Ventricular Tachycardia |
| Torsades de Pointes |

| Abnormality Code | Abnormality Text |
|------------------|------------------------------------------------------|
| 112.5 | Idioventricular Rhythm |
| 113 | Accelerated AV Conduction Pattern |
| 113.5 | Short PR Interval without Ventricular Pre-Excitation |
| 114 | Wolff - Parkinson - White Pattern |
| 115 | Supraventricular Ectopic Beats |
| 115.2 | Frequent Atrial Premature Complexes (>3) |
| 115.3 | Atrial Premature Complexes |
| 115.4 | Supraventricular Tachycardia |
| 115.5 | Ectopic Supraventricular Rhythm |
| 116 | Ventricular Ectopic Beats – Unifocal |
| 117 | Ventricular Ectopic Beats – Multifocal |
| 118 | Pacemaker Rhythm |
| 119 | Ventricular Fibrillation |
| 119.4 | Frequent Ventricular Premature Complexes (>2) |
| 119.5 | Ventricular Premature Complexes |
| 120 | Sinus Arrest |
| 120.5 | Sinus Pause |
| 121 | Sinus Arrhythmia |
| 122 | Nodal Tachycardia |
| 123 | LGL Syndrome |
| 124 | Junctional Escape Complexes |
| 125 | Sino - Atrial Block |
| 199.4 | Ectopy Other |
| 199.5 | Rhythm Other |

#### **Class: PR Intervals**

| Abnormality Code | Abnormality Text |
|------------------|------------------------------------|
| 301 | First Degree AV Block |
| 302 | Second Degree AV Block - Mobitz I |
| 303 | Second Degree AV Block - Mobitz II |
| 304 | Complete AV Block |
| 304.5 | 2:1 AV Block |
| 399.5 | Conduction Other |

ISN/Protocol 178-CL-206A

#### **Class: QT Intervals**

| Abnormality Code | Abnormality Text |
|------------------|------------------------|
| 401 | D 1 1OT I 1 |
| 401 | Prolonged QT Interval |
| 402 | Prolonged QTc interval |

#### Class: P Wave

| Abnormality Code | Abnormality Text |
|------------------|------------------------------------|
| 601 | Right Atrial Enlargement |
| 602 | Left Atrial Enlargement |
| 602.5 | Borderline Left Atrial Enlargement |
| 603 | P-Wave Abnormality |

#### **Class: QRS Complex**

| Abnormality Code | Abnormality Text |
|------------------|-----------------------------------------------|
| 701 | AV Dissociation |
| 702 | Left Anterior Hemiblock |
| 703 | Left Posterior Hemiblock |
| 704 | Right Bundle Branch Block |
| 705 | Incomplete Right Bundle Branch Block |
| 706 | Left Bundle Branch Block |
| 707 | Incomplete Left Bundle Branch Block |
| 708 | Nonspecific Intraventricular Conduction Delay |
| 709 | Bifascicular Block |
| 710 | Left Axis Deviation |
| 711 | Right Axis Deviation |
| 712 | Abnormal QRS Axis |
| 712.5 | Indeterminate Axis |
| 713 | Left Ventricular Hypertrophia |
| 714 | Left Ventricular Hypertrophia by Voltage Only |
| 714.4 | Left Atrial Abnormality |
| 714.5 | Left Ventricular Hypertrophy with Strain |
| 715 | Right Ventricular Hypertrophia |
| 715.5 | Right Atrial Abnormality |
| 716 | Old Myocardial Infarction: Antero Septal |
| 716.4 | Septal MI V1, V2, (V3) |
| 716.5 | Antero Septal MI V1-V4 |

ISN/Protocol 178-CL-206A

| Abnormality Text |
|---------------------------------------------|
| Old Myogardial Inforation: Antara Lateral |
| Old Myocardial Infarction: Antero Lateral |
| Extensive Anterior MI 1, L, V1-V6 |
| Antero Lateral MI V3-V6 |
| Old Myocardial Infarction: Infero Lateral |
| Anterior MI V3, V4 |
| Old Myocardial Infarction: Infero Posterior |
| Inferior MI (2), 3, F |
| Old Myocardial Infarction: Postero Lateral |
| Old Myocardial Infarction: Lateral |
| Lateral MI 1, L, V5, V6 |
| High Lateral MI 1, AVL |
| Low Voltage QRS Complex |
| Poor R-Wave Progression |
| Late R-Wave Transition |
| Early Repolarization - Normal Variant |
| Early R-Wave Transition |
| Morphology Other |
| Myocardial Infarction Other |

## **Class: ST Segment**

| Abnormality Code | Abnormality Text |
|------------------|----------------------------------------------------------|
| 801 | New Myocardial Infarction: Antero Septal |
| 802 | New Myocardial Infarction: Antero Lateral |
| 803 | New Myocardial Infarction: Infero Lateral |
| 804 | New Myocardial Infarction: Infero Posterior |
| 805 | New Myocardial Infarction: Postero Lateral |
| 806 | New Myocardial Infarction: Lateral |
| 807 | Myocardial Infarction - Nontransmural -Acute or Evolving |
| 808 | ST Elevation Consistent with Ischaemia: Anterior |
| 809 | ST Elevation Consistent with Ischaemia: Septal |
| 810 | ST Elevation Consistent with Ischaemia: Lateral |
| 811 | ST Elevation Consistent with Ischaemia: Inferior |
| 812 | ST Elevation Consistent with Ischaemia: Posterior |
| 813 | ST Elevation Consistent with Ischaemia: High Lateral |
| 814 | ST Elevation Consistent with Pericarditis |
| 814.5 | ST Segment Elevated |
| 815 | Non-Specific ST-T Change |

| Abnormality Code | Abnormality Text |
|------------------|-----------------------------------------------------|
| 816 | ST-T Changes - Consistent with Drug Effects |
| 817 | ST Depression: Anterior |
| 818 | ST Depression: Septal |
| 819 | ST Depression: Lateral |
| 820 | ST Depression: Inferior |
| 821 | ST Depression: Posterior |
| 822 | ST Depression: High Lateral |
| 823 | ST Depression - Non-Specific |
| 823.5 | ST Segment Depressed |
| 899.5 | ST Segment Other |
| Class: T Wave | |
| Abnormality Code | Abnormality Text |
| 901 | T-Wave Inversion Suggestive of Non-Q-Wave MI |
| 902 | T-Wave Flattening or Inversion in Two or More Leads |
| 902.4 | T-Wave Flat |
| 902.5 | T-Wave Inverted |
| 903 | Non-Specific T-Wave Changes |
| 904 | T-Wave Inversion Suggestive of Ischaemia |
| 905 | T-Wave Peaking |
| 905.5 | T Wave Other |

#### **Class: Other**

| Abnormality Code | Abnormality Text |
|------------------|--------------------|
| 998 | U-Wave Abnormality |
| 998.5 | U-Wave Other |
| 999 | Other |

## 10.14 Appendix 14: Key Contributors and Approvers

# List of Key Contributors and Approvers

#### **Key Contributors**

The following contributed to or reviewed this Statistical Analysis Plan as relevant to their indicated discipline or role.

#### Primary author (s)



Page 162 of 162

# **Author and Approver Signatories**

(E-signatures are attached at end of document)

